

# STATISTICAL ANALYSIS PLAN

A multicenter, Post-Marketing Surveillance study to Monitor the Safety of Novartis Meningococcal ACWY Conjugate Vaccine (MenACWY-CRM) Administered According to the Prescribing Information to Healthy Subjects from 11 to 55 Years of Age in the Republic of South Korea

**Product Name:** Menveo (MenACWY-CRM)

Protocol No. : V59\_62

Version : V1.0

Date : 06-MAR-2013

| | | Last Update Date |
|---|---|---|
| DCIC | CONFIDENT/AL: | |
| DreamCIS inc. | THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS | 06-MAR-2013 |
| | PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRIHEN PERMISSION OF COMPANY | |
| | THE WIGHEN LEAVINGSION OF CONFAINT. | |
| STATISTICA | LANALYSIS PLAN(VI.0) | |

### **Approvals**







THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

### **Revisions**

| DATE OF<br>REVISION | INDICATION REVISION | REASON FOR CHANGE | AUTHOR<br>NAME |
|---|---|---|---|

THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

## **Table of Contents**

| Revisions | 3 |
|--------------------------------------------------|----|
| 1. Study Objective | 6 |
| 2. Study Method and Study Period | 6 |
| 2.1 Study Period | 6 |
| 2.2 Number of Subjects | 6 |
| 2.3 Study population | 6 |
| 2.3.1 Inclusion criteria | 6 |
| 2.3.2 Exclusion criteria | 7 |
| 2.4 Study Method | 7 |
| 3. Analysis Sets | 10 |
| 3.1 Safety Analysis Sets | 10 |
| 3.2 Efficacy Analysis Set | |
| 4. Endpoints | 12 |
| 4.1 Safety Endpoints | 12 |
| 5. Assessment Criteria | 12 |
| 5.1 Safety Assessment Criteria | 12 |
| 6. Statistical Analyses | 12 |
| 6.1 Baseline Characteristics | 12 |
| 6.2 Safety Analyses | 13 |
| 6.2.1 Adverse Events by Baseline Characteristics | 13 |
| 6.2.2. Analysis of Solicited AE | 14 |
| 6.2.3 Analysis of Unsolicited AE | 14 |
| 7. List of Table and Data Listings | 15 |
| 7.1 Distribution of Subjects | 15 |
| 7.2 Baseline Characteristics | |
| 7.3 Safety Analyses | 16 |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

| 8. Notes |
|-----------|
| Appendix1 |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

## STATISTICAL ANALYSIS PLAN(V1.0)

#### 1. Study Objective

The primary objective of the study is to monitor the safety of a single dose of MenACWY-CRM vaccine in subjects from 11 to 55 years of age, as evaluated by:

- 1. Local and systemic solicited reactions reported from study Day 1(day of vaccination) through study Day 7 post-vaccination
- 2. All unsolicited Adverse Events (AEs) reported from study Day 1(day of vaccination) through study Day 7 post-vaccination
- 3. Medically attended Adverse Events reported from study Day 1 to study termination (Day 29/early termination)
- 4. All Serious Adverse Events (SAEs) reported from study Day 1 to study termination (Day 29/early termination)

### 2. Study Method and Study Period

#### 2.1 Study Period

The trial period shall be from market launch date till approximately 22 May 2018.

#### 2.2 Number of Subjects

A total of approximately 3,300 subjects are planned for enrolment into this study.

Assuming a 10% drop-out rate, this should provide approximately 3,000 evaluable subjects. This sample size meets the post-licensure requirements of the KFDA to provide continued safety monitoring in the Korean population.

#### 2.3 Study population

#### 2.3.1 Inclusion criteria

Individuals eligible for enrolment in this study are those:

1. Male and female subjects from 11 to 55 years of the age at the time of Visit 1(including all 55



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

STATISTICAL ANALYSIS PLAN(V1.0)

years old subjects, up to one day before their 56<sup>th</sup> year birthday), who are scheduled to receive vaccination with MenACWY-CRM conjugate vaccine, according to the local prescribing information and routine clinical practice

- 2. To whom the nature of the study has been described and the subject or subject's parent/legal representative has provided written informed consent
- 3. Whom the investigator believes that the subject can and will comply with the requirements of the protocol
- 4. Who are in good health as determined by the outcome of medical history, physical assessment and clinical judgment of the investigator

#### 2.3.2 Exclusion criteria

Contraindication, special warnings and/or precautions, as evaluated by the investigators, reported in the MenACWY-CRM conjugate vaccine Korean prescribing information. In particular, should not be included in the study a subject who has ever had:

- 1. An allergic reaction to the active substances or any of the other ingredients of the study vaccine; an allergic reaction to diphtheria toxoid;
- 2. An illness with high fever; however, a mild fever or upper respiratory infection (for example cold) itself is not a reason to delay vaccination.

Special care should be taken for subjects having haemophilia or any other problem that may stop your blood from clotting properly, such as persons receiving blood thinners (anticoagulants)

#### 2.4 Study Method

In order to obtain information on Regulatory PMS data after market launch, NVD or delegate will create the Regulatory PMS contract with the relevant clinics/hospitals and the physician in charge of the survey shall implement this Regulatory PMS in subjects that receive MenACWY-CRM in the relevant hospital/clinic since the contract date until the number of contracted survey cases, without omission, is reached.

## Overview of Study Design

This is a multicenter post marketing surveillance study to monitor the safety of MenACWY-CRM



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

administered according to the prescribing information to 3,300 healthy subjects from 11 to 55 years of age in Korea.

Subjects will be enrolled at the time of their visit to a participating clinic or hospital for vaccination with MenACWY-CRM according to the routine clinical care.

At Visit 1 (Day 1), after obtaining consent from the subjects or subjects' parents/legal representative, the vaccination will be administered. Subjects will remain under observation for at least 30 minutes in the clinic after study immunization.

The subjects or subject's parent/legal representative will be then instructed to complete the Diary Card daily, reporting local and systemic reaction and all other AEs occurring within 7 days following immunizations, and medically attended AEs or SAEs occurring up to Day 29.

Subjects will also be instructed to return the completed diaries to the study site at Day 29 as follows:

- During a visit at the study center or
- Using the provided pre-addressed stamped envelope (PASE).

At the investigator discretion, the subject or subject's parent/legal representative will be reminded of the date of the study termination by a phone call at Day 29. If any clarification is required after Diary Card retrieval the site staff will follow up by phone, and any additional finding will be recorded on the subject's medical record.

In case the Diary Card is not retrieved within 10 days after Day 29, subject or subject's parent/legal representative will be contacted by phone to assess the occurrence of adverse events, determine the subject's clinical status and complete study termination. All information will be recorded by the site staff on the subject's medical record and collected in the appropriate section of the CRF.

All SAEs will be monitored until resolution and/or the cause is identified. If a SAE remains unresolved at study termination, a clinical assessment will be made by the investigator and the NVD regional physician to determine whether continued follow up of the SAE is needed.

Table 3.1-1: Safety Assessment Table

| Medical History: | From birth, collected at clinic |
|---|---|
| All significant past diagnoses including all allergies, | visit Day 1 |
| major surgeries requiring inpatient hospitalization, | |
| other significant injuries or hospitalizations, any | |
| conditions requiring prescription or chronic medication | |
| (i.e., >2 weeks in duration), or other significant medical | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

| conditions based on the investigator's judgment. | |
|---|---|
| Immediate reactions: | For at least 30 minutes after |
| Subjects will be assessed for immediate | vaccination |
| hypersensitivity reactions. | |
| Local reactions: | Days 1-7 after vaccination |
| Erythema, induration, pain. | |
| Systemic reactions: | Days 1-7 after vaccination |
| Chills, nausea, malaise, myalgia, arthralgia, headache, | |
| rash, fever. | |
| All unsolicited AEs will be collected | Days 1-7 after vaccination |
| Medically attended Adverse Events: | From Day 1 to study |
| Events that require a physician's visit or an emergency | termination (Day 29/early |
| room visit (events that are managed by telephone or | termination) |
| means other than a face-to-face evaluation by a | |
| clinician do not qualify as medically attended AEs). | |
| Serious AEs: | From Day 1 to study |
| All SAEs will be collected. | termination (Day 29/early |
| | termination) |
| Medications: | From Day 1 to Day 7 |
| Any medications used to treat any solicited local and | |
| systemic reaction and unsolicited AE be collected. | |
| Medications: | From Day 1 to study |
| Any medications used to treat any medically attended | termination (Day 29/early |
| AE or SAE will be collected. | termination) |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

## STATISTICAL ANALYSIS PLAN(V1.0)

#### 1. Analysis Sets

#### 1.1 Safety Analysis Sets

#### Safety Set

All subjects who

- have signed an informed consent form, undergone screening procedure(s) and received a subject number,
- received a study vaccination,
- provided post vaccination safety data.

#### Safety per protocol set

All subjects in the safety Set with the exclusions of the following cases:

- (1) Subjects administered prior to the contract date.
- (2) Subjects who didn't receive MenACWY-CRM.
- (3) Subjects who already receive MenACWY-CRM.
- (4) Follow-up failure: The subjects whose safety information can not be identified due to follow-up loss.
- (5) Not applicable to the indication of study drug [Indication]
  - To prevent invasive meningococcal disease caused by Neisseria meningitides serogroups A, C, Y and W-135 in persons 11 through 55 years of age.
- (6) Subjects who violate of Protocol: Those who do not meet one item at least of the inclusion/exclusion criteria.

[Inclusion criteria]

- 1) Male and female subjects from 11 to 55 years of the age at the time of Visit 1(including all 55 years old subjects, up to one day before their 56<sup>th</sup> year birthday), who are scheduled to receive vaccination with MenACWY-CRM conjugate vaccine, according to the local prescribing information and routine clinical practice.
- 2) To whom the nature of the study has been described and the subject or subject's parent/legal representative has provided written informed consent.
- 3) Whom the investigator believes that the subject can and will comply with the requirements of the protocol.



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

4) Who are in good health as determined by the outcome of medical history, physical assessment and clinical judgment of the investigator.

[Exclusion criteria]

- 1) An allergic reaction to the active substances or any of the other ingredients of the study vaccine; an allergic reaction to diphtheria toxoid;
- 2) An illness with high fever; however, a mild fever or upper respiratory infection (for example cold) itself is not a reason to delay vaccination.
- (7) Subjects who prescribed off-label dosage.
  - Violation of intramuscular injection only (0.5ml)

#### Non-Safety per protocol set

Subjects excluded from safety per protocol set except for subjects who did not receive MenACWY-CRM and follow-up failure.

Based on rules for estimation of each number of safety evaluation cases, the following local regulation and Guideline on Standards for re-examination for new drugs, etc \*\*afaft\* \*\* file\*\* Assistant are excluded from the safety analysis set:

- Guideline on Standards for re-examination for new drugs, etc (Chapter II, no. 3)
  Patient Population for Surveillance
  - A) Patients planned to receive a drug under surveillance by investigator's medical judgment shall be subject.
  - B) Subject who do not use within approved range shall not be included in the subject in principal.
    - X However, if data of subject whose use is beyond approved range is collected, perform analysis as a separate item.
  - C) Describe actual selection methods of subject in detail.

#### 1.2 Efficacy Analysis Set

Not Applicable



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

## STATISTICAL ANALYSIS PLAN(V1.0)

#### 2. Endpoints

## 2.1 Safety Endpoints

Safety will be assessed after administration of study vaccine in terms of the number and percentage of subjects with:

- Local and systemic solicited reactions reported from study Day 1 (day of vaccination) through study Day 7 post-vaccination;
- Unsolicited AEs reported from study Day 1 (day of vaccination) through study Day 7 post-vaccination;
- Medically attended AEs reported from study Day 1 to study termination (Day 29/early termination);
- SAEs reported from study Day 1 to study termination (Day 29/early termination).

#### 3. Assessment Criteria

#### 3.1 Safety Assessment Criteria

Not Applicable

#### 4. Statistical Analyses

#### **4.1 Baseline Characteristics**

Descriptive statistics (mean, standard deviation, median, minimum and maximum) for baseline characteristics such as age, height and weight at enrollment will be calculated in the Safety set and Safety per Protocol set.

The following baseline characteristics will be reported:



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

## STATISTICAL ANALYSIS PLAN(V1.0)

- < Subject Baseline Information >
  - gender, age, ethnic origin, weight, height, past diagnosis, pre-Immunization temperature, temperature location, pregnancy
- < Study Vaccine Information >
  - vaccine site, concomitant medications

### 4.2 Safety Analyses

The number of subjects of  $AE^{\dagger}$  and the number of  $AEs^{\dagger}$  incurred shall be calculated, the incidence rate of  $AEs^{\dagger}$  and its 95% confidence interval will be calculated using the normal approximation on the safety set and safety per protocol set.

† AE : AE includes solicited and unsolicited AE (DAY 1-7), medically attended AE (DAY 1-29) and SAE (DAY 1-29).

### **6.2.1** Adverse Events by Baseline Characteristics

 $AE^{\dagger}s$  (as described below) will be reported (n, %) for the following the baseline characteristics in the safety set and safety per protocol set :

- Age group (11-18, 19-34, 35-55)
- Children group ( $<18, \ge 18$ )
- Gender (male, female)
- Past diagnosis (yes, no)
- Temperature location (axillary, oral, rectal, ear)
- Administration site (left deltoid, right deltoid, other)
- Concomitant medication (yes, no)
- Kidney disorder (yes, no)
- Liver disorder (yes, no)
- Pregnancy (yes, no)

The n(%) of AEs<sup>†</sup> and its 95% confidence interval will be calculated using the normal approximation and analyzed using  $\chi^2$ - test or Fisher's exact test.



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

† AE : AE includes solicited and unsolicited AE (DAY 1-7) and medically attended AE (DAY 1-29) and SAEs.

#### 6.2.2. Analysis of Solicited AE

Frequencies and percentages of subjects experiencing each reaction will be presented for each symptom severity. Summary tables showing the occurrence of any local or systemic reaction overall and at each time point will also be presented (see Table 4.1.3 and 4.2.3).

Post-vaccination reactions reported from Day 1 to Day 7 will be summarized by maximal severity. The severity of local reactions, including injection-site, erythema and induration will be categorized as: none (0 mm), 1 to 25 mm, 26 to 50 mm, 51 to 100 mm, >100 mm.

The severity of pain and systemic reactions occurring up to 7 days after each vaccination will be categorized as None, Mild (present but not interfering with daily activity), Moderate (some interference with daily activity), and Severe (prevents daily activity) except for rash, which will be categorized as None, Urticarial, or other.

Body temperature will be categorized as  $<38^{\circ}$ C (no fever),  $\ge 38^{\circ}$ C (fever) and will summarized by  $0.5^{\circ}$ C increments from  $36.0^{\circ}$ C up to  $\ge 40^{\circ}$ C. Additionally, no fever vs. fever will be reported.

Each local and systemic reaction will also be categorized as none vs. any.

#### 6.2.3 Analysis of Unsolicited AE

All unsolicited AEs and MAAE recorded in the CRF will be mapped to preferred terms using the most recent MedDRA dictionary and classified by System organ class (SOC) and Preferred Terms (PT). Under the classification standard of MedDRA terms, and all AEs excluding the AEs whose causal relation with the study medication is 'Not Related' shall be treated as AEs whose causal relation cannot be excluded {hereafter "Adverse Drug Reaction(ADR)"}.

① The number and percentage of unsolicited AE (Day 1-7) and MAAE (Day 1-29) and SAEs (Day 1-29) according to the serious, severity, frequency, action taken, outcome, relationship to MenACWY-CRM regarding occurred AE will be calculated.



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# **STATISTICAL ANALYSIS PLAN(V1.0)**

- ② Unsolicited AEs (Day 1-7) and MAAE (Day 1-29) and SAEs (Day 1-29) will be classified into the preferred terms according to the serious, severity, frequency, action taken, outcome, relationship to MenACWY-CRM. Also, the number and percentage of each AE (PT) will be calculated.
- ③ The number of subjects and the number of unexpected AE/ADR, SAE/Serious ADR (SADR) and MAAE/ADR will be calculated according to the preferred terms. Also, the incidence rate will be estimated.
- ④ For subjects excluded from safety per protocol set<sup>†</sup>, The number of subjects and the number of unexpected AE/ADR, SAE/Serious ADR (SADR) and MAAE/ADR will be calculated according to the preferred terms. Also, the incidence rate will be estimated.
  - † Subject excluded from safety per protocol set: Except for subjects who didn't receive study vaccination and follow-up failure.

### 5. List of Table and Data Listings

#### 5.1 Distribution of Subjects

- Number of subjects contracted to the study: The number of subjects are to be collected(under contract) as contracted by the investigator
- Number of retrieving completed CRFs: Total number of subjects whose completed CRFs
- Number of safety assessment population: Number of safety assessment population among total number

## **5.2 Baseline Characteristics**

- Mean and standard deviation (SD) or frequency and percentage by gender, age, weight, height, past diagnosis, pre-Immunization temperature, temperature location, pregnancy
- Frequency and percentage by vaccine site, concomitant medications



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

## STATISTICAL ANALYSIS PLAN(V1.0)

#### **5.3 Safety Analyses**

- Incidence rate and the number of AEs according to the baseline characteristics (frequency and percentage)
- The number of the serious, severity, frequency, action taken, outcome, relationship to MenACWY-CRM for Unsolicited AE (DAY 1-7) and MAAE (frequency and percentage)
- The number of AEs for the severity, day, fever to MenACWY-CRM according to individual solicited AE (DAY 1-7) (frequency and percentage)
- Incidence rate and number according to the preferred terms of SAE/SADR, unexpected AE/unexpected ADR, and MAAE/ADR (frequency and percentage)
- For subjects excluded from safety per protocol set<sup>†</sup> incidence rate and number according to the preferred terms of SAE/SADR, unexpected AE/unexpected ADR, and MAAE/ADR (frequency and percentage)
  - † Subject excluded from safety per protocol set: Except for subjects who didn't receive study mediation and follow-up failure

#### 6. Notes

- Each statistical analysis will be carried out with SAS Software version 9.2 or more recent version.
- In the descriptive statistics, mean, SD, minimum, median, and maximum will be calculated for continuous variables, and frequency and percentage for categorical variables.
- Data including sign of inequality such as "≥20", ">20" will be excluded from analysis.
- All test statistics will be the results of two-sided tests with the statistical significant level of 0.05.
- The followings shall be included only in re-examination report:
  - Analysis by type of concomitant medications
  - Item ② of paragraph 6.2.3
  - Estimation of 95% confidence interval for incidence of AEs by background factors



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

## STATISTICAL ANALYSIS PLAN(V1.0)

### Appendix1

## 1. Demographic and baseline values, medication characteristics, specific characteristics

- Baseline characteristics will be reported on the safety set and safety per protocol set.

#### 1.1 Safety Set

Table 1.1.1 Total subject

| Safety Set | Total |
|------------|------------------|
| | No. subjects (%) |
| Total | - |

#### Table 1.1.2 Demographic characteristics

1) (Administration start date)-(birth)+1

| Safety Set | | Total |
|-----------------------|--------------|------------------|
| | | No. subjects (%) |
| Age(years)1) | No. subjects | |
| | mean±std | |
| | median | |
| | min~max | |
| Age(years) | 11-18 | |
| | 19-34 | |
| | 35-55 | |
| | Total | |
| Children group(years) | < 18 | |
| | ≥ 18 | |
| | Total | |
| Ethnic Origin | Asian | |
| | Black | |
| | Caucasian | |
| | Hispanic | |
| | Other | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

| Safety Set | | Total |
|------------------------------------------|--------------|------------------|
| | | No. subjects (%) |
| | Total | |
| Gender | Male | |
| | Female | |
| | Total | |
| Weight(kg) | No. subjects | |
| | mean±std | |
| | median | |
| | min~max | |
| Height(cm) | No. subjects | |
| | mean±std | |
| | median | |
| | min~max | |
| Table 1.1.3 Past diagnosis | | |
| Safety Set | | Total |
| | | No. subjects (%) |
| Yes | | |
| No | | |
| Total | | |
| | , | |
| Table 1.1.4 Pre-Immunization temperature | e | |
| Safety Set | | Total |
| | | No. subjects (%) |
| No. subjects | | |
| mean±std (°C) | | |

median min~max



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

| Table 1.1.5 Temperature Location | |
|------------------------------------|------------------|
| Safety Set | Total |
| | No. subjects (%) |
| Axillary | |
| Oral | |
| Rectal | |
| Ear | |
| Total | |
| Table 1.1.6 Administration Site | |
| Safety Set | Total |
| | No. subjects (%) |
| Left Deltoid | |
| Right Deltoid | |
| Other | |
| Total | |
| Table 1.1.7 Concomitant medication | |
| Safety Set | Total |
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |
| Table 1.1.8 Kidney Disorder | |
| Safety Set | Total |
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

#### Table 1.1.9 Liver disorder

| Safety Set | Total |
|------------|------------------|
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |

#### Table 1.1.10 Pregnancy

| Safety Set | Total |
|------------|------------------|
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |

#### 1.2 Safety Per Protocol Set

### Table 1.2.1 Total subject

| Safety per protocol set | Total |
|-------------------------|------------------|
| | No. subjects (%) |
| Total | |

#### Table 1.2.2 Demographic characteristics

#### 1) (Administration start date)-(birth)+1

| Safety per protocol set | | Total |
|--------------------------|--------------|------------------|
| | | No. subjects (%) |
| Age(years) <sup>1)</sup> | No. subjects | |
| | mean±std | |
| | median | |
| | min~max | |
| Age(years) | 11-18 | |
| | 19-34 | |
| | 35-55 | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

| Safety per protocol set | | Total |
|-------------------------|--------------|------------------|
| | | No. subjects (%) |
| | Total | |
| Children group(years) | < 18 | |
| | ≥ 18 | |
| | Total | |
| Ethnic Origin | Asian | |
| | Black | |
| | Caucasian | |
| | Hispanic | |
| | Other | |
| | Total | |
| Gender | Male | |
| | Female | |
| | Total | |
| Weight(kg) | No. subjects | |
| | mean±std | |
| | median | |
| | min~max | |
| Height(cm) | No. subjects | |
| | mean±std | |
| | median | |
| | min~max | |

### Table 1.2.3 Past diagnosis

| Safety per protocol set | Total |
|-------------------------|------------------|
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |

#### Table 1.2.4 Pre-Immunization temperature

| Safety per protocol set | Total |
|-------------------------|-------|



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

| | No. subjects (%) |
|------------------------------------|------------------|
| No. subjects | |
| mean±std (°C) | |
| median | |
| min~max | |
| Table 1.2.5 Temperature Location | |
| Safety per protocol set | Total |
| | No. subjects (%) |
| Axillary | |
| Oral | |
| Rectal | |
| Ear | |
| Total | |
| Table 1.2.6 Administration Site | |
| Safety per protocol set | Total |
| | No. subjects (%) |
| Left Deltoid | |
| Right Deltoid | |
| Other | |
| Total | |
| Table 1.2.7 Concomitant medication | |
| Safety per protocol set | Total |
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |
| Table 1.2.8 Kidney Disorder | |
| Safety per protocol set | Total |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

| | No. subjects (%) |
|----------------------------|------------------|
| Yes | |
| No | |
| Total | |
| Table 1.2.9 Liver disorder | |
| Safety per protocol set | Total |
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |
| Table 1.2.10 Pregnancy | |
| Safety per protocol set | Total |
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

## STATISTICAL ANALYSIS PLAN(V1.0)

#### 2. Safety Analyses

- AE includes solicited and unsolicited AE (Day 1-7) and medically attended AE (Day 1-29) and SAEs (Day 1-29)
- AE will be reported on the safety set and safety per protocol set.
- SAE/SADR will be reported on the safety set, safety per protocol set and non-safety per protocol set.

#### 2.1 Safety Set

Table 2.1.1 Summary of AE

| Safety Set | No. subjects with AE | 95% CI <sup>†</sup> for the percentage of subjects with AE | No.<br>AEs | Total |
|---|---|---|---|---|
| | n (%) | (Lower , Upper) | n | n (%) |
| Solicited AE | | | | |
| Injection site Reaction | | | | |
| Systemic Reaction | | | | |
| Unsolicited AE | | | | |
| MAAE | | | | |
| Total | | | | |

<sup>† 95%</sup> CI will be calculated using the normal approximation.

Table 2.1.2 Summary of AE by Age (year)

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| 11-18 | | | | |
| 19-34 | | | | X <sup>2</sup> -test or Exact test |
| 35-55 | | | | |
| Total | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

Table 2.1.3 Summary of AE by Children group

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| < 18 years | | | | |
| ≥ 18 years | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

### Table 2.1.4 Summary of AE by Gender

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | (0/) | | (0/) | |
| | n (%) | n | n (%) | |
| Male | | | | |
| Female | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

### Table 2.1.5 Summary of AE by Past diagnosis

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

### Table 2.1.6 Summary of AE by Temperature Location

| Safety Set | No. subjects with AE | No.<br>AEs | Total |
|------------|----------------------|------------|-------|
| | n (%) | n | n (%) |
| Axillary | | | |
| Oral | | | |
| Rectal | | | |
| Ear | | | |
| Total | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

Table 2.1.7 Summary of AE by Administration Site

| Safety Set | No. subjects with AE | No.<br>AEs | Total |
|---------------|----------------------|------------|-------|
| | n (%) | n | n (%) |
| Left Deltoid | | | |
| Right Deltoid | | | |
| Other | | | |
| Total | | | |

#### Table 2.1.8 Summary of AE by Concomitant medication

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

### Table 2.1.9 Summary of AE by Kidney Disorder

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

### Table 2.1.10 Summary of AE by Liver disorder

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

Table 2.1.11 Summary of AE by Pregnancy

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

### 2.2 Safety per protocol set

Table 2.2.1 Summary of AE

| Safety per protocol Set | No. subjects with AE | 95% CI <sup>†</sup> for the percentage of subjects with AE | No.<br>AEs | Total |
|---|---|---|---|---|
| | n (%) | (Lower , Upper) | n | n (%) |
| Solicited AE | | | | |
| Injection site Reaction | | | | |
| Systemic Reaction | | | | |
| Unsolicited AE | | | | |
| MAAE | | | | |
| Total | | | | |

 $<sup>\</sup>dagger$  95% CI will be calculated using the normal approximation.

Table 2.2.2 Summary of AE by Age (year)

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| 11-18 | | | | |
| 19-34 | | | | X <sup>2</sup> -test or Exact test |
| 35-55 | | | | |
| Total | | _ | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

Table 2.2.3 Summary of AE by Children group

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| < 18 years | | | | |
| ≥ 18 years | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

### Table 2.2.4 Summary of AE by Gender

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Male | | | | |
| Female | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

### Table 2.2.5 Summary of AE by Past diagnosis

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

#### Table 2.2.6 Summary of AE by Temperature Location

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total |
|-------------------------|----------------------|------------|-------|
| | n (%) | n | n (%) |
| Axillary | | | |
| Oral | | | |
| Rectal | | | |
| Ear | | | |
| Total | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

STATISTICAL ANALYSIS PLAN(V1.0)

Table 2.2.7 Summary of AE by Administration Site

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total |
|-------------------------|----------------------|------------|-------|
| | n (%) | n | n (%) |
| Left Deltoid | | | |
| Right Deltoid | | | |
| Other | | | |
| Total | | | |

#### Table 2.2.8 Summary of AE by Concomitant medication

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

### Table 2.2.9 Summary of AE by Kidney Disorder

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

### Table 2.2.10 Summary of AE by Liver disorder

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

Table 2.2.11 Summary of AE by Pregnancy

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

## 3. Information of AEs

## 3.1 Safety Set

Table 3.1.1 Summary of solicited AE and unsolicited AE for 7 days after vaccination

| Safety Set | fety Set | | Е |
|----------------|-------------------------|----------------|------------|
| | | Incidence Rate | No. of AEs |
| | | n (%) | n |
| Injection site | Pain | | |
| Reactions | Erythema | | |
| | Induration | | |
| | Sub Total | | |
| Systemic | Chills | | |
| Reactions | Nausea | | |
| | Malaise | | |
| | Myalgia | | |
| | Arthralgia | | |
| | Headache | | |
| | Rash | | |
| | Sub Total | | |
| UNSOLICITED AE | System Organ Class(SOC) | | |
| | Preferred Term(PT) | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

| i. | |
|-------|-----------|
| | Sub Total |
| Total | L |

Table 3.1.2 Summary of medically attended AEs for 28 days after vaccination

| Safety Set | | AE | |
|------------|-------------------------|----------------|------------|
| | | Incidence Rate | No. of AEs |
| | | n (%) | n |
| MAAE | System Organ Class(SOC) | | |
| | Preferred Term(PT) | | |
| Total | - | | |

### 3.2 Safety per protocol set

Table 3.2.1 Summary of solicited AE and unsolicited AE for 7 days after vaccination

| Safety per protocol Set | | AI | E |
|-------------------------|------------|----------------|------------|
| | | Incidence Rate | No. of AEs |
| | | n (%) | n |
| Injection site | Pain | | |
| Reactions | Erythema | | |
| | Induration | | |
| | Sub Total | | |
| Systemic | Chills | | |
| Reactions | Nausea | | |
| | Malaise | | |
| | Myalgia | | |
| | Arthralgia | | |
| | Headache | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

| | Rash |
|----------------|-------------------------|
| | Sub Total |
| UNSOLICITED AE | System Organ Class(SOC) |
| | Preferred Term(PT) |
| | Sub Total |
| Total | |

#### Table 3.2.2 Summary of medically attended AEs for 28 days after vaccination

| Safety per protocol Set | | AI | Ξ |
|---|---|---|---|
| | | Incidence Rate | No. of AEs |
| | | n (%) | n |
| MAAE | System Organ Class(SOC) | | |
| | Preferred Term(PT) | | |
| Total | | | |

## 4. Solicited AE (DAY 1-7)

## 4.1 Safety Set

Table 4.1.1 Summary of Injection site Reaction by Max severity

| Safety Set | | 1* | 2* | 3* | 4* | Total |
|----------------|----------|-------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) | n (%) |
| Injection site | Pain | | | | | |
| Reactions | Erythema | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

| Induration | | | |
|------------|---|---|---|
| | : | : | : |

Table 4.1.2 Summary of Systemic Reaction by Max severity

| Safety Set | | 1* | 2* | 3* | Total |
|------------|------------|-------|-------|-------|-------|
| | _ | n (%) | n (%) | n (%) | n (%) |
| Systemic | Chills | | | | |
| Reactions | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Chills, Nausea, Malaise, Myalgia, Arthralgia, Headache

Table 4.1.3 Summary of Solicited AE by day

| Safety Set | | 30 | min | | 6hr | | 2 | | 3 | | 4 | | 5 | | 6 | | 7 | Т | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) |
| Injection site | Pain | | | | | | | | | | | | | | | | | | |
| Reactions | Erythema | | | | | | | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | | | | | | | |
| | Sub Total | | | | | | | | | | | | | | | | | | |
| Systemic | Chills | | | | - | | | | - | | - | | - | | • | | | • | |
| Reactions | Nausea | | | | | | | | | | | | | | | | | | |
| | Malaise | | | | | | | | | | | | | | | | | | |
| | Myalgia | | | | | | | | | | | | | | | | | | |
| | Arthralgia | | | | | | | | | | | | | | | | | | |
| | Headache | | | | | | | | | | | | | | | | | | |
| | Rash | | | | | | | | | | | | | | | | | | |
| | Sub Total | | | | | | | | | | | | | | | | | | |
| Total | | - | | | - | | - | | | | | | | | | | - | - | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Pain

<sup>\* 1-25(1), 26-50(2), 51-100(3), &</sup>gt;100(4): Erythema, Induration

<sup>\*</sup> Urticarial(1): Rash



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

Table 4.1.4 Summary of Fever

| Safety Set | | Total |
|-----------------|----------|-------|
| | | n (%) |
| | Fever | |
| | No fever | |
| | Total | |
| Temperature(°C) | 36-36.5 | |
| | 36.5-37 | |
| | 37-37.5 | |
| | 37.5-38 | |
| | 38-38.5 | |
| | 38.5-39 | |
| | 39-39.5 | |
| | 39.5-40 | |
| | >40 | |

### 4.2 Safety per protocol set

Table 4.2.1 Summary of Injection site Reaction by Max severity

| Safety per pro | tocol Set | 1* | 2* | 3* | 4* | Total |
|----------------|------------|-------|-------|-------|-------|-------|
| | _ | n (%) | n (%) | n (%) | n (%) | n (%) |
| Injection site | Pain | | | | | |
| Reactions | Erythema | | | | | |
| | Induration | | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Pain

Table 4.2.2 Summary of Systemic Reaction by Max severity

| Safety per proto | col Set | 1* | 2* | 3* | Total |
|------------------|---------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) |
| Systemic | Chills | | | | |
| Reactions | Nausea | | | | |
| | Malaise | | | | |

<sup>\* 1-25(1), 26-50(2), 51-100(3), &</sup>gt;100(4): Erythema, Induration



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

| Myalgia |
|------------|
| Arthralgia |
| Headache |
| Rash |

Table 4.2.3 Summary of Solicited AE by day

| Safety per pro | tocol Set | 30 | ) min | | 6hr | | 2 | | 3 4 | | 4 | | 5 | | 6 | 7 | | Т | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | _ | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) |
| Injection site | Pain | | | | | | | | | | | | | | | | | | |
| Reactions | Erythema | | | | | | | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | | | | | | | |
| | Sub Total | | | | | | | | | | | | | | | | | | |
| Systemic | Chills | | | | | | | | | | | | • | | • | | | | |
| Reactions | Nausea | | | | | | | | | | | | | | | | | | |
| | Malaise | | | | | | | | | | | | | | | | | | |
| | Myalgia | | | | | | | | | | | | | | | | | | |
| | Arthralgia | | | | | | | | | | | | | | | | | | |
| | Headache | | | | | | | | | | | | | | | | | | |
| | Rash | | | | | | | | | | | | | | | | | | |
| | Sub Total | | | | | | | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | | | | | | | |

#### Table 4.2.4 Summary of Fever

| Safety per protocol Set | | Total |
|-------------------------|----------|-------|
| | | n (%) |
| | Fever | |
| | No fever | |
| | Total | |
| Temperature(°C) | 36-36.5 | |
| | 36.5-37 | |
| | 37-37.5 | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Chills, Nausea, Malaise, Myalgia, Arthralgia, Headache

<sup>\*</sup> Urticarial(1): Rash



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

| 37.5-38 | |
|---------|------------------------------------------|
| 38-38.5 | |
| 38.5-39 | |
| 39-39.5 | |
| 39.5-40 | |
| >40 | |
| | 38-38.5<br>38.5-39<br>39-39.5<br>39.5-40 |

## 5. Unsolicited AE (DAY 1-7)

### 5.1 Safety Set

Table 5.1.1 Summary of Unsolicited AE by Expected

| Safety Set | Total |
|---------------|-------------|
| | No. AEs (%) |
| Expected AE | |
| Unexpected AE | |
| Total | |

#### Table 5.1.2 Summary of Unsolicited AE by Serious

| Safety Set | Total |
|------------|-------------|
| | No. AEs (%) |
| Yes | |
| No | |
| Total | |

#### Table 5.1.3 Summary of Unsolicited AE by Severity

| Safety Set | Total |
|------------|-------------|
| | No. AEs (%) |
| Mild | |
| Moderate | |
| Severe | |
| Total | |


THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

Table 5.1.4 Summary of Unsolicited AE by Frequency

| • | 2 1 2 |
|-------------------|-------------|
| Safety Set | Total |
| | No. AEs (%) |
| Single/Continuous | |
| Intermittent | |
| Total | |

Table 5.1.5 Summary of Unsolicited AE by Action Taken

| Safety Set | To | otal |
|--------------------------------|---------|------|
| | No. AEs | (%) |
| None | | |
| Uncertain | | |
| Procedure or physical | | |
| therapy | | |
| Blood or blood products | | |
| Withdrawn from study due to AE | | |
| Prescription drug therapy | | |
| Non-prescription drug therapy | | |
| Hospitalization | | |
| IV fluids | | |
| Physician visit | | |
| Other | | |
| Total | | |

# Table 5.1.6 Summary of Unsolicited AE by Outcome

| Safety Set | Total |
|--------------------------------------|-------------|
| | No. AEs (%) |
| Complete recovery/Return to baseline | |
| Alive with sequelae | |
| Death | |
| Unknown/Lost to follow-up | |
| AE persisting | |
| Total | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

Table 5.1.7 Summary of Unsolicited AE by Relationship to study vaccine

| Safety Set | Total |
|------------------|-------------|
| | No. AEs (%) |
| Not related | |
| Possibly related | |
| Probably related | |
| Total | |

# **5.2** Safety per protocol set

Table 5.2.1 Summary of Unsolicited AE by Expected

| Safety per protocol Set | Total |
|-------------------------|-------------|
| | No. AEs (%) |
| Expected AE | |
| Unexpected AE | |
| Total | |

Table 5.2.2 Summary of Unsolicited AE by Serious

| Safety per protocol Set | Total |
|-------------------------|-------------|
| | No. AEs (%) |
| Yes | |
| No | |
| Total | |

Table 5.2.3 Summary of Unsolicited AE by Severity

| Safety per protocol Set | Total |
|-------------------------|-------------|
| | No. AEs (%) |
| Mild | |
| Moderate | |
| Severe | |
| Total | |

Table 5.2.4 Summary of Unsolicited AE by Frequency



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

| Safety per protocol Set | Total |
|-------------------------|-------------|
| | No. AEs (%) |
| Single/Continuous | |
| Intermittent | |
| Total | |

Table 5.2.5 Summary of Unsolicited AE by Action Taken

| Safety per protocol Set | Total |
|--------------------------------|-------------|
| | No. AEs (%) |
| None | |
| Uncertain | |
| Procedure or physical | |
| Therapy | |
| Blood or blood products | |
| Withdrawn from study due to AE | |
| Prescription drug therapy | |
| Non-prescription drug therapy | |
| Hospitalization | |
| IV fluids | |
| Physician visit | |
| Other | |
| Total | |

## Table 5.2.6 Summary of Unsolicited AE by Outcome

| Safety per protocol Set | Total |
|--------------------------------------|-------------|
| | No. AEs (%) |
| Complete recovery/Return to baseline | |
| Alive with sequelae | |
| Death | |
| Unknown/Lost to follow-up | |
| AE persisting | |
| Total | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

Table 5.2.7 Summary of Unsolicited AE by Relationship to study vaccine

| Safety per protocol Set | Total |
|-------------------------|-------------|
| | No. AEs (%) |
| Not related | |
| Possibly related | |
| Probably related | |
| Total | |

# **6.** MAAE (DAY 1-29)

## **6.1 Safety Set**

Table 6.1.1 Summary of MAAE by Expected

| Safety Set | Total |
|---------------|-------------|
| | No. AEs (%) |
| Expected AE | |
| Unexpected AE | |
| Total | |

# Table 6.1.2 Summary of MAAE by Serious

| Safety Set | Total |
|------------|-------------|
| | No. AEs (%) |
| Yes | |
| No | |
| Total | |

## Table 6.1.3 Summary of MAAE by Severity

| Safety Set | Total |
|------------|-------------|
| | No. AEs (%) |
| Mild | |
| Moderate | |
| Severe | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

| Safety Set | Total |
|------------|-------------|
| | No. AEs (%) |
| Total | |

# Table 6.1.4 Summary of MAAE by Frequency

| Safety Set | Total |
|-------------------|-------------|
| | No. AEs (%) |
| Single/Continuous | |
| Intermittent | |
| Total | |

# Table 6.1.5 Summary of MAAE by Action Taken

| Safety Set | Total |
|--------------------------------|-------------|
| | No. AEs (%) |
| None | |
| Uncertain | |
| Procedure or physical | |
| therapy | |
| Blood or blood products | |
| Withdrawn from study due to AE | |
| Prescription drug therapy | |
| Non-prescription drug therapy | |
| Hospitalization | |
| IV fluids | |
| Physician visit | |
| Other | |
| Total | |

## Table 6.1.6 Summary of MAAE by Outcome

| Safety Set | Total |
|--------------------------------------|-------------|
| | No. AEs (%) |
| Complete recovery/Return to baseline | |
| Alive with sequelae | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

| Safety Set | Total |
|---------------------------|-------------|
| | No. AEs (%) |
| Death | |
| Unknown/Lost to follow-up | |
| AE persisting | |
| Total | |

## Table 6.1.7 Summary of MAAE by Relationship to study vaccine

| Safety Set | Total |
|------------------|-------------|
| | No. AEs (%) |
| Not related | |
| Possibly related | |
| Probably related | |
| Total | |

# **6.2** Safety per protocol set

# Table 6.2.1 Summary of MAAE by Expected

| Safety per protocol Set | Total |
|-------------------------|-------------|
| | No. AEs (%) |
| Expected AE | |
| Unexpected AE | |
| Total | |

# Table 6.2.2 Summary of MAAE by Serious

| Safety per protocol Set | Total |
|-------------------------|-------------|
| | No. AEs (%) |
| Yes | |
| No | |
| Total | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

## Table 6.2.3 Summary of MAAE by Severity

| Safety per protocol Set | Total |
|-------------------------|-------------|
| | No. AEs (%) |
| Mild | |
| Moderate | |
| Severe | |
| Total | |

## Table 6.2.4 Summary of MAAE by Frequency

| Safety per protocol Set | Total |
|-------------------------|-------------|
| | No. AEs (%) |
| Single/Continuous | |
| Intermittent | |
| Total | |

# Table 6.2.5 Summary of MAAE by Action Taken

| Safety per protocol Set | Total |
|--------------------------------|-------------|
| | No. AEs (%) |
| None | |
| Uncertain | |
| Procedure or physical | |
| therapy | |
| Blood or blood products | |
| Withdrawn from study due to AE | |
| Prescription drug therapy | |
| Non-prescription drug therapy | |
| Hospitalization | |
| IV fluids | |
| Physician visit | |
| Other | |
| Total | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

Table 6.2.6 Summary of MAAE by Outcome

| Safety per protocol Set | Total |
|--------------------------------------|-------------|
| | No. AEs (%) |
| Complete recovery/Return to baseline | |
| Alive with sequelae | |
| Death | |
| Unknown/Lost to follow-up | |
| AE persisting | |
| Total | |

## Table 6.2.7 Summary of MAAE by Relationship to study vaccine

| Safety per protocol Set | Total |
|-------------------------|-------------|
| | No. AEs (%) |
| Not related | |
| Possibly related | |
| Probably related | |
| Total | |

# 7. SAE/SADR for 28 days after vaccination

## 7.1 Safety Set

Table 7.1 SAE and SADR

| Safety Set | Se | erious AE | Serious ADR | |
|---|---|---|---|---|
| | Incidence Rate | No. of AEs | Incidence Rate | No. of AEs |
| _ | n (%) | n | n (%) | n |
| System Organ Class(SOC) | | | | |
| Preferred Term(PT) | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

| Total | |
|-------|---|
| | _ |

# 7.2 Safety per protocol set

Table 7.2 SAE and SADR

| Safety per protocol Set | Sei | rious AE | Serious ADR | |
|---|---|---|---|---|
| | Incidence Rate | No. of AEs | Incidence Rate | No. of AEs |
| | n (%) | n | n (%) | n |
| System Organ Class(SOC) | | | | |
| Preferred Term(PT) | | | | |
| Total | | | | |

<sup>\*</sup> MedDRA

# 7.3 Non-Safety per protocol set

Table 7.3 SAE and SADR

| Non- Safety per protocol Set | Serious AE | | Serious ADR | |
|---|---|---|---|---|
| | Incidence Rate | No. of AEs | Incidence Rate | No. of AEs |
| | n (%) | n | n (%) | n |
| System Organ Class(SOC) | | | | |
| Preferred Term(PT) | | | | |
| Total | | | | |

<sup>\*</sup> MedDRA

<sup>\*</sup> MedDRA



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

# 8. Unexpected AE/ADR for 28 days after vaccination

# 8.1 Safety Set

Table 8.1 Unexpected AE and ADR

| Safety Set | Unexpected AE | | Unexpected ADR | |
|---|---|---|---|---|
| | Incidence Rate | No. of AEs | Incidence Rate | No. of AEs |
| | n (%) | n | n (%) | n |
| System Organ Class(SOC) | | | _ | |
| Preferred Term(PT) | | | | |
| Total | | | | |

<sup>\*</sup> MedDRA

# 8.2 Safety per protocol set

Table 8.2 Unexpected AE and ADR

| Safety per protocol Set | Unexpected AE | | Unexpected ADR | |
|---|---|---|---|---|
| | Incidence Rate | No. of AEs | Incidence Rate | No. of AEs |
| | n (%) | n | n (%) | n |
| System Organ Class(SOC) | | | | |
| Preferred Term(PT) | | | | |
| Total | | | | |

<sup>\*</sup> MedDRA



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

## 8.3 Non-Safety per protocol set

Table 8.3 Unexpected AE and ADR

| Non-Safety per protocol Set | Unexpected AE | | Unexpected ADR | |
|---|---|---|---|---|
| | Incidence Rate | No. of AEs | Incidence Rate | No. of AEs |
| | n (%) | n | n (%) | n |
| System Organ Class(SOC) | | | | |
| Preferred Term(PT) | | | | |
| Total | | | | |

<sup>\*</sup> MedDRA

# 9. MAAE/ADR for 28 days after vaccination

# 9.1 Safety Set

Table 9.1 MAAE and ADR

| Safety Set | N | <b>ЛАА</b> Е | ADR | |
|---|---|---|---|---|
| | Incidence Rate | No. of AEs | Incidence Rate | No. of AEs |
| | n (%) | n | n (%) | n |
| System Organ Class(SOC) | | | | |
| Preferred Term(PT) | | | | |
| Total | | | | |

<sup>\*</sup> MedDRA



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

06-MAR-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V1.0)

## 9.2 Safety per protocol set

Table 9.2 MAAE and ADR

| Safety per protocol Set | N | MAAE | ADR | |
|---|---|---|---|---|
| | Incidence Rate | No. of AEs | Incidence Rate | No. of AEs |
| | n (%) | n | n (%) | n |
| System Organ Class(SOC) | | | | |
| Preferred Term(PT) | | | | |
| Total | | | | |

<sup>\*</sup> MedDRA

# 9.3 Non-Safety per protocol set

Table 9.3 MAAE and ADR

| Non- Safety per protocol Set | MAAE | | ADR | |
|---|---|---|---|---|
| | Incidence Rate | No. of AEs | Incidence Rate | No. of AEs |
| | n (%) | n | n (%) | n |
| System Organ Class(SOC) | - | | | |
| Preferred Term(PT) | | | | |
| Total | | | | |

<sup>\*</sup> MedDRA



\_

# STATISTICAL ANALYSIS PLAN

A Multicenter, Post Marketing Surveillance study to Monitor the Safety of Novartis Meningococcal ACWY Conjugate Vaccine (MenACWY-CRM) Administered According to the Prescribing Information to Healthy Subjects from 2 to 55 Years of Age in the Republic of South Korea

Product Name: Menveo (MenACWY-CRM)

Protocol No. : V59\_62

Version : V2.0

Date : 22-NOV-2013



#### CONFIDEI'ffIAL:

THIS DOCUMENT AND JNFORMAT!ON CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY

Last Update Date
22-NOV-2013

# STATISTICAL ANALYSIS PLAN(V2.0)

# **Approvals**

• Author

Biostatistician

PPD ,DreamC!S

Dute





THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

# Revisions

| DATE OF<br>REVISION | INDICATION REVISION | REASON FOR CHANGE | AUTHOR<br>NAME |
|---|---|---|---|
| 22-NOV-2013 | All | Protocol Amendment | PPD |

Last Update Date

# CONFIDENTIAL:

THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

# STATISTICAL ANALYSIS PLAN(V2.0)

# **Table of Contents**

| Revisions | 3 |
|--------------------------------------------------|----|
| 1. Study Objective | 6 |
| 2. Study Method and Study Period | 6 |
| 2.1 Study Period | 6 |
| 2.2 Number of Subjects | 6 |
| 2.3 Study population | 6 |
| 2.3.1 Inclusion criteria | 6 |
| 2.3.2 Exclusion criteria | 7 |
| 2.4 Study Method. | 7 |
| 3. Analysis Sets | 10 |
| 3.1 Safety Analysis Sets | 10 |
| 3.2 Efficacy Analysis Set | 11 |
| 4. Endpoints | 12 |
| 4.1 Safety Endpoints | 12 |
| 5. Assessment Criteria | 12 |
| 5.1 Safety Assessment Criteria | 12 |
| 6. Statistical Analyses | 12 |
| 6.1 Baseline Characteristics | 12 |
| 6.2 Safety Analyses | 13 |
| 6.2.1 Adverse Events by Baseline Characteristics | 13 |
| 6.2.2. Analysis of Solicited AE | 14 |
| 6.2.3 Analysis of Unsolicited AE | 15 |
| 7. List of Table and Data Listings | 16 |
| 7.1 Distribution of Subjects | 16 |
| 7.2 Baseline Characteristics | 16 |
| 7.3 Safety Analyses | 16 |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

| 8. Notes | 17 |
|-----------|----|
| Appendix1 | 18 |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

## 1. Study Objective

The primary objective of the study is to monitor the safety of a single dose of MenACWY-CRM vaccine in subjects from 2 to 55 years of age, as evaluated by:

- 1. Local and systemic solicited adverse events reported from study Day 1 (day of vaccination) through study Day 7 post-vaccination
- 2. All unsolicited Adverse Events (AEs) reported from study Day 1(day of vaccination) through study Day 7 post-vaccination
- 3. Medically attended Adverse Events reported from study Day 1 to study termination (Day 29/early termination)
- 4. All Serious Adverse Events (SAEs) reported from study Day 1 to study termination (Day 29/early termination)

# 2. Study Method and Study Period

## 2.1 Study Period

The trial period shall be from market launch date till approximately 22 May 2018.

## 2.2 Number of Subjects

A total of approximately 3,300 subjects are planned for enrolment into this study.

Assuming a 10% drop-out rate, this should provide approximately 3,000 evaluable subjects. This sample size meets the post-licensure requirements of the MFDS to provide continued safety monitoring in the Korean population.

#### 2.3 Study population

#### 2.3.1 Inclusion criteria

Individuals eligible for enrolment in this study are those:

1. Male and female subjects from 2 to 55 years of the age at the time of Visit 1(including all 55



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

years old subjects, up to one day before their 56<sup>th</sup> year birthday), who are scheduled to receive vaccination with MenACWY-CRM conjugate vaccine, according to the local prescribing information and routine clinical practice

- 2. To whom the nature of the study has been described and the subject or subject's parent/legal representative has provided written informed consent (written assent from minors should be also obtained if required by the relevant IRB);
- 3. Whom the investigator believes that the subject can and will comply with the requirements of the protocol (e.g., completion of the Diary Card);
- 4. Who are in good health as determined by the outcome of medical history, physical assessment and clinical judgment of the investigator

#### 2.3.2 Exclusion criteria

1. Contraindication, special warnings and/or precautions, as evaluated by the investigators, reported in the MenACWY-CRM conjugate vaccine Korean prescribing information.

## 2.4 Study Method

In order to obtain information on Regulatory PMS data after market launch, NVD or delegate will create the Regulatory PMS contract with the relevant clinics/hospitals and the physician in charge of the survey shall implement this Regulatory PMS in subjects that receive MenACWY-CRM in the relevant hospital/clinic since the contract date until the number of contracted survey cases, without omission, is reached.

## Overview of Study Design

This is a multicenter post marketing surveillance study to monitor the safety of MenACWY-CRM administered according to the prescribing information to 3,300 healthy subjects from 2 to 55 years of age in Korea.

Subjects will be enrolled at the time of their visit to a participating clinic or hospital for vaccination with MenACWY-CRM according to the routine clinical care.

At Visit 1 (Day 1), after obtaining consent from the subjects or subjects' parents/legal representative (written assent will be also obtained if required by the relevant IRB), the vaccination will be administered. Subjects will remain under observation for at least 30 minutes in the clinic after study immunization.



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

STATISTICAL ANALYSIS PLAN(V2.0)

The subjects or subject's parent/legal representative will be then instructed to complete the Diary Card daily, reporting local and systemic adverse events and all other AEs occurring within 7 days following immunizations, and medically attended AEs or SAEs occurring up to Day 29.

Subjects will also be instructed to return the completed diaries to the study site at Day 29 as follows:

- During a visit at the study center or
- Using the provided pre-addressed stamped envelope (PASE).

At the investigator discretion, the subject or subject's parent/legal representative will be reminded of the date of the study termination by a phone call at Day 29. If any clarification is required after Diary Card retrieval the site staff will follow up by phone, and any additional finding will be recorded on the subject's medical record.

In case the Diary Card is not retrieved within 10 days after Day 29, subject or subject's parent/legal representative will be contacted by phone to assess the occurrence of adverse events, determine the subject's clinical status and complete study termination. All information will be recorded by the site staff on the subject's medical record and collected in the appropriate section of the CRF.

All SAEs will be monitored until resolution and/or the cause is identified. If a SAE remains unresolved at study termination, a clinical assessment will be made by the investigator and the NVD regional physician to determine whether continued follow up of the SAE is needed.

Table 3.1-1: Safety Assessment Table

| Medical History: | From birth, collected at clinic |
|---|---|
| All significant past diagnoses including all allergies, | visit Day 1 |
| major surgeries requiring inpatient hospitalization, | |
| other significant injuries or hospitalizations, any | |
| conditions requiring prescription or chronic medication | |
| (i.e., >2 weeks in duration), or other significant medical | |
| conditions based on the investigator's judgment. | |
| Immediate reactions: | For at least 30 minutes after |
| Subjects will be assessed for immediate | vaccination |
| hypersensitivity reactions. | |
| Solicited local adverse events: | Days 1-7 after vaccination |
| < 6 years : injection site erythema, injection site | |
| induration, injection site tenderness | |




# THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT

22-NOV-2013

# STATISTICAL ANALYSIS PLAN(V2.0)

THE WRITTEN PERMISSION OF COMPANY.

| ≥ 6 years : injection site erythema, injection site | |
|---|---|
| induration, injection site pain | |
| Solicited systemic adverse events: | Days 1-7 after vaccination |
| < 6 years : change in eating habits, sleepiness, | |
| irritability, rash, vomiting, diarrhea, fever | |
| ≥ 6 years : chills, nausea, malaise, generalized myalgia, | |
| generalized arthralgia, headache, rash, fever | |
| All unsolicited AEs will be collected | Days 1-7 after vaccination |
| Medically attended Adverse Events: | From Day 1 to study |
| Events that require a physician's visit or an emergency | termination (Day 29/early |
| room visit (events that are managed by telephone or | termination) |
| means other than a face-to-face evaluation by a | |
| clinician do not qualify as medically attended AEs). | |
| Serious AEs: | From Day 1 to study |
| All SAEs will be collected. | termination (Day 29/early |
| | termination) |
| Medications: | From Day 1 to Day 7 |
| Any medications used to treat any solicited local and | |
| systemic reaction and unsolicited AE be collected. | |
| Medications: | From Day 1 to study |
| Any medications used to treat any medically attended | termination (Day 29/early |
| AE or SAE will be collected. | termination) |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

## 3. Analysis Sets

## 3.1 Safety Analysis Sets

#### Safety Set

All subjects who

- have signed an informed consent form, undergone screening procedure(s) and received a subject number,
- received a study vaccination,
- provided post vaccination safety data.

#### Safety per protocol set

All subjects in the safety Set with the exclusions of the following cases:

- (1) Subjects administered prior to the contract date.
- (2) Subjects who didn't receive MenACWY-CRM.
- (3) Subjects who already receive MenACWY-CRM.
- (4) Follow-up failure: The subjects whose safety information cannot be identified due to follow-up loss.
- (5) Not applicable to the indication of study drug [Indication]
  - To prevent invasive meningococcal disease caused by Neisseria meningitides serogroups A, C, Y and W-135 in persons 2 through 55 years of age.
- (6) Subjects who violate of Protocol: Those who do not meet one item at least of the inclusion/exclusion criteria.

[Inclusion criteria]

- Male and female subjects from 2 to 55 years of the age at the time of Visit 1(including all 55 years old subjects, up to one day before their 56<sup>th</sup> year birthday), who are scheduled to receive vaccination with MenACWY-CRM conjugate vaccine, according to the local prescribing information and routine clinical practice.
- 2) To whom the nature of the study has been described and the subject or subject's parent/legal representative has provided written informed consent.
- 3) Whom the investigator believes that the subject can and will comply with the requirements of the protocol.



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

4) Who are in good health as determined by the outcome of medical history, physical assessment and clinical judgment of the investigator.

[Exclusion criteria]

- 1) Contraindication, special warnings and/or precautions, as evaluated by the investigators, reported in the MenACWY-CRM conjugate vaccine Korean prescribing information
- (7) Subjects who prescribed off-label dosage.
  - Violation of intramuscular injection only (0.5ml)

### Non-Safety per protocol set

Subjects excluded from safety per protocol set except for subjects who did not receive MenACWY-CRM and follow-up failure.

Based on rules for estimation of each number of safety evaluation cases, the following local regulation and Guideline on Standards for re-examination for new drugs, etc \*\* of MFDS, non-safety analysis set are excluded from the safety analysis set:

- - A) Patients planned to receive a drug under surveillance by investigator's medical judgment shall be subject.
  - B) Subject who do not use within approved range shall not be included in the subject in principal.
    - \* However, if data of subject whose use is beyond approved range is collected, perform analysis as a separate item.
  - C) Describe actual selection methods of subject in detail.

## 3.2 Efficacy Analysis Set

Not Applicable



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

## 4. Endpoints

# 4.1 Safety Endpoints

Safety will be assessed after administration of study vaccine in terms of the number and percentage of subjects with:

- Local and systemic solicited adverse events reported from study Day 1 (day of vaccination) through study Day 7 post-vaccination;
- Unsolicited AEs reported from study Day 1 (day of vaccination) through study Day 7 post-vaccination;
- Medically attended AEs reported from study Day 1 to study termination (Day 29/early termination);
- SAEs reported from study Day 1 to study termination (Day 29/early termination).

#### 5. Assessment Criteria

## **5.1 Safety Assessment Criteria**

Not Applicable

## 6. Statistical Analyses

#### **6.1 Baseline Characteristics**

Descriptive statistics (mean, standard deviation, median, minimum and maximum) for baseline characteristics such as age, height and weight at enrollment will be calculated in the Safety set and Safety per Protocol set.

The following baseline characteristics will be reported:



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

- < Subject Baseline Information >
  - gender, age, ethnic origin, weight, height, past diagnosis, pre-Immunization temperature, temperature location, pregnancy
- < Study Vaccine Information >
  - vaccine site, concomitant medications

## **6.2 Safety Analyses**

The number of subjects of  $AE^{\dagger}$  and the number of  $AEs^{\dagger}$  incurred shall be calculated, the incidence rate of  $AEs^{\dagger}$  and its 95% confidence interval will be calculated using the normal approximation on the safety set and safety per protocol set.

† AE : AE includes solicited and unsolicited AE (DAY 1-7), medically attended AE (DAY 1-29) and SAE (DAY 1-29).

# **6.2.1** Adverse Events by Baseline Characteristics

 $AE^{\dagger}s$  (as described below) will be reported (n, %) for the following the baseline characteristics in the safety set and safety per protocol set :

- Age group (2-10, 11-18, 19-34, 35-55)
- Children group ( $<18, \ge 18$ )
- Gender (male, female)
- Past diagnosis (yes, no)
- Temperature location (axillary, oral, rectal, ear)
- Administration site (left deltoid, right deltoid, other)
- Concomitant medication (yes, no)
- Kidney disorder (yes, no)
- Liver disorder (yes, no)
- Pregnancy (yes, no)

The n(%) of AEs<sup>†</sup> and its 95% confidence interval will be calculated using the normal approximation and analyzed using  $\chi^2$ - test or Fisher's exact test.



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

† AE : AE includes solicited and unsolicited AE (DAY 1-7) and medically attended AE (DAY 1-29) and SAEs.

#### 6.2.2. Analysis of Solicited AE

Frequencies and percentages of subjects experiencing each adverse event will be presented for each symptom severity. Summary tables showing the occurrence of any local or systemic adverse events overall and at each time point will also be presented (see Table 4.1.3 and 4.2.3).

Post-vaccination adverse events reported from Day 1 to Day 7 will be summarized by maximal severity. The severity of local adverse events for subjects < 6 years of age will be categorized as follows. Injection-site erythema and induration: absent (0 to 9 mm), mild (10 to 25 mm), moderate (26 to 50 mm), severe (>50 mm); injection-site tenderness: none, mild (minor light reaction to touch), moderate (cried or protested to touch), severe (cried when injected limb was moved). For subjects  $\geq$  6 years, injection-site erythema and induration absent (1 to 24 mm), mild (25 to 50 mm), moderate (51 to 100 mm), severe (>100 mm); pain: none, mild (present but does not interfere with activity), moderate (interferes with activity), severe (prevents daily activity).

For subjects  $\geq$  6 years of age, the severity of systemic adverse events (i.e., chills, nausea, malaise, generalized myalgia, generalized arthralgia, headache) occurring up to 7 days after each vaccination will be categorized as none, mild (present but not interfering with daily activity), moderate (some interference with daily activity), and severe (prevents daily activity) except for rash, which will be categorized as none, urticarial, or other.

For subjects < 6 years of age, the severity of systemic adverse events occurring up to 7 days after each vaccination will be categorized as follows. Change in eating habits: none (no change in appetite), mild (eating less than normal for 1 to feeds), moderate (missed 1 or 2 feeds), severe (missed more than 2 feeds); sleepiness: none (no change in alertness), mild (shows an increased alertness), moderate (sleeps through feeds), severe (sleeps most of the time and it is hard to arouse him/her); irritability: none (no change in child disposition), mild (requires more cudding and he/she is less playful than usual), moderate (more difficult to settle), severe (unable to console); rash: none, urticarial, or other; vomiting: none, mild (1-2 episodes/24 hours), moderate (>2 episodes/24 hours), severe (requires outpatient hydratation); diarrhea: none (fewer than 2 loose stools/24 hours), mild (2-3 loose stools or < 400 gms/24 hours), moderate (4-5 stools or 400-800 gms/24 hours), severe (6 or more watery stools



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

STATISTICAL ANALYSIS PLAN(V2.0)

or > 800 gms/24 hours or requires outpatient IV hydration).

Body temperature will be categorized as  $<38^{\circ}$ C (no fever),  $\ge 38^{\circ}$ C (fever) and will be summarized by  $0.5^{\circ}$ C increments from  $36.0^{\circ}$ C up to  $\ge 40^{\circ}$ C. Additionally, no fever vs. fever will be reported.

Each local and systemic adverse event will also be categorized as none vs. any.

## **6.2.3** Analysis of Unsolicited AE

All unsolicited AEs and MAAE recorded in the CRF will be mapped to preferred terms using the most recent MedDRA dictionary and classified by System organ class (SOC) and Preferred Terms (PT). Under the classification standard of MedDRA terms, and all AEs excluding the AEs whose causal relation with the study medication is 'Not Related' shall be treated as AEs whose causal relation cannot be excluded {hereafter "Adverse Drug Reaction(ADR)"}.

- ① The number and percentage of unsolicited AE (Day 1-7) and MAAE (Day 1-29) and SAEs (Day 1-29) according to the serious, severity, frequency, action taken, outcome, relationship to MenACWY-CRM regarding occurred AE will be calculated.
- ② Unsolicited AEs (Day 1-7) and MAAE (Day 1-29) and SAEs (Day 1-29) will be classified into the preferred terms according to the serious, severity, frequency, action taken, outcome, relationship to MenACWY-CRM. Also, the number and percentage of each AE (PT) will be calculated.
- ③ The number of subjects and the number of unexpected AE/ADR, SAE/Serious ADR (SADR) and MAAE/ADR will be calculated according to the preferred terms. Also, the incidence rate will be estimated.
- (4) For subjects excluded from safety per protocol set<sup>†</sup>, the number of subjects and the number of unexpected AE/ADR, SAE/Serious ADR (SADR) and MAAE/ADR will be calculated according to the preferred terms. Also, the incidence rate will be estimated.
  - † Subject excluded from safety per protocol set: Except for subjects who didn't receive study vaccination and follow-up failure.



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

STATISTICAL ANALYSIS PLAN(V2.0)

## 7. List of Table and Data Listings

# 7.1 Distribution of Subjects

- Number of subjects contracted to the study: The number of subjects are to be collected(under contract) as contracted by the investigator
- Number of retrieving completed CRFs: Total number of subjects whose completed CRFs
- Number of safety assessment population: Number of safety assessment population among total number

#### 7.2 Baseline Characteristics

- Mean and standard deviation (SD) or frequency and percentage by gender, age, ethnic origin, weight, height, past diagnosis, pre-Immunization temperature, temperature location, pregnancy
- Frequency and percentage by vaccine site, concomitant medications

## 7.3 Safety Analyses

- Incidence rate and the number of AEs according to the baseline characteristics (frequency and percentage)
- The number of the serious, severity, frequency, action taken, outcome, relationship to MenACWY-CRM for Unsolicited AE (DAY 1-7) and MAAE (frequency and percentage)
- The number of AEs for the severity, day, fever to MenACWY-CRM according to individual solicited AE (DAY 1-7) (frequency and percentage)
- Incidence rate and number according to the preferred terms of SAE/SADR, unexpected AE/unexpected ADR, and MAAE/ADR (frequency and percentage)
- For subjects excluded from safety per protocol set<sup>†</sup> incidence rate and number according to the preferred terms of SAE/SADR, unexpected AE/unexpected ADR, and MAAE/ADR (frequency and percentage)
  - † Subject excluded from safety per protocol set: Except for subjects who didn't receive study mediation and follow-up failure



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

## 8. Notes

- Each statistical analysis will be carried out with SAS Software version 9.2 or more recent version.
- In the descriptive statistics, mean, SD, minimum, median, and maximum will be calculated for continuous variables, and frequency and percentage for categorical variables.
- Data including sign of inequality such as "≥20", ">20" will be excluded from analysis.
- All test statistics will be the results of two-sided tests with the statistical significant level of 0.05.
- The followings shall be included only in re-examination report:
  - Analysis by type of concomitant medications
  - Item ② of paragraph 6.2.3
  - Estimation of 95% confidence interval for incidence of AEs by background factors



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# **STATISTICAL ANALYSIS PLAN(V2.0)**

# Appendix1

# 1. Demographic and baseline values, medication characteristics, specific characteristics

- Baseline characteristics will be reported on the safety set and safety per protocol set.

# 1.1 Safety Set

Table 1.1.1 Total subject

| Safety Set | Total |
|------------|------------------|
| | No. subjects (%) |
| Total | |

## Table 1.1.2 Demographic characteristics

#### 1) (Administration start date)-(birth)+1

| Safety Set | | Total |
|--------------------------|--------------|------------------|
| | | No. subjects (%) |
| Age(years) <sup>1)</sup> | No. subjects | |
| | mean±std | |
| | median | |
| | min~max | |
| Age(years) | 2-10 | |
| | 2-5 | |
| | 6-10 | |
| | 11-18 | |
| | 19-34 | |
| | 35-55 | |
| | Total | |
| Children group(years) | < 18 | |
| | ≥ 18 | |
| | Total | |
| Ethnic Origin | Asian | |
| | Black | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

| Safety Set | | Total |
|------------------------------------------|--------------|------------------|
| | | No. subjects (%) |
| | Caucasian | |
| | Hispanic | |
| | Other | |
| | Total | |
| Gender | Male | |
| | Female | |
| | Total | |
| Weight(kg) | No. subjects | |
| | mean±std | |
| | median | |
| | min~max | |
| Height(cm) | No. subjects | |
| | mean±std | |
| | median | |
| | min~max | |
| Table 1.1.3 Past diagnosis | | |
| Safety Set | | Total |
| | | No. subjects (%) |
| Yes | | |
| No | | |
| Total | | |
| Table 1.1.4 Pre-Immunization temperature | e | |
| Safety Set | | Total |
| | | No. subjects (%) |
| No. subjects | | |
| mean±std (°C) | | |
| median | | |

min~max



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

| Table 1.1.5 Temperature Location Safety Set | Total |
|---------------------------------------------|------------------------|
| Safety Set | |
| A '11 | No. subjects (%) |
| Axillary | |
| Oral | |
| Rectal | |
| Ear | |
| Total | |
| Table 1.1.6 Administration Site | |
| Safety Set | Total |
| | No. subjects (%) |
| Left Deltoid | |
| Right Deltoid | |
| Other | |
| Total | |
| | · |
| Table 1.1.7 Concomitant medication | |
| Safety Set | Total |
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |
| Table 1.1.8 Kidney Disorder | |
| Table 1.1.8 Kidney Disorder Safety Set | Total |
| | Total No. subjects (%) |
| Safety Set | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

## Table 1.1.9 Liver disorder

| Safety Set | Total |
|------------|------------------|
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |

## Table 1.1.10 Pregnancy

| Safety Set | Total |
|------------|------------------|
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |

## 1.2 Safety Per Protocol Set

# Table 1.2.1 Total subject

| Safety per protocol set | Total |
|-------------------------|------------------|
| | No. subjects (%) |
| Total | |

## Table 1.2.2 Demographic characteristics

#### 1) (Administration start date)-(birth)+1

| Safety per protocol set | | Total |
|--------------------------|--------------|------------------|
| | | No. subjects (%) |
| Age(years) <sup>1)</sup> | No. subjects | |
| | mean±std | |
| | median | |
| | min~max | |
| Age(years) | 2-10 | |
| | 2-5 | |
| | 6-10 | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

| Safety per protocol set | | Total |
|-------------------------|--------------|------------------|
| | | No. subjects (%) |
| | 11-18 | |
| | 19-34 | |
| | 35-55 | |
| | Total | |
| Children group(years) | < 18 | |
| | ≥ 18 | |
| | Total | |
| Ethnic Origin | Asian | |
| | Black | |
| | Caucasian | |
| | Hispanic | |
| | Other | |
| | Total | |
| Gender | Male | |
| | Female | |
| | Total | |
| Weight(kg) | No. subjects | |
| | mean±std | |
| | median | |
| | min~max | |
| Height(cm) | No. subjects | |
| | mean±std | |
| | median | |
| | min~max | |

# Table 1.2.3 Past diagnosis

| Safety per protocol set | Total |
|-------------------------|------------------|
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

| Safety per protocol set | Total |
|------------------------------------|------------------|
| Safety per protocor set | |
| | No. subjects (%) |
| No. subjects | |
| mean±std (°C) | |
| median | |
| min~max | |
| Table 1.2.5 Temperature Location | |
| Safety per protocol set | Total |
| | No. subjects (%) |
| Axillary | |
| Oral | |
| Rectal | |
| Ear | |
| Total | |
| Table 1.2.6 Administration Site | |
| Safety per protocol set | Total |
| | No. subjects (%) |
| Left Deltoid | |
| Right Deltoid | |
| Other | |
| Total | |
| Table 1.2.7 Concomitant medication | |
| Safety per protocol set | Total |
| | No. subjects (%) |
| Yes | |
| i es | |

Total



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

| Table 1.2.8 Kidney Disorder | |
|-----------------------------|------------------|
| Safety per protocol set | Total |
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |
| Table 1.2.9 Liver disorder | |
| Safety per protocol set | Total |
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |
| Table 1.2.10 Pregnancy | |
| Safety per protocol set | Total |
| | No. subjects (%) |
| Yes | |
| No | |

Total


THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

### STATISTICAL ANALYSIS PLAN(V2.0)

#### 2. Safety Analyses

- AE includes solicited and unsolicited AE (Day 1-7) and medically attended AE (Day 1-29) and SAEs (Day 1-29)
- AE will be reported on the safety set and safety per protocol set.
- SAE/SADR will be reported on the safety set, safety per protocol set and non-safety per protocol set.

#### 2.1 Safety Set

Table 2.1.1 Summary of AE

| Safety Set | No. subjects with AE | 95% CI <sup>†</sup> for the percentage of subjects with AE | No.<br>AEs | Total |
|---|---|---|---|---|
| | n (%) | (Lower , Upper) | n | n (%) |
| Solicited AE (<6years) | | | | |
| Local AE | , | | | |
| Systemic AE | | | | |
| Solicited AE(≥6years) | | | | |
| Local AE | | | | |
| Systemic AE | | | | |
| Unsolicited AE | | | | |
| SAE | | | | |
| MAAE | | | | |
| Death | | | | |
| Total | | | | |

<sup>† 95%</sup> CI will be calculated using the normal approximation.

<sup>\*</sup> Day 1-7: Solicited AE, Unsolicited AE

<sup>\*</sup> Day 1-29: MAAE, SAE, Death



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

Table 2.1.2 Summary of AE by Age (year)

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| 2-10 | | | | |
| 2-5 | | | | |
| 6-10 | | | | |
| 11-18 | | | | X <sup>2</sup> -test or Exact test |
| 19-34 | | | | |
| 35-55 | | | | |
| Total | | | | |

Table 2.1.3 Summary of AE by Age (year)

| Safety Set | No. subjects with AE | No. | Total | p-value |
|-----------------------|----------------------|-----|-------|---------|
| , | J | AEs | | |
| | n (%) | n | n (%) | |
| Solicited AE | | - | | |
| 2-10 | | | | |
| 2-5 | | | | |
| 6-10 | | | | |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |
| Solicited Local AE | | | | |
| 2-10 | | | | |
| 2-5 | | | | |
| 6-10 | | | | |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |
| Solicited Systemic AE | | | Ī | |
| 2-10 | | | | |
| 2-5 | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| 6-10 | | | | |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |
| Unsolicited AE | | | | |
| 2-10 | | | | |
| 11-18 | | | | |
| 19-34 | | | *** | |
| 35-55 | | | # 1 | |
| SAE | | | | |
| 2-10 | | | 11 | |
| 11-18 | | | | |
| 19-34 | | | 1 | |
| 35-55 | | | | |
| MAAE | | | | |
| 2-10 | | | *** | |
| 11-18 | | | # | |
| 19-34 | | | | |
| 35-55 | | | | |
| Death | | | | |
| 2-10 | | | # : | |
| 11-18 | | | # | |
| 19-34 | | | 10 H | |
| 35-55 | | | HI ************************************ | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

Table 2.1.4 Summary of AE by Children group

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| < 18 years | | | | |
| ≥ 18 years | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

### Table 2.1.5 Summary of AE by Gender

| Safety Set | No. subjects with AE | No. | Total | p-value |
|---|---|---|---|---|
| Salety Set | | AEs | | p varae |
| | n (%) | n | n (%) | |
| Male | | | | |
| Female | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

### Table 2.1.6 Summary of AE by Past diagnosis

| Safety Set | No. subjects with AE | No. | Total | p-value |
|---|---|---|---|---|
| | | AEs | | |
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

#### Table 2.1.7 Summary of AE by Temperature Location

| Safety Set | No. subjects with AE | No. AEs | Total |
|------------|----------------------|---------|-------|
| | n (%) | n | n (%) |
| Axillary | | | |
| Oral | | | |
| Rectal | | | |
| Ear | | | |
| Total | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# **STATISTICAL ANALYSIS PLAN(V2.0)**

Table 2.1.8 Summary of AE by Administration Site

| Safety Set | No. subjects with AE | No. | Total |
|---------------|----------------------|-----|-------|
| Salety Set | No. subjects with AE | AEs | Total |
| | n (%) | n | n (%) |
| Left Deltoid | | | |
| Right Deltoid | | | |
| Other | | | |
| Total | | | |

### Table 2.1.9 Summary of AE by Concomitant medication

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

### Table 2.1.10 Summary of AE by Kidney Disorder

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

### Table 2.1.11 Summary of AE by Liver disorder

| Safety Set | No. subjects with AE | No. | Total | p-value |
|---|---|---|---|---|
| surery sec | Tvo. suojoota witai 112 | AEs | Total | p varae |
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# **STATISTICAL ANALYSIS PLAN(V2.0)**

Table 2.1.12 Summary of AE by Pregnancy

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

#### 2.2 Safety per protocol set

Table 2.2.1 Summary of AE

| Safety per protocol Set | No. subjects with AE | 95% CI <sup>†</sup> for the percentage of subjects with AE | No.<br>AEs | Total |
|---|---|---|---|---|
| | n (%) | (Lower , Upper) | n | n (%) |
| Solicited AE (< 6years) | | | | |
| Local AE | | | | |
| Systemic AE | | | | |
| Solicited AE (≥6years) | | | | |
| Local AE | | | | |
| Systemic AE | | | | |
| Unsolicited AE | | | | |
| SAE | | | | |
| MAAE | | | | |
| Death | | | | |
| Total | | | | |

 $<sup>\</sup>dagger$  95% CI will be calculated using the normal approximation.

Table 2.2.2 Summary of AE by Age (year)

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
|---|---|---|---|---|

<sup>\*</sup> Day 1-7: Solicited AE, Unsolicited AE

<sup>\*</sup> Day 1-29: MAAE, SAE, Death



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

| | n (%) | n | n (%) | |
|-------|-------|---|-------|------------------------------------|
| 2-10 | | | | |
| 2-5 | | | | |
| 6-10 | | | | |
| 11-18 | | | | X <sup>2</sup> -test or Exact test |
| 19-34 | | | | |
| 35-55 | | | | |
| Total | | | | |

Table 2.2.3 Summary of AE by Age (year)

| | | No. | | | |
|-----------------------|----------------------|-----|------|----|---------|
| Safety Set | No. subjects with AE | AEs | Tot | al | p-value |
| | n (%) | n | n (' | %) | |
| Solicited AE | | | | | |
| 2-10 | | | | | |
| 2-5 | | | | | |
| 6-10 | | | | | |
| 11-18 | | | | | |
| 19-34 | | | | | |
| 35-55 | | | | | |
| Solicited Local AE | | | | | |
| 2-10 | | | | | |
| 2-5 | | | | | |
| 6-10 | | | | | |
| 11-18 | | | | | |
| 19-34 | | | | | |
| 35-55 | | | | | |
| Solicited Systemic AE | | | | | |
| 2-10 | | | | | |
| 2-5 | | | | | |
| 6-10 | | | | | |
| 11-18 | | | | | |
| 19-34 | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

### STATISTICAL ANALYSIS PLAN(V2.0)

| Safety Set | No. subjects with AE | No. | Total | | p-value |
|----------------|----------------------|-----|-------|---|---------|
| | (0/) | AEs | (0/) | | |
| | n (%) | n | n (%) | ) | |
| 35-55 | | | | | |
| Unsolicited AE | | | | | |
| 2-10 | | | | | |
| 11-18 | | | | | |
| 19-34 | | | | | |
| 35-55 | | | | | |
| SAE | | | | | |
| 2-10 | | | | | |
| 11-18 | | | | | |
| 19-34 | | | | | |
| 35-55 | | | | | |
| MAAE | | | | | |
| 2-10 | | | | | |
| 11-18 | | | | | |
| 19-34 | | | | | |
| 35-55 | | | | | |
| Death | | | | | |
| 2-10 | | | | | |
| 11-18 | | | | | |
| 19-34 | | | | | |
| 35-55 | | | | | |

### Table 2.2.4 Summary of AE by Children group

| Cafeta non mustagal Cat | No. subjects with AE | No. | Total | n volue |
|---|---|---|---|---|
| Safety per protocol Set | No. subjects with AE AEs | Total | p-value | |
| | n (%) | n | n (%) | |
| < 18 years | | | | |
| ≥ 18 years | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

### STATISTICAL ANALYSIS PLAN(V2.0)

Table 2.2.5 Summary of AE by Gender

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Male | | | | |
| Female | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |
| Table 2.2.6 Summary of A | Table 2.2.6 Summary of AE by Past diagnosis | | | |
| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total | p-value |
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

### Table 2.2.7 Summary of AE by Temperature Location

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total |
|---|---|---|---|
| | n (%) | n | n (%) |
| Axillary | | | |
| Oral | | | |
| Rectal | | | |
| Ear | | | |
| Total | | | |
| Table 2.2.8 Summary of AE by Administration Site | | | |

| n (%) Left Deltoid Right Deltoid Other Total | Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total |
|---|---|---|---|---|
| Right Deltoid Other | | n (%) | n | n (%) |
| Other | Left Deltoid | | | |
| | Right Deltoid | | | |
| Total | Other | | | |
| | Total | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

Table 2.2.9 Summary of AE by Concomitant medication

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

#### Table 2.2.10 Summary of AE by Kidney Disorder

| Safety per protocol Set | No. subjects with AE | No. | Total | p-value |
|---|---|---|---|---|
| Salety per protocor set | 1vo. subjects with 7th | AEs | Total | p-varue |
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

#### Table 2.2.11 Summary of AE by Liver disorder

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

#### Table 2.2.12 Summary of AE by Pregnancy

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | (0/) | | (0/) | |
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |



# Last Update Date CONFIDENTIAL: INT AND INFORMATION CONTAINED HEREIN IS 22-NOV-2013

THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

### STATISTICAL ANALYSIS PLAN(V2.0)

### 3. Information of AEs

### 3.1 Safety Set

Table 3.1.1 Summary of solicited AE and unsolicited AE for 7 days after vaccination (<6 years)

| Safety Set | | AI | 3 |
|---|---|---|---|
| | | Incidence Rate | No. of AEs |
| | | n (%) | n |
| Local AE | Tenderness | | |
| | Erythema | | |
| | Induration | | |
| | Sub Total | | <u> </u> |
| Systemic AE | Change in eating habits | g habits Class(SOC) | |
| | Sleepiness | | |
| | Irritability | | |
| | Vomiting | | |
| | Diarrhea | | |
| | Rash | | |
| | Sub Total | | |
| Systemic AE UNSOLICITED AE | System Organ Class(SOC) | | |
| | Preferred Term(PT) | | |
| | Sub Total | | |
| Total | · | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

Table 3.1.2 Summary of solicited AE and unsolicited AE for 7 days after vaccination (≥6years)

| Safety Set | | AI | 3 |
|----------------|-------------------------|----------------|------------|
| | | Incidence Rate | No. of AEs |
| | | n (%) | n |
| Local AE | Pain | | |
| | Erythema | | |
| | Induration | | |
| | Sub Total | | |
| Systemic AE | Chills | | |
| | Nausea | | |
| | Malaise | | |
| | Myalgia | | |
| | Arthralgia | | |
| | Headache | | |
| | Rash | | |
| | Sub Total | | |
| UNSOLICITED AE | System Organ Class(SOC) | | |
| | Preferred Term(PT) | | |
| | Sub Total | | |
| Total | | | |

| DreamCIS Inc. Clinical Investigation Services | | Last Update Date |
|---|---|---|
| | CONFIDENTIAL: THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS | 22 NOV 2012 |
| | PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT 22-NOV | |
| | THE WRITTEN PERMISSION OF COMPANY. | |
| STATISTICA | AL ANALYSIS PLAN(V2.0) | |

Table 3.1.3 Summary of solicited AE and unsolicited AE for 7 days after vaccination (≥6years)

| Safety Set | | | AE(6-1 | 0) | | AE(11-1 | .8) | | AE(19-3 | 4) | | AE(35- | 55) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Incide | nce Rate | No. of<br>AEs | Incidence | Rate | No. of<br>AEs | Incidence | e Rate | No. of<br>AEs | Incidence | e Rate | No. of<br>AEs |
| | | n | (%) | n | n | (%) | n | n | (%) | n | n | (%) | n |
| Local AE | Pain | | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | |
| | Sub Total | | | | | | | | | | | | • |
| Systemic AE | Chills | | | | | | | | | | | | |
| | Nausea | | | | | | | | | | | | |
| | Malaise | | | | | | | | | | | | |
| | Myalgia | | | | | | | | | | | | |
| | Arthralgia | | | | | | | | | | | | |
| | Headache | | | | | | | | | | | | |
| | Rash | | | | | | | | | | | | |
| | Sub Total | , | | | | | | | | | | | |
| UNSOLICITED AE | System Organ Class(SOC) | | | | | | | | | | | | |
| | Preferred Term(PT) | | | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

| Safety Set | | AE(6-10) | | | AE(11-18) | | | AE(19-34) | | | | AE(35-5 | 55) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Incidence Rate | | No. of<br>AEs | Incidence Rate | | No. of<br>AEs | Incidence Rate | | No. of<br>AEs | Incidence | e Rate | No. of<br>AEs |
| | | n | (%) | n | n | (%) | n | n | (%) | n | n | (%) | n |
| | Sub Total | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

Table 3.1.4 Summary of medically attended AEs for 28 days after vaccination

| Safety Set | | AF | 3 |
|------------|-------------------------|----------------|------------|
| | | Incidence Rate | No. of AEs |
| | | n (%) | n |
| MAAE | System Organ Class(SOC) | | |
| | Preferred Term(PT) | | |
| Total | | | |

Table 3.1.5 Summary of medically attended AEs for 28 days after vaccination

| Safety Set | | AE(2-10 | )) | A | AE(11-1 | 8) | A | AE(19-3 | 4) | A | E(35-5 | 5) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Incidence of AEs | | Incidence<br>Rate | | No.<br>of<br>AEs | Incidence<br>Rate | | No.<br>of<br>AEs | Incidence<br>Rate | | No. of AE s |
| | | n (%) | n | n | (%) | n | n | (%) | n | n | (%) | n |
| MAAE | System Organ Class(SOC) Preferred Term(PT) | | | | | | | | | | | |
| Total | | | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

### STATISTICAL ANALYSIS PLAN(V2.0)

### 3.2 Safety per protocol set

Table 3.2.1 Summary of solicited AE and unsolicited AE for 7 days after vaccination (<6 years)

| Safety per protocol Set | | AI | E |
|---|---|---|---|
| | | Incidence Rate | No. of AEs |
| | | n (%) | n |
| Local AE | Tenderness | | |
| | Erythema | | |
| | Induration | eating habits rgan Class(SOC) | |
| | Sub Total | | |
| Systemic AE | Change in eating habits | | |
| | Sleepiness | | |
| | Irritability | | |
| | Vomiting | | |
| | Diarrhea | | |
| | Rash | | |
| | Sub Total | | |
| UNSOLICITED AE | System Organ Class(SOC) | | |
| | Preferred Term(PT) | | |
| | Sub Total | | |
| Total | 1 | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

Table 3.2.2 Summary of solicited AE and unsolicited AE for 7 days after vaccination (≥6 years)

| Safety per protocol Set | | Al | E |
|---|---|---|---|
| | | Incidence Rate | No. of AEs |
| | | n (%) | n |
| Local AE | Pain | | |
| | Erythema | | |
| | Induration | | |
| | Sub Total | | |
| Systemic AE | Chills | | |
| | Nausea | | |
| | Malaise | | |
| | Myalgia | | |
| | Arthralgia | | |
| | Headache | | |
| | Rash | | |
| | Sub Total | | |
| UNSOLICITED AE | System Organ Class(SOC) | | |
| | Preferred Term(PT) | | |
| | Sub Total | | |
| Total | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

Table 3.2.3 Summary of solicited AE and unsolicited AE for 7 days after vaccination (≥6 years)

| Safety per protocol Ser | t | | AE | (6-10) | A | AE(11- | 18) | A | AE(19-3 | 34) | A | AE(35-5 | 55) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Incidence<br>Rate | | No. of AEs | | idence<br>Rate | No.<br>of<br>AEs | | idence<br>Rate | No.<br>of<br>AEs | | dence | No.<br>of<br>AEs |
| | | n | (%) | n | n | (%) | n | n | (%) | n | n | (%) | n |
| Local AE | Pain | | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | | |
| | Induration | | | | | | | | | _ | | | |
| | Sub Total | | | | | | | | | | | | |
| Systemic AE | Chills | | | | | | | | | | | | |
| | Nausea | | | | | | | | | | | | |
| | Malaise | | | | | | | | | | | | |
| | Myalgia | | | | | | | | | | | | |
| | Arthralgia | | | | | | | | | | | | |
| | Headache | | | | | | | | | | | | |
| | Rash | | | | | | | | | _ | | | |
| | Sub Total | 1 | | | | | | | | | | | |
| UNSOLICITED AE | System Organ Class(SOC) | | | | | | | | | | | | |
| | Preferred Term(PT) | | | | | | | | | | | | |
| | Sub Total | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

Table 3.24 Summary of medically attended AEs for 28 days after vaccination

| Safety per protocol Set | | Al | Ε |
|---|---|---|---|
| | | Incidence Rate | No. of AEs |
| | | n (%) | n |
| MAAE | System Organ Class(SOC) | | |
| | Preferred Term(PT) | | |
| Total | | | |

Table 3.2.5 Summary of medically attended AEs for 28 days after vaccination

| Safety Set | | AE(2-10 | AE(11-18) | | 8) | A | AE(19-3 | 34) AE(35-5 | | E(35-5 | 5) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Incidence<br>Rate | No. of | | dence<br>ate | No.<br>of<br>AEs | | dence | No.<br>of<br>AEs | | dence | No.<br>of<br>AE<br>s |
| | | n (%) | n | n | (%) | n | n | (%) | n | n | (%) | n |
| MAAE | System Organ Class(SOC) Preferred Term(PT) | | | | | | | | | | | |
| Total | • | | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# **STATISTICAL ANALYSIS PLAN(V2.0)**

#### 4. Solicited AE (DAY 1-7)

### 4.1 Safety Set

Table 4.1.1 Summary of Local AE Max severity (<6 years)

| Safety Set | | 1* | 2* | 3* | 4* | Total |
|------------|------------|-------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) | n (%) |
| Local AE | Tenderness | | | | | |
| | Erythema | | | | | |
| | Induration | | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Tenderness

Table 4.1.2 Summary of Local AE Max severity (≥6 years)

| Safety Set | | 1* | 2* | 3* | 4* | Total |
|------------|------------|-------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) | n (%) |
| Local AE | Pain | | | | | |
| | Erythema | | | | | |
| | Induration | | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Pain

Table 4.1.3 Summary of Local AE by Max severity

| Safety Set | | 1* | 2* | 3* | 4* | Total |
|-------------|------------|-------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) | n (%) |
| Age (2-5) | Tenderness | | | | | |
| | Erythema | | | | | |
| | Induration | | | | | |
| Age (6-10) | Pain | | | | | |
| | Erythema | | | | | |
| | Induration | | | | | |
| Age (11-18) | Pain | | | | | |

<sup>\* 1-25(1), 26-50(2), 51-100(3), &</sup>gt;100(4): Erythema, Induration

<sup>\* 1-25(1), 26-50(2), 51-100(3), &</sup>gt;100(4): Erythema, Induration



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

| | Erythema | 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 |
|-------------|------------|-----------------------------------------|
| | Induration | |
| Age (19-34) | Pain | |
| | Erythema | |
| | Induration | |
| Age (35-55) | Pain | |
| | Erythema | |
| | Induration | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Pain, Tenderness

Table 4.1.4 Summary of Systemic AE by Max severity(<6 years)

| Safety Set | | 1* | 2* | 3* | Total |
|-------------|-------------------------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) |
| Systemic AE | Change in eating habits | | | | |
| | Sleepiness | | | | |
| | Irritability | | | | |
| | Vomiting | | | | |
| | Diarrhea | | | # 1 | |
| | Rash | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Change in eating habits, Sleepiness, irritability, vomiting, diarrhea,

Table 4.1.5 Summary of Systemic AE by Max severity(≥6 years)

| Safety Set | | 1* | 2* | 3* | Total |
|-------------|------------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) |
| Systemic AE | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |

<sup>\* 1-25(1), 26-50(2), 51-100(3), &</sup>gt;100(4): Erythema, Induration

<sup>\*</sup>None(1), Urticarial(2), Other(3): Rash

 $<sup>* \</sup>ge 38^{\circ}C(1)$ : Fever



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

| | Rusii | I Rash | I D 1 | | Rash |
|------|-------|--------|-------|------|------|
| | | TAGII | Kasn | Rash | |
| Rash | Rash | I D 1 | | | |

Table 4.1.6 Summary of Systemic AE by Max severity

| Safety Set | | 1* | 2* | 3* | Total |
|---|---|---|---|---|---|
| | | n (%) | n (%) | n (%) | n (%) |
| Age (2-5) | Change in eating habits | | | | |
| | Sleepiness | | | | |
| | Irritability | | 1 | | |
| | Vomiting | | | | |
| | Diarrhea | | | | |
| | Rash | | | | |
| Age (6-10) | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |
| Age (11-18) | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |
| Age (19-34) | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | 111111111111111111111111111111111111111 | | |
| | Headache | | | | |
| | Rash | = | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Chills, Nausea, Malaise, Myalgia, Arthralgia, Headache

<sup>\*</sup>None(1), Urticarial(2), Other(3): Rash



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

| Safety Set | | 1* | 2* | 3* | Total |
|-------------|------------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) |
| Age (35-55) | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Chills, Nausea, Malaise, Myalgia, Arthralgia, Headache, Change in eating habits, Sleepiness, irritability, vomiting, diarrhea,

<sup>\*</sup>None(1), Urticarial(2), Other(3): Rash



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

Table 4.1.7 Summary of Solicited AE by day (<6 years)

| Safety Set | | 30 min | 6hr | 2 | 3 | 4 | 5 | 6 | 7 | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| | | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (% |
| Local AE | Tenderness | | | | | | | | | |
| | Erythema | | | | | | | | | |
| | Induration | | | | | | | | | |
| | Sub Total | | | | | | | | | |
| Systemia AE | Change in eating | | | | | | | | | |
| Systemic AE | habits | | | | | | | | | |
| | Sleepiness | | | | | | | | | |
| | Irritability | | | | | | | | | |
| | Vomiting | | | | | | | | | |
| | Diarrhea | | | | | | | | | |
| | Rash | | | | | | | | | |
| | Sub Total | | | | | | | | | |
| Total | | | | | | | | | | |

Table 4.1.8 Summary of Solicited AE by day (≥6 years)

| Safety Set | | 30 | ) min | | 6hr | | 2 | | 3 | | 4 | | 5 | | 6 | | 7 | Т | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) |
| Local AE | Pain | | | | | | | | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | | | | | | | |
| | Sub Total | | | | | | | | | | | | | | | | | | |
| Systemic AE | Chills | | | | | | | | | | | | | | | | | | |
| | Nausea | | | | | | | | | | | | | | | | | | |
| | Malaise | | | | | | | | | | | | | | | | | | |
| | Myalgia | | | | | | | | | | | | | | | | | | |
| | Arthralgia | | | | | | | | | | | | | | | | | | |
| | Headache | | | | | | | | | | | | | | | | | | |
| | Rash | | | | | | | | | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

| | Sub Total | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Total | | | | | | | | | | | | | | | | | | | - |
| Table 4.1.9 S | ummary of S | Solicited . | AE b | y day | y | | | | | | | | | | | | | | =' |
| Safety Set | | | | 30 n | nin | | 5hr | | 2 | | 3 | | 4 | | 5 | | 6 | 7 | Total |
| | | | | n ( | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n (%) | n%) |
| Age (2-5) | Tenderness | | | | | | | | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | | | | | | | |
| Age (6-10) | Pain | | | | | | | | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | | | | | | | |
| Age (11-18) | Pain | | | | | | | | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | | | | | | | |
| Age (19-34) | Pain | | | | | | | | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | | | | | | | |
| Age (35-55) | Pain | | | | | | | | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | | | | | | | |
| | Sub Total | | | | | | | | | | | | | | | | | | |
| Age (2-5) | Change in 6 | eating hab | its | | | | | | | | | | | | | | | | |
| | Sleepiness | | | | | | | | | | | | | | | | | | |
| | Irritability | | | | | | | | | | | | | | | | | | |
| | Vomiting | | | | | | | | | | | | | | | | | | |
| | Diarrhea | | | | | | | | | | | | | | | | | | |
| | Rash | | | | | | | | | | | | | | | | | | |
| Age (6-10) | Chills | | | | | | | | | | | | | | | | | | |
| | Nausea | | | | | | | | | | | | | | | | | | |
| | Malaise | | | | | | | | | | | | | | | | | | |
| | Myalgia | | | | | | | | | | | | | | | | | | |
| | Arthralgia | | | | | | | | | | | | | | | | | | |
| | Headache | | | | | | | | | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

| Safety Set | | 30 | min | | 6hr | | 2 | | 3 | | 4 | | 5 | | 6 | 7 | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n (%) | n%) |
| | Rash | | | | | | | | | | | | | | | | |
| Age (11-18) | Chills | | | | | | | | | | | | | | | | ******* |
| | Nausea | | | | | | | | | | | | | | | | |
| | Malaise | | | | | | | | | | | | | | | | |
| | Myalgia | | | | | | | | | | | | | | | | |
| | Arthralgia | | | | | | | | | | | | | | | | |
| | Headache | | | | | | | | | | | | | | | | |
| | Rash | | | | | | | | | | | | | | | | |
| Age(19-34) | Chills | | | | | | | | | | | | | | | | |
| | Nausea | | | | | | | | | | | | | | | | |
| | Malaise | | | | | | | | | | | | | | | | |
| | Myalgia | | | | | | | | | | | | | | | | |
| | Arthralgia | | | | | | | | | | | | | | | | |
| | Headache | | | | | | | | | | | | | | | | |
| | Rash | | | | | | | | | | | | | | | | |
| Age (35-55) | Chills | | | | | | | | | | | | | | | | |
| | Nausea | | | | | | | | | | | | | | | | |
| | Malaise | | | | | | | | | | | | | | | | |
| | Myalgia | | | | | | | | | | | | | | | | |
| | Arthralgia | | | | | | | | | | | | | | | | |
| | Headache | | | | | | | | | | | | | | | | |
| | Rash | | | | | | | | | | | | | | | | |
| | Sub Total | | | | | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | | | | | |

### Table 4.1.10 Summary of Fever

| Safety Set | | 2- | ·10 | 11- | 18 | 19- | -34 | 35 | -55 | Total |
|------------|----------|----|-----|-----|-----|-----|-----|----|-----|-------|
| | | n | (%) | n | (%) | n | (%) | n | (%) | n (%) |
| | Fever | | | | | | | | | |
| | No fever | | | | | | | | | |
| | Total | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

| Temperature(°C | 36-36.5 |
|----------------|---------|
| | 36.5-37 |
| | 37-37.5 |
| | 37.5-38 |
| | 38-38.5 |
| | 38.5-39 |
| | 39-39.5 |
| | 39.5-40 |
| | >40 |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

### STATISTICAL ANALYSIS PLAN(V2.0)

### 4.2 Safety per protocol set

Table 4.2.1 Summary of local AE by Max severity (<6 years)

| Safety per prot | ocol Set | 1* | 2* | 3* | 4* | Total |
|-----------------|------------|-------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) | n (%) |
| Local AE | Tenderness | | | | | |
| | Erythema | | | | | |
| | Induration | | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Tenderness

Table 4.2.2 Summary of Local AE Max severity (≥6 years)

| | | | | | | I |
|--------------------|------------|-------|-------|-------|-------|-------|
| Safety per protoco | ol Set | 1* | 2* | 3* | 4* | Total |
| | | n (%) | n (%) | n (%) | n (%) | n (%) |
| Local AE | Pain | | | | | |
| | Erythema | | | | | |
| | Induration | | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Pain

Table 4.2.3 Summary of Local AE by Max severity

| Safety per pro | tocol Set | 1* | 2* | 3* | 4* | Total |
|----------------|------------|-------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) | n (%) |
| Age (2-5) | Tenderness | | | | | |
| | Erythema | | | | | |
| | Induration | | | | | |
| Age (6-10) | Pain | | | | | |
| | Erythema | | | | | |
| | Induration | | | | | |
| Age (11-18) | Pain | | | | | |
| | Erythema | | | | | |
| | Induration | | | | | |
| Age (19-34) | Pain | | | | | |

<sup>\* 1-25(1), 26-50(2), 51-100(3), &</sup>gt;100(4): Erythema, Induration

<sup>\* 1-25(1), 26-50(2), 51-100(3), &</sup>gt;100(4): Erythema, Induration



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

| | Erythema | |
|-------------|------------|---|
| | Induration | |
| Age (35-55) | Pain | 1 |
| | Erythema | |
| | Induration | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Pain

Table 4.2.4 Summary of Systemic AE by Max severity (<6 years)

| Safety Set | | 1* | 2* | 3* | Total |
|-------------|-------------------------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) |
| Systemic AE | Change in eating habits | | | | |
| | Sleepiness | | | | |
| | Irritability | | | | |
| | Vomiting | | | | |
| | Diarrhea | | | | |
| | Rash | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Change in eating habits, Sleepiness, irritability, vomiting, diarrhea,

Table 4.2.5 Summary of Systemic AEs by Max severity (≥6 years)

| Safety per proto | col Set | 1* | 2* | 3* | Total |
|------------------|------------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) |
| Systemic AE | Chills | | | | |
| | Nausea | | , | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Chills, Nausea, Malaise, Myalgia, Arthralgia, Headache

<sup>\* 1-25(1), 26-50(2), 51-100(3), &</sup>gt;100(4): Erythema, Induration

<sup>\*</sup>None(1), Urticarial(2), Other(3): Rash

<sup>\*</sup>None(1), Urticarial(2), Other(3): Rash



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

Table 4.2.6 Summary of Systemic AE by Max severity

| Safety per proto | ocol Set | 1* | 2* | 3* | Total |
|---|---|---|---|---|---|
| | | n (%) | n (%) | n (%) | n (%) |
| Age (2-5) | Change in eating habits | | - | | |
| | Sleepiness | | | | |
| | Irritability | | | | |
| | Vomiting | | | | |
| | Diarrhea | | | | |
| | Rash | | | | |
| Age (6-10) | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |
| Age (11-18) | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |
| Age (19-34) | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |
| Age (35-55) | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | # H H H H H H H H H H H H H H H H H H H | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

### STATISTICAL ANALYSIS PLAN(V2.0)

| Safety per protocol | Set | 1* | 2* | 3* | Total |
|---------------------|------------|-------|-------|-------|-------|
| _ | | n (%) | n (%) | n (%) | n (%) |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | 1 | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Chills, Nausea, Malaise, Myalgia, Arthralgia, Headache

Table 4.1.7 Summary of Solicited AE by day (<6 years)

| Safety Set | | 30 | min | | 6hr | | 2 | | 3 | | 4 | | 5 | | 6 | | 7 | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n (%) |
| Local AE | Tenderness | | | | | | | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | | | | | | |
| | Sub Total | | | | | | | | | | | | | | | | | |
| Systemic AE | Change in eating habits | | | | | | | | | | | | | | | | | |
| | Sleepiness | | | | | | | | | | | | | | | | | |
| | Irritability | | | | | | | | | | | | | | | | | |
| | Vomiting | | | | | | | | | | | | | | | | | |
| | Diarrhea | | | | | | | | | | | | | | | | | |
| | Rash | | | | | | | | | | | | | | | | | |
| | Sub Total | | | | | | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | | | | | | |

#### Table 4.2.8 Summary of Solicited AE by day (≥6 years)

| Safety per pro | Safety per protocol Set | | ) min | 6hr | | 2 | | 3 | | 4 | | 5 | | | 6 | | 7 | Т | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) |
| Local AE | Pain | | | | | | | | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | | | | | | | |
| | Sub Total | | | | | | | | | | | | | | | | | | |
| Systemic AE | Chills | | | | | | | | | | | | | | | | | | |
| | Nausea | | | | | | | | | | | | | | | | | | |

<sup>\*</sup>None(1), Urticarial(2), Other(3): Rash



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

| | Malaise |
|-------|------------|
| | Myalgia |
| | Arthralgia |
| | Headache |
| | Rash |
| | Sub Total |
| Total | |

Table 4.2.9 Summary of Solicited AE by day

| Safety Set | | 3 | 0 min | | 6hr | | 2 | | 3 | | 4 | | 5 | | 6 | | 7 | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n (%) |
| Age (2-5) | Tenderness | | | | | | | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | | | | | | |
| Age (6-10) | Pain | | | | | | | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | | | | | | |
| Age (11-18) | Pain | | | | | | | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | | | | | | |
| Age (19-34) | Pain | | | | | | | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | | | | | | |
| Age (35-55) | Pain | | | | | | | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | | | | | | |
| | Sub Total | | | | | | | | | | | | | | | | | |
| Age (2-5) | Change in eating habits | | | | | | | | | | | | | | | | | |
| | Sleepiness | | | | | | | | | | | | | | | | | |
| | Irritability | | | | | | | | | | | | | | | | | |
| | Vomiting | | | | | | | | | | | | | | | | | |
| | Diarrhea | | | | | | | | | | | | | | | | | |
| | Rash | | | | | | | | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

| Safety Set | | 30 min | 6hr | 2 | 3 | 4 | 5 | 6 | 7 | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| | | n (%) n ( | %) n (%) r | ı (%) n (% | ) n (%) n ( | %) n (%) | | | | n (%) |
| Age (6-10) | Chills | | | | | | | | | |
| | Nausea | | | | | | | | | |
| | Malaise | | | | | | | | | |
| | Myalgia | | | | | | | | | |
| | Arthralgia | | | | | | | | | |
| | Headache | | | | | | | | | |
| | Rash | | | | | | | | | |
| Age (11-18) | Chills | | | | | | | | | |
| | Nausea | | | | | | | | | |
| | Malaise | | | | | | | | | |
| | Myalgia | | | | | | | | | |
| | Arthralgia | | | | | | | | | |
| | Headache | | | | | | | | | |
| | Rash | | | | | | | | | |
| Age(19-34) | Chills | | | | | | | | | |
| | Nausea | | | | | | | | | |
| | Malaise | | | | | | | | | |
| | Myalgia | | | | | | | | | |
| | Arthralgia | | | | | | | | | |
| | Headache | | | | | | | | | |
| | Rash | | | | | | | | | |
| Age (35-55) | Chills | | | | | | | | | |
| | Nausea | | | | | | | | | |
| | Malaise | | | | | | | | | |
| | Myalgia | | | | | | | | | |
| | Arthralgia | | | | | | | | | |
| | Headache | | | | | | | | | |
| | Rash | | | | | | | | | |
| | Sub Total | | | | | | | | | |
| Total | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

### STATISTICAL ANALYSIS PLAN(V2.0)

Table 4.2.10 Summary of Fever

| Safety per protocol Set | | 2 | -10 | 1 | 1-18 | | 19 | -34 | 35- | -55 | Total | 1 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | (%) | ı | n (% | 6) | n | (%) | n | (%) | n (% | 5) |
| | Fever | | | | | | | | | | | |
| | No fever | | | | | | | | | | | |
| | Total | | | | | | | | | | | |
| Temperature(°C) | 36-36.5 | | | | | | | | | | | |
| | 36.5-37 | | | | | | | | | | | |
| | 37-37.5 | | | | | | | | | | | |
| | 37.5-38 | | | | | | | | | | | |
| | 38-38.5 | | | | | | | | | | | |
| | 38.5-39 | | | | | | | | | | | |
| | 39-39.5 | | | | | | | | | | | |
| | 39.5-40 | | | | | | | | | | | |
| | >40 | | | | | | | | | | | |

### 5. Unsolicited AE (DAY 1-7)

### 5.1 Safety Set

Table 5.1 Summary of Unsolicited AE

| Safety Set | | 2- | 10 | 11 | -18 | 19-34 | | 35 | -55 | To | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) |
| Expected | Expected AE | | | | | | | | | | |
| | Unexpected AE | | | | | | | | | | |
| Serious | Yes | | | | | | | | | | |
| | No | | | | | | | | | | |
| Severity | Mild | | | | | | | | | | |
| | Moderate | | | | | | | | | | |
| | Severe | | | | | | | | | | |
| Frequency | Single/Continuous | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

| Safety Set | | 2- | 10 | 11 | -18 | 19 | -34 | 35 | -55 | То | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | No. | (%) | No. | (%) | No. | (%) | No. | (%) | No. | (%) |
| | | AEs | (70) | AEs | (70) | AEs | (70) | AEs | (70) | AEs | (70) |
| | Intermittent | | | | | | | | | | |
| Action Taken | None | | | | | | | | | | |
| | Uncertain | | | | | | | | | | |
| | Procedure or physical | | | | | | | | | | |
| | therapy | | | | | | | | | | |
| | Blood or blood products | | | | | | | | | | |
| | Withdrawn from study due to AE | | | | | | | | | | |
| | Prescription drug therapy | | | | | | | | | | |
| | Non-prescription drug therapy | | | | | | | | | | |
| | Hospitalization | | | | | | | | | | |
| | IV fluids | | | | | | | | | | |
| | Physician visit | | | | | | | | | | |
| | Other | | | | | | | | | | |
| Outcome | Complete recovery/Return to baseline | | | | | | | | | | |
| | Alive with sequelae | | | | | | | | | | |
| | Death | | | | | | | | | | |
| | Unknown/Lost to follow-up | | | | | | | | | | |
| | AE persisting | | | | | | | | | | |
| Relationship | | | | | | | | | | | |
| to study | Not related | | | | | | | | | | |
| vaccine | | | | | | | | | | | |
| | Possibly related | | | | | | | | | | |
| | Probably related | | | | | | | | | | |
| Total | | | | | | | | | | | |

### 5.2 Safety per protocol set

### Table 5.2 Summary of Unsolicited AE

| Safety per | 2-10 | 11-18 | 19-34 | 35-55 | Total |
|--------------|------|-------|-------|-------|-------|
| protocol Set | 2-10 | 11-10 | 19-34 | 33-33 | Total |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

| | | No. | (%) | No. | (%) | No. | (%) | No. | (%) | No. | (%) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | AEs | (70) | AEs | (70) | AEs | (70) | AEs | (70) | AEs | (70) |
| Expected | Expected AE | | | | | | | | | | |
| | Unexpected AE | | | | | | | | | | |
| Serious | Yes | | | | | | | | | | |
| | No | | | | | | | | | | |
| Severity | Mild | | | | | | | | | | |
| | Moderate | | | | | | | | | | |
| | Severe | | | | | | | | | | |
| Frequency | Single/Continuous | | | | | | | | | | |
| | Intermittent | | | | | | | | | | |
| Action Taken | None | | | | | | | | | | |
| | Uncertain | | | | | | | | | | |
| | Procedure or physical | | | | | | | | | | |
| | therapy | | | | | | | | | | |
| | Blood or blood products | | | | | | | | | | |
| | Withdrawn from study due to AE | | | | | | | | | | |
| | Prescription drug therapy | | | | | | | | | | |
| | Non-prescription drug therapy | | | | | | | | | | |
| | Hospitalization | | | | | | | | | | |
| | IV fluids | | | | | | | | | | |
| | Physician visit | | | | | | | | | | |
| | Other | | | | | | | | | | |
| Outcome | Complete recovery/Return to baseline | | | | | | | | | | |
| | Alive with sequelae | | | | | | | | | | |
| | Death | | | | | | | | | | |
| | Unknown/Lost to follow-up | | | | | | | | | | |
| | AE persisting | | | | | | | | | | |
| Relationship | | | | | | | | | | | |
| to study | Not related | | | | | | | | | | |
| vaccine | | | | | | | | | | | |
| | Possibly related | | | | | | | | | | |
| | Probably related | | | | | | | | | | |


THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

| Safety per protocol Set | 2- | 10 | 11 | -18 | 19 | -34 | 35 | -55 | То | tal |
|---|---|---|---|---|---|---|---|---|---|---|
| | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) |
| Total | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

# **6.** MAAE (DAY 1-29)

## 6.1 Safety Set

Table 6.1 Summary of MAAE

| Safety Set | | 2- | 10 | 11 | -18 | 19 | -34 | 35 | -55 | To | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) |
| Expected | Expected AE | | | | | | | | | | |
| | Unexpected AE | | | | | | | | | | |
| Serious | Yes | | | | | | | | | | |
| | No | | | | | | | | | | |
| Severity | Mild | | | | | | | | | | |
| | Moderate | | | | | | | | | | |
| | Severe | | | | | | | | | | |
| Frequency | Single/Continuous | | | | | | | | | | |
| | Intermittent | | | | | | | | | | |
| Action<br>Taken | None | | | | | | | | | | |
| | Uncertain | | | | | | | | | | |
| | Procedure or physical | | | | | | | | | | |
| | therapy | | | | | | | | | | |
| | Blood or blood products | | | | | | | | | | |
| | Withdrawn from study due to AE | | | | | | | | | | |
| | Prescription drug therapy | | | | | | | | | | |
| | Non-prescription drug therapy | | | | | | | | | | |
| | Hospitalization | | | | | | | | | | |
| | IV fluids | | | | | | | | | | |
| | Physician visit | | | | | | | | | | |
| | Other | | | | | | | | | | |
| Outcome | Complete recovery/Return to baseline | | | | | | | | | | |
| | Alive with sequelae | | | | | | | | | | |
| | Death | | | | | | | | | | |
| | Unknown/Lost to follow-up | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

| Safety Set | | 2- | 10 | 11 | -18 | 19 | -34 | 35 | -55 | То | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | No. | (0/) | No. | (0/) | No. | (0/) | No. | (0/) | No. | (0/) |
| | | AEs | (%) | AEs | (%) | AEs | (%) | AEs | (%) | AEs | (%) |
| | AE persisting | | | | | | | | | | |
| Relationshi | | | | | | | | | | | |
| p to study | Not related | | | | | | | | | | |
| vaccine | | | | | | | | | | | |
| | Possibly related | | | | | | | | | | |
| | Probably related | | | | | | | | | | |
| Total | | | | | | | | | | | |

## 6.2 Safety per protocol set

Table 6.2 Summary of MAAE

| Safety per protocol Set | | 2- | 10 | 11 | -18 | 19 | -34 | 35 | -55 | Тс | tal |
|---|---|---|---|---|---|---|---|---|---|---|---|
| protocor set | | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) |
| Expected | Expected AE Unexpected AE | | | | | | | | | | |
| Serious | Yes<br>No | | | | | | | | | | |
| Severity | Mild<br>Moderate<br>Severe | | | | | | | | | | |
| Frequency | Single/Continuous Intermittent | | | | | | | | | | |
| Action<br>Taken | None | | | | | | | | | | |
| | Uncertain Procedure or physical | | | | | | | | | | |
| | therapy Blood or blood products | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

| Safety per protocol Set | | 2- | 10 | 11 | -18 | 19 | -34 | 35 | -55 | Тс | tal |
|---|---|---|---|---|---|---|---|---|---|---|---|
| protocor set | | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) |
| | Withdrawn from study due to AE | | | | | | | | | | |
| | Prescription drug therapy | | | | | | | | | | |
| | Non-prescription drug therapy | | | | | | | | | | |
| | Hospitalization | | | | | | | | | | |
| | IV fluids | | | | | | | | | | |
| | Physician visit | | | | | | | | | | |
| | Other | | | | | | | | | | |
| Outcome | Complete recovery/Return to baseline | | | | | | | | | | |
| | Alive with sequelae | | | | | | | | | | |
| | Death | | | | | | | | | | |
| | Unknown/Lost to follow-up | | | | | | | | | | |
| | AE persisting | | | | | | | | | | |
| Relationshi | | | | | | | | | | | |
| p to study | Not related | | | | | | | | | | |
| vaccine | | | | | | | | | | | |
| | Possibly related | | | | | | | | | | |
| | Probably related | | | | | | | | | | |
| Total | | | | | | | | | | | |

| | | Last Update Date |
|---|---|---|
| DreamCIS Inc. | CONFIDENTIAL: THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS | 22-NOV-2013 |
| Clinical Investigation Services | PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY. | 22-NOV-2013 |
| | T ANIATAZOTO DI ANIATA | |

# STATISTICAL ANALYSIS PLAN(V2.0)

## 7. SAE/SADR for 28 days after vaccination

# 7.1 Safety Set

Table 7.1 SAE and SADR

| | | 2- | 10 | | | 11 | -18 | | | 19 | -34 | | | 35 | -55 | | | То | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety Set | Serious | AE | Seriou<br>ADR | | Serious | AE | Seriou<br>ADR | | Serious | <b>Α</b> Ε | Seriou<br>ADR | | Serious | ΑE | Seriou<br>ADR | | Serious | ΑE | Serio<br>ADF | |
| | Inciden<br>ce Rate | N o. of A Es | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | N o . o f A E |
| | ( | | ( | | ( | | ( | | ( | | ( | | ( | | ( | | ( | | ( | S |
| | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n |
| System Organ Class(SOC) | | | | | | | | | | | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

| | | 2- | 10 | | | 11 | -18 | | | 19 | -34 | | | 35 | -55 | | | То | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety Set | Serious | ΑE | Seriou<br>ADR | | Serious | ΑE | Serio<br>ADF | | Serious | ΑE | Seriou<br>ADR | | Serious | ΑE | Seriou<br>ADR | | Serious | ΑE | Serior<br>ADF | |
| | Inciden ce Rate | N o. of A Es | Inciden<br>ce Rate | N<br>o.<br>of<br>A<br>E | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E s | Inciden<br>ce Rate | A<br>E | Inciden<br>ce Rate | N o. of A E | | | Inciden<br>ce Rate | N<br>o.<br>of<br>A<br>E | Inciden<br>ce Rate | | Inciden<br>ce Rate | |
| | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n |
| Preferred Term(PT) | | | | | | MAN (MANIMAN) I I I I I I I I I I I I I I I I I I I | | | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | | | | | | | | |



# STATISTICAL ANALYSIS PLAN(V2.0)

## 7.2 Safety per protocol set

Table 7.2 SAE and SADR

| | | 2- | 10 | | | 11- | -18 | | | | 19 | -34 | | | 35 | -55 | | | To | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety per protocol Set | Serious | <b>A</b> E | Seriou<br>ADR | | Serious | ΑE | | ious<br>DR | | Serious | ΑE | Seriou<br>ADR | | Serious | ΑE | Seriou<br>ADR | | Serious | ΑE | Serio<br>AD | |
| | Inciden<br>ce Rate | N<br>o.<br>of<br>A<br>Es | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | | Incide | e A | o.<br>of<br>A | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | | Incider | |
| | n % | n | n % | n | n % | n | n <sup>0</sup> | ( // r | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n |
| System Organ Class(SOC) | | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

| | | 2- | 10 | | | 11 | -18 | | | | 19 | -34 | | | 35 | -55 | | | То | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety per protocol Set | Serious | ΑE | Seriou<br>ADR | | Serious | AE | ļ | rious<br>DR | | Serious | ΑE | Seriou<br>ADR | | Serious | ΑE | Seriou<br>ADR | | Serious | ΑE | Serio<br>AD | |
| | Inciden<br>ce Rate | N o. of A Es | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | | Incid<br>ce Ra | | N o. of A E | | | Inciden<br>ce Rate | N<br>o.<br>of<br>A<br>E | | | Inciden<br>ce Rate | N<br>o.<br>of<br>A<br>E | Inciden<br>ce Rate | | Inciden<br>ce Rate | |
| | n % | n | n % | n | n % | n | n | (<br>%<br>) | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n |
| Preferred Term(PT) | | | | | | | | | | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | | | | | | | | | |



## 7.3 Non-Safety per protocol set

Table 7.3 SAE and SADR

| - | | 2-10 Serious | | | 11 | -18 | | | 19 | -34 | | | 35 | -55 | | | To | tal | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non- Safety per protocol<br>Set | Serious | ΑE | Seriou<br>ADR | | Serious | ΑE | Seriou<br>ADR | | Serious . | AE | Seriou<br>ADR | | Serious | ΑE | Seriou<br>ADR | | Serious | AE | Serio<br>ADI | |
| | Inciden<br>ce Rate | N o. of A Es | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E | Inciden ce Rate | | Inciden<br>ce Rate | N o. of A E s | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | N o o f A E S |
| | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | |
| System Organ Class(SOC) | | | | | | | : | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

| | | 2- | 10 | | | 11 | -18 | | | | 19 | -34 | | | 35 | -55 | | | То | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non- Safety per protocol<br>Set | Serious | ΑE | Seriou<br>ADR | | Seriou | s <b>A</b> E | | rious<br>.DR | S | Serious | AE | Seriou<br>ADR | | Serious | ΑE | Seriou<br>ADR | | Serious | ΑE | Seriou<br>ADR | |
| | Inciden<br>ce Rate | N o. of A Es | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | | Incide<br>ce Ra | en | N o. of A E s | | | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | |
| | n.% | n | n % | n | n % | n | n | (<br>% | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n |
| Preferred Term(PT) | | | | | | | | | | | NOTE DESCRIPTION OF THE PROPERTY OF THE PROPER | | THE CONTRACTOR OF THE CONTRACT | | THE STATE OF THE S | | | | HOME AND ALL PROPERTY OF THE P | | THE REST OF THE PROPERTY OF TH |
| Total | | | | | | | | | | | | | | | | | | | | | |

| | | Last Update Date |
|---|---|---|
| Proper CTC | CONFIDENTIAL: | |
| DreamCIS Inc. Clinical Investigation Services | THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS | 22-NOV-2013 |
| | PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT | 22 110 1 2013 |
| | THE WRITTEN PERMISSION OF COMPANY. | |
| STATISTICA | L ANALYSIS PLAN(V2.0) | |

## 8. Unexpected AE/ADR for 28 days after vaccination

# 8.1 Safety Set

Table 8.1 Unexpected AE and ADR

Safety Set

| | 2-1 | 10 | | | 11 | -18 | | | 19 | -34 | | | 35 | -55 | | | Tot | al | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Unexpec | ted | Unexped | eted | Unexped | eted | Unexped | eted | Unexped | eted | Unexped | eted | Unexpe | eted | Unexped | eted | Unexpe | eted | Unexpe | cte |
| AE | | ADR | _ | AE | | ADR | _ | AE | | ADR | | AE | | ADR | | AE | | d ADF | ₹ |
| | | | | | | | | | | | | | | | | | | | N |
| | N | | N | | Ν | | N | | Ν | | N | | Ν | | N | | N | | o |
| | 0. | | 0. | | О. | | 0. | | o. | | o. | | o. | | o. | | 0. | | |
| Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Incide | of | Incide | n o |
| ce Rate | A | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | f |
| | Es | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | Α |
| | 123 | | S | | s | | s | | s | | s | | s | | S | | s | | Е |
| | | | | | | | | | | | | | | | | | | | s |

<sup>\*</sup> MedDRA

| | DreamCIS Inc. |
|------|---------------------------------|
| (III | Clinical Investigation Services |

THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

| | n | ( ( ) ( | n | n | ( % | n | n | (<br>% | n | n | (<br>%<br>) | n | n | (<br>%<br>) | n | n | (<br>%<br>) | n | n | (<br>%<br>) | n | n | (<br>%<br>) | n | n | (<br>%<br>) | n | n | (<br>%<br>) | n |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class(SOC) | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Preferred Term(PT) | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | _ |

<sup>\*</sup> MedDRA



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

## 8.2 Safety per protocol set

Table 8.2 Unexpected AE and ADR

| | | | 2-1 | 10 | | | | | 11- | -18 | | | | | 19 | -34 | | | | 35. | -55 | | | | Tot | al | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Un | expe | eted | Un | expec | ted | Une | xpec | ted | Un | expec | eted | Une | xpec | ted | Unexp | ected | Į | Unexpec | ted | Unexpec | cted | Une | expec | ted | Unexp | ecte |
| Safety per protocol Set | | AE | | | ADR | | | ΑE | | | ADR | - | | AE | | AΕ | R | | AE | | ADR | - | | AE | | d AI | OR |
| | | | | | | | | | | | | | | | | | | | | | | | | | | | N |
| | | | N | | | N | | | N | | | N | | | N | | N | | | N | | N | | | N | | О |
| | | | 0. | | | 0. | | | 0. | | | 0. | | | 0. | | 0. | | | 0. | | 0. | | | 0. | | • |
| | Inc | iden | of | Inc | iden | of | Incid | len | of | Inci | den | of | Inci | den | of | Incide | of | Iı | nciden | of | Inciden | of | In | ciden | of | Incid | en o |
| | ce l | nciden<br>ee Rate | A | ce l | Rate | Α | ce R | ate | A | ce F | Rate | Α | ce R | ate | Α | ce Rate | A | c | e Rate | Α | ce Rate | Α | ce I | Rate | Α | ce Rate | e f |
| | | | Es | | | Е | | | Е | | | Е | | | Е | | Е | | | Е | | Е | | | Е | | Α |
| | | | Lo | | | s | | | S | | | s | | | S | | s | | | S | | s | | | S | | Е |
| | | | | | | | | | | | | | | | | | | | | | | | | | | | s |
| | | ( | | | ( | | | ( | | | ( | | | ( | | ( | | | ( | | ( | | | ( | | ( | |
| | n | % | n | n | % | n | n | % | n | n | % | n | n | % | n | n % | n | r | n % | n | n % | n | n | % | n | n % | n |
| | | ) | | | ) | | | ) | | | ) | | | ) | | ) | | | ) | | ) | | | ) | | ) | |
| System Organ Class(SOC) | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Preferred Term(PT) | | | | | | | | | | | | | | | | | | , | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

| | | | 2-1 | 10 | | | | 11 | -18 | | | | 19 | -34 | | | 35 | -55 | | | To | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Ur | expe | eted | Un | expec | ted | Unexpe | cted | Unex | pecte | d | Unexpec | ted | Unexpe | cted | Unexpe | cted | Unexpe | eted | Unexped | eted | Unexpe | cte |
| Safety per protocol Set | | AE | | | ADR | | AE | | A | DR | | AE | | ADI | ξ. | AE | | ADR | | AE | | d AD | R |
| | | iden<br>Rate | N<br>o.<br>of<br>A<br>Es | | iden<br>Rate | N o. of A E | | | Incido<br>ce Ra | en ( | N oo. of A E s | Inciden<br>ce Rate | | Inciden<br>ce Rate | | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E | Incider<br>ce Rate | | | |
| | | | | | | | - | | : | , | | | | <u> </u> | | - | | : , | | | | | S |
| | | % | | | ( | | . 0/ | | | ( | | ( | | ( | | ( | | ( | | ( | | ( | |
| | n | ) | n | n | % | n | n % | n | n ' | ) | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n |
| Total | | | | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

## 8.3 Non-Safety per protocol set

Table 8.3 Unexpected AE and ADR

| | | | 2-1 | 10 | | | | | 11- | -18 | | | | | 19- | -34 | | | 35 | -55 | | | То | tal | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non-Safety per protocol | Un | expec | eted | Une | expec | ted | Une | expec | ted | Une | expec | ted | Une | xpec | ted | Unexpe | cted | Unexpe | cted | Unexpe | cted | Unexpe | cted | Une | xpect | .e |
| Set | | AE | | | ADR | | | ΑE | | | ADR | | | ΑE | | ADI | 1 | AE | | ADF | 1 | AE | | d A | ADR | |
| | | | | | | | | | | | | | | | | | | | | | | | | | | N |
| | | | N | | | N | | | N | | | N | | | N | | N | | N | | N | | N | | | o |
| | | | 0. | | | 0. | | | 0. | | | 0. | | | 0. | | 0. | | 0. | | 0. | | o. | | | |
| | Inc | iden | o.<br>of | Inci | den | of | Inci | den | of | Inci | den | of | Incid | len | of | Inciden | of | Inciden | of | Inciden | of | Incide | n o | f Inc | iden | o |
| | ce l | Rate | A | ce F | Rate | A | ce R | ate | A | ce F | Rate | A | ce Ra | ate | Α | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce R | ate | f |
| | | | Es | | | Е | | | Е | | | Е | | | Е | | Е | | Е | | Е | | Е | | | A |
| | | | Lo | | | s | | | S | | | S | | | s | | s | | s | | s | | s | | | E |
| | | | | | | | | | | | | | | | | | | | | | | | | | | S |
| | | ( | | | ( | | | ( | | | ( | | | ( | | ( | | ( | | ( | | ( | | | ( | |
| | n | % | n | n | % | n | n | % | n | n | % | n | n | % | n | n % | n | n % | n | n % | n | n % | n | n | % | n |
| | | ) | | | ) | | | ) | | | ) | | | ) | | ) | | ) | | ) | | ) | | | ) | |
| System Organ Class(SOC) | | | | | | | | | | | | | | | | | | | | | | | | | | _ |
| Preferred Term(PT) | | | | | | | | | | | | | | | | | | | - | | | | - | | - | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

| | | | 2- | 10 | | | | | 11- | 18 | | | | | 19- | -34 | | | 35 | -55 | | | To | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non-Safety per protocol | Un | expe | cted | Un | expe | eted | Une | xpec | ted | Une | xpec | eted | Unex | xpec | ted | Unexpe | cted | Unexpo | ected | Unexpe | cted | Unexpe | cted | Unex | pecte |
| Set | | AE | 1 | ļ | ADR | | | AE , | | A | ADR | | 1 | AE , | | ADI | ξ | AE | , | ADI | R | AE | 1 | d A | DR |
| | | iden<br>Rate | N o. of A Es | | iden<br>Rate | N<br>o.<br>of<br>A<br>E | Incid<br>ce R | | | Incid<br>ce R | | N o. of A E s | Incid<br>ce Ra | | | Inciden<br>ce Rate | | Inciden<br>ce Rate | | Inciden<br>ce Rate | | Incide<br>ce Rate | | f Inc | N o iden o ate f A E |
| | | ( | | | ( | | | ( | | | ( | | | ( | | ( | | ( | | . ( | | ( | | | ( s |
| | n | % | n | n | % | n | n | % | n | n | % | n | n | % | n | n % | n | n % | n | n % | n | n % | n | n | % n |
| | | ) | | | ) | | | ) | | | ) | | | ) | | ) | | ) | | ) | | ) | | | ) |
| Total | | | | | | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

### 9. MAAE/ADR for 28 days after vaccination

## 9.1 Safety Set

Table 9.1 MAAE and ADR

| | | 2- | 10 | | | 11 | -18 | | | | 19 | -34 | | | 35 | -55 | | | Tot | al | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety Set | MAAl | Ξ | ADR | | MAA | Е | | ADR | | MAA | Е | ADR | 2 | MAA | Е | ADR | - | MAA | Е | AD | R |
| | Inciden<br>ce Rate | N o. of A Es | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | | Inci<br>ce R | | N o. of A E s | Inciden<br>ce Rate | N o. of E | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | N o. of A E | Incider<br>ce Rate | | Incid<br>ce Rat | N o |
| | (% | | ( | | ( | | | ( | | ( | | ( | | ( | | ( | | ( | | ( | |
| | n ) | n | n %<br>) | n | n % | n | n | % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | ó n |
| System Organ Class(SOC) Preferred Term(PT) | THE PERSON NAMED IN COLUMN NAM | | | | | | | | | | | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

| | | MAAE | | 0 | | | 11 | -18 | | | 19 | -34 | | | 35 | -55 | | | Tot | tal | , |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety Set | N | MAAI | 3 | ADR | | MAA | E | ADR | | MAA | E | ADR | | MAAl | E | ADR | | MAAI | Ξ | ADR | |
| | Inci<br>ce F | den<br>Rate | N<br>o.<br>of<br>A<br>Es | Inciden<br>ce Rate | N o. of A E s | Inciden<br>ce Rate | | Inciden<br>ce Rate | | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E | Incider<br>ce Rate | | f Incide<br>ce Rate | |
| | n | (% | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n |
| Total | 111111111111111111111111111111111111111 | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

## 9.2 Safety per protocol set

Table 9.2 MAAE and ADR

| | | | 2-1 | 10 | | | 11 | -18 | | | 19 | -34 | | | 35 | -55 | | | Tot | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety per protocol Set | | MAA | Е | ADR | | MAA | Е | ADF | 2 | MAA | Е | ADR | | MAAl | Е | ADR | | MAA | Е | ADR | |
| | | | | | | | | | | | | | | | | | | | | | N |
| | | | N | | N | | N | | N | | N | | N | | N | | N | | N | | o |
| | | | 0. | | o. | | 0. | | o. | | 0. | | o. | | o. | | 0. | | о. | | |
| | Inc | iden | o.<br>of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | o |
| | ce | Rate | A | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | f |
| | | | Es | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | A |
| | | | La | | s | | s | | s | | s | | s | | s | | s | | s | | Е |
| | | | | | | | | | | | | | | | | | | | | | s |
| | | (% | | ( | | ( | | ( | | ( | | ( | | ( | | ( | | ( | | ( | |
| | n | (,0 | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n |
| . <u> </u> | | , | | ) | | ) | | ) | | ) | | ) | | ) | | ) | | ) | | ) | |
| System Organ Class(SOC) | | | | | | | | | | | | | | | | | | | | | |
| Preferred Term(PT) | | | | | | | | | | | | | | V. | | | | , | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

| | | 2-1 | 10 | | | 11 | -18 | | | 19 | -34 | | | 35 | -55 | | | Tot | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety per protocol Set | MAA | E | ADR | | MAA | E | ADF | <b>\</b> | MAA | E | ADR | | MAAl | E | ADR | | MAA | E | ADR | |
| | Inciden of ce Rate A Es | | Inciden<br>ce Rate | N o. of A E s | Inciden<br>ce Rate | | Inciden<br>ce Rate | | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E s | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | |
| | n (% | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n |
| Total | | | | | _ | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

# STATISTICAL ANALYSIS PLAN(V2.0)

## 9.3 Non-Safety per protocol set

Table 9.3 MAAE and ADR

| 2 | | 2-1 | 10 | | | | | 11-18 | | | | 19-34 | | | | | -55 | Total | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non- Safety per protocol<br>Set | ] | MAA | Е | | ADR | | MA | ΑE | | ADR | | MAA | E | ADI | 2 | MAA | Е | ADR | 1 | MAA | Е | ADR | - |
| | | iden<br>Rate | N o. of A Es | | iden<br>Rate | N o. of A E | Incider | | | eiden<br>Rate | N o. of A E s | Inciden<br>ce Rate | | Inciden<br>ce Rate | | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E s | Incider<br>ce Rate | | Incide<br>ce Rate | |
| | n | (% | n | n | 0/0 | n | n % | n | n | ( % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n |
| System Organ Class(SOC) Preferred Term(PT) | | | | | | | | TO THE RESERVE OF THE PROPERTY | | | | | | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

22-NOV-2013

Last Update Date

| | | | 2-1 | 0 | | | | 11 | -18 | | | | 19 | -34 | | | 35 | -55<br>I | | | Tot | al |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non- Safety per protocol<br>Set | 1 | MAAI | E | | ADR | | MAA | E | | ADR | | MAA | Æ | ADI | ₹ | MAA | E | ADR | | MAAl | Ξ | ADR |
| | | iden<br>Rate | N<br>o.<br>of<br>A<br>Es | | den | | | | | eiden<br>Rate | N o. of A E s | | | Inciden<br>ce Rate | | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E | Incider<br>ce Rate | | Incide<br>ce Rate |
| | n | (%) | n | n | % | n | n % | n | n | ( % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % |
| Total | | | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA



\_

# STATISTICAL ANALYSIS PLAN

A Multicenter, Post Marketing Surveillance study to Monitor the Safety of Novartis Meningococcal ACWY Conjugate Vaccine (MenACWY-CRM) Administered According to the Prescribing Information to Healthy Subjects from 2 to 55 Years of Age in the Republic of South Korea

Product Name: Menveo (MenACWY-CRM)

Protocol No. : V59\_62

Version : V3.0

Effective Date :07-MAY-2014

**EFFECTIVE DATE: 2014-03-04** 



## CON PIDENT!AI. :

THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND JS NOT TO BE DISCLOSED WITHOUT

.I0·APR-2014

Last Update Date

THE WRITTEN PERMISSION OF COMT'ANY

# STATISTICAL ANALYSIS PLAN(V3.0)

### **Approvals**







THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

# STATISTICAL ANALYSIS PLAN(V3.0)

# Revisions

| DATE OF<br>REVISION | INDICATION REVISION | REASON FOR CHANGE | AUTHOR<br>NAME |
|---|---|---|---|
| 22-NOV-2013 | All | Protocol Amendment | PPD |
| | | Modification of tables to include | PPD |
| 10-APR-2014 | Appendix1 | incidence rate of ADR, | |
| | | Fever added to Solicited reaction | |

Last Update Date

### CONFIDENTIAL:

THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

# STATISTICAL ANALYSIS PLAN(V3.0)

## **Table of Contents**

| Revisions | 3 |
|--------------------------------------------------|----|
| 1. Study Objective | 6 |
| 2. Study Method and Study Period | 6 |
| 2.1 Study Period | 6 |
| 2.2 Number of Subjects | 6 |
| 2.3 Study population | 6 |
| 2.3.1 Inclusion criteria | 6 |
| 2.3.2 Exclusion criteria | 7 |
| 2.4 Study Method. | 7 |
| 3. Analysis Sets | 10 |
| 3.1 Safety Analysis Sets | 10 |
| 3.2 Efficacy Analysis Set | 11 |
| 4. Endpoints | 12 |
| 4.1 Safety Endpoints | 12 |
| 5. Assessment Criteria | 12 |
| 5.1 Safety Assessment Criteria | 12 |
| 6. Statistical Analyses | 12 |
| 6.1 Baseline Characteristics | 12 |
| 6.2 Safety Analyses | 13 |
| 6.2.1 Adverse Events by Baseline Characteristics | 13 |
| 6.2.2. Analysis of Solicited AE | 14 |
| 6.2.3 Analysis of Unsolicited AE | 15 |
| 7. List of Table and Data Listings | 16 |
| 7.1 Distribution of Subjects | 16 |
| 7.2 Baseline Characteristics | 16 |
| 7.3 Safety Analyses | 16 |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| 8. Notes | 17 | ! |
|-----------|----|---|
| Appendix1 | 18 | ; |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

STATISTICAL ANALYSIS PLAN(V3.0)

### 1. Study Objective

The primary objective of the study is to monitor the safety of a single dose of MenACWY-CRM vaccine in subjects from 2 to 55 years of age, as evaluated by:

- 1. Local and systemic solicited adverse events reported from study Day 1 (day of vaccination) through study Day 7 post-vaccination
- 2. All unsolicited Adverse Events (AEs) reported from study Day 1(day of vaccination) through study Day 7 post-vaccination
- 3. Medically attended Adverse Events reported from study Day 1 to study termination (Day 29/early termination)
- 4. All Serious Adverse Events (SAEs) reported from study Day 1 to study termination (Day 29/early termination)

### 2. Study Method and Study Period

### 2.1 Study Period

The trial period shall be from market launch date till approximately 22 May 2018.

### 2.2 Number of Subjects

A total of approximately 3,300 subjects are planned for enrolment into this study.

Assuming a 10% drop-out rate, this should provide approximately 3,000 evaluable subjects. This sample size meets the post-licensure requirements of the MFDS to provide continued safety monitoring in the Korean population.

#### 2.3 Study population

#### 2.3.1 Inclusion criteria

Individuals eligible for enrolment in this study are those:

1. Male and female subjects from 2 to 55 years of the age at the time of Visit 1(including all 55



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

# STATISTICAL ANALYSIS PLAN(V3.0)

years old subjects, up to one day before their 56<sup>th</sup> year birthday), who are scheduled to receive vaccination with MenACWY-CRM conjugate vaccine, according to the local prescribing information and routine clinical practice

- 2. To whom the nature of the study has been described and the subject or subject's parent/legal representative has provided written informed consent (written assent from minors should be also obtained if required by the relevant IRB);
- 3. Whom the investigator believes that the subject can and will comply with the requirements of the protocol (e.g., completion of the Diary Card);
- 4. Who are in good health as determined by the outcome of medical history, physical assessment and clinical judgment of the investigator

#### 2.3.2 Exclusion criteria

1. Contraindication, special warnings and/or precautions, as evaluated by the investigators, reported in the MenACWY-CRM conjugate vaccine Korean prescribing information.

### 2.4 Study Method

In order to obtain information on Regulatory PMS data after market launch, NVD or delegate will create the Regulatory PMS contract with the relevant clinics/hospitals and the physician in charge of the survey shall implement this Regulatory PMS in subjects that receive MenACWY-CRM in the relevant hospital/clinic since the contract date until the number of contracted survey cases, without omission, is reached.

### Overview of Study Design

This is a multicenter post marketing surveillance study to monitor the safety of MenACWY-CRM administered according to the prescribing information to 3,300 healthy subjects from 2 to 55 years of age in Korea.

Subjects will be enrolled at the time of their visit to a participating clinic or hospital for vaccination with MenACWY-CRM according to the routine clinical care.

At Visit 1 (Day 1), after obtaining consent from the subjects or subjects' parents/legal representative (written assent will be also obtained if required by the relevant IRB), the vaccination will be administered. Subjects will remain under observation for at least 30 minutes in the clinic after study immunization.



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

# STATISTICAL ANALYSIS PLAN(V3.0)

The subjects or subject's parent/legal representative will be then instructed to complete the Diary Card daily, reporting local and systemic adverse events and all other AEs occurring within 7 days following immunizations, and medically attended AEs or SAEs occurring up to Day 29.

Subjects will also be instructed to return the completed diaries to the study site at Day 29 as follows:

- During a visit at the study center or
- Using the provided pre-addressed stamped envelope (PASE).

At the investigator discretion, the subject or subject's parent/legal representative will be reminded of the date of the study termination by a phone call at Day 29. If any clarification is required after Diary Card retrieval the site staff will follow up by phone, and any additional finding will be recorded on the subject's medical record.

In case the Diary Card is not retrieved within 10 days after Day 29, subject or subject's parent/legal representative will be contacted by phone to assess the occurrence of adverse events, determine the subject's clinical status and complete study termination. All information will be recorded by the site staff on the subject's medical record and collected in the appropriate section of the CRF.

All SAEs will be monitored until resolution and/or the cause is identified. If a SAE remains unresolved at study termination, a clinical assessment will be made by the investigator and the NVD regional physician to determine whether continued follow up of the SAE is needed.

Table 3.1-1: Safety Assessment Table

| Medical History: | From birth, collected at clinic |
|---|---|
| All significant past diagnoses including all allergies, | visit Day 1 |
| major surgeries requiring inpatient hospitalization, | |
| other significant injuries or hospitalizations, any | |
| conditions requiring prescription or chronic medication | |
| (i.e., >2 weeks in duration), or other significant medical | |
| conditions based on the investigator's judgment. | |
| Immediate reactions: | For at least 30 minutes after |
| Subjects will be assessed for immediate | vaccination |
| hypersensitivity reactions. | |
| Solicited local adverse events: | Days 1-7 after vaccination |
| < 6 years : injection site erythema, injection site | |
| induration, injection site tenderness | |



# Last Update Date

### CONFIDENTIAL:

THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

| $\geq$ 6 years : injection site erythema, injection site | |
|---|---|
| induration, injection site pain | |
| Solicited systemic adverse events: | Days 1-7 after vaccination |
| < 6 years : change in eating habits, sleepiness, | |
| irritability, rash, vomiting, diarrhea, fever | |
| ≥ 6 years : chills, nausea, malaise, generalized myalgia, | |
| generalized arthralgia, headache, rash, fever | |
| All unsolicited AEs will be collected | Days 1-7 after vaccination |
| Medically attended Adverse Events: | From Day 1 to study |
| Events that require a physician's visit or an emergency | termination (Day 29/early |
| room visit (events that are managed by telephone or | termination) |
| means other than a face-to-face evaluation by a | |
| clinician do not qualify as medically attended AEs). | |
| Serious AEs: | From Day 1 to study |
| All SAEs will be collected. | termination (Day 29/early |
| | termination) |
| Medications: | From Day 1 to Day 7 |
| Any medications used to treat any solicited local and | |
| systemic reaction and unsolicited AE be collected. | |
| Medications: | From Day 1 to study |
| Any medications used to treat any medically attended | termination (Day 29/early |
| AE or SAE will be collected. | termination) |



# Last Update Date

## CONFIDENTIAL:

THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

# STATISTICAL ANALYSIS PLAN(V3.0)

#### 3. Analysis Sets

### 3.1 Safety Analysis Sets

#### Safety Set

All subjects who

- have signed an informed consent form, undergone screening procedure(s) and received a subject number,
- received a study vaccination,
- provided post vaccination safety data.

#### Safety per protocol set

All subjects in the safety Set with the exclusions of the following cases:

- (1) Subjects administered prior to the contract date.
- (2) Subjects who didn't receive MenACWY-CRM.
- (3) Subjects who already receive MenACWY-CRM.
- (4) Follow-up failure: The subjects whose safety information cannot be identified due to follow-up loss.
- (5) Not applicable to the indication of study drug [Indication]
  - To prevent invasive meningococcal disease caused by Neisseria meningitides serogroups A, C, Y and W-135 in persons 2 through 55 years of age.
- (6) Subjects who violate of Protocol: Those who do not meet one item at least of the inclusion/exclusion criteria.

[Inclusion criteria]

- Male and female subjects from 2 to 55 years of the age at the time of Visit 1(including all 55 years old subjects, up to one day before their 56<sup>th</sup> year birthday), who are scheduled to receive vaccination with MenACWY-CRM conjugate vaccine, according to the local prescribing information and routine clinical practice.
- 2) To whom the nature of the study has been described and the subject or subject's parent/legal representative has provided written informed consent.
- 3) Whom the investigator believes that the subject can and will comply with the requirements of the protocol.



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

# STATISTICAL ANALYSIS PLAN(V3.0)

4) Who are in good health as determined by the outcome of medical history, physical assessment and clinical judgment of the investigator.

[Exclusion criteria]

- 1) Contraindication, special warnings and/or precautions, as evaluated by the investigators, reported in the MenACWY-CRM conjugate vaccine Korean prescribing information
- (7) Subjects who prescribed off-label dosage.
  - Violation of intramuscular injection only (0.5ml)

#### Non-Safety per protocol set

Subjects excluded from safety per protocol set except for subjects who did not receive MenACWY-CRM and follow-up failure.

Based on rules for estimation of each number of safety evaluation cases, the following local regulation and Guideline on Standards for re-examination for new drugs, etc \*\* of MFDS, non-safety analysis set are excluded from the safety analysis set:

- Guideline on Standards for re-examination for new drugs, etc (Chapter II, no. 3)
   Patient Population for Surveillance
  - A) Patients planned to receive a drug under surveillance by investigator's medical judgment shall be subject.
  - B) Subject who do not use within approved range shall not be included in the subject in principal.
    - \* However, if data of subject whose use is beyond approved range is collected, perform analysis as a separate item.
  - C) Describe actual selection methods of subject in detail.

### 3.2 Efficacy Analysis Set

Not Applicable



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

# STATISTICAL ANALYSIS PLAN(V3.0)

### 4. Endpoints

## 4.1 Safety Endpoints

Safety will be assessed after administration of study vaccine in terms of the number and percentage of subjects with:

- Local and systemic solicited adverse events reported from study Day 1 (day of vaccination) through study Day 7 post-vaccination;
- Unsolicited AEs reported from study Day 1 (day of vaccination) through study Day 7 post-vaccination;
- Medically attended AEs reported from study Day 1 to study termination (Day 29/early termination);
- SAEs reported from study Day 1 to study termination (Day 29/early termination).

#### 5. Assessment Criteria

### **5.1 Safety Assessment Criteria**

Not Applicable

### 6. Statistical Analyses

#### **6.1 Baseline Characteristics**

Descriptive statistics (mean, standard deviation, median, minimum and maximum) for baseline characteristics such as age, height and weight at enrollment will be calculated in the Safety set and Safety per Protocol set.

The following baseline characteristics will be reported:



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

# STATISTICAL ANALYSIS PLAN(V3.0)

- < Subject Baseline Information >
  - gender, age, ethnic origin, weight, height, past diagnosis, pre-Immunization temperature, temperature location, pregnancy
- < Study Vaccine Information >
  - vaccine site, concomitant medications

### **6.2 Safety Analyses**

The number of subjects of  $AE^{\dagger}$  and the number of  $AEs^{\dagger}$  incurred shall be calculated, the incidence rate of  $AEs^{\dagger}$  and its 95% confidence interval will be calculated using the normal approximation on the safety set and safety per protocol set.

† AE : AE includes solicited and unsolicited AE (DAY 1-7), medically attended AE (DAY 1-29) and SAE (DAY 1-29).

### **6.2.1** Adverse Events by Baseline Characteristics

 $AE^{\dagger}s$  (as described below) will be reported (n, %) for the following the baseline characteristics in the safety set and safety per protocol set :

- Age group (2-10, 11-18, 19-34, 35-55)
- Children group ( $<18, \ge 18$ )
- Gender (male, female)
- Past diagnosis (yes, no)
- Temperature location (axillary, oral, rectal, ear)
- Administration site (left deltoid, right deltoid, other)
- Concomitant medication (yes, no)
- Kidney disorder (yes, no)
- Liver disorder (yes, no)
- Pregnancy (yes, no)

The n(%) of AEs<sup>†</sup> and its 95% confidence interval will be calculated using the normal approximation and analyzed using  $\chi^2$ - test or Fisher's exact test.



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

# STATISTICAL ANALYSIS PLAN(V3.0)

† AE : AE includes solicited and unsolicited AE (DAY 1-7) and medically attended AE (DAY 1-29) and SAEs.

#### 6.2.2. Analysis of Solicited AE

Frequencies and percentages of subjects experiencing each adverse event will be presented for each symptom severity. Summary tables showing the occurrence of any local or systemic adverse events overall and at each time point will also be presented (see Table 4.1.3 and 4.2.3).

Post-vaccination adverse events reported from Day 1 to Day 7 will be summarized by maximal severity. The severity of local adverse events for subjects < 6 years of age will be categorized as follows. Injection-site erythema and induration: absent (0 to 9 mm), mild (10 to 25 mm), moderate (26 to 50 mm), severe (>50 mm); injection-site tenderness: none, mild (minor light reaction to touch), moderate (cried or protested to touch), severe (cried when injected limb was moved). For subjects  $\geq$  6 years, injection-site erythema and induration absent (1 to 24 mm), mild (25 to 50 mm), moderate (51 to 100 mm), severe (>100 mm); pain: none, mild (present but does not interfere with activity), moderate (interferes with activity), severe (prevents daily activity).

For subjects  $\geq$  6 years of age, the severity of systemic adverse events (i.e., chills, nausea, malaise, generalized myalgia, generalized arthralgia, headache) occurring up to 7 days after each vaccination will be categorized as none, mild (present but not interfering with daily activity), moderate (some interference with daily activity), and severe (prevents daily activity) except for rash, which will be categorized as none, urticarial, or other.

For subjects < 6 years of age, the severity of systemic adverse events occurring up to 7 days after each vaccination will be categorized as follows. Change in eating habits: none (no change in appetite), mild (eating less than normal for 1 to feeds), moderate (missed 1 or 2 feeds), severe (missed more than 2 feeds); sleepiness: none (no change in alertness), mild (shows an increased alertness), moderate (sleeps through feeds), severe (sleeps most of the time and it is hard to arouse him/her); irritability: none (no change in child disposition), mild (requires more cudding and he/she is less playful than usual), moderate (more difficult to settle), severe (unable to console); rash: none, urticarial, or other; vomiting: none, mild (1-2 episodes/24 hours), moderate (>2 episodes/24 hours), severe (requires outpatient hydratation); diarrhea: none (fewer than 2 loose stools/24 hours), mild (2-3 loose stools or < 400 gms/24 hours), moderate (4-5 stools or 400-800 gms/24 hours), severe (6 or more watery stools


THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

#### STATISTICAL ANALYSIS PLAN(V3.0)

or > 800 gms/24 hours or requires outpatient IV hydration).

Body temperature will be categorized as  $<38^{\circ}$ C (no fever),  $\ge 38^{\circ}$ C (fever) and will be summarized by  $0.5^{\circ}$ C increments from  $36.0^{\circ}$ C up to  $\ge 40^{\circ}$ C. Additionally, no fever vs. fever will be reported.

Each local and systemic adverse event will also be categorized as none vs. any.

#### **6.2.3** Analysis of Unsolicited AE

All unsolicited AEs and MAAE recorded in the CRF will be mapped to preferred terms using the most recent MedDRA dictionary and classified by System organ class (SOC) and Preferred Terms (PT). Under the classification standard of MedDRA terms, and all AEs excluding the AEs whose causal relation with the study medication is 'Not Related' shall be treated as AEs whose causal relation cannot be excluded {hereafter "Adverse Drug Reaction(ADR)"}.

- ① The number and percentage of unsolicited AE (Day 1-7) and MAAE (Day 1-29) and SAEs (Day 1-29) according to the serious, severity, frequency, action taken, outcome, relationship to MenACWY-CRM regarding occurred AE will be calculated.
- ② Unsolicited AEs (Day 1-7) and MAAE (Day 1-29) and SAEs (Day 1-29) will be classified into the preferred terms according to the serious, severity, frequency, action taken, outcome, relationship to MenACWY-CRM. Also, the number and percentage of each AE (PT) will be calculated.
- ③ The number of subjects and the number of unexpected AE/ADR, SAE/Serious ADR (SADR) and MAAE/ADR will be calculated according to the preferred terms. Also, the incidence rate will be estimated.
- (4) For subjects excluded from safety per protocol set<sup>†</sup>, the number of subjects and the number of unexpected AE/ADR, SAE/Serious ADR (SADR) and MAAE/ADR will be calculated according to the preferred terms. Also, the incidence rate will be estimated.
  - † Subject excluded from safety per protocol set: Except for subjects who didn't receive study vaccination and follow-up failure.



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

STATISTICAL ANALYSIS PLAN(V3.0)

#### 7. List of Table and Data Listings

#### 7.1 Distribution of Subjects

- Number of subjects contracted to the study: The number of subjects are to be collected(under contract) as contracted by the investigator
- Number of retrieving completed CRFs: Total number of subjects whose completed CRFs
- Number of safety assessment population: Number of safety assessment population among total number

#### 7.2 Baseline Characteristics

- Mean and standard deviation (SD) or frequency and percentage by gender, age, ethnic origin, weight, height, past diagnosis, pre-Immunization temperature, temperature location, pregnancy
- Frequency and percentage by vaccine site, concomitant medications

#### 7.3 Safety Analyses

- Incidence rate and the number of AEs according to the baseline characteristics (frequency and percentage)
- The number of the serious, severity, frequency, action taken, outcome, relationship to MenACWY-CRM for Unsolicited AE (DAY 1-7) and MAAE (frequency and percentage)
- The number of AEs for the severity, day, fever to MenACWY-CRM according to individual solicited AE (DAY 1-7) (frequency and percentage)
- Incidence rate and number according to the preferred terms of SAE/SADR, unexpected AE/unexpected ADR, and MAAE/ADR (frequency and percentage)
- For subjects excluded from safety per protocol set<sup>†</sup> incidence rate and number according to the preferred terms of SAE/SADR, unexpected AE/unexpected ADR, and MAAE/ADR (frequency and percentage)
  - † Subject excluded from safety per protocol set: Except for subjects who didn't receive study mediation and follow-up failure



#### Last Update Date


THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

### STATISTICAL ANALYSIS PLAN(V3.0)

#### 8. Notes

- Each statistical analysis will be carried out with SAS Software version 9.2 or more recent version.
- In the descriptive statistics, mean, SD, minimum, median, and maximum will be calculated for continuous variables, and frequency and percentage for categorical variables.
- Data including sign of inequality such as "≥20", ">20" will be excluded from analysis.
- All test statistics will be the results of two-sided tests with the statistical significant level of 0.05.
- The followings shall be included only in re-examination report:
  - Analysis by type of concomitant medications
  - Item ② of paragraph 6.2.3
  - Estimation of 95% confidence interval for incidence of AEs by background factors



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

### STATISTICAL ANALYSIS PLAN(V3.0)

#### Appendix1

#### 1. Demographic and baseline values, medication characteristics, specific characteristics

- Baseline characteristics will be reported on the safety set and safety per protocol set.

#### 1.1 Safety Set

Table 1.1.1 Total subject

| Safety Set | Total |
|------------|------------------|
| | No. subjects (%) |
| Total | |

#### Table 1.1.2 Demographic characteristics

#### 1) (Administration start date)-(birth)+1

| Safety Set | | Total |
|-----------------------|--------------|------------------|
| | | No. subjects (%) |
| Age(years)1) | No. subjects | |
| | mean±std | |
| | median | |
| | min~max | |
| Age(years) | 2-10 | |
| | 2-5 | |
| | 6-10 | |
| | 11-18 | |
| | 19-34 | |
| | 35-55 | |
| | Total | |
| Children group(years) | < 18 | |
| | ≥ 18 | |
| | Total | |
| Ethnic Origin | Asian | |
| | Black | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| Safety Set | | Total |
|------------------------------------------|--------------|------------------|
| | | No. subjects (%) |
| | Caucasian | |
| | Hispanic | |
| | Other | |
| | Total | |
| Gender | Male | |
| | Female | |
| | Total | |
| Weight(kg) | No. subjects | |
| | mean±std | |
| | median | |
| | min~max | |
| Height(cm) | No. subjects | |
| | mean±std | |
| | median | |
| | min~max | |
| Table 1.1.3 Past diagnosis | | |
| Safety Set | | Total |
| | | No. subjects (%) |
| Yes | | |
| No | | |
| Total | | |
| Table 1.1.4 Pre-Immunization temperature | e | |
| Safety Set | | Total |
| | | No. subjects (%) |
| No. subjects | | |
| mean±std (°C) | | |
| median | | |
| min~max | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| Table 1.1.5 Temperature Location | |
|------------------------------------|------------------|
| Safety Set | Total |
| | No. subjects (%) |
| Axillary | |
| Oral | |
| Rectal | |
| Ear | |
| Total | |
| Table 1.1.6 Administration Site | |
| Safety Set | Total |
| | No. subjects (%) |
| Left Deltoid | |
| Right Deltoid | |
| Other | |
| Total | |
| Table 1.1.7 Concomitant medication | |
| Safety Set | Total |
| Sulety Set | No. subjects (%) |
| Yes | |
| No | |
| Total | |
| Table 1.1.8 Kidney Disorder | |
| Safety Set | Total |
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |
| | 1 |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

### STATISTICAL ANALYSIS PLAN(V3.0)

#### Table 1.1.9 Liver disorder

| Safety Set | Total |
|------------|------------------|
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |

#### Table 1.1.10 Pregnancy

| Safety Set | Total |
|------------|------------------|
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |

#### 1.2 Safety Per Protocol Set

#### Table 1.2.1 Total subject

| Safety per protocol set | Total |
|-------------------------|------------------|
| | No. subjects (%) |
| Total | |

#### Table 1.2.2 Demographic characteristics

#### 1) (Administration start date)-(birth)+1

| Safety per protocol set | | Total |
|--------------------------|--------------|------------------|
| | | No. subjects (%) |
| Age(years) <sup>1)</sup> | No. subjects | |
| | mean±std | |
| | median | |
| | min~max | |
| Age(years) | 2-10 | |
| | 2-5 | |
| | 6-10 | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

# STATISTICAL ANALYSIS PLAN(V3.0)

| Safety per protocol set | | Total |
|-------------------------|--------------|------------------|
| | | No. subjects (%) |
| | 11-18 | |
| | 19-34 | |
| | 35-55 | |
| | Total | |
| Children group(years) | < 18 | |
| | ≥ 18 | |
| | Total | |
| Ethnic Origin | Asian | |
| | Black | |
| | Caucasian | |
| | Hispanic | |
| | Other | |
| | Total | |
| Gender | Male | |
| | Female | |
| | Total | |
| Weight(kg) | No. subjects | |
| | mean±std | |
| | median | |
| | min~max | |
| Height(cm) | No. subjects | |
| | mean±std | |
| | median | |
| | min~max | |

#### Table 1.2.3 Past diagnosis

| Safety per protocol set | Total |
|-------------------------|------------------|
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| Table 1.2.4 Pre-Immunization temperature | |
|------------------------------------------|------------------|
| Safety per protocol set | Total |
| | No. subjects (%) |
| No. subjects | |
| mean±std (°C) | |
| median | |
| min~max | |
| Table 1.2.5 Temperature Location | |
| Safety per protocol set | Total |
| | No. subjects (%) |
| Axillary | |
| Oral | |
| Rectal | |
| Ear | |
| Total | |
| Table 1.2.6 Administration Site | |
| Safety per protocol set | Total |
| | No. subjects (%) |
| Left Deltoid | |
| Right Deltoid | |
| Other | |
| Total | |
| Table 1.2.7 Concomitant medication | |
| Safety per protocol set | Total |
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

## STATISTICAL ANALYSIS PLAN(V3.0)

| Table 1.2.8 Kidney Disorder | |
|-----------------------------|------------------|
| Safety per protocol set | Total |
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |
| Table 1.2.9 Liver disorder | |
| Safety per protocol set | Total |
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |
| Table 1.2.10 Pregnancy | |
| Safety per protocol set | Total |
| | No. subjects (%) |
| Yes | |
| No | |

Total

| | | Last Update Date |
|---|---|---|
| Clinical Investigation Services | THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS | 10-APR-2014 |
| | PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT | 10 111 10 2011 |
| | THE WRITTEN PERMISSION OF COMPANY. | |
| STATISTICAL ANALYSIS PLAN(V3.0) | | |

#### 2. Safety Analyses

- AE includes solicited and unsolicited AE (Day 1-7) and medically attended AE (Day 1-29) and SAEs (Day 1-29)
- AE will be reported on the safety set and safety per protocol set.
- SAE/SADR will be reported on the safety set, safety per protocol set and non-safety per protocol set.

#### 2.1 Safety Set

Table 2.1.1 Summary of AE

| | | 95% CI† for the | | | 95% CI† for the | | |
|---|---|---|---|---|---|---|---|
| Safety set | No. subjects with AE | percentage of | No. AEs | No. subjects with ADR | percentage of | No. ADR | Total |
| | | subjects with AE | | | subjects with ADR | | |
| | n (%) | (Lower , Upper) | n | n (%) | (Lower , Upper) | n | n (%) |
| Solicited AE (< 6 years) | | | | | | | |
| Local AE | | | | | | | |
| Systemic AE | | | | | | | |
| Solicited AE (≥ 6 years) | | | | | | | |
| Local AE | | | | | | | |
| Systemic AE | _ | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| | | 95% CI† for the | | | 95% CI† for the | | |
|---|---|---|---|---|---|---|---|
| Safety set | No. subjects with AE | percentage of | No. AEs | No. subjects with ADR | percentage of | No. ADR | Total |
| | | subjects with AE | | | subjects with ADR | | |
| | n (%) | (Lower ,Upper) | n | n (%) | (Lower ,Upper) | n | n (%) |
| Unsolicited AE | | | | | | | |
| SAE | | | | | | | |
| MAAE | | | | | | | |
| Death | | | | | | | |
| Total | | | | | | | |

<sup>† 95%</sup> CI will be calculated using the normal approximation.

<sup>\*</sup> Day 1-7: Solicited AE, Unsolicited AE

<sup>\*</sup> Day 1-29: MAAE, SAE, Death



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

Table 2.1.2 Summary of AE by Age (year)

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| 2-10 | | | | |
| 2-5 | | | | |
| 6-10 | | | | |
| 11-18 | | | | X <sup>2</sup> -test or Exact test |
| 19-34 | | | | |
| 35-55 | | | | |
| Total | | | | |

Table 2.1.3 Summary of AE by Age (year)

| Safety Set | No. subjects with AE | No. | Total | p-value |
|-----------------------|-----------------------|-----|-------|---------|
| surety set | Tion subjects William | AEs | 10111 | p varae |
| | n (%) | n | n (%) | |
| Solicited AE | | • | | |
| 2-10 | | | | |
| 2-5 | | | | |
| 6-10 | | | | |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |
| Solicited Local AE | | | | |
| 2-10 | | | | |
| 2-5 | | | | |
| 6-10 | | | | |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |
| Solicited Systemic AE | İ | | Ī | |
| 2-10 | | | | |
| 2-5 | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| Safety Set | No. subjects with AE | No.<br>AEs<br>n | Total | p-value |
|---|---|---|---|---|
| 6-10 | | | *************************************** | |
| 11-18 | | | *************************************** | |
| 19-34 | | | *** | |
| 35-55 | | | *************************************** | |
| Unsolicited AE | | | | |
| 2-10 | | | | |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | *** | |
| SAE | | | | |
| 2-10 | | | | |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |
| MAAE | | | | |
| 2-10 | | | | |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |
| ADR | | | | |
| 2-10 | | | 101 11 | |
| 11-18 | | | *************************************** | |
| 19-34 | | | | |
| 35-55 | | | 1111 | |
| Death | | | 1 | |
| 2-10 | | | | |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | *************************************** | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

### STATISTICAL ANALYSIS PLAN(V3.0)

Table 2.1.4 Summary of AE by Children group

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| < 18 years | | | | |
| ≥ 18 years | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

#### Table 2.1.5 Summary of AE by Gender

| Safety Set | No. subjects with AE | No. | Total | p-value |
|---|---|---|---|---|
| Salety Set | No. subjects with AL | AEs AEs | Total | p-varue |
| | n (%) | n | n (%) | |
| Male | | | | |
| Female | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

#### Table 2.1.6 Summary of AE by Past diagnosis

| Safety Set | No. subjects with AE | No. | Total | p-value | |
|---|---|---|---|---|---|
| Salety Set | ivo. subjects with AL | AEs | | AEs P-value | p-varue |
| | n (%) | n | n (%) | | |
| Yes | | | | | |
| No | | | | X <sup>2</sup> -test or Exact test | |
| Total | | | | | |

#### Table 2.1.7 Summary of AE by Temperature Location

| Safety Set | No. subjects with AE | No.<br>AEs | Total |
|------------|----------------------|------------|-------|
| | n (%) | n | n (%) |
| Axillary | | | |
| Oral | | | |
| Rectal | | | |
| Ear | | | |
| Total | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

# STATISTICAL ANALYSIS PLAN(V3.0)

Table 2.1.8 Summary of AE by Administration Site

| Cofoty Cot | No subjects with AE | No. | Total |
|---------------|--------------------------------|-----|-------|
| Safety Set | afety Set No. subjects with AE | | Total |
| | n (%) | n | n (%) |
| Left Deltoid | | | |
| Right Deltoid | | | |
| Other | | | |
| Total | | | |

#### Table 2.1.9 Summary of AE by Concomitant medication

| Safety Set | No. subjects with AE | No. | Total | n volvo | |
|---|---|---|---|---|---|
| Salety Set | ivo. subjects with AL | AEs AEs | | Total | p-value |
| | n (%) | n | n (%) | | |
| Yes | | | | | |
| No | | | | X <sup>2</sup> -test or Exact test | |
| Total | | | | | |

#### Table 2.1.10 Summary of AE by Kidney Disorder

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

#### Table 2.1.11 Summary of AE by Liver disorder

| Safety Set | No. subjects with AE | No. | Total | p-value |
|---|---|---|---|---|
| surery sec | Tvo. suojoota witai 112 | AEs | 10111 | p varae |
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |



10-APR-2014

Table 2.1.12 Summary of AE by Pregnancy

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

| TI. | DreamCIS Inc. Clinical Investigation Services |
|-----|-----------------------------------------------|
| - | Clinical Investigation Services |

THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

STATISTICAL ANALYSIS PLAN(V3.0)

#### 2.2 Safety per protocol set

Table 2.2.1 Summary of AE

| | | | T . | | | | |
|---|---|---|---|---|---|---|---|
| | | 95% CI† for the | | | 95% CI† for the | | |
| Safety per protocol set | No. subjects with AE | percentage of | No. AEs | No. subjects with ADR | percentage of | No. ADR | Total |
| | | subjects with AE | | | subjects with ADR | | |
| | n (%) | (Lower , Upper) | n | n (%) | (Lower , Upper) | n | n (%) |
| Solicited AE (< 6 years) | | | | | | | |
| Local AE | | | | | | | |
| Systemic AE | | | | | | | |
| Solicited AE (≥ 6 years) | | | | | | | |
| Local AE | • | | | | | | |
| Systemic AE | | | | | | | |
| Unsolicited AE | | | | | | | |
| SAE | | | | | | | |
| MAAE | | | | | | | |
| Death | | | | | | | |
| Total | | | | | | | |

<sup>† 95%</sup> CI will be calculated using the normal approximation.

| | | Last Update Date |
|---|---|---|
| Clinical Investigation Services | THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS | 10-APR-2014 |
| | PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT | |
| | THE WRITTEN PERMISSION OF COMPANY. | |
| STATISTICA | L ANALYSIS PLAN(V3.0) | |

<sup>\*</sup> Day 1-7: Solicited AE, Unsolicited AE

<sup>\*</sup> Day 1-29: MAAE, SAE, Death



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

Table 2.2.2 Summary of AE by Age (year)

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| 2-10 | | | | |
| 2-5 | | | | |
| 6-10 | | | | |
| 11-18 | | | | X <sup>2</sup> -test or Exact test |
| 19-34 | | | | |
| 35-55 | | | | |
| Total | | | | |

Table 2.2.3 Summary of AE by Age (year)

| Safety Set | No. subjects with AE | No. | Total | p-value |
|-----------------------|----------------------|-----|-------|---------|
| | | AEs | | |
| | n (%) | n | n (%) | |
| Solicited AE | | | | |
| 2-10 | | | | |
| 2-5 | | | | |
| 6-10 | | | | |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |
| Solicited Local AE | | | | |
| 2-10 | | | | |
| 2-5 | | | | |
| 6-10 | | | | |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |
| Solicited Systemic AE | | | Ī | |
| 2-10 | | | | |
| 2-5 | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| Safety Set | No. subjects with AE | No.<br>AEs<br>n | Total n (%) | p-value |
|---|---|---|---|---|
| 6-10 | | | | |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |
| Unsolicited AE | | | * | |
| 2-10 | | | *** | |
| 11-18 | | | # 1<br># 1<br># 1<br># 1<br># 1 | |
| 19-34 | | | | |
| 35-55 | | | | |
| SAE | | | | |
| 2-10 | | | | |
| 11-18 | | | | |
| 19-34 | | | ************************************** | |
| 35-55 | | | | |
| MAAE | | | | |
| 2-10 | | | 111111111111111111111111111111111111111 | |
| 11-18 | | | | |
| 19-34 | | | *************************************** | |
| 35-55 | | | | |
| ADR | | | | |
| 2-10 | | | | |
| 11-18 | | | # I I I I I I I I I I I I I I I I I I I | |
| 19-34 | | | | |
| 35-55 | | | 11<br>11<br>11<br>11<br>11 | |
| Death | | | | |
| 2-10 | | | | |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

### STATISTICAL ANALYSIS PLAN(V3.0)

Table 2.2.4 Summary of AE by Children group

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| < 18 years | | | | |
| ≥ 18 years | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

#### Table 2.2.5 Summary of AE by Gender

| Safety per protocol Set | No. subjects with AE | No. | Total | p-value |
|---|---|---|---|---|
| | | AEs | | p value |
| | n (%) | n | n (%) | |
| Male | | | | |
| Female | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

#### Table 2.2.6 Summary of AE by Past diagnosis

| Safety per protocol Set | No. subjects with AE | No. | Total | p-value |
|---|---|---|---|---|
| amon, par process and | J | AEs | r | |
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

#### Table 2.2.7 Summary of AE by Temperature Location

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total |
|-------------------------|----------------------|------------|-------|
| | n (%) | n | n (%) |
| Axillary | | | |
| Oral | | | |
| Rectal | | | |
| Ear | | | |
| Total | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

# STATISTICAL ANALYSIS PLAN(V3.0)

Table 2.2.8 Summary of AE by Administration Site

| Cafete nor protocol Cat | No. subjects with AE | No. | Total |
|---|---|---|---|
| Safety per protocol Set | No. subjects with AE | AEs | Total |
| | n (%) | n | n (%) |
| Left Deltoid | | 1<br>1 | |
| Right Deltoid | | | |
| Other | | | |
| Total | | | |

#### Table 2.2.9 Summary of AE by Concomitant medication

| Safaty per protocol Sat | No. subjects with AE | No. | Total | n value |
|---|---|---|---|---|
| Safety per protocol Set | No. subjects with AE | AEs | Total | p-value |
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

#### Table 2.2.10 Summary of AE by Kidney Disorder

| Safety per protocol Set | No. subjects with AE | No. | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

#### Table 2.2.11 Summary of AE by Liver disorder

| Safety per protocol Set | No. subjects with AE | No. | Total | p-value |
|---|---|---|---|---|
| sulety per protocor set | | AEs | 1001 | p value |
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |



### STATISTICAL ANALYSIS PLAN(V3.0)

#### Table 2.2.12 Summary of AE by Pregnancy

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

### STATISTICAL ANALYSIS PLAN(V3.0)

#### 3. Information of AEs

#### 3.1 Safety Set

Table 3.1.1 Summary of solicited AE and unsolicited AE for 7 days after vaccination (<6 years)

| Safety Set | | AF | 3 |
|----------------|-------------------------|----------------|------------|
| | | Incidence Rate | No. of AEs |
| | | n (%) | n |
| Local AE | Tenderness | | |
| | Erythema | | |
| | Induration | | |
| | Sub Total | | |
| Systemic AE | Change in eating habits | | |
| | Sleepiness | | |
| | Irritability | | |
| | Vomiting | | |
| | Diarrhea | | |
| | Rash | | |
| | Fever | | |
| | Sub Total | | |
| UNSOLICITED AE | System Organ Class(SOC) | | |
| | Preferred Term(PT) | | <u> </u> |
| | Sub Total | | |
| Total | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

Table 3.1.2 Summary of solicited AE and unsolicited AE for 7 days after vaccination (≥6years)

| Safety Set | | Al | Е |
|----------------|-------------------------|----------------|------------|
| | | Incidence Rate | No. of AEs |
| | | n (%) | n |
| Local AE | Pain | | |
| | Erythema | | |
| | Induration | | |
| | Sub Total | | |
| Systemic AE | Chills | | |
| | Nausea | | |
| | Malaise | | |
| | Myalgia | | |
| | Arthralgia | | |
| | Headache | | |
| | Rash | | |
| | Fever | | |
| | Sub Total | | |
| UNSOLICITED AE | System Organ Class(SOC) | | |
| | Preferred Term(PT) | | |
| | Sub Total | | |
| Total | | | |

| | | Last Update Date |
|---|---|---|
| Clinical Investigation Services | THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS | 10-APR-2014 |
| | PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT | 10111112011 |
| | THE WRITTEN PERMISSION OF COMPANY. | |
| STATISTICA | L ANALYSIS PLAN(V3.0) | |

Table 3.1.3 Summary of solicited AE and unsolicited AE for 7 days after vaccination (≥6years)

| Safety Set | | | AE(6-1 | 0) | | AE(11-1 | 8) | | AE(19-3 | 4) | | AE(35- | 55) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Incider | nce Rate | No. of<br>AEs | Incidence | Rate | No. of<br>AEs | Incidence | e Rate | No. of<br>AEs | Incidence | e Rate | No. of<br>AEs |
| | | n | (%) | n | n | (%) | n | n | (%) | n | n | (%) | n |
| Local AE | Pain | | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | |
| | Sub Total | | | | | | | | | | | | • |
| Systemic AE | Chills | | | | | | | | | | | | |
| | Nausea | | | | | | | | | | | | |
| | Malaise | | | | | | | | | | | | |
| | Myalgia | | | | | | | | | | | | |
| | Arthralgia | | | | | | | | | | | | |
| | Headache | | | | | | | | | | | | |
| | Rash | | | | | | | | | | | | |
| | Fever | | | | | | | | | | | | |
| | Sub Total | , | | | | | | | | | | | |
| UNSOLICITED AE | System Organ Class(SOC) | | | | | | | | | | | | |
| | Preferred Term(PT) | | | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| Safety Set | | | AE(6-10) | | AE(11-18) | | AE(19-34) | | | AE(35-55) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Inaida | ence Rate | No. of | Incidence | Doto | No. of | Incidence | . Doto | No. of | Incidence | Data | No. of |
| | | Hiciae | ince Kate | AEs | Incidence Rate AEs | | meidence | e Kate | AEs | merdence | Rate | AEs | |
| | | n | (%) | n | n | (%) | n | n | (%) | n | n | (%) | n |
| | Sub Total | | | | | | | | | | | | |
| Total | • | | | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

Table 3.1.4 Summary of medically attended AEs for 28 days after vaccination

| Safety Set | | AF | 3 |
|------------|-------------------------|----------------|------------|
| | | Incidence Rate | No. of AEs |
| | | n (%) | n |
| MAAE | System Organ Class(SOC) | | |
| | Preferred Term(PT) | | |
| Total | | | |

Table 3.1.5 Summary of medically attended AEs for 28 days after vaccination

| Safety Set | | AE(2-10 | )) | A | λE(11-1 | 8) | A | AE(19-3 | 34) AE(35- | | E(35-5 | 5) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Incidence<br>Rate | No. of | | dence<br>ate | No.<br>of<br>AEs | | dence | No.<br>of<br>AEs | | dence | No.<br>of<br>AE<br>s |
| | | n (%) | n | n | (%) | n | n | (%) | n | n | (%) | n |
| MAAE | System Organ Class(SOC) Preferred Term(PT) | | | | | | | | | | | |
| Total | | | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

### STATISTICAL ANALYSIS PLAN(V3.0)

#### 3.2 Safety per protocol set

Table 3.2.1 Summary of solicited AE and unsolicited AE for 7 days after vaccination (<6 years)

| Safety per protocol Set | | Al | E |
|---|---|---|---|
| | | Incidence Rate | No. of AEs |
| | | n (%) | n |
| Local AE | Tenderness | | |
| | Erythema | | |
| | Induration | | |
| | Sub Total | | |
| Systemic AE | Change in eating habits | | |
| | Sleepiness | | |
| | Irritability | | |
| | Vomiting | | |
| | Diarrhea | | |
| | Rash | | |
| | Fever | | |
| | Sub Total | | |
| UNSOLICITED AE | System Organ Class(SOC) | | |
| | Preferred Term(PT) | | |
| | Sub Total | | |
| Total | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

Table 3.2.2 Summary of solicited AE and unsolicited AE for 7 days after vaccination (≥6 years)

| Safety per protocol Set | | AI | Ξ |
|---|---|---|---|
| | | Incidence Rate | No. of AEs |
| | | n (%) | n |
| Local AE | Pain | | |
| | Erythema | | |
| | Induration | | |
| | Sub Total | | |
| Systemic AE | Chills | | |
| | Nausea | | |
| | Malaise | | |
| | Myalgia | | |
| | Arthralgia | | |
| | Headache | | |
| | Rash | | |
| | Fever | | |
| | Sub Total | | |
| UNSOLICITED AE | System Organ Class(SOC) | | |
| | Preferred Term(PT) | | |
| | Sub Total | | |
| Total | | | |




THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Table 3.2.3 Summary of solicited AE and unsolicited AE for 7 days after vaccination (≥6 years)

| Safety per protocol Ser | t | | AE( | (6-10) | Ā | AE(11-1 | 18) | A | AE(19-3 | 34) | A | AE(35-5 | 55) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | dence<br>ate | No. of AEs | | ncidence<br>of<br>Rate | No.<br>of<br>AEs | | idence<br>Rate | No.<br>of<br>AEs | | dence | No.<br>of<br>AEs |
| | | n | (%) | n | n | (%) | n | n | (%) | n | n | (%) | n |
| Local AE | Pain | | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | _ | |
| | Sub Total | | | | | | | | | | | | |
| Systemic AE | Chills | | | | | | | | | | | | |
| | Nausea | | | | | | | | | | | | |
| | Malaise | | | | | | | | | | | | |
| | Myalgia | | | | | | | | | | | | |
| | Arthralgia | | | | | | | | | | | | |
| | Headache | | | | | | | | | | | | |
| | Rash | | | | | | | | | | | | |
| | Fever | | | | | | | | | | | | |
| | Sub Total | | | | | | | | | | | | |
| UNSOLICITED AE | System Organ Class(SOC) | | | | | | | | | | | | |
| | Preferred Term(PT) | | | | | | | | | | | | |
| | Sub Total | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

Table 3.24 Summary of medically attended AEs for 28 days after vaccination

| Safety per protocol Set | | AI | 3 |
|---|---|---|---|
| | | Incidence Rate | No. of AEs |
| | | n (%) | n |
| MAAE | System Organ Class(SOC) | | |
| | Preferred Term(PT) | | |
| Total | I | | |

Table 3.2.5 Summary of medically attended AEs for 28 days after vaccination

| Safety Set | | AE(2-10 | )) | A | AE(11-1 | 8) | A | AE(19-3 | 34) AE(35-: | | E(35-5 | 5) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Incidence<br>Rate | No.<br>of<br>AEs | | dence<br>ate | No.<br>of<br>AEs | | dence | No.<br>of<br>AEs | | dence<br>ate | No.<br>of<br>AE<br>s |
| | | n (%) | n | n | (%) | n | n | (%) | n | n | (%) | n |
| MAAE | System Organ Class(SOC) Preferred Term(PT) | | | | | | | | | | | |
| Total | | | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

## **STATISTICAL ANALYSIS PLAN(V3.0)**

#### 4. Solicited AE (DAY 1-7)

#### 4.1 Safety Set

Table 4.1.1 Summary of Local AE Max severity (<6 years)

| Safety Set | | 1* | 2* | 3* | 4* | Total |
|------------|------------|-------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) | n (%) |
| Local AE | Tenderness | | | | | |
| | Erythema | | | | | |
| | Induration | | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Tenderness

Table 4.1.2 Summary of Local AE Max severity (≥6 years)

| Safety Set | | 1* | 2* | 3* | 4* | Total |
|------------|------------|-------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) | n (%) |
| Local AE | Pain | | | | | |
| | Erythema | | | | | |
| | Induration | | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Pain

Table 4.1.3 Summary of Local AE by Max severity

| Safety Set | | 1* | 2* | 3* | 4* | Total |
|-------------|------------|-------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) | n (%) |
| Age (2-5) | Tenderness | | | | | |
| | Erythema | | | | | |
| | Induration | | | | | |
| Age (6-10) | Pain | | | | | |
| | Erythema | | | | | |
| | Induration | | | | | |
| Age (11-18) | Pain | | | | | |

<sup>\* 1-25(1), 26-50(2), 51-100(3), &</sup>gt;100(4): Erythema, Induration

<sup>\* 1-25(1), 26-50(2), 51-100(3), &</sup>gt;100(4): Erythema, Induration



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| | Erythema | # |
|-------------|------------|---------------------------------------|
| | Induration | |
| Age (19-34) | Pain | |
| | Erythema | |
| | Induration | |
| Age (35-55) | Pain | |
| | Erythema | |
| | Induration | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Pain, Tenderness

Table 4.1.4 Summary of Systemic AE by Max severity(<6 years)

| Safety Set | | 1* | 2* | 3* | Total |
|-------------|-------------------------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) |
| Systemic AE | Change in eating habits | | | | |
| | Sleepiness | | | | |
| | Irritability | | | | |
| | Vomiting | | | | |
| | Diarrhea | | | | |
| | Rash | | | | |
| | Fever | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Change in eating habits, Sleepiness, irritability, vomiting, diarrhea,

Table 4.1.5 Summary of Systemic AE by Max severity(≥6 years)

| Safety Set | | 1* | 2* | 3* | Total |
|-------------|------------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) |
| Systemic AE | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |

<sup>\* 1-25(1), 26-50(2), 51-100(3), &</sup>gt;100(4): Erythema, Induration

<sup>\*</sup>None(1), Urticarial(2), Other(3): Rash

 $<sup>* \</sup>ge 38^{\circ}C(1)$ : Fever



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| Headache |
|----------|
| Rash |
| Fever |

Table 4.1.6 Summary of Systemic AE by Max severity

| Safety Set | | 1* | 2* | 3* | Total |
|-------------|-------------------------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) |
| Age (2-5) | Change in eating habits | | | | |
| | Sleepiness | | : | | |
| | Irritability | | | | |
| | Vomiting | | | | |
| | Diarrhea | | | | |
| | Rash | | | | |
| | Fever | | | | |
| Age (6-10) | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |
| | Fever | | | | |
| Age (11-18) | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |
| | Fever | | | | |
| Age (19-34) | Chills | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Chills, Nausea, Malaise, Myalgia, Arthralgia, Headache

<sup>\*</sup>None(1), Urticarial(2), Other(3): Rash

 $<sup>* \</sup>ge 38^{\circ}C(1)$ : Fever


THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| Safety Set | | 1* | 2* | 3* | Total |
|-------------|------------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |
| | Fever | | | | |
| Age (35-55) | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |
| | Fever | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Chills, Nausea, Malaise, Myalgia, Arthralgia, Headache, Change in eating habits, Sleepiness, irritability, vomiting, diarrhea,

<sup>\*</sup>None(1), Urticarial(2), Other(3): Rash

<sup>\*</sup>  $\geq$  38°C(1): Fever



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

Table 4.1.7 Summary of Solicited AE by day (<6 years)

| Safety Set | | 30 min | 6 | 6hr | | 2 | | 3 | | 4 | | 5 | | 6 | | 7 | Т | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (% |
| Local AE | Tenderness | | | | | | | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | | | | | | |
| | Sub Total | | | | | | | | | | | | | | | | | |
| C AE | Change in eating | | | | | | | | | | | | | | | | | |
| Systemic AE | Systemic AE habits | | | | | | | | | | | | | | | | | |
| | Sleepiness | | | | | | | | | | | | | | | | | |
| | Irritability | | | | | | | | | | | | | | | | | |
| | Vomiting | | | | | | | | | | | | | | | | | |
| | Diarrhea | | | | | | | | | | | | | | | | | |
| | Rash | | | | | | | | | | | | | | | | | |
| | Fever | | | | | | | | | | | | | | | | | |
| | Sub Total | | | | | | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | | | | | | |

Table 4.1.8 Summary of Solicited AE by day (≥6 years)

| Safety Set | | 30 | ) min | | 6hr | | 2 | | 3 | | 4 | | 5 | | 6 | | 7 | Т | `otal |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) |
| Local AE | Pain | | | | | | | | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | | | | | | | |
| | Sub Total | | | | | | | | | | | | | | | | | • | |
| Systemic AE | Chills | | | | | | | | | | | | | | | | | | |
| | Nausea | | | | | | | | | | | | | | | | | | |
| | Malaise | | | | | | | | | | | | | | | | | | |
| | Myalgia | | | | | | | | | | | | | | | | | | |
| | Arthralgia | | | | | | | | | | | | | | | | | | |
| | Headache | | | | | | | | | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| Sub Total |
|-----------|
| Rash |

Table 4.1.9 Summary of Solicited AE by day

| Safety Set | | 30 | ) min | | 6hr | | 2 | | 3 | | 4 | | 5 | | 6 | 7 | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n (%) | n%) |
| Age (2-5) | Tenderness | | | | | | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | | | | | |
| Age (6-10) | Pain | | | | | | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | | | | | |
| Age (11-18) | Pain | | | | | | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | | | | | |
| Age (19-34) | Pain | | | | | | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | | | | | |
| Age (35-55) | Pain | | | | | | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | | | | | |
| | Sub Total | | | | | | | | | | | | | | | | |
| Age (2-5) | Change in eating habits | | | | | | | | | | | | | | | | |
| | Sleepiness | | | | | | | | | | | | | | | | |
| | Irritability | | | | | | | | | | | | | | | | |
| | Vomiting | | | | | | | | | | | | | | | | |
| | Diarrhea | | | | | | | | | | | | | | | | |
| | Rash | | | | | | | | | | | | | | | * | |
| | Fever | | | | | | | | | | | | | | | | |
| Age (6-10) | Chills | | | | | | | | | | | | | | | | |
| | Nausea | | | | | | | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| Safety Set | | 30 min | 6hr | 2 | 3 | 4 | 5 | 6 | 7 | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| | | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n%) |
| | Malaise | | | | | | | | | |
| | Myalgia | | | | | | | | | |
| | Arthralgia | | | | | | | | | |
| | Headache | | | | | | | | | |
| | Rash | | | | | | | | | |
| | Fever | | | | | | | | | |
| Age (11-18) | Chills | | | | | | | | | |
| | Nausea | | | | | | | | | |
| | Malaise | | | | | | | | | |
| | Myalgia | | | | | | | | | |
| | Arthralgia | | | | | | | | | |
| | Headache | | | | | | | | | |
| | Rash | | | | | | | | | |
| | Fever | | | | | | | | | |
| Age(19-34) | Chills | | | | | | | | | |
| | Nausea | | | | | | | | | |
| | Malaise | | | | | | | | | |
| | Myalgia | | | | | | | | | |
| | Arthralgia | | | | | | | | | |
| | Headache | | | | | | | | | |
| | Rash | | | | | | | | | |
| | Fever | | | | | | | | | |
| Age (35-55) | Chills | | | | | | | | | *************************************** |
| | Nausea | | | | | | | | | |
| | Malaise | | | | | | | | | |
| | Myalgia | | | | | | | | | |
| | Arthralgia | | | | | | | | | |
| | Headache | | | | | | | | | |
| | Rash | | | | | • | | | | |
| | Fever | | | | | | | | | |
| | Sub Total | | <u> </u> | | <u> </u> | <u> </u> | | <u>.</u> | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

# STATISTICAL ANALYSIS PLAN(V3.0)

| Safety Set | 30 | min | | 6hr | | 2 | | 3 | | 4 | | 5 | | 6 | 7 | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n (%) | n%) |
| Total | | | | | | | | | | | | | | | | |

#### Table 4.1.10 Summary of Fever

| Safety Set | | 2- | 10 | 11 | -18 | 19 | -34 | 35 | -55 | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| | | n | (%) | n | (%) | n | (%) | n | (%) | n (%) |
| | Fever | | | | | | | | | |
| | No fever | | | | | | | | | |
| | Total | | | | | | | | | |
| Temperature(°C) | 36-36.5 | | | | | | | | | |
| | 36.5-37 | | | | | | | | | |
| | 37-37.5 | | | | | | | | | |
| | 37.5-38 | | | | | | | | | |
| | 38-38.5 | | | | | | | | | |
| | 38.5-39 | | | | | | | | | |
| | 39-39.5 | | | | | | | | | |
| | 39.5-40 | | | | | | | | | |
| | >40 | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

### STATISTICAL ANALYSIS PLAN(V3.0)

#### 4.2 Safety per protocol set

Table 4.2.1 Summary of local AE by Max severity (<6 years)

| Safety per prot | ocol Set | 1* | 2* | 3* | 4* | Total |
|-----------------|------------|-------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) | n (%) |
| Local AE | Tenderness | | | | | |
| | Erythema | | | | | |
| | Induration | | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Tenderness

Table 4.2.2 Summary of Local AE Max severity (≥6 years)

| Safety per protocol | Set | 1* | 2* | 3* | 4* | Total |
|---------------------|------------|-------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) | n (%) |
| Local AE | Pain | | | | | |
| | Erythema | | | | | |
| | Induration | | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Pain

Table 4.2.3 Summary of Local AE by Max severity

| Safety per pro | tocol Set | 1* | 2* | 3* | 4* | Total |
|----------------|------------|-------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) | n (%) |
| Age (2-5) | Tenderness | | | | | |
| | Erythema | | | | | |
| | Induration | | | | | |
| Age (6-10) | Pain | | | | | |
| | Erythema | | | | / | |
| | Induration | | | | | |
| Age (11-18) | Pain | | | | | |
| | Erythema | | | | | |
| | Induration | | | | | |
| Age (19-34) | Pain | | | | | |

<sup>\* 1-25(1), 26-50(2), 51-100(3), &</sup>gt;100(4): Erythema, Induration

<sup>\* 1-25(1), 26-50(2), 51-100(3), &</sup>gt;100(4): Erythema, Induration



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| | Erythema |
|-------------|------------|
| | Induration |
| Age (35-55) | Pain |
| | Erythema |
| | Induration |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Pain

Table 4.2.4 Summary of Systemic AE by Max severity (<6 years)

| Safety Set | | 1* | 2* | 3* | Total |
|-------------|-------------------------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) |
| Systemic AE | Change in eating habits | | | | |
| | Sleepiness | | | | |
| | Irritability | | | | |
| | Vomiting | | | | |
| | Diarrhea | | | | |
| | Rash | | | | |
| | Fever | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Change in eating habits, Sleepiness, irritability, vomiting, diarrhea,

Table 4.2.5 Summary of Systemic AEs by Max severity (≥6 years)

| Safety per proto | col Set | 1* | 2* | 3* | Total |
|------------------|------------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) |
| Systemic AE | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |
| | Fever | | | | |

 $<sup>*\</sup> Mild (1),\ Moderate (2),\ Severe (3): Chills,\ Nausea,\ Malaise,\ Myalgia,\ Arthralgia,\ Headache$ 

<sup>\* 1-25(1), 26-50(2), 51-100(3), &</sup>gt;100(4): Erythema, Induration

<sup>\*</sup>None(1), Urticarial(2), Other(3): Rash

<sup>\*</sup>  $\geq$  38°C(1) : Fever



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

# STATISTICAL ANALYSIS PLAN(V3.0)

\*None(1), Urticarial(2), Other(3): Rash

 $* \ge 38^{\circ}C(1)$ : Fever

Table 4.2.6 Summary of Systemic AE by Max severity

| Safety per protoc | col Set | 1* | 2* | 3* | Total |
|---|---|---|---|---|---|
| | | n (%) | n (%) | n (%) | n (%) |
| Age (2-5) | Change in eating habits | | | | |
| | Sleepiness | | | | |
| | Irritability | | | | |
| | Vomiting | | | | |
| | Diarrhea | | | | |
| | Rash | | | | |
| | Fever | | | | |
| Age (6-10) | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | # P P P P P P P P P P P P P P P P P P P | |
| | Fever | | | | |
| Age (11-18) | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |
| | Fever | | | | |
| Age (19-34) | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| Safety per proto | col Set | 1* | 2* | 3* | Total |
|------------------|------------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) |
| | Headache | | | | |
| | Rash | | | | |
| | Fever | | | | |
| Age (35-55) | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |
| | Fever | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Chills, Nausea, Malaise, Myalgia, Arthralgia, Headache

Table 4.1.7 Summary of Solicited AE by day (<6 years)

| Safety Set | | 30 | ) min | ( | 6hr | | 2 | | 3 | | 4 | | 5 | | 6 | | 7 | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n (%) |
| Local AE | Tenderness | | | | | | | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | | | | | | |
| | Sub Total | | | | | | | | | | | | | | | | | |
| Systemic AE | Change in eating habits | | | | | | | | | | | | | | | | | |
| | Sleepiness | | | | | | | | | | | | | | | | | |
| | Irritability | | | | | | | | | | | | | | | | | |
| | Vomiting | | | | | | | | | | | | | | | | | |
| | Diarrhea | | | | | | | | | | | | | | | | | |
| | Rash | | | | | | | | | | | | | | | | | |
| | Fever | | | | | | | | | | | | | | | | | |
| | Sub Total | | | | | | | | | <u> </u> | • | | | | | | | |
| Total | • | | | | | | | | | | | | | | | | | |

<sup>\*</sup>None(1), Urticarial(2), Other(3): Rash

 $<sup>* \</sup>ge 38^{\circ}C(1)$ : Fever



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

Table 4.2.8 Summary of Solicited AE by day (≥6 years)

| Safety per pro | tocol Set | 30 | ) min | | 6hr | | 2 | | 3 | | 4 | | 5 | | 6 | | 7 | Т | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) |
| Local AE | Pain | | | | | | | | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | | | | | | | |
| _ | Sub Total | | | | | | | | | | | | | | | | | | |
| Systemic AE | Chills | | | | | | | | | | | | | | | | | | |
| | Nausea | | | | | | | | | | | | | | | | | | |
| | Malaise | | | | | | | | | | | | | | | | | | |
| | Myalgia | | | | | | | | | | | | | | | | | | |
| | Arthralgia | | | | | | | | | | | | | | | | | | |
| | Headache | | | | | | | | | | | | | | | | | | |
| | Rash | | | | | | | | | | | | | | | | | | |
| | Fever | | | | | | | | | | | | | | | | | | |
| | Sub Total | | | | | | | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | | | | | | | |

Table 4.2.9 Summary of Solicited AE by day

| Safety Set | | 30 min | 6hr | 2 | 3 | 4 | 5 | 6 | 7 | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| | | n (%) n ( | %) n (%) n | (%) n (% | n (%) n (° | %) n (%) | | | | n (%) |
| Age (2-5) | Tenderness | | | | | | | | | |
| | Erythema | | | | | | | | | |
| | Induration | | | | | | | | | |
| Age (6-10) | Pain | | | | | | | | | |
| | Erythema | | | | | | | | | |
| | Induration | | | | | | | | | |
| Age (11-18) | Pain | | | | | | | | | |
| | Erythema | | | | | | | | | |
| | Induration | | | | | | | | | |
| Age (19-34) | Pain | | | | | | | | | |
| | Erythema | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| Safety Set | | 30 min | 6hr | 2 | 3 | 4 | 5 | 6 | 7 | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| | | n (%) n ( | %) n (%) r | ı (%) n (% | ) n (%) n ( <sup>6</sup> | %) n (%) | | | | n (%) |
| | Induration | | | | | | | | | |
| Age (35-55) | Pain | | | | | | | | | |
| | Erythema | | | | | | | | | |
| | Induration | | | | | | | | | |
| | Sub Total | | | | | | | | | |
| Age (2-5) | Change in eating habits | | | | | | | | | |
| | Sleepiness | | | | | | | | | |
| | Irritability | | | | | | | | | |
| | Vomiting | | | | | | | | | |
| | Diarrhea | | | | | | | | | |
| | Rash | | | | | | | | | |
| | Fever | | | | | | | | | |
| Age (6-10) | Chills | | | | | | | | | |
| | Nausea | | | | | | | | | |
| | Malaise | | | | | | | | | |
| | Myalgia | | | | | | | | | |
| | Arthralgia | | | | | | | | | |
| | Headache | | | | | | | | | |
| | Rash | | | | | | | | | |
| | Fever | | | | | | | | | |
| Age (11-18) | Chills | | | | | | | | | |
| | Nausea | | | | | | | | | |
| | Malaise | | | | | | | | | |
| | Myalgia | | | | | | | | | |
| | Arthralgia | | | | | | | | | |
| | Headache | | | | | | | | | |
| | Rash | | | | | | | | | |
| | Fever | | | | | | | | | |
| Age(19-34) | Chills | | | | | | | | | |
| | Nausea | | | | | | | | | |
| | Malaise | | | | | | | | | |




THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

| Safety Set | | 30 min | 6hr | 2 | 3 | 4 | 5 | 6 | 7 | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| | | n (%) n ( | %) n (%) r | ı (%) n (% | ) n (%) n ( | %) n (%) | | | | n (%) |
| | Myalgia | | | | | | | | | |
| | Arthralgia | | | | | | | | | |
| | Headache | | | | | | | | | |
| | Rash | | 5 | | | | | | | |
| | Fever | | | | | | | | | |
| Age (35-55) | Chills | | | | | | | | | |
| | Nausea | | | | | | | | | |
| | Malaise | | | | | | | | | |
| | Myalgia | | | | | | | | | |
| | Arthralgia | | | | | | | | | |
| | Headache | | | | | | | | | |
| | Rash | | | | | | | | | |
| | Fever | | | | | | | | | |
| | Sub Total | | | | | | | | | |
| Total | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

# STATISTICAL ANALYSIS PLAN(V3.0)

Table 4.2.10 Summary of Fever

| Safety per protocol Set | | 2 | -10 | 11- | 18 | 19- | -34 | 35 | -55 | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| | | n | (%) | n | (%) | n | (%) | n | (%) | n (%) |
| | Fever | | | | | | | | | |
| | No fever | | | | | | | | | |
| | Total | | | | | | | | | |
| Temperature(°C) | 36-36.5 | | | | | | | | | |
| | 36.5-37 | | | | | | | | | |
| | 37-37.5 | | | | | | | | | |
| | 37.5-38 | | | | | | | | | |
| | 38-38.5 | | | | | | | | | |
| | 38.5-39 | | | | | | | | | |
| | 39-39.5 | | | | | | | | | |
| | 39.5-40 | | | | | | | | | |
| | >40 | | | | | | | | | |

### 5. Unsolicited AE (DAY 1-7)

#### 5.1 Safety Set

Table 5.1 Summary of Unsolicited AE

| Safety Set | | 2- | 10 | 11 | -18 | 19 | -34 | 35 | -55 | To | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) |
| Expected | Expected AE | | | | | | | | | | |
| | Unexpected AE | | | | | | | | | | |
| Serious | Yes | | | | | | | | | | |
| | No | | | | | | | | | | |
| Severity | Mild | | | | | | | | | | |
| | Moderate | | | | | | | | | | |
| | Severe | | | | | | | | | | |
| Frequency | Single/Continuous | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| Safety Set | | 2- | 10 | 11 | -18 | 19 | -34 | 35 | -55 | То | tal |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) |
| | Intermittent | | | | | | | | | | |
| Action Taken | None | | | | | | | | | | |
| | Uncertain | | | | | | | | | | |
| | Procedure or physical | | | | | | | | | | |
| | therapy | | | | | | | | | | |
| | Blood or blood products | | | | | | | | | | |
| | Withdrawn from study due to AE | | | | | | | | | | |
| | Prescription drug therapy | | | | | | | | | | |
| | Non-prescription drug therapy | | | | | | | | | | |
| | Hospitalization | | | | | | | | | | |
| | IV fluids | | | | | | | | | | |
| | Physician visit | | | | | | | | | | |
| | Other | | | | | | | | | | |
| Outcome | Complete recovery/Return to baseline | | | | | | | | | | |
| | Alive with sequelae | | | | | | | | | | |
| | Death | | | | | | | | | | |
| | Unknown/Lost to follow-up | | | | | | | | | | |
| | AE persisting | | | | | | | | | | |
| Relationship | | | | | | | | | | | |
| to study | Not related | | | | | | | | | | |
| vaccine | | | | | | | | | | | |
| | Possibly related | | | | | | | | | | |
| | Probably related | | | | | | | | | | |
| Total | | | | | | | | | | | |




THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

# STATISTICAL ANALYSIS PLAN(V3.0)

#### 5.2 Safety per protocol set

Table 5.2 Summary of Unsolicited AE

| Safety per | | 2- | -10 | 11 | -18 | 19 | -34 | 35 | -55 | То | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|
| protocol Set | | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) |
| Expected | Expected AE | | | | | | | | | | |
| | Unexpected AE | | | | | | | | | | |
| Serious | Yes | | | | | | | | | | |
| | No | | | | | | | | | | |
| Severity | Mild | | | | | | | | | | |
| | Moderate | | | | | | | | | | |
| | Severe | | | | | | | | | | |
| Frequency | Single/Continuous | | | | | | | | | | |
| | Intermittent | | | | | | | | | | |
| Action Taken | None | | | | | | | | | | |
| | Uncertain | | | | | | | | | | |
| | Procedure or physical | | | | | | | | | | |
| | therapy | | | | | | | | | | |
| | Blood or blood products | | | | | | | | | | |
| | Withdrawn from study due to AE | | | | | | | | | | |
| | Prescription drug therapy | | | | | | | | | | |
| | Non-prescription drug therapy | | | | | | | | | | |
| | Hospitalization | | | | | | | | | | |
| | IV fluids | | | | | | | | | | |
| | Physician visit | | | | | | | | | | |
| | Other | | | | | | | | | | |
| Outcome | Complete recovery/Return to baseline | | | | | | | | | | |
| | Alive with sequelae | | | | | | | | | | |
| | Death | | | | | | | | | | |
| | Unknown/Lost to follow-up | | | | | | | | | | |
| | AE persisting | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| Safety per protocol Set | | 2- | 10 | 11 | -18 | 19 | -34 | 35 | -55 | То | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|
| r | | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) |
| Relationship<br>to study<br>vaccine | Not related Possibly related Probably related | | | | | | | | | | |
| Total | | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

# STATISTICAL ANALYSIS PLAN(V3.0)

### **6.** MAAE (DAY 1-29)

### 6.1 Safety Set

Table 6.1 Summary of MAAE

| Safety Set | | 2- | 10 | 11 | -18 | 19 | -34 | 35 | -55 | To | tal |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) |
| Expected | Expected AE | | | | | | | | | | |
| | Unexpected AE | | | | | | | | | | |
| Serious | Yes | | | | | | | | | | |
| | No | | | | | | | | | | |
| Severity | Mild | | | | | | | | | | |
| | Moderate | | | | | | | | | | |
| | Severe | | | | | | | | | | |
| Frequency | Single/Continuous | | | | | | | | | | |
| | Intermittent | | | | | | | | | | |
| Action<br>Taken | None | | | | | | | | | | |
| | Uncertain | | | | | | | | | | |
| | Procedure or physical | | | | | | | | | | |
| | therapy | | | | | | | | | | |
| | Blood or blood products | | | | | | | | | | |
| | Withdrawn from study due to AE | | | | | | | | | | |
| | Prescription drug therapy | | | | | | | | | | |
| | Non-prescription drug therapy | | | | | | | | | | |
| | Hospitalization | | | | | | | | | | |
| | IV fluids | | | | | | | | | | |
| | Physician visit | | | | | | | | | | |
| | Other | | | | | | | | | | |
| Outcome | Complete recovery/Return to baseline | | | | | | | | | | |
| | Alive with sequelae | | | | | | | | | | |
| | Death | | | | | | | | | | |
| | Unknown/Lost to follow-up | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

# STATISTICAL ANALYSIS PLAN(V3.0)

| Safety Set | | 2- | 10 | 11 | -18 | 19 | -34 | 35 | -55 | То | tal |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | No. | (0/) | No. | (0/) | No. | (0/) | No. | (0/) | No. | (0/) |
| | | AEs | (%) | AEs | (%) | AEs | (%) | AEs | (%) | AEs | (%) |
| | AE persisting | | | | | | | | | | |
| Relationshi | | | | | | | | | | | |
| p to study | Not related | | | | | | | | | | |
| vaccine | | | | | | | | | | | |
| | Possibly related | | | | | | | | | | |
| | Probably related | | | | | | | | | | |
| Total | | | | | | | | | | | |

### 6.2 Safety per protocol set

Table 6.2 Summary of MAAE

| Safety per protocol Set | | 2- | 10 | 11 | -18 | 19 | -34 | 35 | -55 | Тс | tal |
|---|---|---|---|---|---|---|---|---|---|---|---|
| protocor set | | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) |
| Expected | Expected AE Unexpected AE | | | | | | | | | | |
| Serious | Yes<br>No | | | | | | | | | | |
| Severity | Mild<br>Moderate<br>Severe | | | | | | | | | | |
| Frequency | Single/Continuous Intermittent | | | | | | | | | | |
| Action<br>Taken | None | | | | | | | | | | |
| | Uncertain Procedure or physical | | | | | | | | | | |
| | therapy Blood or blood products | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| Safety per protocol Set | | 2- | 10 | 11 | -18 | 19 | -34 | 35 | -55 | То | tal |
|---|---|---|---|---|---|---|---|---|---|---|---|
| protocor set | | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) |
| | Withdrawn from study due to AE | | | | | | | | | | |
| | Prescription drug therapy | | | | | | | | | | |
| | Non-prescription drug therapy | | | | | | | | | | |
| | Hospitalization | | | | | | | | | | |
| | IV fluids | | | | | | | | | | |
| | Physician visit | | | | | | | | | | |
| | Other | | | | | | | | | | |
| Outcome | Complete recovery/Return to baseline | | | | | | | | | | |
| | Alive with sequelae | | | | | | | | | | |
| | Death | | | | | | | | | | |
| | Unknown/Lost to follow-up | | | | | | | | | | |
| | AE persisting | | | | | | | | | | |
| Relationshi | | | | | | | | | | | |
| p to study | Not related | | | | | | | | | | |
| vaccine | | | | | | | | | | | |
| | Possibly related | | | | | | | | | | |
| | Probably related | | | | | | | | | | |
| Total | | | | | | | | | | | |

| | | Last Update Date |
|---|---|---|
| Clinical Investigation Services | THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS | 10-APR-2014 |
| | PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT | 1011112011 |
| | THE WRITTEN PERMISSION OF COMPANY. | |
| STATISTICA | AL ANALYSIS PLAN(V3.0) | |

### 7. SAE/SADR for 28 days after vaccination

### 7.1 Safety Set

Table 7.1 SAE and SADR

| | | 2- | 10 | | | 11 | -18 | | | 19 | -34 | | | 35 | -55 | | | То | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety Set | Serious | ΑE | Seriou<br>ADR | | Serious | AE | Seriou<br>ADR | | Serious | ΑE | Seriou<br>ADR | | Serious | ΑE | Seriou<br>ADR | | Serious | AE | Serio<br>ADF | |
| | | | | | | | | | | | | | | | | | | | | N |
| | | N | | N | | N | | N | | N | | N | | N | | N | | N | | О |
| | | o. | | 0. | | 0. | | 0. | | 0. | | 0. | | 0. | | О. | | О. | | |
| | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | О |
| | ce Rate | Α | ce Rate | A | ce Rate | A | ce Rate | A | ce Rate | A | ce Rate | Α | ce Rate | A | ce Rate | Α | ce Rate | A | ce Rate | f |
| | | Es | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | Α |
| | | | | S | | S | | S | | S | | S | | S | | S | | s | | Е |
| | | | | | | | | | | | | | | | | | | | | S |
| | ( | | ( | | ( | | ( | | ( | | ( | | ( | | ( | | ( | | ( | |
| | n % | n | n %<br>) | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n |
| System Organ Class(SOC) | | | | | | | | | | | - | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| | | 2- | 10 | | | 11 | -18 | | | 19 | -34 | | | 35 | -55 | | | То | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety Set | Serious | ΑE | Seriou<br>ADR | | Serious | ΑE | Serio<br>ADF | | Serious | ΑE | Seriou<br>ADR | | Serious | <b>Α</b> Ε | Seriou<br>ADR | | Serious | ΑE | Serior<br>ADF | |
| | Inciden ce Rate | N o. of A Es | Inciden<br>ce Rate | N<br>o.<br>of<br>A<br>E | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E s | Inciden<br>ce Rate | A<br>E | Inciden<br>ce Rate | N o. of A E | | | Inciden<br>ce Rate | N<br>o.<br>of<br>A<br>E | Inciden<br>ce Rate | | Inciden<br>ce Rate | |
| | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n |
| Preferred Term(PT) | | | | | | MAN (MANIMAN) I I I I I I I I I I I I I I I I I I I | | | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | | | | | | | | |



### 7.2 Safety per protocol set

Table 7.2 SAE and SADR

| | | 2- | 10 | | | 11 | -18 | | | 19 | -34 | | | 35 | -55 | | | То | tal | | _ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety per protocol Set | Serious | ΑE | Seriou<br>ADR | | Serious | ΑE | Seriou<br>ADR | | Serious | ΑE | Seriou<br>ADR | | Serious | ΑE | Seriou<br>ADR | | Serious | AE | | ous<br>DR | _ |
| | | | | | | | | | | | | | | | | | | | | N | 1 |
| | | | | N | | N | | N | | N | | N | | N | | N | | N | | o | , |
| | | N | | 0. | | 0. | | 0. | | o. | | o. | | o. | | o. | | o. | | | |
| | Inciden | 0. | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Incide | n o | ) |
| | ce Rate | of | ce Rate | Α | ce Rate | A | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Ra | ite f | f |
| | | A | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | A | L. |
| | | Es | | s | | s | | s | | S | | s | | s | | s | | s | | Е | į |
| | | | | | | | | | | | | | | | | | | | | s | i |
| | ( | | ( | | ( | | ( | | ( | | ( | | ( | | ( | | ( | | | ( | _ |
| | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n | % n | l |
| | ) | | ) | | ) | | ) | | ) | | ) | | ) | | ) | | ) | | | ) | _ |
| System Organ Class(SOC) | | | | | | | <u>.</u> | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| | | 2- | 10 | | | 11 | -18 | | | | 19 | -34 | | | 35 | -55 | | | То | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety per protocol Set | Serious | ΑE | Seriou<br>ADR | | Serious | AE | ļ | riou<br>ADR | | Serious | ΑE | Seriou<br>ADR | | Serious | ΑE | Seriou<br>ADR | | Serious | ΑE | Serio<br>ADI | |
| | Inciden ce Rate | N<br>o.<br>of<br>A<br>Es | Inciden<br>ce Rate | N<br>o.<br>of<br>A<br>E | Inciden<br>ce Rate | | Incid<br>ce Ra | | N o. of A E | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E | | N<br>o.<br>of<br>A<br>E | Inciden<br>ce Rate | N<br>o.<br>of<br>A<br>E | Inciden<br>ce Rate | | Inciden<br>ce Rate | |
| | n % | n | n % | n | n % | n | n | (<br>%<br>) | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n |
| Preferred Term(PT) | | | | | | | | | | | A CONTRACTOR OF THE PROPERTY O | | AND I ARREST COMMENTS OF THE THE STATE OF TH | | | | | | | | |
| Total | | | | | | | | | | | | | | | | | | | | | |



### 7.3 Non-Safety per protocol set

Table 7.3 SAE and SADR

| | | 2- | 10 | | | 11 | -18 | | | 19 | -34 | | | 35 | -55 | | | To | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non- Safety per protocol<br>Set | Serious | ΑE | Seriou<br>ADR | | Serious | ΑE | Seriou<br>ADR | | Serious | ΑE | Seriou<br>ADR | | Serious | ΑE | Seriou<br>ADR | | Serious | ΑE | Serio<br>ADI | |
| | Inciden<br>ce Rate | N o. of A Es | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | | Inciden<br>ce Rate | N<br>o.<br>of<br>A<br>E | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o o f A E |
| | n % | n | n % | n | n % | n | n % | n | (<br>n % | n | n % | n | n % | n | n % | n | n % | n | n % | s n |
| System Organ Class(SOC) | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| - | | 2- | 10 | | | 11 | -18 | | | 19 | -34 | | | 35 | -55 | | | То | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non- Safety per protocol<br>Set | Serious | ΑE | Seriou<br>ADR | | Serious | ΑE | Serio<br>AD | | Serious | ΑE | Seriou<br>ADR | | Serious | <b>Α</b> Ε | Seriou<br>ADR | | Serious | ΑE | Serio<br>ADF | |
| | Inciden<br>ce Rate | N<br>o.<br>of<br>A<br>Es | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E s | | | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | |
| | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n |
| Preferred Term(PT) | | | | | | | | | | WIND IN THE STATE OF THE STATE | | | | | | | | | | |
| Total | | | | | | | | | | | | | | | | | | | | |

| | | Last Update Date |
|---|---|---|
| Proper CTC | CONFIDENTIAL: | |
| DreamCIS Inc. Clinical Investigation Services | THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS | 10-APR-2014 |
| | PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT | 10 / 11 10 2011 |
| | THE WRITTEN PERMISSION OF COMPANY. | |
| STATISTICA | L ANALYSIS PLAN(V3.0) | |

### 8. Unexpected AE/ADR for 28 days after vaccination

### 8.1 Safety Set

Table 8.1 Unexpected AE and ADR

Safety Set

| | 2-1 | 10 | | | 11. | 18 | | | 19 | -34 | | | 35- | -55 | | | Tot | al | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Unexpec | eted | Unexped | eted | Unexped | ted | Unexpec | eted | Unexped | eted | Unexped | eted | Unexped | eted | Unexped | eted | Unexped | eted | Unexped | ete |
| AE | | ADR | | AE | | ADR | - | AE | | ADR | - | AE | | ADR | | AE | | d ADR | t |
| | | | | | | | | | | | | | | | | | | | N |
| | N | | N | | N | | N | | N | | N | | N | | N | | N | | o |
| | 0. | | О. | | О. | | o. | | 0. | | o. | | 0. | | o. | | 0. | | • |
| Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Incide | of | Incider | 10 |
| ce Rate | A | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | f |
| | Es | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | A |
| | LS | | S | | s | | S | | s | | s | | s | | s | | s | | Е |
| | | | | | | | | | | | | | | | | | | | S |

<sup>\*</sup> MedDRA

| 0 | DreamCIS Inc. |
|------|---------------------------------|
| (III | Clinical Investigation Services |

THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| | n | (<br>% | n | n | (<br>%<br>) | n | n | (<br>%<br>) | n | n | (<br>%<br>) | n | n | (<br>%<br>) | n | n | (<br>%<br>) | n | n | (<br>%<br>) | n | n | (<br>%<br>) | n | n | (<br>%<br>) | n | n | (<br>%<br>) | n |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class(SOC) | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Preferred Term(PT) | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA

| | | Last Update Date |
|---|---|---|
| DreamCIS Inc. Clinical Investigation Services | CONFIDENTIAL: THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT | 10-APR-2014 |
| | THE WRITTEN PERMISSION OF COMPANY. | |
| | T ANIAT MOTO DE ANIAMA | |

# STATISTICAL ANALYSIS PLAN(V3.0)

### 8.2 Safety per protocol set

Table 8.2 Unexpected AE and ADR

| | | | 2- | 10 | | | | | 11- | -18 | | | | | 19- | -34 | | | 35 | -55 | | | | Tot | al | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Un | expe | eted | Un | expec | ted | Une | xpec | ted | Un | expec | ted | Unex | pect | ted | Unexpe | cted | Unexpe | ected | Unexpe | ected | Un | expec | ted | Unex | secte |
| Safety per protocol Set | | AE | | | ADR | | | AE | | | ADR | | A | E | | ADF | 1 | AE | , | AD | R | | AE | | d A | OR |
| | | | | | | N | | | <b>N</b> T | | | NT | | | NI | | NT | | NI | | N | | | NI | | N |
| | | | N | | | 0. | | | N | | | N | | | N | | N | | N | | N | | | N | | О |
| | Inc | iden | 0. | Inci | den | o.<br>of | Incid | den | o.<br>of | Inc | iden | o.<br>of | Incide | n | o.<br>of | Inciden | o.<br>of | Inciden | o. | Inciden | o.<br>of | Iı | ncider | 0. | · Inci | den o |
| | | Rate | of | | Rate | A | ce R | | | ce I | | A | ce Ra | | | ce Rate | A | ce Rate | | | | | Rate | A | ce Ra | |
| | | | of | | Е | | | Е | | | Е | | | Е | | Е | | Е | | Е | | | Е | | Α | |
| | | | ate ce l | | S | | | S | | | s | | | s | | S | | s | | s | | | S | | Е | |
| | | Es | | | | | | | | | | | | | | | | | | | | | | | S | |
| | | ( | | | ( | | | ( | | | ( | | | ( | | ( | | ( | | ( | | | ( | | | |
| | n | % | n | n | % | n | n | % | n | n | % | n | n <sup>0</sup> | 6 | n | n % | n | n % | n | n % | n | n | % | n | n % | 6 n |
| | | ) | | | ) | | | ) | | | ) | | | ) | | ) | | ) | | ) | | | ) | | | |
| System Organ Class(SOC) | | | | | | | | | | ! | | | | | | | | | | 1 | | | | | | |
| Preferred Term(PT) | | | | | | | | | | | | | | | | | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| | | | 2- | 10 | | | | | 11- | -18 | | | | 19 | -34 | | | | 35- | -55 | | | To | al | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Un | expe | cted | Un | expe | eted | Unex | pecte | ed | Unexp | ected | U | nexpec | eted | Unexp | ected | Une | expec | eted | Unexpe | eted | Unexpe | eted | Unex | pecte |
| Safety per protocol Set | | AE | | | ADR | | I | ΛE , | | AD | R | | AE | | AD | R | | AE | | ADR | | AE | 1 | d A | .DR |
| | | iden<br>Rate | N o. of A Es | : | iden<br>Rate | N o. of A | Incid-<br>ce Ra | en de | | Inciden | | | ciden<br>Rate | | Incider | | | | | Inciden<br>ce Rate | N o. of A E | Incide<br>ce Rate | | f Inc | N o iden o ate f A |
| | | | | | S | | | S | | S | | | S | | S | | | S | | S | | S | | E<br>s | |
| | | ( | | | ( | | | ( | | ( | | | ( | | ( | | | ( | | ( | | ( | | | ( |
| | n | % | n | n | % | n | n | % | n | n % | n | n | % | n | n % | n | n | % | n | n % | n | n % | n | n | % n |
| | | ) | | | ) | | | ) | | ) | | | ) | | ) | | | ) | | ) | | ) | | | ) |
| Total | | | | | | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

# STATISTICAL ANALYSIS PLAN(V3.0)

### 8.3 Non-Safety per protocol set

Table 8.3 Unexpected AE and ADR

| | | | 2-1 | 10 | | | 11 | -18 | | | | | 19- | 34 | | | 35 | -55 | | | To | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non-Safety per protocol | Un | expe | eted | Unexp | ected | Unex | pected | Uı | nexpec | ted | Unex | ecte | d | Unexpec | ted | Unexpec | ted | Unexpe | eted | Unexpe | eted | Unex | ecte |
| Set | | AE | | AD | R | A | Æ | | ADR | | A | Е | | ADR | | AE | | ADR | _ | AE | | d Al | OR |
| | | of | | Inciden<br>ce Rate | | Incide<br>ce Ra | | | ciden<br>Rate | N o. of A E | Incide ce Rat | n o | | Inciden<br>ce Rate | N o. of A E | Inciden ce Rate | | Inciden<br>ce Rate | N o. of | Incider<br>ce Rate | | f Incid | A |
| | | | | | S | | S | | | S | | | S | | S | | S | | S | | S | | E |
| | | ( | | ( | | | ( | - | ( | | | | | ( | | ( | | ( | | ( | | ( | |
| | n | % | n | n % | n | n 9 | ⁄o n | n | % | n | n % | 6 I | n | n % | n | n % | n | n % | n | n % | n | n % | 'n |
| | | ) | | ) | | | ) | | ) | | | | | ) | | ) | | ) | | ) | | ) | |
| System Organ Class(SOC) | 1 | | | | | | | • | | | | į | - { | | | | | | | | | | |
| Preferred Term(PT) | | | | | | | | | | | | | | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| | | | 2- | 10 | | | | | 11- | 18 | | | | | 19- | -34 | | | 35 | -55 | | | To | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non-Safety per protocol | Un | expe | cted | Un | expe | eted | Une | xpec | ted | Une | xpec | eted | Unex | xpec | ted | Unexpe | cted | Unexpo | ected | Unexpe | cted | Unexpe | cted | Unex | pecte |
| Set | | AE | 1 | ļ | ADR | | | AE , | | A | ADR | | 1 | AE , | | ADI | ξ | AE | , | ADI | R | AE | 1 | d A | DR |
| | | iden<br>Rate | N o. of A Es | | iden<br>Rate | N<br>o.<br>of<br>A<br>E | Incid<br>ce R | | | Incid<br>ce R | | N o. of A E s | Incid<br>ce Ra | | | Inciden<br>ce Rate | | Inciden<br>ce Rate | | Inciden<br>ce Rate | | Incide<br>ce Rate | | f Inc | N o c iden o A E |
| | | ( | | | ( | | | ( | | | ( | | | ( | | ( | | ( | | . ( | | ( | | | ( s |
| | n | % | n | n | % | n | n | % | n | n | % | n | n | % | n | n % | n | n % | n | n % | n | n % | n | n | % n |
| | | ) | | | ) | | | ) | | | ) | | | ) | | ) | | ) | | ) | | ) | | | ) |
| Total | | | | | | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA

| | | Last Update Date |
|---|---|---|
| Clinical Investigation Services | THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT | 10-APR-2014 |
| | THE WRITTEN PERMISSION OF COMPANY. | |
| | I ANIAT VICTO DI ANIATO O | |

# STATISTICAL ANALYSIS PLAN(V3.0)

### 9. MAAE/ADR for 28 days after vaccination

### 9.1 Safety Set

Table 9.1 MAAE and ADR

| | | 2- | 10 | | | 11 | -18 | | | | 19 | -34 | | | 35 | -55 | | | Tot | al | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety Set | MAAl | Ξ | ADR | | MAA | Е | | ADR | | MAA | Е | ADR | 2 | MAA | Е | ADR | - | MAA | Е | AD | R |
| | Inciden<br>ce Rate | N o. of A Es | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | | Inci<br>ce R | | N o. of A E s | Inciden<br>ce Rate | N o. of E | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | N o. of A E | Incider<br>ce Rate | | Incid<br>ce Rat | N o |
| | (% | | ( | | ( | | | ( | | ( | | ( | | ( | | ( | | ( | | ( | |
| | n ) | n | n %<br>) | n | n % | n | n | % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | ó n |
| System Organ Class(SOC) Preferred Term(PT) | THE PERSON NAMED IN COLUMN NAM | | | | | | | | | | | | | | | | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| | | | 2-1 | 0 | | | 11 | -18 | | | 19 | -34 | | | 35 | -55 | Total | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety Set | MAAI | | 3 | ADR | | MAA | E | ADR | | MAAE | | ADR | | MAAE | | ADR | | MAAE | | ADR | |
| | Inci<br>ce F | den<br>Rate | of | Inciden | | | | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E | Incider<br>ce Rate | | f Incide<br>ce Rate | |
| | n | (% | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n |
| Total | | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

# STATISTICAL ANALYSIS PLAN(V3.0)

### 9.2 Safety per protocol set

Table 9.2 MAAE and ADR

| | 2-10 | | | | | | -18 | | -34 | | 35 | -55 | | | tal | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety per protocol Set | | MAAE | | ADR | | MAA | Е | ADF | 2 | MAA | Е | ADR | | MAAl | Е | ADR | | MAA | Е | ADR | |
| | | | | | | | | | | | | | | | | | | | | | N |
| | | | N | | N | | N | | N | | N | | N | | N | | N | | N | | o |
| | | | 0. | | o. | | 0. | | o. | | 0. | | o. | | o. | | 0. | | o. | | |
| | Inc | iden | o.<br>of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | of | Inciden | o |
| | ce | ce Rate | | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | Α | ce Rate | f |
| | | | A<br>Es | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | Α |
| | | | La | | s | | s | | s | | s | | s | | s | | s | | s | | Е |
| | | | | | | | | | | | | | | | | : | | | | | s |
| | | (% | | ( | | ( | | ( | | ( | | ( | | ( | | ( | | ( | | ( | |
| | n | (,0 | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n |
| . <u> </u> | | , | | ) | | ) | | ) | | ) | | ) | | ) | | ) | | ) | | ) | |
| System Organ Class(SOC) | | | | | | | | | | | | | | | | | | | | | |
| Preferred Term(PT) | | | | | | | | | | | | | | V. | | | | , | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

| | | | 2-1 | 0 | | -18 | | | | -34 | 35-55 | | | | | Total | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety per protocol Set | MAAE | | E | ADR | | MAA | E | A | ADR | | MAAE | | ADR | | MAAE | | [4] | ADR | | MAAE | | E ADR | | _ |
| | | iden<br>Rate | N o. of A | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | | Incide<br>ce Ra | | f<br>£ | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E | Incid<br>ce Ra | | | Inciden<br>ce Rate | N o. of A E s | Incider<br>ce Rat | | f Ir | ociden<br>e Rate | |
| | | | | | | | | | | | | | | | | | | | | | | | | s |
| | | (% | | ( | | ( | | | ( | | ( | | ( | | | ( | | ( | | ( | | | ( | |
| | n | ) | n | n % | n | n % | n | n | % n | 1 | n % | n | n % | n | n | % | n | n % | n | n % | n | n | % | n |
| | | | | ) | | ) | | | ) | | ) | | ) | | | ) | | ) | | ) | | | ) | |
| Total | | | | | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

# STATISTICAL ANALYSIS PLAN(V3.0)

### 9.3 Non-Safety per protocol set

Table 9.3 MAAE and ADR

| | | 2-10 | | | | | | 11 | -18 | | | | 19 | -34 | | | 35 | -55 | | | Tot | al | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non- Safety per protocol<br>Set | MAAE | | ADR | | MAAE | | | ADR | | MAAE | | ADR | | MAAE | | ADR | | MAAE | | ADR | | | |
| | | iden<br>Rate | N o. of A Es | | iden<br>Rate | N o. of A E | Incider | | | ciden<br>Rate | N o. of A E | Inciden<br>ce Rate | | Inciden<br>ce Rate | | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E s | Incide<br>ce Rate | | Incide<br>ce Rate | |
| | n | (% | n | n | 0/0 | n | n % | n | n | (<br>%<br>) | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n |
| System Organ Class(SOC) Preferred Term(PT) | | | | | | | | 10 1 | | | | | THE COLUMN TO THE PARTY OF THE | | | | | | | | | | |


THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

# STATISTICAL ANALYSIS PLAN(V3.0)

| | | | 2-1 | 0 | | | | 11- | -18 | | | | 19 | -34 | | | 35 | -55 | | | Tot | al | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non- Safety per protocol<br>Set | ı | MAAI | E | A | ADR | | MAA | E | AI | OR | | MAAE | Ξ | ADR | | MAA | E | ADR | | MAA | Ε | ADR | |
| | | iden<br>Rate | N<br>o.<br>of<br>A<br>Es | Incic<br>ce R | | N o. of A E | | | Incide<br>ce Rat | | f | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E | Inciden ce Rate | | Inciden<br>ce Rate | N o. of A E s | Incider<br>ce Rate | | f Incide | f<br>A<br>E |
| | n | (%) | n n | n | % | n | n % | n | n % | 60 n | | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n |
| Total | | | | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

STATISTICAL ANALYSIS PLAN(V3.0)

#### 10. AE/ADR for 28 days after vaccination

### 10.1 Safety Set

Table 10.1 AE and ADR

| | | 2-1 | 0 | | | 11 | -18 | | | 19 | -34 | | | 35 | -55 | | | To | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety Set | AE | | ADR | - | AE | | ADR | - | AE | | ADR | - | AE | | ADR | _ | AE | | ADR | - |
| | Inciden<br>ce Rate | N<br>o.<br>of<br>A<br>Es | Inciden<br>ce Rate | | Inciden<br>ce Rate | | Inciden<br>ce Rate | N<br>o.<br>of<br>A<br>E | | | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E s | Inciden<br>ce Rate | | Inciden<br>ce Rate | f |
| | n (% | n | n% | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n |
| System Organ Class(SOC) | | | | | | | | | | | | | | | : | | | | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

# STATISTICAL ANALYSIS PLAN(V3.0)

| | | 2-1 | .0 | | | | 11- | -18 | | | | | 19- | -34 | | | | 35- | .55 | | | | To | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety Set | AE | | A | DR | | AE | | | ADR | - | | AE | | AD | ₹ | | ΑE | | AI | )R | | AE | | AD | R |
| Preferred Term(PT) | AE iden Rate | N o. of A Es | Incid | N o. of the A E s | Inc | ciden Rate | | Inci | den | N o. of A E s | Incid<br>ce R | den | A<br>E<br>s | Inciden ce Rate | N o. of A E s | Incid<br>ce R | len | | Incide ce Rat | n ( | N o. of A E s | Inciden ce Rate ( n % ) | ************************************** | Incider<br>ce Rate | N o o o f f e E s |
| Total | | | | | | | | | | | | | | | | | | | | | | | | | |



# STATISTICAL ANALYSIS PLAN(V3.0)

### 10.2 Safety per protocol Set

Table 10.2 AE and ADR

| | | 2-1 | .0 | | | 11 | -18 | | | 19 | -34 | | | 35 | -55 | | | То | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety per protocol Set | AE | | ADR | | AE | | ADR | = | AE | | ADR | | AE | | ADR | - | AE | | Al | OR |
| | Inciden<br>ce Rate | N o. of A | Inciden<br>ce Rate | N<br>o.<br>of<br>A | Inciden<br>ce Rate | | Inciden<br>ce Rate | | | | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | | Incid<br>ce Ra | te f |
| | | Es | | S | | S | | S | | S | | S | | S | | S | | S | | A<br>E<br>s |
| | n (% | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n | ( n<br>% n |
| System Organ Class(SOC) | | | | | | | : | | | | | | | | : | | | | | |

<sup>\*</sup> MedDRA



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

# STATISTICAL ANALYSIS PLAN(V3.0)

| | | | 2-1 | .0 | | | | 11- | -18 | | | | | 19- | -34 | | | 35 | -55 | | | To | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety per protocol Set | | AE | | Al | DR | | AE | | A | ADR | | | ΑE | | ADI | ι | AE | | ADR | 1 | AE | | ADR | <b>\</b> |
| | | iden<br>Rate | N<br>o.<br>of<br>A<br>Es | Incide<br>ce Rat | N o. on of the A E s | Incid<br>ce R | den | | Incid<br>ce R | | N o. of A E s | Incid<br>ce Ra | | | Inciden<br>ce Rate | N o. of A E s | Inciden<br>ce Rate | N o. | Inciden<br>ce Rate | N o. of A E s | Inciden<br>ce Rate | | Inciden<br>ce Rate | f |
| | n | (%<br>) | n | n % | | n | % | n | n | %<br>) | n | n | % | n | n % | n | n % | n | n % | n | n % | n | n % | n |
| Preferred Term(PT) | | | | | | | | | | | | | | | | | | | | | | | | All the second s |
| Total | | | | | | | | | | | | | | | | | | | | | | | | |



### \* MedDRA

### 10.3 Non-Safety per protocol Set

Table 10.3 AE and ADR

| | | 2-1 | .0 | | | 11 | -18 | | | 19 | -34 | | | 35 | -55 | | | Tot | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non-Safety per protocol Set | AE | | ADR | | AE | | ADR | = | AE | | ADR | | AE | | ADR | | AE | | AD | R |
| | Inciden<br>ce Rate | N<br>o.<br>of<br>A<br>Es | Inciden<br>ce Rate | N o. of A E | Inciden ce Rate | | Inciden<br>ce Rate | | | | Inciden<br>ce Rate | N o. of A E | Inciden<br>ce Rate | | Inciden<br>ce Rate | N<br>o.<br>of<br>A<br>E | Inciden ce Rate | | Incide<br>ce Rat | f<br>A<br>E |
| | n (% | n | n% | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | ó m |
| System Organ Class(SOC) | | | | | | | :<br>! | | | | : | | | | | | | | | = |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

10-APR-2014

Last Update Date

# STATISTICAL ANALYSIS PLAN(V3.0)

| | | 2-1 | 0 | | | | | 11- | -18 | | | | 19 | -34 | | | | 35 | -55 | | | | Tot | tal | | _ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non-Safety per protocol Set | AE | | | ADR | | | ΑE | | | ADR | | AF | | A | DR | | AE | | AE | R | | AE | | Α | DR | |
| Preferred Term(PT) | iden<br>Rate<br>(% | N o. of A Es | ce I | iden<br>Rate | N o. of A E s | Incid<br>ce R | | | Inci<br>ce R | | N o. of A E s | Inciden<br>ce Rate | 1 | Incide<br>ce Ra | en te | N o. of A E s | Inciden ce Rate ( n % ) | | Incider<br>ce Rate<br>(<br>n % | E s | In ce | ciden<br>Rate | 1 | Incid<br>ce R | den<br>.ate | N o f A E s |
| Total | | | | | | | | | | | | | | | | | | | | | | | AMALIAN AND A | | | |

| | | Last Update Date |
|---|---|---|
| Clinical Investigation Services | THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS | 10-APR-2014 |
| | PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT | 10 7H K 2011 |
| | THE WRITTEN PERMISSION OF COMPANY. | |
| STATISTICA | L ANALYSIS PLAN(V3.0) | |

\* MedDRA

### V59\_62\_SAP(V3.0) Revisions

| Indication Revision | SAP (V2.0) | SAP (V3.0) | Reason for change |
|---|---|---|---|
| Appendix 1 Table 2.1.1, Table 2.1.3 Table 2.2.1, Table 2.2.3 | | Add ADR | Reflected by NVD Korea comments |
| Appendix 1 Table $3.1.1 \sim \text{Table } 3.1.3$ Table $3.2.1 \sim \text{Table } 3.2.3$ Table $4.1.4 \sim \text{Table } 4.1.9$ Table $4.2.4 \sim \text{Table } 4.2.9$ | | Add Fever | Reflected by NVD Korea comments |
| Appendix 1 Table 10.1 ~ Table 10.3 | | Add AE/ADR Table | Reflected by NVD Korea comments |



# STATISTICAL ANALYSIS PLAN

A Multicenter Post Marketing Surveillance Study to Monitor the Safety of GSK Meningococcal ACWY Conjugate Vaccine (MenACWY-CRM) Administered According to the Prescribing Information to Healthy Subjects from 2 months to 55 Years of Age in the Republic of South Korea

Product Name: Menveo (MenACWY-CRM)

Protocol No. : V59 62

Version : V4.0

**Effective Date** : 2016-01-29

| | | Last Update Date |
|---|---|---|
| dreamc1s | CONFIDENTIAL: THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY. | 26-JAN-2016 |
| STATISTICA | L ANALYSIS PLAN(V4.0) | |

### **Approvals**





THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

26-JAN-2016

Last Update Date

# STATISTICAL ANALYSIS PLAN(V4.0)

### Revisions

| DATE OF<br>REVISION | INDICATION REVISION | REASON FOR CHANGE | AUTHOR<br>NAME |
|---|---|---|---|
| 22-NOV-2013 | All | Protocol Amendment | PPD |
| 10-APR-2014 | Appendix1 | Modification of tables to include incidence rate of ADR, Fever added to Solicited reaction | PPD |
| 26-JAN-2016 | All | Protocol Amendment | PPD |

THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

26-JAN-2016

Last Update Date

# STATISTICAL ANALYSIS PLAN(V4.0)

### **Table of Contents**

| Revisions | 3 |
|--------------------------------------------------|----|
| 1. Study Objective | 6 |
| 2. Study Method and Study Period | 6 |
| 2.1 Study Period | 6 |
| 2.2 Number of Subjects | 6 |
| 2.3 Study population | 6 |
| 2.3.1 Inclusion criteria | 6 |
| 2.3.2 Exclusion criteria | 7 |
| 2.4 Study Method | 7 |
| 3. Analysis Sets | 10 |
| 3.1 Safety Analysis Sets | 10 |
| 3.2 Efficacy Analysis Set | 12 |
| 4. Endpoints | 12 |
| 4.1 Safety Endpoints | 12 |
| 5. Assessment Criteria | 12 |
| 5.1 Safety Assessment Criteria | 12 |
| 6. Statistical Analyses | 13 |
| 6.1 Baseline Characteristics | 13 |
| 6.2 Safety Analyses | 13 |
| 6.2.1 Adverse Events by Baseline Characteristics | 13 |
| 6.2.2. Analysis of Solicited AE | 14 |
| 6.2.3 Analysis of Unsolicited AE | 15 |
| 7. List of Table and Data Listings | 16 |
| 7.1 Distribution of Subjects | 16 |
| 7.2 Baseline Characteristics | 16 |
| 7.3 Safety Analyses | 17 |





THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

26-JAN-2016

Last Update Date

STATISTICAL ANALYSIS PLAN(V4.0)

#### 1. Study Objective

The primary objective of the study is to monitor the safety of a single dose of MenACWY-CRM vaccine in subjects from 2 months to 55 years of age, as evaluated by:

- Local and systemic solicited adverse events reported from study Day 1 (day of vaccination) through study Day 7 post-vaccination.
- All unsolicited Adverse Events (AEs) reported from study Day 1 (day of vaccination) through study Day 7 post-vaccination.
- Medically attended Adverse Events reported from study Day 1 to study termination (Day 29/early termination).
- All Serious Adverse Events (SAEs) reported from study Day 1 to study termination (Day 29/early termination).

#### 2. Study Method and Study Period

#### 2.1 Study Period

The trial period shall be from market launch date till approximately 22 May 2018.

#### 2.2 Number of Subjects

A total of approximately 3,960 subjects are planned for enrolment into this study.

Assuming a 10% drop-out rate, this should provide approximately 3,000 evaluable subjects in the cohort 2 to 55 years of age and 600 in the cohort 2 to 23 months of age. This sample size meets the post-licensure requirements of the MFDS to provide continued safety monitoring in the Korean population.

#### 2.3 Study population

#### 2.3.1 Inclusion criteria

Individuals eligible for enrolment in this study are those:



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

26-JAN-2016

Last Update Date

### STATISTICAL ANALYSIS PLAN(V4.0)

- 1. Male and female subjects from 2 months to 55 years of the age at the time of vaccination (including all 55 years of age subjects, up to one day before their 56<sup>th</sup> year birthday), who are scheduled to receive vaccination with MenACWY-CRM conjugate vaccine, according to the local prescribing information and routine clinical practice
- 2. To whom the nature of the study has been described and the subject or subject's parent/legal representative has provided written informed consent (written assent from minors should be also obtained if required by the relevant IRB);
- 3. Whom the investigator believes that the subject can and will comply with the requirements of the protocol (e.g., completion of the Diary Card);
- 4. Who are in good health as determined by the outcome of medical history, physical assessment and clinical judgment of the investigator

#### 2.3.2 Exclusion criteria

- 1. Contraindication, special warnings and/or precautions, as evaluated by the investigators, reported in the MenACWY-CRM conjugate vaccine Korean prescribing information.
- 2. Infants who were already enrolled in this trial for previous vaccination.

#### 2.4 Study Method

In order to obtain information on Regulatory PMS data after-market launch, or delegate will create the Regulatory PMS contract with the relevant clinics/hospitals and the physician in charge of the survey shall implement this Regulatory PMS in subjects that receive MenACWY-CRM in the relevant hospital/clinic since the contract date until the number of contracted survey cases, without omission, is reached.

#### Overview of Study Design

This is a multicenter post marketing surveillance study to monitor the safety of MenACWY-CRM administered according to the prescribing information to 3,960 healthy subjects from 2 months to 55 years of age in Korea.

Subjects will be enrolled at the time of their visit to a participating clinic or hospital for vaccination with MenACWY-CRM according to the routine clinical care.



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

26-JAN-2016

Last Update Date

### STATISTICAL ANALYSIS PLAN(V4.0)

At Visit 1 (Day 1), after obtaining consent from the subjects or subjects' parents/legal representative (and Assent Form, if required by the relevant IRB), the vaccination will be administered. Subjects will remain under observation for at least 30 minutes in the clinic after study immunization.

The subjects or subject's parent/legal representative will be then instructed to complete the Diary Card daily, reporting local and systemic adverse events and all other AEs occurring within 7 days following immunizations, and medically attended AEs or SAEs occurring up to Day 29 within the surveillance period after each study vaccination.

Subjects will also be instructed to return the completed diaries to the study site at Day 29 as follows:

- During a visit at the study center or
- Using the provided pre-addressed stamped envelope (PASE).

At the investigator discretion, the subject or subject's parent/legal representative will be reminded of the date of the study termination by a phone call at Day 29. If any clarification is required after Diary Card retrieval the site staff will follow up by phone, and any additional finding will be recorded on the subject's medical record.

In case the Diary Card is not retrieved within 10 days after Day 29, subject or subject's parent/legal representative will be contacted by phone to assess the occurrence of adverse events, determine the subject's clinical status and complete study termination. All information will be recorded by the site staff on the subject's medical record and collected in the appropriate section of the CRF.

All SAEs will be monitored until resolution and/or the cause is identified. If a SAE remains unresolved at study termination, a clinical assessment will be made by the investigator and the GSK regional physician to determine whether continued follow up of the SAE is needed.

Table 3.1-1: Safety Assessment Table

| Medical History: | From birth, collected at clinic visit |
|---|---|
| All significant past diagnoses including all allergies, major | Day 1 |
| surgeries requiring inpatient hospitalization, other significant | |
| injuries or hospitalizations, any conditions requiring | |
| prescription or chronic medication (i.e., >2 weeks in duration), | |
| or other significant medical conditions based on the | |
| investigator's judgment. | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

26-JAN-2016

Last Update Date

# STATISTICAL ANALYSIS PLAN(V4.0)

| Immediate reactions: | For at least 30 minutes after |
|---|---|
| Subjects will be assessed for immediate hypersensitivity | vaccination |
| reactions. | |
| Solicited local adverse events: | Days 1-7 after vaccination |
| < 6 years : injection site erythema, injection site induration, | |
| injection site tenderness | |
| $\geq$ 6 years : injection site erythema, injection site induration, | |
| injection site pain | |
| Solicited systemic adverse events: | Days 1-7 after vaccination |
| < 6 years : change in eating habits, sleepiness, irritability, rash, | |
| vomiting, diarrhea, fever | |
| ≥ 6 years : chills, nausea, malaise, generalized myalgia, | |
| generalized arthralgia, headache, rash, fever | |
| All unsolicited AEs will be collected | Days 1-7 after vaccination |
| Medically attended Adverse Events: From Day 1 to study termin | |
| Events that require a physician's visit or an emergency room | (Day 29/early termination) |
| visit (events that are managed by telephone or means other than | |
| a face-to-face evaluation by a clinician do not qualify as | |
| medically attended AEs). | |
| Serious AEs: | From Day 1 to study termination |
| All SAEs will be collected. | (Day 29/early termination) |
| Medications: | From Day 1 to Day 7 |
| Any medications used to treat any solicited local and systemic | |
| reaction and unsolicited AE be collected. | |
| Medications: | From Day 1 to study termination |
| Any medications used to treat any medically attended AE or | (Day 29/early termination) |
| SAE will be collected. | |

| | CONFIDENTIAL: |
|------------|-----------------------------------------------------------|
| dreamcis | THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS |
| or comicio | PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT |
| | THE WRITTEN PERMISSION OF COMPANY. |

Last Update Date

26-JAN-2016

### STATISTICAL ANALYSIS PLAN(V4.0)

#### 3. Analysis Sets

#### 3.1 Safety Analysis Sets

#### Safety Set

All subjects who

- have signed an informed consent form, undergone screening procedure(s) and received a subject number,
- received a study vaccination,
- provided post vaccination safety data.

#### Safety per protocol set

All subjects in the safety Set with the exclusions of the following cases:

- (1) Subjects administered prior to the contract date.
- (2) Subjects who didn't receive MenACWY-CRM.
- (3) Follow-up failure: The subjects whose safety information cannot be identified due to follow-up loss.
- (4) Not applicable to the indication of study drug [Indication]
  - To prevent invasive meningococcal disease caused by Neisseria meningitides serogroups A, C, Y and W-135 in persons 2 months through 55 years of age.
- (5) Subjects who violate of Protocol: Those who do not meet one item at least of the inclusion/exclusion criteria.

[Inclusion criteria]

- 1) Male and female subjects from 2 months to 55 years of the age at the time of Visit 1 (including all 55 years old subjects, up to one day before their 56<sup>th</sup> year birthday), who are scheduled to receive vaccination with MenACWY-CRM conjugate vaccine, according to the local prescribing information and routine clinical practice.
- 2) To whom the nature of the study has been described and the subject or subject's parent/legal representative has provided written informed consent.
- 3) Whom the investigator believes that the subject can and will comply with the requirements of the protocol.
- 4) Who are in good health as determined by the outcome of medical history, physical



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

26-JAN-2016

Last Update Date

STATISTICAL ANALYSIS PLAN(V4.0)

assessment and clinical judgment of the investigator.

[Exclusion criteria]

- 1) Contraindication, special warnings and/or precautions, as evaluated by the investigators, reported in the MenACWY-CRM conjugate vaccine Korean prescribing information
- 2) Infants who were already enrolled in this trial for previous vaccination.
- (6) Subjects who prescribed off-label dosage:
  - Vaccine schedule for children from 2 to 23 months of age :
    - Infants 2 to 6 months of age: Three doses of MenACWY-CRM, each of 0.5 ml, is to be given with an interval of at least 2 months; the fourth dose schedule be administered during the second year of life with an interval of at least 6 months after the third dose.
    - Infants 7 to 23 months of age: MenACWY-CRM is to be administered as two doses, each as single dose (0.5ml), with the second dose administered in the second year of life and at least three months after the first dose.
  - 2 to 55 years of age: MenACWY-CRM is to be administered as a single dose (0.5ml).
  - \* The infant from 2 to 23 months of age may enroll at any point, in the vaccination series, including those subjects who may already initiated vaccination series. According to parental consents, these subjects may be followed up for 29 days within the surveillance period after subsequent vaccination(s) at the same study site.

#### Non-Safety per protocol set

Subjects excluded from safety per protocol set except for subjects who did not receive MenACWY-CRM and follow-up failure.

Based on rules for estimation of each number of safety evaluation cases, the following local regulation and Guideline on Standards for re-examination for new drugs, etc of MFDS, non-safety analysis set are excluded from the safety analysis set:

Guideline on Standards for re-examination for new drugs, etc (Chapter II, no. 3) Patient Population for Surveillance:

- A) Patients planned to receive a drug under surveillance by investigator's medical ju dgment shall be subject.
- B) Subject who do not use within approved range shall not be included in the subject in principal.

However, if data of subject whose use is beyond approved range is collected, p erform analysis as a separate item.

| | | Last Update Date |
|---|---|---|
| dreamcis | CONFIDENTIAL: THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS | 26-JAN-2016 |
| | PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY. | 20-JAIN-2010 |
| STATISTICAL ANALYSIS PLAN(V4.0) | | |

C) Describe actual selection methods of subject in detail.

### 3.2 Efficacy Analysis Set

Not Applicable

#### 4. Endpoints

### 4.1 Safety Endpoints

Safety will be assessed after administration of study vaccine in terms of the number and percentage of subjects with:

- Local and systemic solicited adverse events reported from study Day 1 (day of vaccination) through study Day 7 post-vaccination;
- Unsolicited AEs reported from study Day 1 (day of vaccination) through study Day 7 postvaccination;
- Medically attended AEs reported from study Day 1 to study termination (Day 29/early termination);
- SAEs reported from study Day 1 to study termination (Day 29/early termination).

#### 5. Assessment Criteria

#### **5.1 Safety Assessment Criteria**

Not Applicable



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

26-JAN-2016

Last Update Date

### STATISTICAL ANALYSIS PLAN(V4.0)

#### 6. Statistical Analyses

#### **6.1 Baseline Characteristics**

Descriptive statistics (mean, standard deviation, median, minimum and maximum) for baseline characteristics such as age, height and weight at enrollment will be calculated in the Safety set and Safety per Protocol set.

The following baseline characteristics will be reported:

- < Subject Baseline Information >
  - gender, age, ethnic origin, children group, weight, height, past diagnosis, kidney disorder, liver disorder, pre-Immunization temperature, temperature location, pregnancy
- < Study Vaccine Information >
  - vaccine site, number of previous Menveo, study vaccination number, concomitant medications

### **6.2 Safety Analyses**

The number of subjects of AE<sup>†</sup> and the number of AEs<sup>†</sup> incurred shall be calculated, the incidence rate of AEs<sup>†</sup> and its 95% confidence interval will be calculated using the normal approximation on the safety set and safety per protocol set.

† AE : AE includes solicited and unsolicited AE (DAY 1-7), medically attended AE (DAY 1-29) and SAE (DAY 1-29).

#### **6.2.1** Adverse Events by Baseline Characteristics

 $AE^{\dagger}s$  (as described below) will be reported (n %) for the following baseline characteristics in the safety set and safety per protocol set :

- Age group (2-23 months, 2-10, 11-18, 19-34, 35-55)
- Children group ( $<18, \ge 18$ )
- Gender (male, female)
- Past diagnosis (yes, no)



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

26-JAN-2016

Last Update Date

STATISTICAL ANALYSIS PLAN(V4.0)

- Temperature location (axillary, oral, rectal, ear)
- Administration site (left deltoid, right deltoid, left thigh, right thigh, other)
- Concomitant medication (yes, no)
- Kidney disorder (yes, no)
- Liver disorder (yes, no)
- Pregnancy (yes, no)
- Number of previous Menveo (0, 1, 2, 3)
- Study vaccination number (1, 2, 3, 4)

The n(%) of AEs<sup>†</sup> and its 95% confidence interval will be calculated using the normal approximation and analyzed using  $\chi^2$ - test. If more than 20% of expected frequencies of the cell counts are less than 5, Fisher's exact test will be used instead of the chi-square test.

† AE : AE includes solicited and unsolicited AE (DAY 1-7), medically attended AE (DAY 1-29) and SAE (DAY 1-29).

#### **6.2.2.** Analysis of Solicited AE

Frequencies and % of subjects experiencing each adverse event will be presented for each symptom severity. Summary tables showing the occurrence of any local or systemic reaction overall and at each time point will also be presented (see Appendix 1 Table 4.1.3 and 4.2.3).

Post-vaccination adverse events reported from Day 1 to Day 7 will be summarized by maximal severity. The severity of local adverse events for subjects < 6 years of age will be categorized as follows. Injection-site erythema and induration: absent (0 to 9 mm), mild (10 to 25 mm), moderate (26 to 50 mm), severe (> 50 mm); injection-site tenderness: none, mild (minor light reaction to touch), moderate (cried or protested to touch), severe (cried when injected limb was moved). For subjects  $\ge$  6 years, injection-site erythema and induration absent (1 to 24 mm), mild (25 to 50 mm), moderate (51 to 100 mm), severe (>100 mm); pain: none, mild (present but does not interfere with activity), moderate (interferes with activity), severe (prevents daily activity).

For subjects  $\geq$  6 years of age, the severity of systemic adverse events (i.e., chills, nausea, malaise, generalized myalgia, generalized arthralgia, headache) occurring up to 7 days after each vaccination will be categorized as none, mild (present but not interfering with daily activity), moderate (some interference with daily activity), and severe (prevents daily activity) except for rash, which will be



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

26-JAN-2016

Last Update Date

### STATISTICAL ANALYSIS PLAN(V4.0)

categorized as none, urticarial, or other.

For subjects < 6 years of age, the severity of systemic adverse events occurring up to 7 days after each vaccination will be categorized as follows. Change in eating habits: none (no change in appetite), mild (eating less than normal for 1 to feeds), moderate (missed 1 or 2 feeds), severe (missed more than 2 feeds); sleepiness: none (no change in alertness), mild (shows an increased alertness), moderate (sleeps through feeds), severe (sleeps most of the time and it is hard to arouse him/her); irritability: none (no change in child disposition), mild (requires more cudding and he/she is less playful than usual), moderate (more difficult to settle), severe (unable to console); rash: none, urticarial, or other; vomiting: none, mild (1-2 episodes/24 hours), moderate (>2 episodes/24 hours), severe (requires outpatient hydratation); diarrhea: none (fewer than 2 loose stools/24 hours), mild (2-3 loose stools or < 400 gms/24 hours), moderate (4-5 stools or 400-800 gms/24 hours), severe (6 or more watery stools or > 800 gms/24 hours or requires outpatient IV hydration).

Body temperature will be categorized as  $<38^{\circ}$ C (no fever),  $\ge 38^{\circ}$ C (fever) and will be summarized by  $0.5^{\circ}$ C increments from  $36.0^{\circ}$ C up to  $\ge 40^{\circ}$ C. Additionally, no fever vs. fever will be reported.

Each local and systemic adverse event will also be categorized as none vs. any.

#### 6.2.3 Analysis of Unsolicited AE

All unsolicited AEs and MAAE recorded in the CRF will be mapped to preferred terms using the most recent MedDRA dictionary and classified by System organ class (SOC) and Preferred Terms (PT). Under the classification standard of MedDRA terms, and all AEs excluding the AEs whose causal relation with the study medication is 'Not Related' shall be treated as AEs whose causal relation cannot be excluded {hereafter "Adverse Drug Reaction(ADR)"}.

- ① The frequency and percentage of unsolicited AE (Day 1-7) and MAAE (Day 8-29) according to the expected, serious, severity, frequency, action taken, outcome, relationship to MenACWY-CRM regarding occurred AE will be calculated.
- ② The frequency of unsolicited AEs (Day 1-7) and MAAE (Day 8-29) will be classified into the preferred terms according to the expected, serious, severity, frequency, action taken, outcome, relationship to MenACWY-CRM.
- 3 The number of subjects and percentage of SAE/Serious ADR (SADR), unexpected AE/ADR,



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

26-JAN-2016

Last Update Date

### STATISTICAL ANALYSIS PLAN(V4.0)

MAAE/ADR, unsolicited AE/ADR and continuous solicited AE/ADR will be calculated according to the preferred terms. And the number of subjects and percentage by study vaccination number of SAE/Serious ADR (SADR), unexpected AE/ADR, MAAE/ADR, unsolicited AE/ADR and continuous solicited AE/ADR will be calculated according to the preferred terms in infants 2 to 23 months.

(4) For subjects excluded from safety per protocol set<sup>†</sup>, the number of subjects and the percentage of SAE/Serious ADR (SADR), unexpected AE/ADR, MAAE/ADR, unsolicited AE/ADR and continuous solicited AE/ADR will be calculated according to the preferred terms. And the number of subjects and percentage by study vaccination number of SAE/Serious ADR (SADR), unexpected AE/ADR, MAAE/ADR, unsolicited AE/ADR and continuous solicited AE/ADR will be calculated according to the preferred terms in infants 2 to 23 months.

Subject excluded from safety per protocol set: Except for subjects who didn't receive study vaccination and follow-up failure.

#### 7. List of Table and Data Listings

### 7.1 Distribution of Subjects

- Number of subjects contracted to the study: The number of subjects are to be collected(under contract) as contracted by the investigator.
- Number of retrieving completed CRFs: Total number of subjects whose completed CRFs.
- Number of safety assessment population: Number of safety assessment population among total number.

#### 7.2 Baseline Characteristics

- Mean and standard deviation (SD) or frequency and percentage by gender, age, ethnic origin, weight, height, past diagnosis, pre-Immunization temperature, temperature location, pregnancy
- Frequency and percentage by vaccine site, number of previous Menveo, study vaccination number, concomitant medications.

# dreamcis


THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

26-JAN-2016

Last Update Date

STATISTICAL ANALYSIS PLAN(V4.0)

#### 7.3 Safety Analyses

- Incidence rate and the number of AEs according to the baseline characteristics (frequency and percentage).
- The number of the expected serious, severity, frequency, action taken, outcome, relationship to MenACWY-CRM for Unsolicited AE (DAY 1-7) and MAAE (DAY 8-29) (frequency and percentage).
- The number of AEs for the severity, day, fever to MenACWY-CRM according to individual solicited AE (DAY 1-7) (frequency and percentage)..
- Incidence rate and number according to the preferred terms of SAE/SADR, unexpected AE/ADR, MAAE/ADR, unsolicited AE/ADR and continuous solicited AE/ADR (frequency and percentage)
- For subjects excluded from safety per protocol set<sup>†</sup> incidence rate and number according to the preferred terms of SAE/SADR, unexpected AE/ADR, MAAE/ADR, unsolicited AE/ADR and continuous solicited AE/ADR (frequency and percentage).

Subject excluded from safety per protocol set: Except for subjects who didn't receive study mediation and follow-up failure.

#### 8. Notes

- Each statistical analysis will be carried out with SAS Software version 9.4 or more recent version.
- In the descriptive statistics, mean, SD, minimum, median, and maximum will be calculated for continuous variables, and frequency and percentage for categorical variables.
- Data including sign of inequality such as "≥20", ">20" will be excluded from analysis.
- All test statistics will be the results of two-sided tests with the statistical significant level of 0.05.
- The followings shall be included only in re-examination report:
  - Analysis by type of concomitant medications
  - Item ② of paragraph 6.2.3
  - Estimation of 95% confidence interval for incidence of AEs by background factors

# Appendix 1

| 1. D | Demographic and baseline values, medication characteristics, specific characteristics | 6 |
|---|---|---|
| | 1.1 Safety Set | 6 |
| | Table 1.1.1 Total subject | 6 |
| | Table 1.1.2 Demographic characteristics | 6 |
| | Table 1.1.3 Past diagnosis | 7 |
| | Table 1.1.4 Pre-Immunization temperature | 7 |
| | Table 1.1.5 Temperature Location | 8 |
| | Table 1.1.6 Administration Site | 8 |
| | Table 1.1.7 Concomitant medication | 8 |
| | Table 1.1.8 Kidney Disorder | 8 |
| | Table 1.1.9 Liver disorder | 10 |
| | Table 1.1.10 Pregnancy | 10 |
| | Table 1.1.11 Number of previous MenACWY | 10 |
| | Table 1.1.12 Study vaccination number | 10 |
| | 1.2 Safety Per Protocol Set | 12 |
| | Table 1.2.1 Total subject | 12 |
| | Table 1.2.2 Demographic characteristics | 12 |
| | Table 1.2.3 Past diagnosis | 13 |
| | Table 1.2.4 Pre-Immunization temperature | 13 |
| | Table 1.2.5 Temperature Location | 14 |
| | Table 1.2.6 Administration Site | 14 |
| | Table 1.2.7 Concomitant medication | 14 |
| | Table 1.2.8 Kidney Disorder | 15 |
| | Table 1.2.9 Liver disorder | 15 |
| | Table 1.2.10 Pregnancy | 15 |
| | Table 1.2.11 Number of previous MenACWY | 15 |
| | Table 1.2.12 Study vaccination number | 16 |
| 2. S | afety Analyses | 17 |
| | 2.1 Safety Set | |
| | Table 2.1.1 Summary of AE | 17 |
| | Table 2.1.2 Summary of AE by Age (month, year) | 19 |
| | Table 2.1.3 Summary of AE by Age (month, year) | 19 |
| | Table 2.1.4 Summary of AE by Children group | 21 |

| Table 2.1.5 Summary of AE by Gender | 22 |
|---|---|
| Table 2.1.6 Summary of AE by Past diagnosis | 22 |
| Table 2.1.7 Summary of AE by Temperature Location | 22 |
| Table 2.1.8 Summary of AE by Administration Site | 23 |
| Table 2.1.9 Summary of AE by Concomitant medication | 23 |
| Table 2.1.10 Summary of AE by Kidney Disorder | 23 |
| Table 2.1.11 Summary of AE by Liver disorder | 24 |
| Table 2.1.12 Summary of AE by Pregnancy | 24 |
| Table 2.1.13 Summary of AE by Number of previous MenACWY | 24 |
| Table 2.1.14 Summary of AE by Study vaccination number | 24 |
| 2.2 Safety per protocol set | 26 |
| Table 2.2.1 Summary of AE | 26 |
| Table 2.2.2 Summary of AE by Age (month, year) | 28 |
| Table 2.2.3 Summary of AE by Age (year) | 28 |
| Table 2.2.4 Summary of AE by Children group | 30 |
| Table 2.2.5 Summary of AE by Gender | 30 |
| Table 2.2.6 Summary of AE by Past diagnosis | 31 |
| Table 2.2.7 Summary of AE by Temperature Location | 31 |
| Table 2.2.8 Summary of AE by Administration Site | 31 |
| Table 2.2.9 Summary of AE by Concomitant medication | 32 |
| Table 2.2.10 Summary of AE by Kidney Disorder | 32 |
| Table 2.2.11 Summary of AE by Liver disorder | 32 |
| Table 2.2.12 Summary of AE by Pregnancy | 32 |
| Table 2.2.13 Summary of AE by Number of previous MenACWY | 33 |
| Table 2.2.14 Summary of AE by Study vaccination number | 33 |
| formation of AEs | 34 |
| 3.1 Safety Set | 34 |
| Table 3.1.1 Summary of solicited AE and unsolicited AE for 7 days after vaccinati | ion (<6 years)34 |
| Table 3.1.2 Summary of solicited AE and unsolicited AE for 7 days after vaccinati | ion (<6 years)35 |
| Table 3.1.3 Summary of solicited AE and unsolicited AE for 7 days after vacci | ination by study |
| vaccination number (2-23months) | 36 |
| Table 3.1.4 Summary of solicited AE and unsolicited AE for 7 days after vaccinati | on (≥ 6years)38 |
| Table 3.1.5 Summary of solicited AE and unsolicited AE for 7 days after vaccinati | on (≥6years) 39 |
| Table 3.1.7 Summary of medically attended AEs for 8 days to 28 days after vaccin | ation 41 |
| Table 3.1.8 Summary of medically attended AEs for 8 days to 28 days after vacc | ination by study |
| vaccination number (2-23 months) | 42 |

| Table 3.2.1 Summary of solicited AE and unsolicited AE for 7 days after vaccination (<6 | 5 years)43 |
|---|---|
| Table 3.2.2 Summary of solicited AE and unsolicited AE for 7 days after vaccination (<6 | 5 years)44 |
| Table 3.2.3 Summary of solicited AE and unsolicited AE for 7 days after vaccination | by study |
| vaccination number (2-23months) | 45 |
| Table 3.2.4 Summary of solicited AE and unsolicited AE for 7 days after vaccination (≥6 | years)47 |
| Table 3.2.5 Summary of solicited AE and unsolicited AE for 7 days after vaccination (≥6 | years)48 |
| Table 3.2.6 Summary of medically attended AEs for 8 days to 28 days after vaccination. | 50 |
| Table 3.2.7 Summary of medically attended AEs for 8 days to 28 days after vaccination . | 51 |
| Table 3.2.8 Summary of medically attended AEs for 8 days to 28 days after vaccination | ı by study |
| vaccination number (2-23 months) | 52 |
| 4. Solicited AE (DAY 1-7) | 53 |
| 4.1 Safety Set | 53 |
| Table 4.1.1 Summary of Local AE Max severity (<6 years) | 53 |
| Table 4.1.2 Summary of Local AE Max severity (≥6 years) | 53 |
| Table 4.1.3 Summary of Local AE by Max severity | 53 |
| Table 4.1.4 Summary of Systemic AE by Max severity (<6 years) | 54 |
| Table 4.1.5 Summary of Systemic AE by Max severity(≥6 years) | 55 |
| Table 4.1.6 Summary of Systemic AE by Max severity | 55 |
| Table 4.1.7 Summary of Solicited AE by day (<6 years) | 57 |
| Table 4.1.8 Summary of Solicited AE by day (≥6 years) | 58 |
| Table 4.1.9 Summary of Solicited AE by day | 58 |
| Table 4.1.10 Summary of Fever | 61 |
| 4.2 Safety per protocol set | 62 |
| Table 4.2.1 Summary of local AE by Max severity (<6 years) | 62 |
| Table 4.2.2 Summary of Local AE Max severity (≥6 years) | 62 |
| Table 4.2.3 Summary of Local AE by Max severity | 62 |
| Table 4.2.4 Summary of Systemic AE by Max severity (<6 years) | 63 |
| Table 4.2.5 Summary of Systemic AEs by Max severity (≥6 years) | 64 |
| Table 4.2.6 Summary of Systemic AE by Max severity | 64 |
| Table 4.2.7 Summary of Solicited AE by day (<6 years) | 66 |
| Table 4.2.8 Summary of Solicited AE by day (≥6 years) | 66 |
| Table 4.2.9 Summary of Solicited AE by day | 67 |
| Table 4.2.10 Summary of Fever | 69 |
| 5. Unsolicited AE (DAY 1-7) | 70 |
| 5.1 Safety Set | 70 |
| Table 5.1.1 Summary of Unsolicited AE | |
| 5.2 Safety per protocol set | |
| Table 5.2.1 Summary of Unsolicited AE | <b>3</b> ·/· <b>12</b> 3 <sup>2</sup> |

| 6. MAAE (DAY 8-29) | 74 |
|---|---|
| 6.1 Safety Set | 74 |
| Table 6.1.1 Summary of MAAE | 74 |
| 6.2 Safety per protocol set | 76 |
| Table 6.2.1 Summary of MAAE | 76 |
| 7. SAE/SADR for 28 days after vaccination | 78 |
| 7.1 Safety Set | 78 |
| Table 7.1.1 SAE and SADR | 78 |
| Table 7.1.1.1 SAE and SADR by study vaccination (2-23 months) | 80 |
| 7.2 Safety per protocol set | 81 |
| Table 7.2.1 SAE and SADR | 81 |
| Table 7.2.1.1 SAE and SADR by study vaccination (2-23 months) | 83 |
| 7.3 Non-Safety per protocol set | 84 |
| Table 7.3.1 SAE and SADR | 84 |
| Table 7.3.1.1 SAE and SADR by study vaccination (2-23 months) | 86 |
| 8. Unexpected AE/ADR for 28 days after vaccination | 87 |
| 8.1 Safety Set | 87 |
| Table 8.1.1 Unexpected AE and ADR | 87 |
| Table 8.1.1.1 Unexpected AE and ADR by study vaccination number (2-23 months) | 90 |
| 8.2 Safety per protocol set | 91 |
| Table 8.2.1 Unexpected AE and ADR | 91 |
| Table 8.2.1.1 Unexpected AE and ADR by study vaccination number (2-23 months) | 93 |
| 8.3 Non-Safety per protocol set | 94 |
| Table 8.3.1 Unexpected AE and ADR | 94 |
| Table 8.3.1.1 Unexpected AE and ADR by study vaccination number (2-23 months) | 96 |
| 9. MAAE/ADR for 8 days to 28 days after vaccination | 97 |
| 9.1 Safety Set | 97 |
| Table 9.1.1 MAAE and ADR | 97 |
| Table 9.1.1.1 MAAE and ADR by study vaccination number (2-23months) | 99 |
| 9.2 Safety per protocol set | 100 |
| Table 9.2.1 MAAE and ADR | 100 |
| Table 9.2.1.1 MAAE and ADR by study vaccination number (2-23months) | 102 |
| 9.3 Non-Safety per protocol set | 103 |
| Table 9.3.1 MAAE and ADR | 103 |
| Table 9.3.1.1 MAAE and ADR by study vaccination number (2-23months) | |
| 10. Unsolicited AE/ADR for 28 days after vaccination | |
| 10.1 Safety Set | |
| Table 10.1.1 Unsolicited AE and ADR | |
| Tube 10.1.1 Chomology ID and 1 DA | 4/.123° |

| Table 10.1.1.1 Unsolicited AE and ADR by study vaccination number (2-23 months) | 108 |
|---|---|
| 10.2 Safety per protocol Set | 109 |
| Table 10.2.1 Unsolicited AE and ADR | 109 |
| Table 10.2.1.1 Unsolicited AE and ADR by study vaccination number (2-23 months) | 111 |
| Table 10.3.1 Unsolicited AE and ADR | 112 |
| Table 10.3.1.1 Unsolicited AE and ADR by study vaccination number (2-23 months) | 114 |
| 11.1 Safety Set | 115 |
| Table 11.1.1 Continuous Solicited AE | 115 |
| Table 11.1.1.1 Continuous Solicited AE by study vaccination number (2-23 months) | 117 |
| 11.2 Safety per protocol set | 118 |
| Table 11.2.1 Continuous Solicited AE | 118 |
| Table 11.2.1.1 Continuous Solicited AE by study vaccination number (2-23 months) | 120 |
| 11.3 Non-Safety per protocol set | 121 |
| Table 11.3.1 Continuous Solicited AE | 121 |
| Table 11.3.1.1 Continuous Solicited AE by study vaccination number (2-23 months) | 123 |

### 1. Demographic and baseline values, medication characteristics, specific characteristics

- Baseline characteristics will be reported on the safety set and safety per protocol set.

### 1.1 Safety Set

Table 1.1.1 Total subject

| Safety Set | Total |
|------------|------------------|
| | No. subjects (%) |
| Total | |

Table 1.1.2 Demographic characteristics

#### 1) (Administration start date)-(birth)+1

| Safety Set | | Total |
|-----------------------|--------------|------------------|
| | | No. subjects (%) |
| Age(years)1) | No. subjects | |
| | mean±std | |
| | median | |
| | min~max | |
| Age(months, years) | 2-23 months | |
| | 2-10 years | |
| | 2-5 years | |
| | 6-10 years | |
| | 11-18 years | |
| | 19-34 years | |
| | 35-55 years | |
| | > 55 years | |
| | Total | <u> </u> |
| Children group(years) | < 18 | |
| | ≥ 18 | |
| | Total | |
| Ethnic Origin | Asian | |
| | Black | |

| Safety Set | | Total |
|------------|--------------|------------------|
| | | No. subjects (%) |
| | Caucasian | |
| | Hispanic | |
| | Other | |
| | Total | |
| Gender | Male | |
| | Female | |
| | Total | |
| Weight(kg) | No. subjects | |
| | mean±std | |
| | median | |
| | min~max | |
| Height(cm) | No. subjects | |
| | mean±std | |
| | median | |
| | min~max | |

### Table 1.1.3 Past diagnosis

| Safety Set | Total |
|------------|------------------|
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |

# Table 1.1.4 Pre-Immunization temperature

| Safety Set | Total |
|---------------|------------------|
| | No. subjects (%) |
| No. subjects | |
| mean±std (°C) | |
| median | |
| min~max | |

Table 1.1.5 Temperature Location

| Safety Set | Total |
|------------|------------------|
| | No. subjects (%) |
| Axillary | |
| Oral | |
| Rectal | |
| Ear | |
| Total | |

### Table 1.1.6 Administration Site

| Safety Set | Total |
|---------------------------|------------------|
| | No. subjects (%) |
| Left Deltoid | |
| Right Deltoid | |
| Left Thigh (Infant only) | |
| Right Thigh (Infant only) | |
| Other | |
| Total | |

### Table 1.1.7 Concomitant medication

| Safety Set | Total |
|------------|------------------|
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |

### Table 1.1.8 Kidney Disorder

| Safety Set | Total |
|------------|------------------|
| | No. subjects (%) |
| Yes | |

| No |
|-------|
| Total |

Table 1.1.9 Liver disorder

| Safety Set | Total |
|------------|------------------|
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |

# Table 1.1.10 Pregnancy

| Safety Set | Total |
|------------|------------------|
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |

# Table 1.1.11 Number of previous MenACWY

| Safety Set | Total |
|------------|------------------|
| | No. subjects (%) |
| 0 | |
| 1 | |
| 2 | |
| 3 | |
| Total | |

# Table 1.1.12 Study vaccination number

| Safety Set | Total |
|------------|------------------|
| | No. subjects (%) |
| 1 | |
| 2 | |
| 3 | |
| 4 | |
| E + 1 | |
|-------|--|
| Total | |
| 10111 | |

# 1.2 Safety Per Protocol Set

Table 1.2.1 Total subject

| Safety per protocol set | Total |
|-------------------------|------------------|
| | No. subjects (%) |
| Total | |

# Table 1.2.2 Demographic characteristics

#### 1) (Administration start date)-(birth)+1

| Safety per protocol set | | Total |
|-------------------------|--------------|------------------|
| | | No. subjects (%) |
| Age(years)1) | No. subjects | |
| | mean±std | |
| | median | |
| | min~max | |
| Age(months, years) | 2-23 months | |
| | 2-10 years | |
| | 2-5 years | |
| | 6-10 years | |
| | 11-18 years | <u> </u> |
| | 19-34 years | |
| | 35-55 years | |
| | Total | |
| Children group(years) | < 18 | |
| | ≥ 18 | |
| | Total | <u> </u> |
| Ethnic Origin | Asian | |
| | Black | |
| | Caucasian | |
| | Hispanic | |
| | Other | |
| | Total | |
| Gender | Male | |
| | | I |

| Safety per protocol set | | Total |
|-------------------------|--------------|------------------|
| | | No. subjects (%) |
| | Female | |
| | Total | |
| Weight(kg) | No. subjects | |
| | mean±std | |
| | median | |
| | min~max | |
| Height(cm) | No. subjects | |
| | mean±std | |
| | median | |
| | min~max | |

#### Table 1.2.3 Past diagnosis

| Safety per protocol set | Total |
|-------------------------|------------------|
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |

# Table 1.2.4 Pre-Immunization temperature

| Safety per protocol set | Total |
|-------------------------|------------------|
| | No. subjects (%) |
| No. subjects | |
| mean±std (°C) | |
| median | |
| min~max | |

Table 1.2.5 Temperature Location

| Safety per protocol set | Total |
|-------------------------|------------------|
| | No. subjects (%) |
| Axillary | |
| Oral | |
| Rectal | |
| Ear | |
| Total | |

#### Table 1.2.6 Administration Site

| Safety per protocol set | Total |
|---------------------------|------------------|
| | No. subjects (%) |
| Left Deltoid | |
| Right Deltoid | |
| Left Thigh (Infant only) | |
| Right Thigh (Infant only) | |
| Other | |
| Total | |

#### Table 1.2.7 Concomitant medication

| Safety per protocol set | Total |
|-------------------------|------------------|
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |

Table 1.2.8 Kidney Disorder

| Safety per protocol set | Total |
|-------------------------|------------------|
| _ | No. subjects (%) |
| Yes | |
| No | |
| Total | |

#### Table 1.2.9 Liver disorder

| Safety per protocol set | Total |
|-------------------------|------------------|
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |

# Table 1.2.10 Pregnancy

| Safety per protocol set | Total |
|-------------------------|------------------|
| | No. subjects (%) |
| Yes | |
| No | |
| Total | |

# Table 1.2.11 Number of previous MenACWY

| Safety per protocol Set | Total |
|-------------------------|------------------|
| | No. subjects (%) |
| 0 | |
| 1 | |
| 2 | |
| 3 | |
| Total | |

Table 1.2.12 Study vaccination number

| Safety per protocol Set | Total |
|-------------------------|------------------|
| | No. subjects (%) |
| 1 | |
| 2 | |
| 3 | |
| 4 | |
| Total | |

#### 2. Safety Analyses

- AE includes solicited and unsolicited AE (Day 1-7) and medically attended AE (Day 1-29) and SAEs (Day
- AE will be reported on the safety set and safety per protocol set.
- SAE/SADR will be reported on the safety set, safety per protocol set and non-safety per protocol set.

#### 2.1 Safety Set

Table 2.1.1 Summary of AE

| | 95% CI† for the | | | 95% CI† for |
|---|---|---|---|---|
| No. subjects with AE | percentage of | No. AEs | No. subjects with ADR | percentage of |
| | subjects with AE | | | subjects with A |
| n (%) | (Lower , Upper) | n | n (%) | (Lower ,Upp |
| | | No. subjects with AE percentage of subjects with AE | No. subjects with AE percentage of subjects with AE No. AEs | No. subjects with AE percentage of subjects with AE No. AEs No. subjects with ADR |

| | | 95% CI† for the | | | 95% CI† for the | | |
|---|---|---|---|---|---|---|---|
| Safety set | No. subjects with AE | percentage of | No. AEs | No. subjects with ADR | percentage of | No. ADR | Total |
| | | subjects with AE | | | subjects with ADR | | |
| | n (%) | (Lower, Upper) | n | n (%) | (Lower , Upper) | n | n (%) |
| Unsolicited AE | | | | | | | |
| SAE | | | | | | | |
| MAAE | | | | | | | |
| Death | | | | | | | |
| Total | | | | | | | |

<sup>† 95%</sup> CI will be calculated using the normal approximation.

<sup>\*</sup> Day 1-7: Solicited AE, Unsolicited AE

<sup>\*</sup> Day 1-29: SAE, Death

<sup>\*</sup> Day 8-29: MAAE

Table 2.1.2 Summary of AE by Age (month, year)

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| 2-23 months | | | | |
| 2-10 | | | | |
| 2-5 | | | | |
| 6-10 | | | | X <sup>2</sup> -test or Exact test |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |
| > 55 | | | | |
| Total | | | | |

Table 2.1.3 Summary of AE by Age (month, year)

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Solicited AE | | | | |
| 2-23 months | | | | |
| 2-10 | | | | |
| 2-5 | | | | |
| 6-10 | | | | X <sup>2</sup> -test or Exact test |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |
| > 55 | | | | |
| Solicited Local AE | | | | |
| 2-23 months | | | | |
| 2-10 | | | | |
| 2-5 | | | | X <sup>2</sup> -test or Exact test |
| 6-10 | | | | |
| 11-18 | | | | |
| 19-34 | | | | |

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| 35-55 | | Î | | |
| > 55 | | | | |
| Solicited Systemic AE | | | | |
| 2-23 months | | | | |
| 2-10 | | | | |
| 2-5 | | | | |
| 6-10 | | | | X <sup>2</sup> -test or Exact test |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |
| ≥56 | | | | |
| Unsolicited AE | | | | |
| 2-23 months | | | | |
| 2-10 | | | | |
| 2-5 | | | | |
| 6-10 | | | | X <sup>2</sup> -test or Exact test |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |
| ≥56 | | | | |
| SAE | | | | |
| 2-23 months | | | | |
| 2-10 | | | | |
| 2-5 | | | | |
| 6-10 | | | | X <sup>2</sup> -test or Exact test |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |
| ≥56 | | | | |
| MAAE | | | | |
| 2-23 months | | | | *** |
| 2-10 | | | | X <sup>2</sup> -test or Exact test |
| 2-5 | | | | |

| Safety Set | No. subjects with AE | No. | Total | p-value |
|---|---|---|---|---|
| | | AEs | | |
| | n (%) | n | n (%) | |
| 6-10 | | | | |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |
| ≥56 | | | | |
| ADR | | | | |
| 2-23 months | | | | |
| 2-10 | | | | |
| 2-5 | | | | |
| 6-10 | | | | X <sup>2</sup> -test or Exact test |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |
| ≥56 | | | | |
| Death | | | | |
| 2-23 months | | | | |
| 2-10 | | | | |
| 2-5 | | | | |
| 6-10 | | | | X <sup>2</sup> -test or Exact test |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |
| ≥56 | | | | |

Table 2.1.4 Summary of AE by Children group

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| < 18 years | | | | |
| ≥ 18 years | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

Table 2.1.5 Summary of AE by Gender

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Male | | | | |
| Female | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

#### Table 2.1.6 Summary of AE by Past diagnosis

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

# Table 2.1.7 Summary of AE by Temperature Location

| Safety Set | No. subjects with AE | No.<br>AEs<br>n | Total n (%) | p-value |
|---|---|---|---|---|
| Axillary | | | | |
| Oral | | | | X <sup>2</sup> -test or Exact test |
| Rectal | | | | |
| Ear | | | | |
| Total | | | | |

Table 2.1.8 Summary of AE by Administration Site

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Left Deltoid | | | | |
| Right Deltoid | | | | X <sup>2</sup> -test or Exact test |
| Left Thigh (Infant only) | | | | |
| Right Thigh (Infant only) | | | | |
| Other | | | | |
| Total | | | | |

# Table 2.1.9 Summary of AE by Concomitant medication

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

# Table 2.1.10 Summary of AE by Kidney Disorder

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

Table 2.1.11 Summary of AE by Liver disorder

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

Table 2.1.12 Summary of AE by Pregnancy

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

Table 2.1.13 Summary of AE by Number of previous MenACWY

| Safety Set | No. subjects with AE | No.<br>AEs<br>n | Total<br>n (%) | p-value |
|---|---|---|---|---|
| 0 | | | | |
| 1 | | | | X <sup>2</sup> -test or Exact test |
| 2 | | | | |
| 3 | | | | |
| Total | | | | |

Table 2.1.14 Summary of AE by Study vaccination number

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|------------|----------------------|------------|-------|---------|
| | n (%) | n | n (%) | |
| 1 | | | | |

| Safety Set | No. subjects with AE | No. | Total | p-value |
|---|---|---|---|---|
| Safety Set | No. subjects with AE | AEs | Total | |
| | n (%) | n | n (%) | |
| 2 | | | | X <sup>2</sup> -test or Exact test |
| 3 | | | | |
| 4 | | | | |
| Total | | | | |

#### 2.2 Safety per protocol set

Table 2.2.1 Summary of AE

| Safety per protocol set | No. subjects with AE | 95% CI† for the percentage of subjects with AE | No. AEs | No. subjects with ADR | 95% CI† for the percentage of subjects with ADR | No. ADR | Total |
|---|---|---|---|---|---|---|---|
| | n (%) | (Lower , Upper) | n | n (%) | (Lower , Upper) | n | n (%) |
| Solicited AE (2-23 months) | | | | | | | |
| Local AE | | | | | | | |
| Systemic AE | | | | | | | |
| Solicited AE (2-5 years) | | | | | | | |
| Local AE | | | | | | | |
| Systemic AE | | | | | | | |
| Solicited AE (≥ 6 years) | | | | | | | |
| Local AE | | | | | | | |
| Systemic AE | | | | | | | |
| Unsolicited AE | | | | | | | |
| SAE | | | | | | | |
| MAAE | | | | | | | |
| Death | | | | | | | |
| Total | | | | | | | |

<sup>† 95%</sup> CI will be calculated using the normal approximation.

<sup>\*</sup> Day 1-7: Solicited AE, Unsolicited AE

<sup>\*</sup> Day 1-29: SAE, Death

<sup>\*</sup> Day 8-29: MAAE

Table 2.2.2 Summary of AE by Age (month, year)

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| 2-23 months | | | | |
| 2-10 | | | | |
| 2-5 | | | | |
| 6-10 | | | | |
| 11-18 | | | | X <sup>2</sup> -test or Exact test |
| 19-34 | | | | |
| 35-55 | | | | |
| Total | | | | |

Table 2.2.3 Summary of AE by Age (year)

| Safety Set | No. subjects with AE | No. | Total | p-value |
|---|---|---|---|---|
| | n (%) | AEs<br>n | n (%) | |
| Solicited AE | n (/0) | | 11 (70) | |
| 2-23 months | | | | |
| 2-10 | | | | |
| 2-5 | | | | W2 |
| 6-10 | | | | X <sup>2</sup> -test or Exact test |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |
| Solicited Local AE | | | | |
| 2-23 months | | | | |
| 2-10 | | | | |
| 2-5 | | | | X <sup>2</sup> -test or Exact test |
| 6-10 | | | | A*-test of Exact test |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |
| Solicited Systemic AE | | | | |

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| 2-23 months | | | | X <sup>2</sup> -test or Exact test |
| 2-10 | | | | |
| 2-5 | | | | |
| 6-10 | | | | |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |
| Unsolicited AE | | | | |
| 2-23 months | | | | |
| 2-10 | | | | |
| 2-5 | | | | |
| 6-10 | | | | X <sup>2</sup> -test or Exact test |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |
| SAE | | | | |
| 2-23 months | | | | |
| 2-10 | | | | |
| 2-5 | | | | |
| 6-10 | | | | X <sup>2</sup> -test or Exact test |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |
| MAAE | | | | |
| 2-23 months | | | | |
| 2-10 | | | | |
| 2-5 | | | | |
| 6-10 | | | | X <sup>2</sup> -test or Exact test |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |
| ADR | | | | |
| 2-23 months | | | | X <sup>2</sup> -test or Exact test |

| Safety Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| 2-10 | | | | |
| 2-5 | | | | |
| 6-10 | | | | |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |
| Death | | | | |
| 2-23 months | | | | |
| 2-10 | | | | |
| 2-5 | | | | X <sup>2</sup> -test or Exact test |
| 6-10 | | | | X²-test or Exact test |
| 11-18 | | | | |
| 19-34 | | | | |
| 35-55 | | | | |

# Table 2.2.4 Summary of AE by Children group

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| < 18 years | | | | |
| ≥ 18 years | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

# Table 2.2.5 Summary of AE by Gender

| Safety per protocol Set | No. subjects with AE | No. | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Male | | | | |
| Female | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

Table 2.2.6 Summary of AE by Past diagnosis

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

# Table 2.2.7 Summary of AE by Temperature Location

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Axillary | | | | |
| Oral | | | | X <sup>2</sup> -test or Exact test |
| Rectal | | | | |
| Ear | | | | |
| Total | | | | |

#### Table 2.2.8 Summary of AE by Administration Site

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Left Deltoid | | | | |
| Right Deltoid | | | | X <sup>2</sup> -test or Exact test |
| Left Thigh (Infant only) | | | | |
| Right Thigh (Infant only) | | | | |
| Other | | | | |
| Total | | | | |

Table 2.2.9 Summary of AE by Concomitant medication

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

Table 2.2.10 Summary of AE by Kidney Disorder

| Safety per protocol Set | No. subjects with AE | No. | Total | p-value |
|---|---|---|---|---|
| | No. subjects with AL | AEs | | |
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

Table 2.2.11 Summary of AE by Liver disorder

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

Table 2.2.12 Summary of AE by Pregnancy

| Safety per protocol Set | No. subjects with AE | No. | Total | p-value |
|---|---|---|---|---|
| | 140. Subjects with AL | AEs | | |
| | n (%) | n | n (%) | |
| Yes | | | | |
| No | | | | X <sup>2</sup> -test or Exact test |
| Total | | | | |

Table 2.2.13 Summary of AE by Number of previous MenACWY

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| 0 | | | | |
| 1 | | | | X <sup>2</sup> -test or Exact test |
| 2 | | | | |
| 3 | | | | |
| Total | | | | |

Table 2.2.14 Summary of AE by Study vaccination number

| Safety per protocol Set | No. subjects with AE | No.<br>AEs | Total | p-value |
|---|---|---|---|---|
| | n (%) | n | n (%) | |
| 1 | | | | |
| 2 | | | | X <sup>2</sup> -test or Exact test |
| 3 | | | | |
| 4 | | | | |
| Total | | | | |

#### 3. Information of AEs

# 3.1 Safety Set

Table 3.1.1 Summary of solicited AE and unsolicited AE for 7 days after vaccination (<6 years)

| Safety Set | | AF | 3 |
|----------------|---------------------------|----------------|------------|
| | | Incidence Rate | No. of AEs |
| | | n (%) | n |
| Local AE | Local AE | | |
| | Injection site tenderness | | |
| | Injection site erythema | | |
| | Injection site induration | | |
| Systemic AE | Systemic AE | | |
| | Change in eating habits | | |
| | Sleepiness | | |
| | Irritability | | |
| | Vomiting | | |
| | Diarrhea | | |
| | Rash | | |
| | Fever | | |
| UNSOLICITED AE | System Organ Class(SOC) | | |
| | Preferred Term(PT) | | |
| | Sub Total | | |
| Total | • | | |

Table 3.1.2 Summary of solicited AE and unsolicited AE for 7 days after vaccination (<6 years)

| Safety Set | | AE(2-23 mon | ths) N=0 | AE(2-5year | s) N=0 |
|---|---|---|---|---|---|
| | | Incidence | No. of | Incidence | No. of |
| | | Rate | AEs | Rate | AEs |
| | | n (%) | n | n (%) | n |
| Local AE | Local AE | | | | |
| | Pain | | | | |
| | Erythema | | | | |
| | Induration | | | | |
| Systemic AE | Systemic AE | | | | |
| | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |
| | Fever | | | | |
| | Sub Total | | | | |
| UNSOLICITED AE | System Organ Class(SOC) | | | | |
| | Preferred Term(PT) | | | | |
| | Sub Total | | | | |
| Total | | | | | |

Table 3.1.3 Summary of solicited AE and unsolicited AE for 7 days after vaccination by study vaccination number (2-23months)

| Safety Set | | 1 N=0 | | 2 N=0 | | 3 N=0 | | 4 N=0 | |
|---|---|---|---|---|---|---|---|---|---|
| | | Incidence Rate | No. of | Incidence Rate | No. of | Incidence Rate | No. of | Incidence Rate | No. |
| | | | AEs | | AEs | | AEs | | of |
| | | | | | | | | | AEs |
| | | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Local AE | Local AE | | | | | | | | |
| | Pain | | | | | | | | |
| | Erythema | | | | | | | | |
| | Induration | | | | | | | | |
| Systemic AE | Systemic AE | | | | | | | | |
| | Chills | | | | | | | | |
| | Nausea | | | | | | | | |
| | Malaise | | | | | | | | |
| | Myalgia | | | | | | | | |
| | Arthralgia | | | | | | | | |
| | Headache | | | | | | | | |
| | Rash | | | | | | | | |
| | Fever | | | | | | | | |
| | Sub Total | | | | | | | | |
| UNSOLICITED AE | System Organ Class(SOC) | | | | | | | | |
| | Preferred Term(PT) | | | | | | | | |

| Safety Set | 1 N=0 | | 2 N=0 | | 3 N=0 | • | 4 N=0 | |
|---|---|---|---|---|---|---|---|---|
| | Incidence Rate | No. of | Incidence Rate | No. of | Incidence Rate | No. of | Incidence Rate | No. |
| | | AEs | | AEs | | AEs | | of |
| | | | | | | | | AEs |
| | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Sub Total | | <u> </u> | | | | <u> </u> | | |
| Total | | | | | | | | |

Table 3.1.4 Summary of solicited AE and unsolicited AE for 7 days after vaccination ( $\geq$  6 years)

| Safety Set | | Al | Ξ. |
|----------------|-------------------------|----------------|------------|
| | | Incidence Rate | No. of AEs |
| | | n (%) | n |
| Local AE | Local AE | | |
| | Pain | | |
| | Erythema | | |
| | Induration | | |
| Systemic AE | Systemic AE | | |
| | Chills | | |
| | Nausea | | |
| | Malaise | | |
| | Myalgia | | |
| | Arthralgia | | |
| | Headache | | |
| | Rash | | |
| | Fever | | |
| UNSOLICITED AE | System Organ Class(SOC) | | |
| | Preferred Term(PT) | | |
| | Sub Total | | |
| Total | • | | |

Table 3.1.5 Summary of solicited AE and unsolicited AE for 7 days after vaccination (≥6years)

| G 2 G | | AE(6- | 10) | Al | E(11- | 18) | A | E(19- | 34) | A | E(35- | 55) | A | E(≥5 | 56) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety Set | | N= | 0 | | N=0 | 1 | | N=0 | | | N=0 | 1 | | N=0 | |
| | | Inciden | No | Inci | iden | No | Inc | iden | No | Inc | iden | No | Inci | den | No |
| | | ce Rate | | ce F | Rate | | ce I | Rate | | ce l | Rate | | ce F | Rate | |
| | | | of | | | of | | | of | | | of | | | of |
| | | | Α | | | A | | | Α | | | A | | | Α |
| | | | Es | | | Es | | | Es | | | Es | | | Es |
| | | ( | | | ( | | | ( | | | ( | | | ( | |
| | | n % | n | n | % | n | n | % | n | n | % | n | n | % | n |
| | | ) | | | ) | | | ) | | | ) | | | ) | |
| Local AE | Local AE | | | | | | | | | | | | | | |
| | Pain | • | | | | | | | | | •••• | | | | |
| | Erythema | | | | | | | | | | | | | | |
| | Induration | | | | | | | | | | | | | | |
| Systemic AE | Systemic AE | | | | | | | | | | | | | | |
| | Chills | • | | | | | | | | | | | | | |
| | Nausea | | | | | | | | | | | | | | |
| | Malaise | | | | | | | | | | | | | | |
| | Myalgia | | | | | | | | | | | | | | |
| | Arthralgia | | | | | | | | | | | | | | |
| | Headache | | | | | | | | | | | | | | |
| | Rash | | | | | | | | | | | | | | |
| | Fever | | | | | | | | | | | | | | |
| | Sub Total | | | | | | | | | | | | | | |
| UNSOLICITE | System Organ | | | | | | | | | | | | | | |
| D AE | Class(SOC) | | | | | | | | | | | | | | |
| | Preferred Term(PT) | | | | | | | | İ | | | | | | İ |
| | Sub Total | - | | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | | | |

Table 3.1.6 Summary of medically attended AEs for 8 days to 28 days after vaccination

| Safety Set | | AF | E |
|------------|-------------------------|----------------|------------|
| | | Incidence Rate | No. of AEs |
| | | n (%) | n |
| MAAE | System Organ Class(SOC) | | |
| | Preferred Term(PT) | | |
| Total | | | |

Table 3.1.7 Summary of medically attended AEs for 8 days to 28 days after vaccination

| Safety Se | t | AE(2-23mo | onths) | AE(2-10) | N=0 | AE(11-18) | N=0 | AE(19-34) | N=0 | AE(35-55) | N=0 | AE(≥56) N | N=0 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Saicty Sc | ı | N=0 | | | | | | | | | | | |
| | | Incidence | No. | Incidence | No. | Incidence | No. | Incidence | No. | Incidence | No. | Incidence | No |
| | | Rate | of | Rate | of | Rate | of | Rate | of | Rate | of | Rate | |
| | | | AEs | | AEs | | AEs | | AEs | | AEs | | of |
| | | | | | | | | | | | | | A |
| | | | | | | | | | | | | | Es |
| | | n (%) | n | n (%) | n | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| MAAE | System Organ Class(SOC) | | | | | | | | | | | | |
| | Preferred Term(PT) | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | |

Table 3.1.8 Summary of medically attended AEs for 8 days to 28 days after vaccination by study vaccination number (2-23 months)

| Safety Set | | 1 N=0 | | 2 N=0 | | 3 N=0 | | 4 N=0 | |
|---|---|---|---|---|---|---|---|---|---|
| | | Incidence Rate | No. of | Incidence Rate | No. of | Incidence Rate | No. of | Incidence Rate | No. |
| | | | AEs | | AEs | | AEs | | of |
| | | | | | | | | | AEs |
| | | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| MAAE | System Organ Class(SOC) | | | | | | | | |
| | Preferred Term(PT) | | | | | | | | |
| Total | | | | | | | | | |

# 3.2 Safety per protocol set

Table 3.2.1 Summary of solicited AE and unsolicited AE for 7 days after vaccination (<6 years)

| Safety per protocol Set | | AF | Ξ |
|---|---|---|---|
| | | Incidence Rate | No. of AEs |
| | | n (%) | n |
| Local AE | Local AE | | |
| | Injection site tenderness | | |
| | Injection site erythema | | |
| | Injection site induration | | |
| Systemic AE | Systemic AE | | |
| | Change in eating habits | | |
| | Sleepiness | | |
| | Irritability | | |
| | Vomiting | | |
| | Diarrhea | | |
| | Rash | | |
| | Fever | | |
| UNSOLICITED AE | System Organ Class(SOC) | | |
| | Preferred Term(PT) | | |
| | Sub Total | | |
| Total | | | |

Table 3.2.2 Summary of solicited AE and unsolicited AE for 7 days after vaccination (<6 years)

| Safety per protocol Set | | AE(2-23 mon | ths) N=0 | AE(2-5year | s) N=0 |
|---|---|---|---|---|---|
| | | Incidence | No. of | Incidence | No. of |
| | | Rate | AEs | Rate | AEs |
| | | n (%) | n | n (%) | n |
| Local AE | Local AE | | | | |
| | Pain | | | | |
| | Erythema | | | | |
| | Induration | | | | |
| Systemic AE | Systemic AE | | | | |
| | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |
| | Fever | | | | |
| | Sub Total | | | | |
| UNSOLICITED AE | System Organ Class(SOC) | | | | |
| | Preferred Term(PT) | | | | |
| | Sub Total | | | | <u> </u> |
| Total | | | | | |

Table 3.2.3 Summary of solicited AE and unsolicited AE for 7 days after vaccination by study vaccination number (2-23months)

| Safety per protocol Set | | 1 N=0 | | 2 N=0 | | 3 N=0 | | 4 N=0 | |
|---|---|---|---|---|---|---|---|---|---|
| | | Incidence Rate | No. of | Incidence Rate | No. of | Incidence Rate | No. of | Incidence Rate | No. |
| | | | AEs | | AEs | | AEs | | of |
| | | | | | | | | | AEs |
| | | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Local AE | Local AE | | | | | | | | |
| | Pain | | | | | | | | |
| | Erythema | | | | | | | | |
| | Induration | | | | | | | | |
| Systemic AE | Systemic AE | | | | | | | | |
| | Chills | | | | | | | | |
| | Nausea | | | | | | | | |
| | Malaise | | | | | | | | |
| | Myalgia | | | | | | | | |
| | Arthralgia | | | | | | | | |
| | Headache | | | | | | | | |
| | Rash | | | | | | | | |
| | Fever | | | | | | | | |
| | Sub Total | | | | | | | | |
| UNSOLICITED AE | System Organ Class(SOC) | | | | | | | | |
| | Preferred Term(PT) | | | | | | | | |

| Safety per protocol Set | 1 N=0 | | 2 N=0 | | 3 N=0 | | 4 N=0 | |
|---|---|---|---|---|---|---|---|---|
| | Incidence Rate | No. of | Incidence Rate | No. of | Incidence Rate | No. of | Incidence Rate | No. |
| | | AEs | | AEs | | AEs | | of |
| | | | | | | | | AEs |
| | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Sub Total | | | | | | i<br>i | | I |
| Total | | | | | | | | |
Table 3.2.4 Summary of solicited AE and unsolicited AE for 7 days after vaccination (≥6 years)

| Safety per protocol Set | | AI | 3 |
|---|---|---|---|
| | | Incidence Rate | No. of AEs |
| | | n (%) | n |
| Local AE | Local AE | | |
| | Pain | | |
| | Erythema | | |
| | Induration | | |
| Systemic AE | Systemic AE | | |
| | Chills | | |
| | Nausea | | |
| | Malaise | | |
| | Myalgia | | |
| | Arthralgia | | |
| | Headache | | |
| | Rash | | |
| | Fever | | |
| UNSOLICITED AE | System Organ Class(SOC) | | |
| | Preferred Term(PT) | | |
| | Sub Total | | |
| Total | · | | |

Table 3.2.5 Summary of solicited AE and unsolicited AE for 7 days after vaccination (≥6 years)

| Safety per protocol Set | | AE(6-10) N | 1=0 | AE(11-18) N | N=0 | AE(19-34) N | V=0 | AE(35-55) N | N=0 |
|---|---|---|---|---|---|---|---|---|---|
| | | Incidence Rate | No. of | Incidence Rate | No. of | Incidence Rate | No. of | Incidence Rate | No. of |
| | | | AEs | | AEs | | AEs | | AEs |
| | | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Local AE | Local AE | | | | | | | | |
| | Pain | | | | | | | | |
| | Erythema | | | | | | | | |
| | Induration | | | | | | | | |
| Systemic AE | Systemic AE | | | | | | | | |
| | Chills | | | | | | | | |
| | Nausea | | | | | | | | |
| | Malaise | | | | | | | | |
| | Myalgia | | | | | | | | |
| | Arthralgia | | | | | | | | |
| | Headache | | | | | | | | |
| | Rash | | | | | | | | |
| | Fever | | | | | | | | |
| | Sub Total | | | | | | | | |
| UNSOLICITED AE | System Organ Class(SOC) | | | | | | | | |
| | Preferred Term(PT) | | | | | | <u> </u> | | |

| Safety per protocol Set | AE(6-10) N | AE(6-10) N=0 | | AE(11-18) N=0 | | N=0 | AE(35-55) N=0 | |
|---|---|---|---|---|---|---|---|---|
| | Incidence Rate | No. of | Incidence Rate | No. of | Incidence Rate | No. of | Incidence Rate | No. of |
| | | AEs | | AEs | | AEs | | AEs |
| | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Sub Total | | | | | | | | |
| Total | | | | | | | | |

Table 3.2.6 Summary of medically attended AEs for 8 days to 28 days after vaccination

| Safety per protocol S | et | AI | 3 |
|---|---|---|---|
| | | Incidence Rate | No. of AEs |
| | | n (%) | n |
| MAAE | System Organ Class(SOC) | | |
| | Preferred Term(PT) | | |
| Total | | | |

Table 3.2.7 Summary of medically attended AEs for 8 days to 28 days after vaccination

| Safety per | protocol Set | AE(2-23months | s) N=0 | AE(2-10) | N=0 | AE(11-18) | N=0 | AE(19-34) | N=0 | AE(35-55) | N=0 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Incidence Rate | No. | Incidence | No. | Incidence | No. | Incidence | No. | Incidence | No. |
| | | | of | Rate | of | Rate | of | Rate | of | Rate | of |
| | | | AEs | | AEs | | AEs | | AEs | | AEs |
| | | n (%) | n | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| MAAE | System Organ Class(SOC) | | | | | | | | | | |
| | Preferred Term(PT) | - | | | | | | | | | |
| Total | | | | | | | | | | | |

Table 3.2.8 Summary of medically attended AEs for 8 days to 28 days after vaccination by study vaccination number (2-23 months)

| Safety per | protocol Set | 1 | N=0 | | 2 | N=0 | | | 3 N=0 | | | 4 N=0 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Incidence | Rate | No. of | Incidence R | late | No. of | Incider | nce Rate | No. of | Incide | nce Rate | No. of |
| | | | | AEs | | | AEs | | | AEs | | | AEs |
| | | n (% | 6) | n | n (% | ) | n | n | (%) | n | n | (%) | n |
| MAAE | System Organ Class(SOC) | | | | | | | | | | | | |
| | Preferred Term(PT) | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | |

#### 4. Solicited AE (DAY 1-7)

Table 4.1.1 Summary of Local AE Max severity (<6 years)

| Safety Set | | 1*<br>n (%) | 2*<br>n (%) | 3*<br>n (%) | 4*<br>n (%) | Total n (%) |
|---|---|---|---|---|---|---|
| Local AE | Injection site tenderness Injection site erythema | | | | | |
| | Injection site induration | | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Injection site tenderness

Table 4.1.2 Summary of Local AE Max severity (≥6 years)

| Safety Set | | 1* | 2* | 3* | 4* | Total |
|---|---|---|---|---|---|---|
| | | n (%) | n (%) | n (%) | n (%) | n (%) |
| Local AE | Injection site pain | | | | | |
| | Injection site erythema | | | | | |
| | Injection site induration | | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Injection site pain

Table 4.1.3 Summary of Local AE by Max severity

| Safety Set | | 1* | 2* | 3* | 4* | Total |
|---|---|---|---|---|---|---|
| | | n (%) | n (%) | n (%) | n (%) | n (%) |
| Age (2-23 months) | Injection site tenderness | | | | | |
| | Injection site erythema | | | | | |
| | Injection site induration | | | | | |
| Age (2-5) | Injection site tenderness | | | | | |
| | Injection site erythema | | | | | |
| | Injection site induration | | | | | |
| Age (6-10) | Injection site pain | | | | | |

<sup>\* 0-9(1), 10-25(2), 26-50(3), &</sup>gt;50(4): Injection site erythema, Injection site induration

<sup>\* 1-24(1), 25-50(2), 51-100(3), &</sup>gt;100(4): Injection site erythema, Injection site induration

| Safety Set | | 1* | 2* | 3* | 4* | Total |
|---|---|---|---|---|---|---|
| | | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Injection site erythema | | | | | |
| | Injection site induration | | | | | |
| Age (11-18) | Injection site pain | | | | | |
| | Injection site erythema | | | | | |
| | Injection site induration | | | | | |
| Age (19-34) | Injection site pain | | | | | |
| | Injection site erythema | | | | | |
| | Injection site induration | | | | | |
| Age (35-55) | Injection site pain | | | | | |
| | Injection site erythema | | | | | |
| | Injection site induration | | | | | |
| Age (≥56) | Injection site pain | | | | | |
| | Injection site erythema | | | | | |
| | Injection site induration | | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Injection site tenderness, Injection site pain

Table 4.1.4 Summary of Systemic AE by Max severity (<6 years)

| Safety Set | | 1* | 2* | 3* | Total |
|-------------|-------------------------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) |
| Systemic AE | Change in eating habits | | | | |
| | Sleepiness | | | | |
| | Irritability | | | | |
| | Vomiting | | | | |
| | Diarrhea | | | | |
| | Rash | | | | |
| | Fever | | | | |

 $<sup>*\</sup> Mild (1),\ Moderate (2),\ Severe (3): Change\ in\ eating\ habits,\ Sleepiness,\ irritability,\ vomiting,\ diarrhea,$ 

<sup>\* 0-9(1), 10-25(2), 26-50(3),</sup> >50(4) : Injection site erythema, Injection site induration (Age < 6 years)

<sup>\* 1-24(1), 25-50(2), 51-100(3),</sup> >100(4): Injection site erythema, Injection site induration (Age  $\geq$  6 years)

<sup>\*</sup> None(1), Urticarial(2), Other(3): Rash

 $<sup>* \</sup>ge 38^{\circ}C(1)$ : Fever

Table 4.1.5 Summary of Systemic AE by Max severity(≥6 years)

| Safety Set | | 1* | 2* | 3* | Total |
|-------------|------------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) |
| Systemic AE | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |
| | Fever | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Chills, Nausea, Malaise, Myalgia, Arthralgia, Headache

Table 4.1.6 Summary of Systemic AE by Max severity

| Safety Set | | 1* | 2* | 3* | Total |
|---|---|---|---|---|---|
| | | n (%) | n (%) | n (%) | n (%) |
| Age (2-23 months) | Change in eating habits | | | | |
| | Sleepiness | | | | |
| | Irritability | | | | |
| | Vomiting | | | | |
| | Diarrhea | | | | |
| | Rash | | | | |
| | Fever | | | | |
| Age (2-5) | Change in eating habits | | | | |
| | Sleepiness | | | | |
| | Irritability | | | | |
| | Vomiting | | #<br>=<br>=<br>= | | |
| | Diarrhea | | | | |
| | Rash | | | | |
| | Fever | | | | |
| Age (6-10) | Chills | | | | |
| | Nausea | | | | |

<sup>\*</sup>None(1), Urticarial(2), Other(3): Rash

 $<sup>* \</sup>ge 38^{\circ}C(1)$ : Fever

| Safety Set | | 1* | 2* | 3* | Total |
|-------------|------------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |
| | Fever | | | | |
| Age (11-18) | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |
| | Fever | | | | |
| Age (19-34) | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |
| | Fever | | | | |
| Age (35-55) | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |
| | Fever | | | | |
| Age (≥56) | Chills | | | | |
| - , / | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |

| Safety Set | | 1* | 2* | 3* | Total |
|------------|------------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |
| | Fever | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Chills, Nausea, Malaise, Myalgia, Arthralgia, Headache, Change in eating habits, Sleepiness, irritability, vomiting, diarrhea,

Table 4.1.7 Summary of Solicited AE by day (<6 years)

| Safety Set | | 30 min | 6hr | 2 days | 3 days | 4 days | 5 days | 6 days | 7 days | Tot | al |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n ( | (%<br>) |
| Solicited AE | Local AE | | | | | | | | | | |
| | Injection site | | | | | | | | ************************************** | | |
| | tenderness | | | | | | | | | | |
| | Injection site | | | | | | | | | | |
| | erythema | | | | | | | | | | |
| | Injection site | | | | | | # | | | | |
| | induration | | | | | | | | | | |
| | Systemic AE | | | | | | | | | | |
| | Change in eating | | | | | | | | | | |
| | habits Sleepiness | | | | | | | | | | |
| | Irritability | | | | | | | | | | |
| | Vomiting | | | | | | | | | | |
| | Diarrhea | | | | | | | | | | |
| | Rash | | | | | | | | | | |
| | Fever | | | | | | | | | | |
| Total | L | | | | | | | | | | |

<sup>\*</sup>None(1), Urticarial(2), Other(3): Rash

 $<sup>* \</sup>ge 38$ °C(1): Fever

Table 4.1.8 Summary of Solicited AE by day (≥6 years)

| Safety Set | | 30 min | 6hr | 2 days | 3 days | 4 days | 5 days | 6 days | 7 days | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| | | n (% | n (% | n (% | n (% | n (% | n (% | n (% | n (% | n (% |
| Solicited<br>AE | Local AE | | | | | | | | | |
| | Injection site pain | | | | | | | | | |
| | Injection site | | | | | | | | | |
| | erythema | | | | | | | | | |
| | Injection site | | | | | | | | | |
| | induration | | | | | | | | | |
| | Systemic AE | | | | | | | | | |
| | Chills | | | | | | | | | |
| | Nausea | | | | | | | | | |
| | Malaise | | | | | | | | | |
| | Myalgia | | | | | | | | | |
| | Arthralgia | | | | | | | | | |
| | Headache | | | | | | | | | |
| | Rash | | | | | | | | | |
| | Fever | | | | | | | | | |
| Total | | | | | | | | | | |

Table 4.1.9 Summary of Solicited AE by day

| Safety Set | Safety Set | | 6hı | ſ | 2 days | 3 days | 4 days | 5 days | 6 days | 7 days | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n (%) | n | (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n%) |
| Age (2-23 months) | Injection site tenderness | | | | | | | | | | |
| | Injection site erythema | | | | | | | | | | |
| | Injection site induration | | | | | | | | | | |
| Age (2-5) | Injection site tenderness | | | | | | | | | | |
| | Injection site erythema | | | | | | | | | | |
| | Injection site induration | | | | | | | | | | |
| Age (6-10) | Injection site pain | | | | | | | | | | |
| | Injection site erythema | | | | | | | | | | |

| Safety Set | | 30 min | 6hr | | 2 days | 3 days | 4 days | 5 days | 6 days | 7 days | Tota |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n (%) | n | (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n%) |
| | Injection site induration | | | | | | | | | | |
| Age (11-18) | Injection site pain | | | | | | | | | | |
| | Injection site erythema | | | | | | | | | | |
| | Injection site induration | | | | | | | | | | |
| Age (19-34) | Injection site pain | | | | | | | | | | |
| | Injection site erythema | | | | | | | | | | |
| | Injection site induration | | | | | | | | | | |
| Age (35-55) | Injection site pain | | | | | | | | | | |
| | Injection site erythema | | | | | | | | | | |
| | Injection site induration | | | | | | | | | | |
| Age (≥56) | Injection site pain | | | | | | | | | | |
| | Injection site erythema | | | | | | | | | | |
| | Injection site induration | | | | | | | | | | |
| | Sub Total | | | | | | | | | | |
| Age (2-23 months) | Change in eating habits | | | | | | | | | | |
| | Sleepiness | | | | | | | | | | |
| | Irritability | | | | | | | | | | |
| | Vomiting | | | | | | | | | | |
| | Diarrhea | | | | | | | | | | |
| | Rash | | | | | | | | | | |
| | Fever | | | | | | | | | | |
| Age (2-5) | Change in eating habits | | | | | | | | | | |
| | Sleepiness | | | | | | | | | | |
| | Irritability | | | | | | | | | | |
| | Vomiting | | | | | | | | | | |
| | Diarrhea | | | | | | | | | | |
| | Rash | | | | | | | | | | |
| | Fever | | | | | | | | | | |
| Age (6-10) | Chills | | | | | | | | | | |
| | Nausea | | | | | | | | | | |
| | Malaise | | | | | | | | | | |
| | Myalgia | | | | | | | | | | |
| | Arthralgia | | | | | | | | | | |

| Safety Set | | 30 min | 6h | nr | 2 days | 3 days | 4 days | 5 days | 6 days | 7 days | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n (%) | n | (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n%) |
| | Headache | | | | | | | | | | |
| | Rash | | | | | | | | | | |
| | Fever | | | | | | | | | | |
| Age (11-18) | Chills | | | | | | | | | | |
| | Nausea | | | | | | | | | | |
| | Malaise | | | | | | | | | | |
| | Myalgia | | | | | | | | | | |
| | Arthralgia | | | | | | | | | | |
| | Headache | | | | | | | | | | |
| | Rash | | | | | | | | | | |
| | Fever | | | | | | | | | | |
| Age(19-34) | Chills | | | | | | | | | | |
| | Nausea | | | | | | | | | | |
| | Malaise | | | | | | | | | | |
| | Myalgia | | | | | | | | | | |
| | Arthralgia | | | | | | | | | | |
| | Headache | | | | | | | | | | |
| | Rash | | | | | | | | | | |
| | Fever | | | | | | | | | | |
| Age (35-55) | Chills | | | | | | | | | | |
| | Nausea | | | | | | | | | | |
| | Malaise | | | | | | | | | | |
| | Myalgia | | | | | | | | | | |
| | Arthralgia | | | | | | | | | | |
| | Headache | | | | | | | | | | |
| | Rash | | | | | | | | | | |
| | Fever | | | | | | | | | | |
| Age (≥56) | Chills | | | | | | | | | | |
| | Nausea | | | | | | | | | | |
| | Malaise | | | | | | | | | • | |
| | Myalgia | | | | | | | | | | |
| | Arthralgia | | | | | | | | | | |
| | Headache | | | | | | | | | | |
| | Rash | | | | | | | | | | |

| Safety Set | | 30 | min | 6h | r | 2 | days | 3 | days | 4 | days | 5 | days | 6 | days | 7 days | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n (%) | n%) |
| | Fever | | | | | | | | | | | | | | | | |
| | Sub Total | | | | | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | | | | | |

Table 4.1.10 Summary of Fever

| Safety Set | | 2-<br>23mo | onths | 2-10 | | 11-18 | | 19-34 | 1 | 35-55 | ; | ≥ 56 | | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n (%) |
| | Fever | | | | | | | | | | | | | |
| | No fever | | | | | | | | | | | | | |
| | Total | | | | | | | | | | | | | |
| Temperature(°C) | 36-36.5 | | | | | | | | | | | | | |
| | 36.5-37 | | | | | | | | | | | | | |
| | 37-37.5 | | | | | | | | | | | | | |
| | 37.5-38 | | | | | | | | | | | | | |
| | 38-38.5 | | | | | | | | | | | | | |
| | 38.5-39 | | | | | | | | | | | | | |
| | 39-39.5 | | | | | | | | | | | | | |
| | 39.5-40 | | | | | | | | | | | | | |
| | >40 | | | | | | | | | | | | | |

Table 4.2.1 Summary of local AE by Max severity (<6 years)

| Safety per protoc | ool Set | 1*<br>n (%) | 2*<br>n (%) | 3*<br>n (%) | 4*<br>n (%) | Total<br>n (%) |
|---|---|---|---|---|---|---|
| Local AE | Injection site tenderness Injection site erythema Injection site induration | | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Injection site tenderness

Table 4.2.2 Summary of Local AE Max severity (≥6 years)

| Safety per prot | Safety per protocol Set | | 2* | 3* | 4* | Total |
|---|---|---|---|---|---|---|
| | | n (%) | n (%) | n (%) | n (%) | n (%) |
| Local AE | Injection site pain | | | | | |
| | Injection site erythema | | | | | |
| | Injection site induration | | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Injection site pain

Table 4.2.3 Summary of Local AE by Max severity

| Safety per protocol Se | t | 1* | ķ | | 2* | | 3* | 4 | .* | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| | | n | (%) | n | (%) | n | (%) | n | (%) | n (%) |
| Age (2-23 months) | Injection site tenderness | | | | | | | | | |
| | Injection site erythema | | | | | | | | | |
| | Injection site induration | | | | | | | | | |
| Age (2-5) | Injection site tenderness | | | | | | | | | |
| | Injection site erythema | | | | | | | | | |
| | Injection site induration | | | | | | | | | |
| Age (6-10) | Injection site pain | | | | | | | | | |
| | Injection site erythema | | | | | | | | | |
| | Injection site induration | | | | | | | | | |

<sup>\* 0-9(1), 10-25(2), 26-50(3), &</sup>gt;50(4): Injection site erythema, Injection site induration

<sup>\* 1-24(1), 25-50(2), 51-100(3), &</sup>gt;100(4): Injection site erythema, Injection site induration

| Safety per protocol | Set | 1* | 2* | 3* | 4* | Total |
|---|---|---|---|---|---|---|
| | | n (%) | n (%) | n (%) | n (%) | n (%) |
| Age (11-18) | Injection site pain | | | | | |
| | Injection site erythema | | | | | |
| | Injection site induration | | | | 3 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 | |
| Age (19-34) | Injection site pain | | | | | |
| | Injection site erythema | | | | | |
| | Injection site induration | | | | | |
| Age (35-55) | Injection site pain | | | | | |
| | Injection site erythema | | | | | |
| | Injection site induration | | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Injection site tenderness, Injection site pain

Table 4.2.4 Summary of Systemic AE by Max severity (<6 years)

| Safety per protoco | l Set | 1* | 2* | 3* | Total |
|--------------------|-------------------------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) |
| Systemic AE | Change in eating habits | | | | |
| | Sleepiness | | | | |
| | Irritability | | | | |
| | Vomiting | | | | |
| | Diarrhea | | | | |
| | Rash | | | | |
| | Fever | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Change in eating habits, Sleepiness, irritability, vomiting, diarrhea,

<sup>\* 0-9(1), 10-25(2), 26-50(3), &</sup>gt;50(4): Injection site erythema, Injection site induration (Age < 6 years)

<sup>\* 1-24(1), 25-50(2), 51-100(3),</sup> >100(4): Injection site erythema, Injection site induration (Age  $\geq$  6 years)

<sup>\*</sup>None(1), Urticarial(2), Other(3): Rash

 $<sup>* \</sup>ge 38$ °C(1): Fever

Table 4.2.5 Summary of Systemic AEs by Max severity (≥6 years)

| Safety per protoc | col Set | 1* | 2* | 3* | Total |
|-------------------|------------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) |
| Systemic AE | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |
| | Fever | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Chills, Nausea, Malaise, Myalgia, Arthralgia, Headache

Table 4.2.6 Summary of Systemic AE by Max severity

| Safety per protocol Set | | 1* | 2* | 3* | Total |
|---|---|---|---|---|---|
| | | n (%) | n (%) | n (%) | n (%) |
| Age (2-23 months) | Change in eating habits | | | | |
| | Sleepiness | | | | |
| | Irritability | | | | |
| | Vomiting | | | | |
| | Diarrhea | | | | |
| | Rash | | | | |
| | Fever | | | | |
| Age (2-5) | Change in eating habits | | | | |
| | Sleepiness | | | | |
| | Irritability | | | | |
| | Vomiting | | | | |
| | Diarrhea | | | | |
| | Rash | | | | |
| | Fever | | | | |
| Age (6-10) | Chills | | | | |
| | Nausea | | | | |

<sup>\*</sup>None(1), Urticarial(2), Other(3): Rash

 $<sup>* \</sup>ge 38^{\circ}C(1)$ : Fever

| Safety per protoco | ol Set | 1* | 2* | 3* | Total |
|--------------------|------------|-------|-------|-------|-------|
| | | n (%) | n (%) | n (%) | n (%) |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |
| | Fever | | | | |
| Age (11-18) | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |
| | Fever | | | | |
| Age (19-34) | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |
| | Fever | | | | |
| Age (35-55) | Chills | | | | |
| | Nausea | | | | |
| | Malaise | | | | |
| | Myalgia | | | | |
| | Arthralgia | | | | |
| | Headache | | | | |
| | Rash | | | | |
| | Fever | | | | |

<sup>\*</sup> Mild(1), Moderate(2), Severe(3): Chills, Nausea, Malaise, Myalgia, Arthralgia, Headache, Change in eating habits, Sleepiness, irritability, vomiting, diarrhea,

<sup>\*</sup>None(1), Urticarial(2), Other(3): Rash

 $<sup>* \</sup>ge 38$ °C(1): Fever

Table 4.2.7 Summary of Solicited AE by day (<6 years)

| Safety per prot | tocol Set | 30 min | 6hr | 2 days | 3 days | 4 days | 5 days | 6 days | 7 days | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| | | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (% |
| Solicited AE | Local AE | | | | | | | | | |
| | Injection site | | | | | | | | | |
| | tenderness | | | | | | | | | |
| | Injection site | | | | | | | | | |
| | erythema | | | | | | | | | |
| | Injection site | | | | | | | | | |
| | induration | | | | | | | | | |
| | Systemic AE | | | | | | | | | |
| | Change in eating | | | | | | | | | |
| | habits Sleepiness | | | | | | | | | |
| | Irritability | | | | | | | | | |
| | Vomiting | | | | | | | | | |
| | Diarrhea | | | | | | | | | |
| | Rash | | | | | | | | | |
| | Fever | | | | | | | | | |
| Total | | | | | | | | | | |

Table 4.2.8 Summary of Solicited AE by day (≥6 years)

| Safety per p | rotocol Set | 30 min | 6hr | 2 days | 3 days | 4 days | 5 days | 6 days | 7 days | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| | | n (% | n (% | n (% | n (% | n (% | n (% | n (% | n (% | n (% |
| Solicited<br>AE | Local AE | | | | | | | | | |
| | Injection site pain | | | | | | | | | |
| | Injection site erythema Injection site | | | | | | | | | |
| | induration | | | | | | | | | |
| | Systemic AE | | | | | | | | | |

| | Chills |
|-------|------------|
| | Nausea |
| | Malaise |
| | Myalgia |
| | Arthralgia |
| | Headache |
| | Rash |
| | Fever |
| Total | |

Table 4.2.9 Summary of Solicited AE by day

| Safety per proto | ocol Set | 30 | min | | 6hr | 2 days | 3 days | 4 days | 5 days | 6 days | 7 days | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | (%) | n | (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n%) |
| Age (2-23 months) | Injection site tenderness | | | | | | | | H H H H H H H H H H H H H H H H H H H | | | |
| | Injection site erythema | | | | | | | | | | | |
| | Injection site induration | | | | | | | | | | | |
| Age (2-5) | Injection site tenderness | | | | | | | | | | | |
| | Injection site erythema | | | | | | | | | | | |
| | Injection site induration | | | | | | | | | | | |
| Age (6-10) | Injection site pain | | | | | | | | | | | |
| | Injection site erythema | | | | | | | | | | | |
| | Injection site induration | | | | | | | | | | | |
| Age (11-18) | Injection site pain | | | | | | | | | | | |
| | Injection site erythema | | | | | | | | | | | |
| | Injection site induration | | | | | | | | | | | |
| Age (19-34) | Injection site pain | | | | | | | | | | | |
| | Injection site erythema | | | | | | | | | | | |
| | Injection site induration | | | | | | | | | | | |
| Age (35-55) | Injection site pain | | | | | | | | | | | |
| | Injection site erythema | | | | | | | | | | | |
| | Injection site induration | | | | | | | | | | | |
| Age (2-23 months) | Change in eating habits | | | | | | | | | | | |
| | Sleepiness | | | | | | | | | | | |

| Safety per prot | ocol Set | 30 | 0 min | | 6hr | 2 days | 3 days | 4 days | 5 days | 6 days | 7 days | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | (%) | n | (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n%) |
| | Irritability | | | | | | | | | | | |
| | Vomiting | | | | | | | | | | | |
| | Diarrhea | | | | | | | | | | | |
| | Rash | | | | | | | | | | | |
| | Fever | | | | | | | | | | | |
| Age (2-5) | Change in eating habits | | | | | | | | | | | |
| | Sleepiness | | | | | | | | | | | |
| | Irritability | | | | | | | | | | | |
| | Vomiting | | | | | | | | | | | |
| | Diarrhea | | | | | | | | | | | |
| | Rash | | | | | | | | | | | |
| | Fever | | | | | | | | | | | |
| Age (6-10) | Chills | | | | | | | | | | | |
| | Nausea | | | | | | | | | | | |
| | Malaise | | | | | | | | | | | |
| | Myalgia | | | | | | | | | | | |
| | Arthralgia | | | | | | | | | | | |
| | Headache | | | | | | | | | | | |
| | Rash | | | | | | | | | | | |
| | Fever | | | | | | | | | | | |
| Age (11-18) | Chills | | | | | | | | | | | |
| | Nausea | | | | | | | | | | | |
| | Malaise | | | | | | | | | | | |
| | Myalgia | | | | | | | | | | | |
| | Arthralgia | | | | | | | | | | | |
| | Headache | | | | | | | | | | | |
| | Rash | | | | | | | | | | | |
| | Fever | | | | | | | | | | | |
| Age (19-34) | Chills | | | | | | | | | | | |
| | Nausea | | | | | | | | | | | |
| | Malaise | | | | | | | | | | | |
| | Myalgia | | | | | | | | | | | |
| | Arthralgia | | | | | | | | | | | |
| | Headache | | | | | | | | | | | |

| Safety per prot | ocol Set | 30 | min | | 6hr | 2 days | 3 days | 4 days | 5 days | 6 days | 7 days | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | (%) | n | (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n%) |
| | Rash | | | | | | | | | | | |
| | Fever | | | | | | | | | | | |
| Age (35-55) | Chills | | | | | | | | | | | |
| | Nausea | | | | | | | | | | | |
| | Malaise | | | | | | | | | | | |
| | Myalgia | | | | | | | | | | | |
| | Arthralgia | | | | | | | | | | | |
| | Headache | | | | | | | | | | | |
| | Rash | | | | | | | | | | | |
| | Fever | | | | | | | | | | | |
| | Sub Total | | | | | | | | | | | |
| Total | | | | | | | | | | | | |

Table 4.2.10 Summary of Fever

| Safety per protocol Set | | 2-23months<br>n (%) | 2-10<br>n (%) | 11-18<br>n (%) | 19-34<br>n (%) | 35-55<br>n (%) | Total<br>n (%) |
|---|---|---|---|---|---|---|---|
| | Fever | | | | | | |
| | No fever | | | | | | |
| | Total | | | | | | |
| Temperature(°C) | 36-36.5 | | | | | | |
| | 36.5-37 | | | | | | |
| | 37-37.5 | | | | | | |
| | 37.5-38 | | | | | | |
| | 38-38.5 | | | | | | |
| | 38.5-39 | | | | | | |
| | 39-39.5 | | | | | | |
| | 39.5-40 | | | | | | |
| | >40 | | | • | | | |

# 5. Unsolicited AE (DAY 1-7)

Table 5.1.1 Summary of Unsolicited AE

| Safety Set | | 2-23 n | nonths | 2-1 | 0 | 11 | -18 | 19 | -34 | 35 | 5-55 | ≥ | 56 | T | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | No.<br>AEs | (%) | No. AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) |
| Expected | Expected AE | | | | | | | | | | | | | | |
| | Unexpected AE | | | | | | | | | | | | | | |
| Serious | Yes | | | | | | | | | | | | | | |
| | No | | | | | | | | | | | | | | |
| Severity | Mild | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | |
| Frequency | Single/Continuous | | | | | | | | | | | | | | |
| | Intermittent | | | | | | | | | | | | | | |
| Action Taken | None | | | | | | | | | | | | | | |
| | Uncertain | | | | | | | | | | | | | | |
| | Procedure or physical therapy | | | | | | | | | | | | | | |
| | Blood or blood products | | | | | | | | | | | | | | |
| | Withdrawn from study due to AE | | | | | | | | | | | | | | |
| | Prescription drug therapy | | | | | | | | | | | | | | |

| Safety Set | | 2-23 n | nonths | 2-1 | 0 | 11 | -18 | 19 | -34 | 35 | 5-55 | ≥ | 56 | To | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | No. | (%) | No. AEs | (%) | No. | (%) | No. | (%) | No. | (%) | No. | (%) | No. | (%) |
| | | AEs | (, , | 110.7125 | (70) | AEs | (, , | AEs | (, , | AEs | (, , | AEs | | AEs | (, , |
| | Non-prescription drug therapy | | | | | | | | | | | | | | |
| | Hospitalization | | | | | | | | | | | | | | |
| | IV fluids | | | | | | | | | | | | | | |
| | Physician visit | | | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | | | |
| Outcome | Complete recovery/Return to baseline | | | | | | | | | | | | | | |
| | Alive with sequelae | | | | | | | | | | | | | | |
| | Death | | | | | | | | | | | | | | |
| | Unknown/Lost to follow-up | | | | | | | | | | | | | | |
| | AE persisting | | | | | | | | | | | | | | |
| Relationship to | Network | | | | | | | | | | | | | | |
| study vaccine | Not related | | | | | | | | | | | | | | |
| | Possibly related | | | | | | | | | | | | | | |
| | Probably related | | | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | | | |

Table 5.2.1 Summary of Unsolicited AE

| Safety per protocol<br>Set | | 2-23 | months | 2-1 | 0 | 1 | 1-18 | 19 | 9-34 | 3. | 5-55 | T | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <b>5.</b> | | No.<br>AEs | (%) | No. AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) |
| Expected | Expected AE | | | | | | | | | | | | |
| | Unexpected AE | | | | | | | | | | | | |
| Serious | Yes | | | | | | | | | | | | |
| | No | | | | | | | | | | | | |
| Severity | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Frequency | Single/Continuous | | | | | | | | | | | | |
| | Intermittent | | | | | | | | | | | | |
| Action Taken | None | | | | | | | | | | | | |
| | Uncertain | | | | | | | | | | | | |
| | Procedure or physical therapy | | | | | | | | | | | | |
| | Blood or blood products | | | | | | | | | | | | |
| | Withdrawn from study due to AE | | | | | | | | | | | | |
| | Prescription drug therapy | | | | | | | | | | | | |
| | Non-prescription drug therapy | | | | | | | | | | | | |

| Safety per protocol<br>Set | | 2-23 | months | 2-1 | 0 | 1 | 1-18 | 1 | 9-34 | 35 | 5-55 | Т | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | No.<br>AEs | (%) | No. AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) |
| | Hospitalization IV fluids Physician visit | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | |
| Outcome | Complete recovery/Return to baseline Alive with sequelae Death Unknown/Lost to follow-up AE persisting | | | | | | | | | | | | |
| Relationship to study vaccine | Not related Possibly related Probably related | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | |

# 6. MAAE (DAY 8-29)

Table 6.1.1 Summary of MAAE

| Safety Set | | 2-23 m | onths | 2-1 | 0 | 11 | -18 | 19 | <b>)-34</b> | 35 | 5-55 | ≥ | 56 | To | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | No.<br>AEs | (%) | No. AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) |
| Expected | Expected AE | | | | | | | | | | | | | | |
| | Unexpected AE | | | | | | | | | | | | | | |
| Serious | Yes | | | | | | | | | | | | | | |
| | No | | | | | | | | | | | | | | |
| Severity | Mild | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | |
| Frequency | Single/Continuous | | | | | | | | | | | | | | |
| | Intermittent | | | | | | | | | | | | | | |
| Action Taken | None | | | | | | | | | | | | | | |
| | Uncertain | | | | | | | | | | | | | | |
| | Procedure or physical therapy | | | | | | | | | | | | | | |
| | Blood or blood products | | | | | | | | | | | | | | |
| | Withdrawn from study due to AE | | | | | | | | | | | | | | |
| | Prescription drug therapy | | | | | | | | | | | | | | |

| Safety Set | | 2-23 r | nonths | 2-1 | 0 | 11 | -18 | 19 | -34 | 35 | 5-55 | ≥ | 56 | To | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | No. | (%) | No. AEs | (%) | No. | (%) | No. | (%) | No. | (%) | No. | (%) | No. | (%) |
| | | AEs | () | 110.1125 | (/*) | AEs | (* -) | AEs | () | AEs | () | AEs | . , | AEs | () |
| | Non-prescription drug therapy | | | | | | | | | | | | | | |
| | Hospitalization | | | | | | | | | | | | | | |
| | IV fluids | | | | | | | | | | | | | | |
| | Physician visit | | | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | | | |
| Outcome | Complete recovery/Return to baseline | | | | | | | | | | | | | | |
| | Alive with sequelae | | | | | | | | | | | | | | |
| | Death | | | | | | | | | | | | | | |
| | Unknown/Lost to follow-up | | | | | | | | | | | | | | |
| | AE persisting | | | | | | | | | | | | | | |
| Relationship to | Netherland | | | | | | | | | | | | | | |
| study vaccine | Not related | | | | | | | | | | | | | | |
| | Possibly related | | | | | | | | | | | | | | |
| | Probably related | | | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | | | |

Table 6.2.1 Summary of MAAE

| Safety per protocol<br>Set | | 2-23 | months | 2-1 | 0 | 1 | 1-18 | 19 | 9-34 | 3. | 5-55 | T | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <b>5.</b> | | No.<br>AEs | (%) | No. AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) | No.<br>AEs | (%) |
| Expected | Expected AE | | | | | | | | | | | | |
| | Unexpected AE | | | | | | | | | | | | |
| Serious | Yes | | | | | | | | | | | | |
| | No | | | | | | | | | | | | |
| Severity | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Frequency | Single/Continuous | | | | | | | | | | | | |
| | Intermittent | | | | | | | | | | | | |
| Action Taken | None | | | | | | | | | | | | |
| | Uncertain | | | | | | | | | | | | |
| | Procedure or physical therapy | | | | | | | | | | | | |
| | Blood or blood products | | | | | | | | | | | | |
| | Withdrawn from study due to AE | | | | | | | | | | | | |
| | Prescription drug therapy | | | | | | | | | | | | |
| | Non-prescription drug therapy | | | | | | | | | | | | |

| Safety per protocol<br>Set | | 2-23 months | 2-10 | 11-18 | 19-34 | 35-55 | Total |
|---|---|---|---|---|---|---|---|
| | | No. (%)<br>AEs | No. AEs (%) | No.<br>(%)<br>AEs | No.<br>(%)<br>AEs | No.<br>(%)<br>AEs | No.<br>(%)<br>AEs |
| | Hospitalization IV fluids Physician visit Other | | | | | | |
| Outcome | Complete recovery/Return to baseline Alive with sequelae Death Unknown/Lost to follow-up AE persisting | | | | | | |
| Relationship to study vaccine | Not related Possibly related Probably related | | | | | | |
| Total | | | | | | | |

### 7. SAE/SADR for 28 days after vaccination

Table 7.1.1 SAE and SADR

| | 2- | -23 r | nonths | | | 2- | 10 | | | 11 | -18 | | | 19 | -34 | | | 35 | -55 | | | ≥5 | 56 | | | To | tal | _ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety Set | Seriou<br>AE | S | Seriou<br>ADR | S | Serious<br>AE | S | Seriou:<br>ADR | S | Seriou<br>AE | S | Seriou<br>ADR | S | Seriou<br>AE | S | Seriou<br>ADR | S | Serious<br>AE | 5 | Serious<br>ADR | S | Serious<br>AE | S | Seriou<br>ADR | s | Serio<br>us A | - 1 | Serio<br>us<br>ADR | |
| | | | | | | | | | | | | - | | | | | | | | | | | | N | | N | | N |
| | | N | | N | | N | | N | | N | | N | | N | | N | | N | | N | | N | | o | | 0 | | o |
| | | o | | 0 | | o | | o | | o | | o | | o | | o | | o | | О | | o | | | Inc | ٠ | Inc | |
| | Incid | | Incid | | Incid | • | Incid | • | Incid | | Incid | | Incid | | Incid | • | Incid | • | Incid | • | Incid | | Incid | | ide | | ide | |
| | ence | o<br>f | ence | o<br>f | ence | o<br>f | ence | o<br>f | ence | 0<br>f | ence | o<br>f | ence | o<br>f | ence | o<br>f | ence | o<br>f | ence | o<br>f | ence | 0<br>f | ence | 0 | nc | | | 0 |
| | Rate | ı<br>A | Rate | A | Rate | ı<br>A | Rate | ı<br>A | Rate | ı<br>A | Rate | A | Rate | ı<br>A | Rate | ı<br>A | Rate | ı<br>A | Rate | ı<br>A | Rate | ı<br>A | Rate | 1 | e<br>Ra | - | e<br>Ra | 1 |
| | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | A | | | | A |
| | | s | | s | | s | | s | | s | | s | | s | | s | | s | | s | | s | | Е | | Е | | Е |
| | | | | | | | | | | | | | | | | | | | | | | | | s | | s | | S |
| | ( | | ( | | | | | | ( | | ( | | ( | | | | ( | | ( | | ( | | | | ( | | ( | _ |
| | n % | n | n % | n | n | | | n | n % | n | n % | n | n % | | | n | n % | n | n % | n | n % | | | n | n <sup>o</sup> | ⁄6 n | n % n | |
| | ) | | ) | | | | | | ) | | ) | | ) | | | | ) | | ) | | ) | | | | ) | | ) | _ |
| System Organ | 1 | | | | | | | | | <u> </u> | | | | | : | | | | =<br>=<br>=<br>=<br>= | | | | | | | | | |

| | 2. | -23 r | nonths | | | 2- | 10 | | | 11- | -18 | | | 19- | -34 | | | 35- | -55 | | | ≥5 | 56 | | | Tota | al | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety Set | Seriou<br>AE | ıs | Seriou<br>ADR | S | Serious<br>AE | 3 | Serious<br>ADR | 3 | Serious<br>AE | 5 | Serious<br>ADR | S | Serious<br>AE | S | Seriou<br>ADR | s | Serious<br>AE | 5 | Serious<br>ADR | S | Seriou:<br>AE | 5 | Serious<br>ADR | S | Serio<br>us Al | E | Serio<br>us<br>ADR | |
| Class(SOC) Preferred Term(PT) | Incid ence Rate | N o o f A A E s | Incid<br>ence<br>Rate | N o o f A E s | Incid ence Rate | N<br>o<br>o<br>f<br>A<br>E<br>s | Incid<br>ence<br>Rate | N o . o f A E s | Incid ence Rate ( n % | N o f A E s | Incid ence Rate ( n % | N o . o f A E s | Incid ence Rate | N o f A E s | Incid<br>ence<br>Rate | N o o f A E s | Incid ence Rate | N o o f A E s | Incid<br>ence<br>Rate | N o c f A E s | Incid ence Rate | N o . o f A E s | Incid<br>ence<br>Rate | N o o f A A E s | Inc ide nc e Ra te | N<br>o<br>o<br>f<br>A<br>E | Inc<br>ide<br>nc<br>e<br>Ra | N o o f E E s |
| Total | | | | | | | | | | | | | | | | | | | | | | | | | | 1 | | _ |

### \* MedDRA

Table 7.1.1.1 SAE and SADR by study vaccination (2-23 months)

| | | | 11 | N=0 | | | | | 2 N | 1=0 | | | | | 3 N | V=0 | | | | | 4 N | 1=0 | | | | Тс | otal | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety Set | Ser | ious | ΑE | Sei<br>AE | rious<br>DR | | Serie | ous AE | | Serious | s AD | )R | Ser | rious | <b>Α</b> Ε | Ser | rious<br>PR | | Ser | ious . | <b>Α</b> Ε | Serious<br>ADR | | Ser | ious . | <b>Α</b> Ε | Ser<br>AD | ious<br>R | |
| | | | N | | | N | | | | | | | | | N | | | N | | | N | | N | | | N | | | N |
| | Inc | ide | o. | Inc | ide | o. | | 1 | N. C | T 1 | | N. C | Inc | ide | o. | Inci | ide | o. | Inc | ide | o. | Incide | o. | Inci | ide | o. | Inc | ide | o. |
| | nce | : | of | nce | e | of | | dence | | Inciden | ice | No. of | nce | , | of | nce | , | of | nce | | of | nce | of | nce | | of | nce | ; | of |
| | Rat | e A | Rate | Å | | | Rate | ; | AEs | Rate | | AEs | Rat | te A I | Rate 1 | A | | | Rat | e A I | Rate 1 | <b>A</b> | | Rat | e A I | Rate 1 | A | | |
| | | | Es | | | Es | | | | | | | | | Es | | | Es | | | Es | | Es | | | Es | | | Es |
| | | ( | | | ( | | | | | | | | | ( | | | ( | | | ( | | | | | ( | | | ( | |
| | n | % | n | n | % | n | n | | | | | n | n | % | n | n | % | n | n | % | | | n | n | % | n | n | % | n |
| | | ) | | | ) | | | | | | | | | ) | | | ) | | | ) | | | | | ) | | | ) | |
| System Organ | | | İ | | | | | | | | | | | | İ | | | İ | | ļ | | | | | | İ | | | |
| Class(SOC) | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Preferred | *************************************** | | | | | | | | | | | | | | | | | | | _ | | | | | | | | | |
| Term(PT) | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Total | | | | _ | | | | | | | | | | | | | | | | | | | | | | | _ | | |

#### \* MedDRA

Table 7.2.1 SAE and SADR

| | 2 | 2-23 months | | | | 2-10 | | | | 11-18 | | | | 19-34 | | | | 35-55 | | | | Total | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety per protocol set | Serious | Serious | | Serious | | Serious | | Serious | | Serious | | Serious | | Serious | | Serious | | Serious | | 5 | Serious | | Serious | |
| | AE | | ADR | | AE | | ADR | | AE | | ADR | | AE | | ADR | | AE | | ADR | | AE | | ADR | |
| | Incid<br>ence<br>Rate | N 0 0 f A A E S | Incid<br>ence<br>Rate | N 0 0 f A E E s | Incid<br>ence<br>Rate | N o. o f A E | Incid<br>ence<br>Rate | N o o f A A E | Incid<br>ence<br>Rate | N o o f A A E | Incid<br>ence<br>Rate | N O O F A A E S | Incid<br>ence<br>Rate | N 0 0 f A A E s | Incid<br>ence<br>Rate | N o o f A E | Incid<br>ence<br>Rate | N o o f A E | Incid<br>ence<br>Rate | N o f A E | Incid<br>ence<br>Rate | N o o f A E | Incid<br>ence<br>Rate | N o f A E s |
| | ( | | ( | | | | | | ( | | ( | | ( | | | | ( | | ( | | ( | | ( | |
| | n % | n | n % | n | n | | | n | n % | n | n % | n | n % | | | n | n % | n | n % | n | n % | n | n % | n |
| | ) | | ) | | | | | | ) | | ) | | ) | | | | ) | | ) | | ) | | ) | |
| System Organ | | | | | | | | | | | | | | | | | | | | | | | | |
| Class(SOC) | | | | | | | | | | | | | | | | | | !<br>!<br>!<br>! | | | | <u> </u> | : | |

| | 2 | -23 n | nonths | | 2-10 | | | | 11-18 | | | | 19-34 | | | | 35-55 | | | | Total | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety per protocol set | Serious | | Serious | | Serious | | Serious | | Serious | | Serious | | Serious | | Serious | | Serious | | Serious | | Serious | | Serious | |
| | AE | | ADR | | AE | | ADR | | AE | | ADR | | AE | | ADR | | AE | | ADR | <u> </u> | AE | | ADR | |
| | Incid<br>ence<br>Rate | N 0 | Incid<br>ence<br>Rate | N 0 0 f A A E S | Incid<br>ence<br>Rate | f | Incid<br>ence<br>Rate | N o o f A A E S | Incid<br>ence<br>Rate | N o o f f A A E E s | Incid<br>ence<br>Rate | N o o f A A E S | Incid<br>ence<br>Rate | N o o f A A E S | Incid<br>ence<br>Rate | N o f A E s | Incid<br>ence<br>Rate | N o o f A E | Incid<br>ence<br>Rate | N o . o f A E s | Incid<br>ence<br>Rate | N o f A E s | Incid<br>ence<br>Rate | N 0 |
| | n % | n | n % | n | n | | | n | n % | n | n % | n | n % | | | n | n % | n | n % | n | n % | n | n % | n |
| Preferred Term(PT) | | | | EII | | | | | | | | | · · · · | | | | | MI TETTI I TETTI I I TOTO DE LA COLONIA DE L | | THE RESERVE OF THE PROPERTY OF | | | | AND THE CONTRACT OF THE CONTRA |
| Total | | | | | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA
Table 7.2.1.1 SAE and SADR by study vaccination (2-23 months)

| | | | 1 N | V=0 | | | | | 2 N | 1=0 | | | | | 3 N | V=0 | | | | | 4 N | 1=0 | | | | Тс | tal | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety per protocol set | Ser | ious . | ΑE | Ser<br>AI | rious<br>DR | | Serie | ous AE | , | Serio | ous AE | )R | Se | rious | <b>Α</b> Ε | Ser<br>AD | rious<br>DR | | Ser | ious . | ΑE | Serious<br>ADR | | Seri | ous 2 | ΑE | Ser | | |
| protocol set Ir no F System Organ | | | N | | | N | | | | | | | | | N | | | N | | | N | | N | | | N | | | N |
| | Inc | ide | 0. | Inc | cide | 0. | , . | 1 | N. C | | | N C | Inc | eide | o. | Inc | ide | o. | Inc | ide | о. | Incide | О. | Inci | de | o. | Inci | de | 0. |
| | nce | : | of | nce | e | of | | dence | No. of | | | No. of | nce | e | of | nce | • | of | nce | ; | of | nce | of | nce | | of | nce | | of |
| | Ra | ite | Α | Ra | te | Α | Rate | ; | AEs | Rate | | AEs | R | ate | Α | Rat | te | Α | Ra | ite | Α | Rate | Α | Rat | te | A | Rat | e | A |
| | | | Es | | | Es | | | | | | | | | Es | | | Es | | | Es | | Es | | | Es | | | Es |
| | | ( | | : | ( | | | | | | | | | ( | | | ( | | | ( | | | | | ( | | | ( | |
| | n | % | n | n | % | n | n | | | | | n | n | % | n | n | % | n | n | % | | | n | n | % | n | n | % | n |
| | | ) | | | ) | | | | | | | | | ) | | | ) | | | ) | | | | | ) | | | ) | |
| System Organ | | | | | | | | | | | | | | | | | | | | | | | | | | | | | 1 |
| Class(SOC) | | | | | | l | | | | | | | | | | | | | | | | | | | | | | | |
| Preferred | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Term(PT) | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| | | | | | | | | | | | | # | | | | | | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | | | | İ | | | | | | | | | | | | | |
| * MedDR A | | | | 1 | | | • | | | | | | • | | | 1 | | | | | | | | • | | | i | | |

<sup>\*</sup> MedDRA

# 7.3 Non-Safety per protocol set

Table 7.3.1 SAE and SADR

| | | 2-2 | 23 m | nonths | | | 2- | 10 | | | 11- | -18 | | | 19 | -34 | | | 35- | -55 | | | ≥5 | 56 | | | То | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non-Safety pe<br>protocol set | Seri<br>AE | ous | | Seriou<br>ADR | S | Serious<br>AE | 5 | Serious<br>ADR | S | Seriou<br>AE | S | Serio<br>ADR | ıs | Seriou<br>AE | S | Seriou<br>ADR | S | Serious<br>AE | S | Serious<br>ADR | S | Seriou<br>AE | s | Seriou<br>ADR | ıs | Seri<br>us A | | Seri<br>us<br>AD | |
| | Incidence Rate | d | N o f A E | Incid<br>ence<br>Rate | N o o f A E | Incid<br>ence<br>Rate | N o o f A A E E s | Incid<br>ence<br>Rate | N o o f A A E | Incid<br>ence<br>Rate | N o o f A E E s | Incid<br>ence<br>Rate | N 0 0 f A E s | Incid<br>ence<br>Rate | N o o f A E E s | Rate | N o o f f A E | Incid<br>ence<br>Rate | N 0 0 6 f A E 5 s | Incid<br>ence<br>Rate | N o o f A A E s | Incid<br>ence<br>Rate | N o o f A E s | Incid<br>ence<br>Rate | N $O$ $O$ $f$ $E$ $S$ | Inc ide nc e Ra | o | Inc<br>ide<br>nc<br>e<br>Ra<br>te | N o o f A A E s |
| System Organ Class(SOC) Preferred Term(PT) | | 9/0 | n | (<br>n % | m | n | | | n | n % | n n | (<br>n % | o n | n % | | | n | n % | n | n % | n | (<br>n %<br>) | | | n | (n ) | % n | (n % | H 100 1 |

| | | 2- | -23 n | nonths | | | 2- | 10 | | | 11 | 18 | | | 19- | 34 | | | 35- | ·55 | | | ≥5 | 6 | | , | Total | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non-Safety protocol set | per | Seriou<br>AE | S | Seriou:<br>ADR | S | Seriou:<br>AE | S | Seriou<br>ADR | S | Seriou<br>AE | s | Seriou:<br>ADR | 8 | Seriou<br>AE | S | Serious<br>ADR | 8 | Serious<br>AE | 5 | Serious<br>ADR | 8 | Seriou<br>AE | .S | Seriou<br>ADR | S | Serio<br>us AI | us | |
| | | Incid ence Rate | N o o f A E s | Incid<br>ence<br>Rate | N o o f A E s | Incid ence Rate | N o . o f A E s | Incid<br>ence<br>Rate | N o c f A E s | Incid ence Rate | N o c f A E s | Incid<br>ence<br>Rate | N o . o f A E s | Incid ence Rate ( n % | N o o f A A E s | Incid<br>ence<br>Rate | N o f A E s | Incid ence Rate | N o . o f A E s | Incid ence Rate ( n % | N o f A E s | Incid ence Rate ( n % | N o o f A E s | Incid<br>ence<br>Rate | N o o f A E s n | Inc ide nc e Ra te | N o . Inc ide o nc f e Ra A te E s | N o o f A E s |
| Total | | | | | | | | | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA

Table 7.3.1.1 SAE and SADR by study vaccination (2-23 months)

| | | | 1 1 | <b>V=</b> 0 | | | | | 2 N | 1=0 | | | | | 3 N | <b>1</b> =0 | | | | | 4 N | 1=0 | | | | Тс | tal | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non-Safety per protocol set | Ser | ious . | ΑE | Ser<br>AI | rious<br>DR | | Seri | ous AE | , | Serio | ous AE | )R | Se | rious | <b>Α</b> Ε | Ser | ious<br>R | | Sei | rious . | ΑE | Serious<br>ADR | | Seri | ous A | ΑE | Ser | ious<br>R | |
| In no | | | N | | | N | | | | | | | | | N | | | N | | | N | | N | | | N | | | N |
| | Inc | ide | 0. | Inc | eide | 0. | | | | | | | Inc | eide | o. | Inc | ide | o. | Inc | ide | О. | Incide | 0. | Inci | de | 0. | Inc | ide | 0. |
| | nce | : | of | nce | e | of | | dence | No. of | | | No. of | nce | e | of | nce | | of | nce | • | of | nce | of | nce | | of | nce | | of |
| | Ra | ite | Α | Ra | te | Α | Rate | ; | AEs | Rate | | AEs | R | ate | Α | Rat | e | Α | Ra | ate | Α | Rate | Α | Rat | te | A | Rat | e | Α |
| | | | Es | | | Es | | | | | | | | | Es | | | Es | | | Es | | Es | | | Es | | | Es |
| | | ( | | | ( | | | | | | | | | ( | | | ( | | | ( | | | İ | | ( | | | ( | |
| | n | % | n | n | % | n | n | | | | | n | n | % | n | n | % | n | n | % | | | n | n | % | n | n | % | n |
| | | ) | | | ) | | | | | | | | | ) | | | ) | | | ) | | | | | ) | | | ) | |
| System Organ | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Class(SOC) | | | | | | | | | | | | | | | İ | | | | | | | | | | | | | | |
| Preferred | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Term(PT) | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | | | | İ | | | | | | | | | | | | | |
| * MedDR A | | | | 1 | | | • | | | | | | | | | | | | | | | | | | | | <b> </b> | | |

<sup>\*</sup> MedDRA

### 8. Unexpected AE/ADR for 28 days after vaccination

Table 8.1.1 Unexpected AE and ADR

| | 2- | -23 1 | months | | | 2- | 10 | | | 11- | -18 | | | 19 | -34 | | | 35 | -55 | | | ≥5 | 56 | | | To | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety Set | Unexp<br>ed AE | | Unexp | | Unexpe | ect | Unexpo | | Unexp<br>ed AE | ect | Unexpo | | Unexp<br>ed AE | | Unexpo | | Unexpeed AE | | Unexpo | | Unexp<br>ed AE | | Unexp<br>cted<br>ADR | e | Unexpected d AF | , | Une<br>pect<br>d<br>ADI | e |
| | | N | | N | | N | | N | | N | | N | | N | | N | | N | | N | | N | | N<br>o | | N<br>o | | N<br>o |
| | | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | | | Inc | | Inc | |
| | Incid | 0 | Incid | o | Incid | 0 | Incid | 0 | Incid | 0 | Incid | 0 | Incid | 0 | Incid | 0 | Incid | 0 | Incid | 0 | Incid | 0 | Incid | o | ide<br>nc | : | ide<br>nc | О |
| | ence<br>Rate | f | Rate | f | Rate | f | Rate | f | ence<br>Rate | f | ence<br>Rate | f | ence<br>Rate | f | Rate | f | ence<br>Rate | f | ence<br>Rate | f | ence<br>Rate | f | ence<br>Rate | f | e | : | e | f |
| | | A<br>E | | A<br>E | | A<br>E | | A<br>E | | A<br>E | | A<br>E | | A<br>E | | A<br>E | | A<br>E | | A<br>E | | A<br>E | | A | Ra<br>te | A | Ra<br>te | Α |
| | | S | | s | | S | | S | | S | | s | | S | | S | | s | | S | | S | | E | | E<br>s | | E<br>s |
| | ( | | ( | | ( | | ( | | ( | | ( | | ( | | ( | | ( | | ( | | ( | | ( | 3 | ( | 3 | ( | |
| | n % | n | n % | ó n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | n | n % | ∕o n | n % | 1 |

| | 2- | -23 r | nonths | | | 2- | 10 | | | 11 | -18 | | | 19 | -34 | | | 35- | 55 | | | ≥5 | 56 | | | То | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety Set | Unexp | | Unexp | | Unexpe | ect | Unexp | | Unexp<br>ed AE | ect | Unexp | | Unexpo | ect | Unexpo | | Unexpected AE | ct | Unexpo | | Unexp<br>ed AE | | Unexp<br>cted<br>ADR | e | Unexpected d AF | e | Une<br>pect<br>d<br>AD | te |
| | | | | | | | | | | | | | | | | | | | | | | | | N | | N | | N |
| | Incid<br>ence<br>Rate | N 0 0 f A E | Incid<br>ence<br>Rate | N o o f A E E s | Incid<br>ence<br>Rate | o o f A E E s | Incid<br>ence<br>Rate | N 0 0 f A E s | Incid<br>ence<br>Rate | N 0 0 f A A E s | Incid<br>ence<br>Rate | N o o f A A E S | Incid<br>ence<br>Rate | N o f A E | Incid<br>ence<br>Rate | N o o f A E | Incid<br>ence<br>Rate | N o o f A E s | Incid<br>ence<br>Rate | N | Incid<br>ence<br>Rate | N 0 0 f A E S | Incid<br>ence<br>Rate | 0 · | Inc ide nc e Ra | o<br>f | Inc<br>ide<br>nc<br>e<br>Ra<br>te | o o f |
| | n % | o n | n % | n | n | | | n | n % | n | n % | n | n % | | | n | n % | n | n % | n | n % | | | n | n 9 | | n % | |
| System Organ Class(SOC) Preferred Term(PT) | | MATERIAL DESCRIPTION OF THE PROPERTY OF THE PR | | | | | | THE RESERVE THE PROPERTY OF TH | | | | | | | | | | | | | | | | | | | | |

| | 2- | -23 r | nonths | | | 2- | 10 | | | 11 | -18 | | | 19- | -34 | | | 35 | -55 | | | ≥5 | 56 | | | Total | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety Set | Unexp<br>ed AE | | Unexp | | Unexp | | Unexp | | Unexp<br>ed AE | | Unexp | | Unexp<br>ed AE | ect | Unexp | | Unexpo | ect | Unexp | | Unexp<br>ed AE | | Unexpo<br>cted<br>ADR | e | Une<br>pect<br>d Al | pect<br>e d | te |
| | Incid<br>ence<br>Rate | N 0 0 f A E | Incid<br>ence<br>Rate | N 0 0 f A E | Incid<br>ence<br>Rate | N 0 0 f A E E s | Incid<br>ence<br>Rate | N 0 0 f A E s | Incid<br>ence<br>Rate | N 0 0 f A E S | Incid<br>ence<br>Rate | N 0 0 f A E S | Incid<br>ence<br>Rate | N 0 0 f A E S | Incid<br>ence<br>Rate | N o o f A E E s | Incid<br>ence<br>Rate | N o o f A E | Incid<br>ence<br>Rate | N 0 0 f A A E s | Incid<br>ence<br>Rate | N 0 0 f A E s | Incid<br>ence<br>Rate | f<br>A | Inc<br>ide<br>nc<br>e<br>Ra<br>te | o . Inc ide o nc f e Ra A te E | N o o f A A |
| | ( | | | | - | | | | ( | | ( | | ( | | | | | | ( | | ( | | | S | ( | s | S |
| | n % | o n | n % | n | n | | | n | n % | n | n % | n | n % | | | n | n % | n | n % | n | n % | | | n | n ' | % n n % | |
| Total | | | | | | | | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA

Table 8.1.1.1 Unexpected AE and ADR by study vaccination number (2-23 months)

| | | | 1 1 | N=0 | | | | | 2 1 | V=0 | | | | 3 N | <b>V=</b> 0 | | | | | 4 N | 1=0 | | | | То | otal | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Un | expec | ted | Un | expec | ted | Une | expec | ted | Unexpec | ted | Un | expec | ted | Ur | nexpect | ted | Un | expec | ted | Unexpec | ted | Un | expec | ted | Un | xpec | ted |
| Safety Set | AE | Į. | | ΑI | OR | | AE | | | ADR | | AF | Ξ | | AI | DR | | AE | , | | ADR | | AE | | | AD | R | |
| | | | N | | | N | | | N | | N | | | N | | | N | | | N | | N | | | N | | | N |
| | Inc | iden | 0. | Inc | eiden | 0. | Inc | iden | 0. | Inciden | 0. | Inc | ciden | о. | Inc | ciden | 0. | Inc | iden | 0. | Inciden | 0. | Inc | iden | О. | Inc | den | о. |
| | | Rate | of | | Rate | of | | Rate | of | ce Rate | of | | Rate | of | : | Rate | of | | Rate | of | ce Rate | of | | Rate | of | | late | of |
| | | raic | Α | | ruic | A | | cuic | Α | Cortato | Α | | raic | Α | | rate | A | | rtuto | Α | Cortato | Α | | cuic | Α | | cuic | Α |
| | | | Es | | | Es | | | Es | | Es | | | Es | | | Es | | | Es | | Es | | | Es | | | Es |
| | | ( | | | ( | | | ( | | | | | ( | | | ( | | | ( | | | | | ( | | | ( | |
| | n | % | n | n | % | n | n | % | | | n | n | % | n | n | % | n | n | % | | | n | n | % | n | n | % | n |
| | | ) | | | ) | | | ) | | | | | ) | | | ) | | | ) | | | | | ) | | | ) | |
| System Organ | | | | | | | | | | | | | | 1 | | | | | | | | | | | | | | ! |
| Class(SOC) | | | | | | | | | | | İ | | | | | | | | | | | | | | | | | |
| Preferred | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Term(PT) | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Total | | | | | | | | | | ĺ | İ | | | İ | ĺ | | | | | | ĺ | | | | İ | ĺ | | İ |

<sup>\*</sup> MedDRA

### 8.2 Safety per protocol set

Table 8.2.1 Unexpected AE and ADR

| | 2- | -23 r | nonths | | | 2- | 10 | | | 11 | -18 | | | 19 | -34 | | | 35 | -55 | | | To | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Unexpe | ect | Unexpe | ecte | Unexpe | ecte | Unexpo | ect | Unexpe | ect | Unexpo | ect | Unexpe | ct | Unexpe | ct | Unexpe | ect | Unexpe | ect | Unexpe | ect | Unexp | iec |
| Safety per protocol set | ed AE | | d ADR | | d AE | | ed ADI | R | ed AE | | ed ADI | } | ed AE | | ed ADR | _ | ed AE | | ed ADI | 3 | ed AE | | ted AI | )R |
| | Incid<br>ence<br>Rate | N o o f A A E S | Incid<br>ence<br>Rate | N 0 0 f A A E S | Incid<br>ence<br>Rate | f | Incid<br>ence<br>Rate | N 0 0 F F E S | Incid<br>ence<br>Rate | N 0 0 f A E E s | Incid<br>ence<br>Rate | N o f A E | Incid<br>ence<br>Rate | N o f A E s | Incid<br>ence<br>Rate | N o o f A E s | Incid<br>ence<br>Rate | N o o f A E E s | Incid<br>ence<br>Rate | N o o f A A E S | Incid<br>ence<br>Rate | N o o f f A E | Incid<br>ence<br>Rate | N o o f F A A E S |
| | n % | n | n % | n | n | | | n | n % | n | n % | n | n % | | | n | n % | n | n % | n | n % | n | n % | 6 n |
| System Organ Class(SOC) Preferred Term(PT) | | | | | | | THE REAL PROPERTY OF THE PROPE | 0.01.1.1.1.1.1.1.1.1.1.1.1.1.1.1.1.1.1. | | | | | | | | | | | | THE RESERVE OF THE PROPERTY OF | | | | |

| | 2- | -23 r | nonths | | | 2- | 10 | | | 11- | 18 | | | 19 | -34 | | | 35 | -55 | | | То | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Unexpe | ect | Unexpe | ecte | Unexpe | ecte | Unexpe | ect | Unexpe | ect | Unexp | ect | Unexpe | ect | Unexpe | ct | Unexpe | ect | Unexp | ect | Unexp | pect | Une | крес |
| Safety per protocol set | ed AE | | d ADR | | d AE | | ed ADI | 2 | ed AE | | ed ADI | <b>?</b> | ed AE | | ed ADR | 1 | ed AE | | ed AD | R | ed AE | <u> </u> | ted A | ADR |
| | Incid<br>ence<br>Rate | N 0 0 0 f A A E S | Incid<br>ence<br>Rate | N 0 0 f A A E s | Incid<br>ence<br>Rate | f | Incid<br>ence<br>Rate | N 0 0 f A A E s | Incid<br>ence<br>Rate | N o o f A E s | Incid<br>ence<br>Rate | N 0 0 f A E s | Incid<br>ence<br>Rate | N o o f A A E s | Incid<br>ence<br>Rate | N o . o f A E s | Incid<br>ence<br>Rate | N o o f A A E E s | Incid<br>ence<br>Rate | N o o f A A E s | Incid<br>ence<br>Rate | N o f A E s | Incidence<br>Rate | f |
| | n % | n | n % | n | n | | | n | n % | n | n % | n | n % | | | n | n % | n | n % | n | n % | | n | % n |
| Total | | | | | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA

Table 8.2.1.1 Unexpected AE and ADR by study vaccination number (2-23 months)

| | | | 1 N | V=0 | | | | | 2 N | 1=0 | | | | 3 N | 1=0 | | | | 4 N | N=0 | | | | То | otal | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety per protocol | Une | expec | ted | Un | expec | ted | Un | expec | ted | Unexpect | ted | Un | expec | ted | Unexpe | cted | U | nexpec | ted | Unexpec | ted | Un | expec | ted | Un | expec | ted |
| set | AE | | | AD | PR | | AE | | | ADR | | AE | , | | ADR | | A | .E | | ADR | | AE | | | AD | R | |
| | | | N | | | N | | | N | | N | | | N | | N | | | N | | N | | | N | | | N |
| | Inc | iden | o. | Inc | iden | 0. | Inc | iden | 0. | Inciden | o. | Inc | iden | 0. | Inciden | 0. | T., | nciden | 0. | Inciden | o. | Ina | iden | o. | Inc | iden | 0. |
| | | | of | | | of | | | of | | of | | | of | | of | | | of | | of | | | of | | | of |
| | ce i | Rate | Α | ce | Rate | Α | ce. | Rate | Α | ce Rate | Α | ce. | Rate | Α | ce Rate | Α | CE | e Rate | Α | ce Rate | Α | ce | Rate | Α | ce | Rate | Α |
| | | | Es | | | Es | | | Es | | Es | | | Es | | Es | | | Es | | Es | | | Es | | | Es |
| | | ( | | | ( | | | ( | | | | | ( | | ( | | | ( | | | | | ( | | | ( | |
| | n | % | n | n | % | n | n | % | | | n | n | % | n | n % | n | n | % | | | n | n | % | n | n | % | n |
| | | ) | | | ) | | | ) | | | | | ) | | ) | | | ) | | | | | ) | | | ) | |
| System Organ | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Class(SOC) | | | | | | | | | İ | | İ | | | | | İ | | | | | | | | | | | |
| Preferred | | | | | | | | | | | | *************************************** | | | | | | | | : | | | | | | | |
| Term(PT) | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | | | İ | | | | | | | | | | | | |
| * MedDR A | | | | 1 | | | | | | | | | | | | + | 1 | | | 1 | | 1 | | | 1 | | $\vdash$ |

<sup>\*</sup> MedDRA

# 8.3 Non-Safety per protocol set

Table 8.3.1 Unexpected AE and ADR

| | | 2. | -23 n | nonths | | | 2- | 10 | | | 11 | -18 | | | 19 | -34 | | | 35 | -55 | | | ≥: | 56 | | | Tot | al | _ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non-Safety<br>protocol set | per | Unexp<br>ed AE | | Unex | | Unexp<br>ed AE | | Unexp | | Unexped AF | | Unexp | | Unexp | | Unexp | | Unexp | | Unexp | | Unexp | | Unexp<br>cted<br>ADR | e | Unex pected d AE | <b>.</b> | Unex pected d ADR | е |
| | | | | | | | | | | | | | | | | | | | | | | | | | N | | N | | N |
| | | | N | | N | | N | | N | | N | | N | | N | | N | | N | | N | | N | | o | | o | | o |
| | | | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | | | Inc | | Inc | • |
| | | Incid | | Incid | | Incid | | Incid | | Incid | | Incid | | Incid | | Incid | | Incid | | Incid | | Incid | | Incid | | ide | | ide | |
| | | ence | o<br>f | ence | o<br>f | ence | o<br>f | ence | o<br>f | ence | o<br>f | ence | o<br>f | ence | o<br>f | ence | o<br>f | ence | o<br>f | ence | o<br>f | ence | o<br>f | ence | o<br>f | nc<br>e | f | | o<br>f |
| | | Rate | A | Rate | A | Rate | A | Rate | A | Rate | A | Rate | A | Rate | A | Rate | A | Rate | A | Rate | A | Rate | A | Rate | 1 | Ra | : | Ra | 1 |
| | | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | A | | : | te | A |
| | | | s | | s | | s | | s | | s | | S | | s | | s | | s | | s | | s | | Е | | Е | | Е |
| | | | | | | | | | | | | | | | | | | | | | | | | | s | | s | | s |
| | | ( | | ( | | | | | | ( | | ( | | ( | | | | ( | | ( | | ( | | | | ( | | ( | |
| | | n % | n | n 9 | o n | n | | | n | n % | o n | n % | o n | n % | | | n | n % | n | n % | 6 n | n % | | | n | n 🦠 | 6 n | n % n | Ĺ |
| | | ) | | ) | | | | | | ) | | ) | | ) | | | | ) | | ) | | ) | | | | ) | | ) | _ |
| System | Organ | | | | | | | | | | | | | | | | | | | | | | | | - | | | | |
| Class(SOC) | | | | : | | | | | | | | | | | | | | | | | | | | | | | | | |

| | 2. | -23 n | nonths | | | 2- | 10 | | | 11 | -18 | | | 19- | -34 | | | 35. | -55 | | | ≥5 | 56 | | | То | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non-Safety per<br>protocol set | Unexp | | Unexp | | Unexpo | | Unexp | | Unexp<br>ed AE | | Unexp | | Unexpe | | Unexpo | | Unexpe | ect | Unexpo | | Unexp | | Unexp<br>cted<br>ADR | e | Une<br>pect<br>d Al | e | Une:<br>pecto<br>d<br>ADF | e |
| | | N | | N | | N | | N | | N | | N | | N | | N | | N | | N | | N | | N<br>o | | N<br>o | : | N<br>o |
| | Incid<br>ence<br>Rate | 0 | Incid<br>ence<br>Rate | o o f A E | Incid | o o f A E E s | Incid<br>ence<br>Rate | o o f A A E E s | Incid<br>ence<br>Rate | o o f A E | Incid<br>ence<br>Rate | o o f A E | Incid<br>ence<br>Rate | o o f A E S | Incid<br>ence<br>Rate | o o f A A E | Incid<br>ence<br>Rate | o o f A E s | Incid<br>ence<br>Rate | o o f A A E S | Incid<br>ence<br>Rate | o f E | Incid<br>ence<br>Rate | | Inc ide nc e Ra te | o<br>f | Inc ide nc e Ra te | o f E S |
| | n % | n | n % | o n | n | | | n | n % | n | n % | n | n % | | | n | n % | n | n % | n | n % | | | n | n ' | | (<br> n % <br> | <b>(1)</b> |
| Preferred Term(PT) | | THE RESERVE OF THE PROPERTY OF | | | | NOTICE OF THE STATE OF THE STAT | | | | THE RESERVE THE PROPERTY OF TH | | THE RESERVE OF THE PROPERTY OF | | | | | | | | | | | | A THE THE PERSON OF THE PERSON | | | | |
| Total | | | | | | | | | | | | | | | | | | | | | | | | | | | | |

### \* MedDRA

Table 8.3.1.1 Unexpected AE and ADR by study vaccination number (2-23 months)

| | Inciden of ce Rate A Es Es E | | | | | 2 N | 1=0 | | | | 3 N | 1=0 | | | | | 4 N | 1=0 | | | | Тс | otal | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non-Safety per | Une | expec | ted | Une | expec | ted | Une | expec | ted | Unexpect | ted | Un | expec | ted | Un | nexpect | ted | Une | expect | ed | Unexpec | ted | Un | expec | ted | Une | xpec | ted |
| protocol set | Unexpected Unexpected AE ADR N N N N N N N N N N N N N N N N N N N | | | AE | | | ADR | | AE | ) | | AΓ | OR | | AE | | | ADR | | AE | | | ADI | 2 | | | | |
| | | | N | | | N | | | N | | N | | | N | | | N | | | N | | N | | | N | | | N |
| | Inci | don | 0. | Inci | idan | 0. | Inci | den | 0. | Inciden | o. | Inc | iden | 0. | Inc | ciden | 0. | Inc | iden | o. | Inciden | o. | Inc | iden | o. | Inci | dan | 0. |
| | | | of | | | of | ce I | | of | ce Rate | of | | Rate | of | | Rate | of | | Rate | of | ce Rate | of | | Rate | of | ce R | | of |
| | ce r | Cate | Α | Ce r | Xaie | Α | Ce i | Cale | A | ce Kale | Α | Ce. | Kate | Α | | Nate | A | Ce I | Naic | A | ce Kale | Α | Cel | Xate | Α | CCN | ale | A |
| | | | Es | | | Es | | | Es | | Es | | | Es | | | Es | | | Es | | Es | | | Es | | | Es |
| | | Unexpected AE Inciden ce Rate A Es | | | ( | | | ( | | | | | ( | | | ( | | | ( | | | | | ( | | | ( | |
| | n | Unexpected AE Inciden ce Rate ( Es | | n | % | n | n | % | | | n | n | % | n | n | % | n | n | % | | | n | n | % | n | n | % | n |
| | | ) | | | ) | | | ) | | | | | ) | | | ) | | | ) | | | | | ) | | | ) | |
| System Organ | | | | | | | | | İ | | | | | | | | | | | | | | | | İ | | | |
| Class(SOC) | | | | | | <b> </b> | | | l | | | | | | | | | | | | | | | | | | | |
| Preferred | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Term(PT) | | | | | | | | | | : | | | | | | | | | | | | | | | | | | |
| | | Inciden of the ce Rate A E | | | | | | | | | | | | | | | | | | | | | | | | | | |
| | Inciden ce Rate A Es | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| | | Unexpected AE N o. Inciden ce Rate A Es | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Total | Unexpected Unexpected AE ADR Inciden of ce Rate A Es ( | | | | | | | | | | | | | ĺ | | | | | | | | | | | ĺ | | | |

#### \* MedDRA

### 9. MAAE/ADR for 8 days to 28 days after vaccination

Table 9.1.1 MAAE and ADR

| | 2- | -23 n | nonths | | | 2- | 10 | | | 11- | -18 | | | 19 | -34 | | | 35- | -55 | | | <u>&gt;</u> | 56 | | | То | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety Set | MAAI | Е | ADR | | MAAl | E | ADR | | MAAI | Ξ | ADR | | MAAl | Ξ | ADR | | MAAE | | ADR | | MAA | Е | ADR | | MAA | Е | ADF | <u> </u> |
| | | | | | | | | | | | | | | | | | | | | | | | : | N | | | | N |
| | | N | | N | | N | | N | | N | | N | | N | | N | | N | | N | | N | | o | | N | | o |
| | | o | | o | | o | | o | | o | | o | | o | | o | | o | | 0 | | o | | • | | o | | • |
| | Incid | | Incid | | Incid | | Inci | | Inci | • | Inci | | Inci | | Inci | | Inci | | Inci | | Inci | | Inci | | Inci . | Inci | | |
| | ence | О | | О | ence | o | denc | o | denc | o | denc | o | denc | o | denc | o | denc | o | denc | 0 | denc | o | denc | o | den | О | den | o |
| | Rate | f | Rate | f | Rate | f | e | f | e | f | e | f | e | f | е | f | e | f | e | f | e | f | e | f | ce | f | ce | f |
| | | A | | Α | | A | Rate | A | Rate | Α | Rate | Α | Rate | A | Rate | Α | Rate | A | Rate | A | Rate | Α | Rate | | Rate A | A R | ate | |
| | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | E | | Е | | Е | | Α | | Е | | Α |
| | | s | | s | | S | | s | | s | | s | | s | | S | | S | | S | | s | | Е | | s | | Е |
| | | | | | | | | | | | | | | | | | | | | | | | <u> </u> | s | | | | S |
| | ( | | ( | | ( | | ( | | ( | | ( | | ( | | ( | | ( | | ( | | ( | | ( | | ( | | ( | |
| | n % | n | n % | n | n % | n | n % | n | n % | nı | 1 % n | | n % | nı | 1 % n | | n % | n i | ı%n | | n % | n | n % | n | n % | n | n % | ⁄0 n |
| | ) | | ) | | ) | | ) | | ) | | ) | | ) | | ) | | ) | | ) | | ) | | ) | | ) | | ) | |

| N | | 2- | 23 n | nonths | | | 2- | 10 | | | 11 | -18 | | | 19 | -34<br>I | | | 35- | -55<br>I | | | ≥ | 56 | | | То | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| N | Safety Set | MAAI | | ADR | | MAAl | E | ADR | | MAAI | 3 | ADR | | MAAl | E | ADR | | MAAl | Ξ | ADR | | MAA | Ę | ADR | | MAA | Е | AD | R |
| ( ( ( ( ( ( ( n % n n % n n n % n n n m % n n n m m n n m m n m m n m m n m m n m m n m m n m m m m m m m m m m m m m m m m m m m m | | ence | o<br>f<br>A | Incid<br>ence<br>Rate | o o f A | ence<br>Rate | o | Inci<br>denc<br>e | o<br>o<br>f<br>A<br>E | denc<br>e | o<br>o<br>f<br>A<br>E | Inci<br>denc<br>e<br>Rate | o o f A | denc<br>e | o o f | Inci<br>denc<br>e | o<br>o<br>f<br>A | Inci<br>denc<br>e<br>Rate | o<br>o<br>f<br>A<br>E | Inci<br>denc<br>e<br>Rate | o o | denc<br>e | o o f A | Inci<br>denc<br>e<br>Rate | o<br>o<br>f | den<br>ce | o<br>Inci<br>o<br>A R | den<br>ce<br>ate | |
| | System Organ Class(SOC) Preferred Term(PT) | n % | n | (<br>n%<br>) | n | n | | | n | | n ı | | | ( n % ) | | | | ( n % ) | nr | | | n % | | | | n % | n | n ' | 9%nn) |

<sup>\*</sup> MedDRA

Table 9.1.1.1 MAAE and ADR by study vaccination number (2-23months)

| | MAAE ADR MAAE N o. Inciden of ce Rate ( n % n n ) | | | | | | | | 2 N | V=0 | | | | 3 N | 1=0 | | | | | 4 N | 1=0 | | | | То | otal | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety Set | MA | AAE | | AD | R | | MA | AE | | ADR | | MA | AAE | | AD | R | | MA | AE | | ADR | | MA | AE | | AD | R | |
| | | | N | | | N | | | N | | N | | | N | | | N | | | N | | N | | | N | | | N |
| | | | of<br>A | | | o.<br>of<br>A | | iden<br>Rate | o.<br>of<br>A | Inciden<br>ce Rate | o.<br>of<br>A | | iden<br>Rate | o.<br>of<br>A | | iden<br>Rate | o.<br>of | | iden<br>Rate | o.<br>of<br>A | Inciden<br>ce Rate | o.<br>of<br>A | | iden<br>Rate | o.<br>of<br>A | | iden<br>Rate | o.<br>of<br>A |
| | | | Es | | | Es | | | Es | | Es | | | Es | | | Es | | | Es | | Es | | | Es | | | Es |
| | n | ( % | n | n | ( % | n | n | ( % | | | n | n | (<br>% | n | n | (<br>% | n | n | (<br>% | | | n | n | (<br>% | n | n | ( % | n |
| | | ) | | | ) | | | ) | | | | | ) | | | ) | | | ) | | | | | ) | | | ) | |
| System Organ Class(SOC) Preferred Term(PT) | | | NATIONAL THE CONTRACTOR OF THE | | | 10 10 10 10 10 10 10 10 | | | AND THE RESERVE OF THE PROPERTY OF THE PROPERT | | | | | A DATE OF THE PROPERTY OF THE | | | TO THE RESERVE OF THE PROPERTY | | | | | | - | | | | | |
| Total | | | | | | | | | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA

# 9.2 Safety per protocol set

Table 9.2.1 MAAE and ADR

| | 2- | -23 r | nonths | | | 2- | 10 | | | 11- | -18 | | | 19 | -34 | | | 35 | -55 | | | То | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety per protocol Set | Incid o Incid o ence f Rate A E s s | | | | MAAE | Į. | ADR | | MAAE | , | ADR | | MAAE | | ADR | | MAAE | | ADR | | MAAE | 3 | ADR | |
| | ence | o o f | ence | N 0 c f A E s | Incid<br>ence<br>Rate | N o. o f A E | Incid<br>ence<br>Rate | N o f A E E s | Incid<br>ence<br>Rate | N 0 0 f A A E S | Incid<br>ence<br>Rate | N o o f A E E s | Incid<br>ence<br>Rate | N o f A E | Incid<br>ence<br>Rate | N o o f A E | Incid<br>ence<br>Rate | N o o f A E s | Incid<br>ence<br>Rate | N o c f A E S | Incid<br>ence<br>Rate | N o o f A E | Incid<br>ence<br>Rate | N o o f A E s |
| System Organ Class(SOC) Preferred Term(PT) | | n | n % | | n | en e | | n | (<br>n %<br>) | n | (<br>n % | * The same of the | (<br>n %<br>) | | | n | ( n % ) | n | (<br>n % | | ( n % | n | n % | n |

| | 2- | -23 n | nonths | | | 2- | 10 | | | 11 | -18 | | | 19 | -34 | | | 35 | -55<br>! | | | То | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety per protocol Set | MAAE | | ADR | | MAAE | | ADR | | MAAE | | ADR | | MAAE | | ADR | | MAAE | | ADR | | MAAE | Ξ | ADR | |
| | Incid<br>ence<br>Rate | N | Incid<br>ence<br>Rate | N 0 0 f A E E s | Incid<br>ence<br>Rate | f | Incid<br>ence<br>Rate | N o o f A E E s | Incid<br>ence<br>Rate | N 0 0 f A A E s | Incid<br>ence<br>Rate | N 0 0 f A E E s | Incid<br>ence<br>Rate | N o f A E | Incid<br>ence<br>Rate | N o o f A E s | Incid<br>ence<br>Rate | N o o f A E | Incid<br>ence<br>Rate | N 0 0 f A E s | Incid<br>ence<br>Rate | N o o f A E s | Incid<br>ence<br>Rate | N o o f E E s |
| Total | n % | n | n % | n | n | | | n | n % | n | n % | n | n % | | | n | n % | n | n % | n | n % | n | n % | n |

<sup>\*</sup> MedDRA

Table 9.2.1.1 MAAE and ADR by study vaccination number (2-23months)

| | | | 1 N | V=0 | | | | | 2 N | 1=0 | | | | 3 N | 1=0 | ) | | | | 4 N | 1=0 | | | | То | otal | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety Per Protocol<br>Set | MA | MAAE Inciden ce Rate ( | | AD | R | | MA | AE | | ADR | | MA | AAE | | A | .DR | | MA | AE | | ADR | | MA | AAE | | ADF | t | |
| | | Inciden ce Rate A E | | | iden<br>Rate | N o. of A Es | | iden<br>Rate | N o. of A Es | Inciden<br>ce Rate | N o. of A Es | | iden<br>Rate | N o. of A Es | | nciden<br>e Rate | N o. of A Es | Inci<br>ce R | | N o. of A Es | Inciden<br>ce Rate | N o. of A Es | | iden<br>Rate | N o. of A Es | Incid<br>ce R | | N o. of A Es |
| | n | | n | n | (<br>%<br>) | n | n | (<br>%<br>) | | | n | n | (<br>%<br>) | n | n | ( %<br>%<br>) | n | n | (<br>%<br>) | | | n | n | (<br>%<br>) | n | n | (<br>%<br>) | n |
| System Organ Class(SOC) Preferred Term(PT) | | | | | | | | | | | | | | | | | | | | | | | • | | | | | |
| Total | | | | | | | | | | | | | | | _ | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA

### 9.3 Non-Safety per protocol set

Table 9.3.1 MAAE and ADR

| | 2- | -23 n | nonths | | | 2- | 10 | | | 11 | -18 | | | 19- | -34 | | | 35- | -55 | | | <u>&gt;</u> | 56 | | | Tota | al | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non-Safety per protocol set | MAAl | Е | ADR | | MAAI | Е | ADR | | MAAl | Е | ADR | | MAAl | Ξ | ADR | | MAAI | 3 | ADR | | MAA | Е | ADR | | MAA | Е | ADR | |
| | | N | | N | | N | | N | | N | | N | | N | | N | | N | | N | | N | | N<br>o | | N | | N<br>o |
| | Incid | | Incid | 0 . 0 | Incid | | Inci<br>denc | o | Inci | · · · | Inci<br>denc | | Inci<br>denc | | Inci | | Inci<br>denc | | Inci<br>denc | | Inci | | Inci<br>denc | | Inci . | | den | |
| | ence<br>Rate | f<br>A | ence<br>Rate | f A | ence<br>Rate | f | e<br>Rate | f<br>A | e | f | e<br>Rate | o<br>f<br>A | e<br>Rate | f | denc<br>e<br>Rate | o<br>f<br>A | e<br>Rate | | e<br>Rate | o<br>f<br>A | denc<br>e<br>Rate | | e<br>Rate | f | | f | ce | o<br>f |
| | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | Е | | A | | Е | | A |
| | | S | | S | | S | | S | | S | | S | | S | | S | | S | | S | | S | | E<br>s | | s | | E<br>s |
| | ( | | ( | | | | | | ( | | ( | | ( | | | | ( | | ( | | ( | | | | ( | | ( | |
| | n % | n | n % | n | n ¶ | | | n | n % | n | n % n | | n % | | | | n % | n r | 1 % n | | n % | | | n | n % | n | n % | n |
| System Organ | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Class(SOC) | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Preferred Term(PT) | | | | | 10 HOROLOGICA (1981) | | | | | | | | | | | | | | | | | | | | | | | |

| | | 2- | 23 n | nonths | | | 2- | 10 | | | 11 | -18 | | | 19- | 34 | | | 35- | -55 | | | ≥ | 56 | | | Tot | al | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non-Safety protocol set | per | MAAI | Ξ | ADR | | MAAI | Е | ADR | | MAAI | Ξ | ADR | | MAAl | E) | ADR | | MAAF | 3 | ADR | | MAA | Е | ADR | | MAA | Е | ADR | |
| protocorset | | Incid<br>ence<br>Rate | N o o f A A E s | Incid<br>ence<br>Rate | N o f A E s | Incid<br>ence<br>Rate | o<br>f | Inci<br>denc<br>e<br>Rate | N o f A E | Inci<br>denc<br>e<br>Rate | f | Inci<br>denc<br>e<br>Rate | N 0 0 f A E S S | Inci<br>denc<br>e<br>Rate | o<br>f | Inci<br>denc | N o f A E | Inci<br>denc<br>e<br>Rate | N o f A E s | Inci<br>denc<br>e<br>Rate | N o f A E s | Inci<br>denc<br>e<br>Rate | f | Inci<br>denc<br>e<br>Rate | N o o f A A E s | | o<br>f | den<br>ce | N o o f |
| | | n % | n | n % | n | n G | | | n | n % | n ı | n % n | | n % | | | | n % | n r | (<br>n % n<br>) | | n % | | | n | n % | n | n % | n |
| Total | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA

Table 9.3.1.1 MAAE and ADR by study vaccination number (2-23months)

| | MAAE ADR Inciden ce Rate ( n % n n n % ) | | | | | | | 2 N | 1=0 | | | | 3 N | 1=0 | | | | | 4 N | 1=0 | | | | То | otal | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non-Safety per protocol set | MAAE Inciden ce Rate A E ( n % n | | AD | R | | MA | AAE | | ADR | | MA | AAE | | AD | )R | | MA | ΑE | | ADR | | MA | AAE | | ADI | _ | |
| | | o.<br>of<br>A | | | N o. of | | iden<br>Rate | N o. of A Es | Inciden<br>ce Rate | N o. of A Es | | eiden<br>Rate | N o. of A Es | | iden<br>Rate | N o. of A Es | Inci- | | N o. of A Es | Inciden<br>ce Rate | N o. of A Es | | iden<br>Rate | N o. of A Es | Incid<br>ce R | | N o. of A Es |
| | | n | n | (<br>%<br>) | n | n | (<br>%<br>) | | | n | n | (<br>%<br>) | n | n | (<br>%<br>) | n | n | (<br>%<br>) | | | n | n | (<br>%<br>) | n | n | (<br>%<br>) | n |
| System Organ Class(SOC) Preferred Term(PT) | | | | , | | | | | | | | | | | | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA

### 10. Unsolicited AE/ADR for 28 days after vaccination

Table 10.1.1 Unsolicited AE and ADR

| | 2- | -23 r | nonths | | | 2- | 10 | | | 11 | -18 | | | 19- | 34 | | | 35- | -55 | | | ≥ | 56 | | | Tot | al | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety set | AE | , | AD | R | AE | | ADI | χ. | AE | | ADI | ~ | AE | | ADF | $\sim$ | AE | | ADF | ξ. | AE | | ADR | | AE | | ADI | 3 |
| | Incid<br>ence<br>Rate | N o o f f A E S | Incid<br>ence<br>Rate | N o o f A A E S | Incid<br>ence<br>Rate | N o o f A E E s | Inci<br>denc<br>e<br>Rate | N o . o f A E E s | Inci<br>denc<br>e<br>Rate | N o o f A E s | Inci<br>denc<br>e<br>Rate | N o c f A E s | Inci<br>denc<br>e<br>Rate | N o o f A E s | Inci<br>denc | N 0 0 f A A E S | Inci<br>denc<br>e<br>Rate | | Inci<br>denc<br>e<br>Rate | N o o f A E s | e | f | Inci<br>denc<br>e<br>Rate | N o o o f f E S | Inci . den ce Rate 4 | o<br>f | den<br>ce<br>ate | |
| System Organ Class(SOC) Preferred Term(PT) | (<br>n % | *** | (<br>n % n | ************************************** | | | | The same of the sa | (<br>n % | n 1 | (<br>n % n | | (<br>n % | | | | (<br>n % | n r | (<br>1 % n<br>) | | n % | 1110 - 1100 - 1001 - 100 - 1001 - | | Δ | n % | n | ( n % | 5 n |

| | 2- | 23 n | nonths | | | 2- | 10 | | | 11 | -18 | | | 19 | -34 | | | 35- | -55<br>I | | | ≥ | 56 | | | То | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety set | AE | | ADI | Ŗ | AE | | ADI | ₹ | AE | | ADF | <b>!</b> | AE | | ADF | ? | AE | | ADI | ₹ | AE | | ADR | | AE | | ADI | _ |
| | Incid<br>ence<br>Rate | N<br>o<br>o | Incid | N o o f | Incid<br>ence<br>Rate | N<br>o | Inci<br>denc | N<br>o | Inci<br>denc<br>e | N<br>o | | N<br>o<br>o | Inci | N<br>o | | N<br>0 | Inci | N<br>o | | N<br>o<br>o | Inci<br>denc<br>e | N<br>o | | N<br>o | Inci .<br>den | N<br>o<br>Inci | | o<br>o |
| | | A<br>E<br>s | | A<br>E<br>s | | A<br>E<br>s | Rate | A<br>E<br>s | Rate | A<br>E<br>s | Rate | A<br>E<br>s | Rate | A<br>E<br>s | Rate | A<br>E<br>s | Rate | A<br>E<br>s | Rate | A<br>E<br>s | Rate | A<br>E<br>s | Rate | A<br>E<br>s | Rate A | AR<br>E<br>s | | A<br>E |
| | n % | n r | (<br>1 % n | | | | | | n % | n ı | (<br>1 % n | | (<br>n %<br>) | | | | n % | n r | (<br>1 % n | | n % | | | n | n % | n | n % | n |
| Total | | | | | | | | | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA

Table 10.1.1.1 Unsolicited AE and ADR by study vaccination number (2-23 months)

| | | | 1 N | <b>1</b> =0 | | | | | 2 N | V=0 | | | | 3 N | 1=0 | | | | | 4 N | 1=0 | | | | То | otal | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety set | | AE | | | ADR | | | ΑE | | ADR | 1 | | AE | | | ADR | | | ΑE | | ADR | | | AE | | | ADR | ξ |
| | | | N | | | N | | | N | | N | | | N | | | N | | | N | | N | | | N | | | N |
| | | iden<br>Rate | o.<br>of<br>A<br>Es | ce I | iden<br>Rate | o.<br>of<br>A<br>Es | | iden<br>Rate | o.<br>of<br>A<br>Es | Inciden<br>ce Rate | o.<br>of<br>A<br>Es | | eiden<br>Rate | o.<br>of<br>A<br>Es | | iden<br>Rate | o.<br>of<br>A<br>Es | Incid<br>ce R | | o.<br>of<br>A<br>Es | Inciden<br>ce Rate | o.<br>of<br>A<br>Es | | iden<br>Rate | o.<br>of<br>A<br>Es | | iden<br>Rate | o. of A |
| | n | (<br>%<br>) | n | n | (<br>% | n | n | (<br>%<br>) | | | n | n | (<br>%<br>) | n | n | ( % | n | n | (<br>%<br>) | | | n | n | (<br>%<br>) | n | n | (<br>% | n |
| System Organ Class(SOC) Preferred Term(PT) | | | | | , | | | | | | | | | | | 1 | | | | | | | | | | | , | |
| Total | | | | | | | | | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA

### 10.2 Safety per protocol Set

Table 10.2.1 Unsolicited AE and ADR

| | 2. | -23 n | nonths | | | 2- | 10 | | | 11 | -18 | | | 19 | -34 | | | 35 | -55 | | | То | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety per protocol set | AE | | ADI | 2 | AE | | ADI | ١ | AE | | ADF | } | AE | | ADR | | AE | | ADF | 1 | AE | | ADI | R |
| | Incid<br>ence<br>Rate | N 0 0 F A A E E S | Incid<br>ence<br>Rate | N o o f A E s | Incid<br>ence<br>Rate | | Incid<br>ence<br>Rate | N o f A E s | Incid<br>ence<br>Rate | N 0 0 f A E E s | Incid<br>ence<br>Rate | N 0 0 f A E E s | Incid<br>ence<br>Rate | N o f A E | Incid<br>ence<br>Rate | N o o f A E | Incid<br>ence<br>Rate | N o o f A E | Incid<br>ence<br>Rate | N o o f A E s | Incid<br>ence<br>Rate | N o o f A E | Incid<br>ence<br>Rate | N 0 0 6 f A A E S |
| System Organ Class(SOC) Preferred Term(PT) | (<br>n % | m | (<br>n % | · | n | | | n | n % | n | n % | n | (<br>n % | | | 1 | (<br>n %<br>) | n | (<br>n % | n | n % | n | (<br>n % | n |

| | 2-23 months | | | | | 2- | 10 | | | 11 | -18 | | | 19 | -34<br>I | | | 35 | -55<br>I | | | To | tal | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety per protocol set | AE | I | ADR | | AE | | ADF | <b>!</b> | AE | | ADF | | ΑE | ı | ADR | | AE | | AD | R | AE | | A | DR <sub>.</sub> | |
| | Incid<br>ence<br>Rate | N 0 0 f A A E s | Incid<br>ence<br>Rate | N 0 0 f A E s | Incid<br>ence<br>Rate | f | Incid<br>ence<br>Rate | N o f A E | Incid<br>ence<br>Rate | N 0 0 f A E S | Incid<br>ence<br>Rate | N 0 0 f A E s | Incid<br>ence<br>Rate | N 0 0 f A E S | Incid<br>ence<br>Rate | N 0 . 0 f A E s | Incid<br>ence<br>Rate | N 0 0 f A A E S | Incid<br>ence<br>Rate | N o o f A E | Incid<br>ence<br>Rate | N o o f A E | Inci<br>ence<br>Rate | id e | N o f A E |
| | (<br>n % | n | n % | n | n | | | n | (<br>n % | n | n % | n | n % | | | 1 | n % | n | n % | n | n % | n | n | % | n |
| Total | | | | | | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA

Table 10.2.1.1 Unsolicited AE and ADR by study vaccination number (2-23 months)

| | | | 1 N | <b>1=</b> 0 | | | | | 2 N | 1=0 | | | | 3 N | <b>1</b> =0 | ) | | | 4 | N=0 | | | | То | otal | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety Per Protocol<br>set | | ΑE | | | ADF | ₹ | | ΑE | | ADR | L | | AE | | | ADR | | A | Е | ADI | ₹ | | AE | | P | DR | |
| | | iden<br>Rate | N o. of A Es | Inci<br>ce F | | N o. of | | iden<br>Rate | N o. of A Es | Inciden<br>ce Rate | N<br>o.<br>of<br>A<br>Es | | eiden<br>Rate | N o. of A Es | | nciden<br>e Rate | N o. of A Es | Incider<br>ce Rate | of | ce Rate | N o. of A Es | | iden<br>Rate | N o. of A Es | Incid<br>ce Ra | | N o. of A Es |
| | n | (<br>%<br>) | n | n | (<br>%<br>) | n | n | (<br>%<br>) | | | n | n | (<br>%<br>) | n | n | ( % | n | n % | | | n | n | (<br>%<br>) | n | n | (<br>%<br>) | n |
| System Organ Class(SOC) Preferred Term(PT) | | | | | | | | | | | | | | | | | | | | | | - | | | | | |
| Total | | | | | | | | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA

### 10.3 Non-Safety per protocol Set

Table 10.3.1 Unsolicited AE and ADR

| | 2- | -23 r | nonths | | | 2- | 10 | | | 11 | -18 | | | 19 | -34 | | | 35- | -55 | | | <u>&gt;</u> | 56 | | | Tot | al | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non-Safety per protocol set | AE | : | ADI | ₹ | AE | | ADI | ₹ | AE | | ADI | ₹ | AE | | ADI | ₹ | AE | | ADF | 2 | AE | | ADR | Ŀ | AE | | ADF | 3 |
| | | N | | N | | N | | N | | N | | N | | N | | N | | N | | N | | N | | N<br>o | | N | | N |
| | | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | | | | o | | |
| | Incid | 0 | - | 0 | Incid | 0 | Inci<br>denc | 0 | Inci<br>denc | o | Inci<br>denc | 0 | Inci<br>denc | 0 | Inci<br>denc | 0 | Inci<br>denc | 0 | Inci<br>denc | 0 | Inci<br>denc | o | Inci<br>denc | o | Inci .<br>den | | den | o |
| | Rate | f<br>A | Rate | f<br>A | Rate | | e<br>Rate | f<br>A | e<br>Rate | | e<br>Rate | f<br>A | e<br>Rate | f<br>A | e<br>Rate | f<br>A | e<br>Rate | f<br>A | e<br>Rate | f<br>A | e<br>Rate | | e<br>Rate | f | ce<br>Rate | f<br>A Re | | f |
| | | Е | | Е | | Е | | Е | | Е | 1 | Е | 11000 | Е | | Е | | Е | | Е | 1 | Е | | Α | | Е | | Α |
| | | S | | S | | S | | S | | S | | S | | S | | S | | S | | S | | S | | E<br>s | | S | | E |
| | n % | n | n % | n | | | | n | (<br>n % | | (<br>nn% | 6 n | (<br>n % | | | n | (<br>n % | | (<br>n n % | ó n | (<br>n % | | | n | (<br>n % | n | n % | n n |
| | ) | | ) | | | | | | ) | | ) | | ) | | | | ) | | ) | | ) | | | | ) | | ) | |
| System Organ | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Class(SOC) | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Preferred Term(PT) | | | | | | | | | | | | | | | | | | | | | | | | | | | | |

| | | 2- | -23 r | nonths | | | 2- | 10 | | | 11 | -18 | | | 19 | -34 | | | 35- | -55 | | | <u>&gt;</u> | 56 | | | Tota | al | _ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non-Safety protocol set | per | AE | | ADI | 2 | AE | | ADI | } | AE | | ADI | ~ | AE | | ADF | ₹ | AE | | ADI | ₹ | AE | | ADR | <b>\</b> | AE | | ADR | \<br>! |
| | | Incid<br>ence<br>Rate | N 0 0 f A E S | Incid<br>ence<br>Rate | N 0 0 f A A E s | Incid<br>ence<br>Rate | f | Inci<br>denc<br>e<br>Rate | N 0 0 f A E s | Inci<br>denc<br>e<br>Rate | o<br>f | Inci<br>denc<br>e<br>Rate | N 0 . 0 f A E S | Inci<br>denc<br>e<br>Rate | f | Inci<br>denc<br>e<br>Rate | N 0 0 f A E S | Inci<br>denc<br>e<br>Rate | f | Inci<br>denc<br>e<br>Rate | N 0 0 f A E S | Inci<br>denc<br>e<br>Rate | f | Inci<br>denc<br>e<br>Rate | N o · · · o f | Inci . den ce Rate A | o<br>f | ce | N 0 0 f |
| | | (<br>n %<br>) | n | (<br>n % | n | | | | n | (<br>n % | | nn% | o n | (<br>n % | | | n | (<br>n % | | (<br>nn%<br>) | o n | n % | Mile on the control of the control o | | S | n % | n | (<br>n % | S |
| Total | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA

Table 10.3.1.1 Unsolicited AE and ADR by study vaccination number (2-23 months)

| | | 1 N | N=0 | | | 2 1 | N=0 | | | | 3 N | I=0 | | | 4 1 | N=0 | | | | То | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non-Safety per protocol set | AE | | ADI | ₹ | A | Ξ | ADR | <b>t</b> | | AE | | ADF | ₹ | A | Ε | ADR | ł. | | AE | | AΣ | R |
| | Inciden ce Rate | N o. of A Es | Inciden<br>ce Rate | N o. of A Es | Inciden | of | Inciden<br>ce Rate | N o. of | | eiden<br>Rate | N o. of A Es | Inciden<br>ce Rate | N o. of A Es | Incider | of | Inciden<br>ce Rate | N o. of A Es | Incid<br>ce Ra | | N o. of A Es | Inciden | of |
| | n % | | n % | n | n % | | | n | n | (<br>%<br>) | | (<br>n % | n | n % | | | n | n | (<br>%<br>) | | n % | |
| System Organ Class(SOC) Preferred Term(PT) | | | | | | | | | | | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA

### 11. Continuous Solicited AE (After 7 days)

Table 11.1.1 Continuous Solicited AE

| | 2- | -23 r | nonths | | | 2- | 10 | | | 11 | -18 | | | 19- | 34 | | | 35- | -55 | | | ≥ | 56 | | | Tot | al | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety set | AE | , | AD | R | AE | | ADI | χ. | AE | | ADI | ~ | AE | | ADF | $\sim$ | AE | | ADF | ξ. | AE | | ADR | | AE | | ADI | 3 |
| | Incid<br>ence<br>Rate | N o o f f A E S | Incid<br>ence<br>Rate | N o o f A A E S | Incid<br>ence<br>Rate | N o o f A E E s | Inci<br>denc<br>e<br>Rate | N o . o f A E E s | Inci<br>denc<br>e<br>Rate | N o o f A E s | Inci<br>denc<br>e<br>Rate | N o c f A E s | Inci<br>denc<br>e<br>Rate | N o o f A E s | Inci<br>denc | N 0 0 f A A E S | Inci<br>denc<br>e<br>Rate | | Inci<br>denc<br>e<br>Rate | N o o f A E s | e | f | Inci<br>denc<br>e<br>Rate | N o o o f f E S | Inci . den ce Rate 4 | o<br>f | den<br>ce<br>ate | |
| System Organ Class(SOC) Preferred Term(PT) | (<br>n % | *** | (<br>n % n | ************************************** | | | | The same of the sa | (<br>n % | n 1 | (<br>n % n | | (<br>n % | | | | (<br>n % | n r | (<br>1 % n<br>) | | n % | 1110 - 1100 - 1001 - 100 - 1001 - | | Δ | n % | n | ( n % | 5 n |

| | 2- | -23 n | nonths | | | 2- | 10 | | | 11 | -18 | | | 19 | -34 | | | 35- | -55 | | | ≥ | 56 | | | То | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety set | AE | | ADI | Ŗ | AE | | ADI | ? | AE | | ADF | ~ | AE | | ADF | ? | AE | | ADI | ₹ | AE | | ADR | | AE | | ADI | —<br>} |
| Safety set | Incid ence Rate | N o o f A E E s | Incid<br>ence<br>Rate | N o f A E s | Incid<br>ence<br>Rate | N o o f | Inci<br>denc | N o o f A E s | Inci<br>denc<br>e<br>Rate | N o o f A E s | Inci<br>denc<br>e<br>Rate | N<br>o<br>o | Inci denc e Rate | N<br>o<br>o | Inci<br>denc | N o | Inci<br>denc<br>e<br>Rate | N 0 0 0 f A E E s | Inci<br>denc<br>e<br>Rate | | Inci<br>denc<br>e<br>Rate | N<br>o<br>o | Inci<br>denc<br>e<br>Rate | N 0 | Inci . | N o lnci | den<br>ce<br>ate | N O O f E S S |
| Total | ) | | ) | | | | | The state of the s | ) | | ) | | ) | | | A THE RESIDENCE AND A STREET OF THE PROPERTY O | ) | | ) | | | | | | | | ) | |

<sup>\*</sup> MedDRA

Table 11.1.1.1 Continuous Solicited AE by study vaccination number (2-23 months)

| | | | 1 N | <b>V=</b> 0 | | | | | 2 N | V=0 | | | | 3 N | 1=0 | | | | | 4 N | 1=0 | | | | То | otal | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety Set | | ΑE | | | ADR | | | ΑE | | ADR | | | AE | | | ADR | | , | <b>Λ</b> E | | ADR | - | | AE | | | ADR | 2 |
| | | | N | | | N | | | N | | N | | | N | | | N | | | N | | N | | | N | | | N |
| | | iden<br>Rate | o. of A Es | ce I | den | o.<br>of<br>A<br>Es | | iden<br>Rate | o. of A Es | Inciden<br>ce Rate | o.<br>of<br>A<br>Es | | eiden<br>Rate | o.<br>of<br>A<br>Es | Incid<br>ce R | | o.<br>of<br>A<br>Es | Incide ce Ra | en<br>te | o.<br>of<br>A<br>Es | Inciden<br>ce Rate | o.<br>of<br>A<br>Es | | iden<br>Rate | o.<br>of<br>A<br>Es | | iden<br>Rate | o.<br>of<br>A<br>Es |
| | n | (<br>%<br>) | n | n | (<br>%<br>) | n | n | (<br>%<br>) | | | n | n | (<br>%<br>) | n | n | (<br>% | n | n | <b>%</b> | | | n | n | (<br>%<br>) | n | n | (<br>%<br>) | n |
| System Organ Class(SOC) Preferred Term(PT) | - | | | | | | | | | | | | | | | | | | | | | | | | | | , | |
| Total | | | | | | | | | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA

### 11.2 Safety per protocol set

Table 11.2.1 Continuous Solicited AE

| | 2 | -23 r | nonths | | | 2- | 10 | | | 11 | -18 | | | 19 | -34 | | | 35 | -55 | | | To | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety per protocol set | AE | | ADF | ₹ | AE | , | ADI | 2 | AE | | ADI | ₹ | AE | , | ADR | | AE | | ADF | t | AE | | ADR | |
| | Incid<br>ence<br>Rate | N 0 | Incid<br>ence<br>Rate | N 0 0 f A A E s | Incid<br>ence<br>Rate | N o. o f A E | Incid<br>ence<br>Rate | N o o f A E s | Incid<br>ence<br>Rate | N o o f A E E s | Incid<br>ence<br>Rate | N 0 c f A E E s | Incid<br>ence<br>Rate | N o o f A E E s | Incid<br>ence<br>Rate | N o f A E s | Incid<br>ence<br>Rate | N o f A E | Incid<br>ence<br>Rate | N o o f A E s | Incid<br>ence<br>Rate | N o o f A E | Incid<br>ence<br>Rate | N o o f A E s |
| System Organ Class(SOC) Preferred Term(PT) | ( n % ) | n | (<br>n % | <u> </u> | n | | | n | n % | n | (<br>n % | | (<br>n % | | | n | (<br>n %<br>) | n | (<br>n % | | (<br>n %<br>) | n | (<br>n % | m |
| | 2- | -23 n | nonths | | | 2- | 10 | | | 11 | -18 | | | 19 | -34 | | | 35 | <b>-</b> 55 | | | То | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety per protocol set | AE | | AD | R | AE | ) | ADI | <b>?</b> | AE | | ADF | 2 | AE | | ADR | | AE | | ADI | 2 | Al | Ξ | AD | R |
| | Incid<br>ence<br>Rate | N 0 0 f A E s | Incid<br>ence<br>Rate | N o o f A E s | Incid<br>ence<br>Rate | | Incid<br>ence<br>Rate | N o o f A E E s | Incid<br>ence<br>Rate | N 0 . 0 f A E s | Incid<br>ence<br>Rate | N 0 0 f A E s | Incid<br>ence<br>Rate | N o o f A E s | Incid<br>ence<br>Rate | N o o f A E s | Incid<br>ence<br>Rate | N o o f A E | ence<br>Rate | N o o f A E s | Incid<br>ence<br>Rate | N o o f A A E S | Incid<br>ence<br>Rate | N o f A E |
| Total | n % | n | n % | <u> </u> | n | | | n | n % | n | n % | n | n % | | | n | n % | n | n % | n | n % | n | n % | 6 n |

<sup>\*</sup> MedDRA

Table 11.2.1.1 Continuous Solicited AE by study vaccination number (2-23 months)

| | | | 1 N | V=0 | | | | | 2 N | 1=0 | | | | 3 N | 1=0 | | | | | 4 N | 1=0 | | | | То | otal | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety Per Protocol<br>Set | | AE | | | ADR | l. | | AE | | ADR | | | AE | | A | DR | | | AE | | ADR | - | | AE | | | ADR | |
| | ce] | iden<br>Rate | N<br>o.<br>of<br>A<br>Es | ce F | den<br>Rate | N o. of A Es | ce l | iden<br>Rate | N<br>o.<br>of<br>A<br>Es | Inciden<br>ce Rate | N o. of A Es | ce | iden<br>Rate | N o. of A Es | Incide<br>ce Ra | te | N o. of A Es | Inci<br>ce R | Rate | N o. of A Es | Inciden<br>ce Rate | N o. of A Es | ce ] | iden<br>Rate | N o. of A Es | Inci<br>ce F | ate | N o. of A Es |
| | n | % | n | n | % | n | n | % | | | n | n | % | n | n ( | 6 | n | n | % | | | n | n | % | n | n | % | n |
| System Organ Class(SOC) Preferred Term(PT) | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA

# 11.3 Non-Safety per protocol set

Table 11.3.1 Continuous Solicited AE

| | 2 | -23 1 | nonths | | | 2- | 10 | | | 11 | -18 | | | 19 | -34 | | | 35- | -55 | | | <u>&gt;</u> | 56 | | | Tot | al | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non-Safety per protocol set | AH | Ē | ADI | 2 | AE | Į. | ADI | R | AE | | ADI | ₹ | AE | | ADF | <b>t</b> | AE | | ADF | 3 | AE | | ADR | L | AE | | ADI | 3 |
| | Incid<br>ence<br>Rate | N o o f A E s | Incid<br>ence<br>Rate | N o o f A A E | Incid<br>ence<br>Rate | f | Inci<br>denc<br>e<br>Rate | N 0 0 f A E E s | Inci<br>denc<br>e<br>Rate | f | Inci<br>denc<br>e<br>Rate | N 0 0 f A A E | Inci<br>denc<br>e<br>Rate | o<br>f | Inci<br>denc<br>e<br>Rate | N o . o f A E s | Inci<br>denc<br>e<br>Rate | N o f A E | Inci<br>denc<br>e<br>Rate | N o o f A E s | Inci<br>denc<br>e<br>Rate | | Inci<br>denc<br>e<br>Rate | N o o f | Inci . den ce Rate | o<br>f | den<br>ce | N o o f |
| System Organ Class(SOC) Preferred Term(PT) | ( n % ) | | (<br>n %<br>) | n | | | | n | (<br>n % | | (<br>nn%<br>) | | (<br>n % | 3 | | n | (<br>n %<br>) | 3 | (<br>nn%<br>) | | ( n % ) | | | s s | (<br>n % | | n % | S |

| Non-Safety per protocol set Incidence Rate | d c | ADI | R N 0 0 | AE | N | ADF | N | AE | N | ADF | N | AE | | ADR | | AE | | ADF | <b>\</b> | AE | | ADR | N | AE | | ADI | R<br>N |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ence | d c | Incid | o | Incid | О | | | | N | | N | | | | | | | | | | | : | N | | | | N |
| | F | Rate | f A E s | ence<br>Rate | o<br>f | Inci<br>denc<br>e<br>Rate | o<br>o<br>f<br>A<br>E | Inci<br>denc<br>e<br>Rate | o<br>f | Inci<br>denc<br>e<br>Rate | o<br>o | Inci<br>denc<br>e<br>Rate | o<br>f | Inci<br>denc | N o o f A E s | Inci<br>denc<br>e<br>Rate | f | Inci<br>denc | N o o f A A E S | Inci<br>denc<br>e<br>Rate | f | Inci<br>denc<br>e<br>Rate | o o f | | o<br>f | den<br>ce | o |
| n % | ( | (<br>n % | n | | | | n | (<br>n %<br>) | | (<br>nn%<br>) | | (<br>n % | | | n | (<br>n %<br>) | | (<br>nn% | | n % | | | n | (<br>n % | | ( n % | s<br>n |

<sup>\*</sup> MedDRA

Table 11.3.1.1 Continuous Solicited AE by study vaccination number (2-23 months)

| | | | 1 N | 1=0 | | | | | 2 N | 1=0 | | | | 3 N | 1=0 | | | 4 N | N=0 | | | | То | otal | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Non-Safety Per<br>Protocol Set | | AE | | | ADR | t | | ΑE | | ADR | | | AE | | ΑI | )R | AE | | ADR | | | AE | | | ADR | Ł |
| | | eiden<br>Rate | N o. of A Es | | iden<br>Rate | N o. of A Es | | iden<br>Rate | N o. of A Es | Inciden<br>ce Rate | N o. of A Es | | eiden<br>Rate | N o. of A Es | Incider<br>ce Rate | of | Inciden<br>ce Rate | N o. of A Es | Inciden<br>ce Rate | N o. of A Es | | iden<br>Rate | N o. of A Es | | iden<br>Rate | N o. of A Es |
| | n | (<br>%<br>) | n | n | (<br>%<br>) | n | n | ( % | A 1000 1000 1000 1000 1000 1000 1000 10 | | n | n | (<br>%<br>) | n | n % | n | (<br>n %<br>) | | | n | n | (<br>%<br>) | n | n | (<br>%<br>) | n |
| System Organ Class(SOC) Preferred Term(PT) | | | | | | | | | To the state of th | | | | | | <i>'</i> | | | | | | | | | | | THE REPORT OF THE PROPERTY OF |
| Total | | | | | | | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> MedDRA



# STATISTICAL ANALYSIS PLAN

A Multicenter Post Marketing Surveillance Study to Monitor the Safety of GSK Meningococcal ACWY Conjugate Vaccine (MenACWY-CRM)
Administered According to the Prescribing Information to Healthy
Subjects from 2 months to 55 Years of Age in the Republic of South Korea

Product Name : Menveo (MenACWY-CRM)

Protocol No. : V59\_62

Version : V5.0

Effective Date : 28-JUL-2016

| | | Last Update Date |
|---|---|---|
| | CONFIDENTIAL: | |
| <b>"</b> ":rea <u>r.tt\."</u> f<;;, | THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY | 07-JUL-2016 |
| STATISTICAL ANALYSIS PLAN(V5.0) | | |

# **Approvals**







THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

07-JUL-2016

Last Update Date

# STATISTICAL ANALYSIS PLAN(V5.0)

### **Revisions**

| DATE OF<br>REVISION | INDICATION REVISION | REASON FOR CHANGE | AUTHOR<br>NAME |
|---|---|---|---|
| 22-NOV-2013 | All | Protocol Amendment | PPD |
| 10-APR-2014 | Appendix1 | Modification of tables to include incidence rate of ADR, Fever added to Solicited reaction | PPD |
| 26-JAN-2016 | All | Protocol Amendment | PPD |
| 07-JUL-2016 | 6.3 Additional Analyses for DDS (Data Disclosure Shell) 7.4 Additional Analyses for DDS (Data Disclosure Shell) | Add the DDS(Data Disclosure Shell) analysis Add the DDS(Data Disclosure Shell) analysis Add the DDS(Data Disclosure | PPD |
| 07 301 2010 | 8. Notes | Shell) analysis in re-examination report | |
| | Appendix1 | Add the DDS(Data Disclosure<br>Shell) analysis | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

07-JUL-2016

Last Update Date

# STATISTICAL ANALYSIS PLAN(V5.0)

### **Table of Contents**

| Revisions | 3 |
|---------------------------------------------------------|----|
| 1. Study Objective | 6 |
| 2. Study Method and Study Period | 6 |
| 2.1 Study Period | 6 |
| 2.2 Number of Subjects | 6 |
| 2.3 Study population | 6 |
| 2.3.1 Inclusion criteria | 6 |
| 2.3.2 Exclusion criteria | 7 |
| 2.4 Study Method | 7 |
| 3. Analysis Sets | 10 |
| 3.1 Safety Analysis Sets | 10 |
| 3.2 Efficacy Analysis Set | 12 |
| 4. Endpoints | 12 |
| 4.1 Safety Endpoints | 12 |
| 5. Assessment Criteria | 12 |
| 5.1 Safety Assessment Criteria | 12 |
| 6. Statistical Analyses | 13 |
| 6.1 Baseline Characteristics | 13 |
| 6.2 Safety Analyses | 13 |
| 6.2.1 Adverse Events by Baseline Characteristics | 13 |
| 6.2.2. Analysis of Solicited AE | 14 |
| 6.2.3 Analysis of Unsolicited AE | 15 |
| 6.3 Additional Analyses for DDS (Data Disclosure Shell) | 16 |
| 7. List of Table and Data Listings | 16 |
| 7.1 Distribution of Subjects | 16 |
| 7.2 Baseline Characteristics | 17 |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

07-JUL-2016

Last Update Date

# STATISTICAL ANALYSIS PLAN(V5.0)

| 8 N | Notes | 18 |
|-----|---------------------------------------------------------|------|
| | 7.4 Additional Analyses for DDS (Data Disclosure Shell) | . 17 |
| | 7.3 Safety Analyses | . 17 |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

07-JUL-2016

Last Update Date

STATISTICAL ANALYSIS PLAN(V5.0)

### 1. Study Objective

The primary objective of the study is to monitor the safety of a single dose of MenACWY-CRM vaccine in subjects from 2 months to 55 years of age, as evaluated by:

- Local and systemic solicited adverse events reported from study Day 1 (day of vaccination) through study Day 7 post-vaccination.
- All unsolicited Adverse Events (AEs) reported from study Day 1 (day of vaccination) through study Day 7 post-vaccination.
- Medically attended Adverse Events reported from study Day 1 to study termination (Day 29/early termination).
- All Serious Adverse Events (SAEs) reported from study Day 1 to study termination (Day 29/early termination).

### 2. Study Method and Study Period

### 2.1 Study Period

The trial period shall be from market launch date till approximately 22 May 2018.

### 2.2 Number of Subjects

A total of approximately 3,960 subjects are planned for enrolment into this study.

Assuming a 10% drop-out rate, this should provide approximately 3,000 evaluable subjects in the cohort 2 to 55 years of age and 600 in the cohort 2 to 23 months of age. This sample size meets the post-licensure requirements of the MFDS to provide continued safety monitoring in the Korean population.

### 2.3 Study population

### 2.3.1 Inclusion criteria

Individuals eligible for enrolment in this study are those:

# dreamc:s


THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

07-JUL-2016

Last Update Date

# STATISTICAL ANALYSIS PLAN(V5.0)

- 1. Male and female subjects from 2 months to 55 years of the age at the time of vaccination (including all 55 years of age subjects, up to one day before their 56<sup>th</sup> year birthday), who are scheduled to receive vaccination with MenACWY-CRM conjugate vaccine, according to the local prescribing information and routine clinical practice
- 2. To whom the nature of the study has been described and the subject or subject's parent/legal representative has provided written informed consent (written assent from minors should be also obtained if required by the relevant IRB);
- 3. Whom the investigator believes that the subject can and will comply with the requirements of the protocol (e.g., completion of the Diary Card);
- 4. Who are in good health as determined by the outcome of medical history, physical assessment and clinical judgment of the investigator

### 2.3.2 Exclusion criteria

- 1. Contraindication, special warnings and/or precautions, as evaluated by the investigators, reported in the MenACWY-CRM conjugate vaccine Korean prescribing information.
- 2. Infants who were already enrolled in this trial for previous vaccination.

### 2.4 Study Method

In order to obtain information on Regulatory PMS data after-market launch, or delegate will create the Regulatory PMS contract with the relevant clinics/hospitals and the physician in charge of the survey shall implement this Regulatory PMS in subjects that receive MenACWY-CRM in the relevant hospital/clinic since the contract date until the number of contracted survey cases, without omission, is reached.

### Overview of Study Design

This is a multicenter post marketing surveillance study to monitor the safety of MenACWY-CRM administered according to the prescribing information to 3,960 healthy subjects from 2 months to 55 years of age in Korea.

Subjects will be enrolled at the time of their visit to a participating clinic or hospital for vaccination with MenACWY-CRM according to the routine clinical care.



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

07-JUL-2016

Last Update Date

STATISTICAL ANALYSIS PLAN(V5.0)

At Visit 1 (Day 1), after obtaining consent from the subjects or subjects' parents/legal representative (and Assent Form, if required by the relevant IRB), the vaccination will be administered. Subjects will remain under observation for at least 30 minutes in the clinic after study immunization.

The subjects or subject's parent/legal representative will be then instructed to complete the Diary Card daily, reporting local and systemic adverse events and all other AEs occurring within 7 days following immunizations, and medically attended AEs or SAEs occurring up to Day 29 within the surveillance period after each study vaccination.

Subjects will also be instructed to return the completed diaries to the study site at Day 29 as follows:

- During a visit at the study center or
- Using the provided pre-addressed stamped envelope (PASE).

At the investigator discretion, the subject or subject's parent/legal representative will be reminded of the date of the study termination by a phone call at Day 29. If any clarification is required after Diary Card retrieval the site staff will follow up by phone, and any additional finding will be recorded on the subject's medical record.

In case the Diary Card is not retrieved within 10 days after Day 29, subject or subject's parent/legal representative will be contacted by phone to assess the occurrence of adverse events, determine the subject's clinical status and complete study termination. All information will be recorded by the site staff on the subject's medical record and collected in the appropriate section of the CRF.

All SAEs will be monitored until resolution and/or the cause is identified. If a SAE remains unresolved at study termination, a clinical assessment will be made by the investigator and the GSK regional physician to determine whether continued follow up of the SAE is needed.

Table 3.1-1: Safety Assessment Table

| Medical History: | From birth, collected at clinic visit |
|---|---|
| All significant past diagnoses including all allergies, major | Day 1 |
| surgeries requiring inpatient hospitalization, other significant | |
| injuries or hospitalizations, any conditions requiring | |
| prescription or chronic medication (i.e., >2 weeks in duration), | |
| or other significant medical conditions based on the | |
| investigator's judgment. | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

07-JUL-2016

Last Update Date

# STATISTICAL ANALYSIS PLAN(V5.0)

| Immediate reactions: | For at least 30 minutes after |
|---|---|
| Subjects will be assessed for immediate hypersensitivity | vaccination |
| reactions. | |
| Solicited local adverse events: | Days 1-7 after vaccination |
| < 6 years : injection site erythema, injection site induration, | |
| injection site tenderness | |
| $\geq$ 6 years : injection site erythema, injection site induration, | |
| injection site pain | |
| Solicited systemic adverse events: | Days 1-7 after vaccination |
| < 6 years : change in eating habits, sleepiness, irritability, rash, | |
| vomiting, diarrhea, fever | |
| $\geq$ 6 years : chills, nausea, malaise, generalized myalgia, | |
| generalized arthralgia, headache, rash, fever | |
| All unsolicited AEs will be collected | Days 1-7 after vaccination |
| Medically attended Adverse Events: | From Day 1 to study termination |
| Events that require a physician's visit or an emergency room | (Day 29/early termination) |
| visit (events that are managed by telephone or means other than | |
| a face-to-face evaluation by a clinician do not qualify as | |
| medically attended AEs). | |
| Serious AEs: | From Day 1 to study termination |
| All SAEs will be collected. | (Day 29/early termination) |
| Medications: | From Day 1 to Day 7 |
| Any medications used to treat any solicited local and systemic | |
| reaction and unsolicited AE be collected. | |
| Medications: | From Day 1 to study termination |
| Any medications used to treat any medically attended AE or | (Day 29/early termination) |
| SAE will be collected. | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

07-JUL-2016

Last Update Date

# STATISTICAL ANALYSIS PLAN(V5.0)

### 3. Analysis Sets

### 3.1 Safety Analysis Sets

### Safety Set

All subjects who

- have signed an informed consent form, undergone screening procedure(s) and received a subject number,
- received a study vaccination,
- provided post vaccination safety data.

### Safety per protocol set

All subjects in the safety Set with the exclusions of the following cases:

- (1) Subjects administered prior to the contract date.
- (2) Subjects who didn't receive MenACWY-CRM.
- (3) Follow-up failure: The subjects whose safety information cannot be identified due to follow-up loss.
- (4) Not applicable to the indication of study drug [Indication]
  - To prevent invasive meningococcal disease caused by Neisseria meningitides serogroups A, C, Y and W-135 in persons 2 months through 55 years of age.
- (5) Subjects who violate of Protocol: Those who do not meet one item at least of the inclusion/exclusion criteria.

[Inclusion criteria]

- 1) Male and female subjects from 2 months to 55 years of the age at the time of Visit 1 (including all 55 years old subjects, up to one day before their 56<sup>th</sup> year birthday), who are scheduled to receive vaccination with MenACWY-CRM conjugate vaccine, according to the local prescribing information and routine clinical practice.
- 2) To whom the nature of the study has been described and the subject or subject's parent/legal representative has provided written informed consent.
- 3) Whom the investigator believes that the subject can and will comply with the requirements of the protocol.
- 4) Who are in good health as determined by the outcome of medical history, physical

# dreamc:s

#### **CONFIDENTIAL**:

THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

07-JUL-2016

Last Update Date

# STATISTICAL ANALYSIS PLAN(V5.0)

assessment and clinical judgment of the investigator.

[Exclusion criteria]

- 1) Contraindication, special warnings and/or precautions, as evaluated by the investigators, reported in the MenACWY-CRM conjugate vaccine Korean prescribing information
- 2) Infants who were already enrolled in this trial for previous vaccination.
- (6) Subjects who prescribed off-label dosage:
  - Vaccine schedule for children from 2 to 23 months of age :
    - Infants 2 to 6 months of age: Three doses of MenACWY-CRM, each of 0.5 ml, is to be given with an interval of at least 2 months; the fourth dose schedule be administered during the second year of life with an interval of at least 6 months after the third dose.
    - Infants 7 to 23 months of age: MenACWY-CRM is to be administered as two doses, each as single dose (0.5ml), with the second dose administered in the second year of life and at least three months after the first dose.
  - 2 to 55 years of age: MenACWY-CRM is to be administered as a single dose (0.5ml).
  - \* The infant from 2 to 23 months of age may enroll at any point, in the vaccination series, including those subjects who may already initiated vaccination series. According to parental consents, these subjects may be followed up for 29 days within the surveillance period after subsequent vaccination(s) at the same study site.

### Non-Safety per protocol set

Subjects excluded from safety per protocol set except for subjects who did not receive MenACWY-CRM and follow-up failure.

Based on rules for estimation of each number of safety evaluation cases, the following local regulation and Guideline on Standards for re-examination for new drugs, etc of MFDS, non-safety analysis set are excluded from the safety analysis set:

Guideline on Standards for re-examination for new drugs, etc (Chapter II, no. 3) Patient Population for Surveillance:

- A) Patients planned to receive a drug under surveillance by investigator's medical ju dgment shall be subject.
- B) Subject who do not use within approved range shall not be included in the subject in principal.

However, if data of subject whose use is beyond approved range is collected, p erform analysis as a separate item.



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

07-JUL-2016

Last Update Date

STATISTICAL ANALYSIS PLAN(V5.0)

C) Describe actual selection methods of subject in detail.

### 3.2 Efficacy Analysis Set

Not Applicable

### 4. Endpoints

### 4.1 Safety Endpoints

Safety will be assessed after administration of study vaccine in terms of the number and percentage of subjects with:

- Local and systemic solicited adverse events reported from study Day 1 (day of vaccination) through study Day 7 post-vaccination;
- Unsolicited AEs reported from study Day 1 (day of vaccination) through study Day 7 post-vaccination;
- Medically attended AEs reported from study Day 1 to study termination (Day 29/early termination);
- SAEs reported from study Day 1 to study termination (Day 29/early termination).

### 5. Assessment Criteria

### 5.1 Safety Assessment Criteria

Not Applicable



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

07-JUL-2016

Last Update Date

# STATISTICAL ANALYSIS PLAN(V5.0)

### 6. Statistical Analyses

### **6.1 Baseline Characteristics**

Descriptive statistics (mean, standard deviation, median, minimum and maximum) for baseline characteristics such as age, height and weight at enrollment will be calculated in the Safety set and Safety per Protocol set.

The following baseline characteristics will be reported:

- < Subject Baseline Information >
  - gender, age, ethnic origin, children group, weight, height, past diagnosis, kidney disorder, liver disorder, pre-Immunization temperature, temperature location, pregnancy
- < Study Vaccine Information >
  - vaccine site, number of previous Menveo, study vaccination number, concomitant medications

### **6.2 Safety Analyses**

The number of subjects of AE<sup>†</sup> and the number of AEs<sup>†</sup> incurred shall be calculated, the incidence rate of AEs<sup>†</sup> and its 95% confidence interval will be calculated using the normal approximation on the safety set and safety per protocol set.

† AE : AE includes solicited and unsolicited AE (DAY 1-7), medically attended AE (DAY 1-29) and SAE (DAY 1-29).

### 6.2.1 Adverse Events by Baseline Characteristics

 $AE^{\dagger}s$  (as described below) will be reported (n %) for the following baseline characteristics in the safety set and safety per protocol set :

- Age group (2-23 months, 2-10, 11-18, 19-34, 35-55)
- Children group ( $<18, \ge 18$ )
- Gender (male, female)
- Past diagnosis (yes, no)



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

07-JUL-2016

Last Update Date

# STATISTICAL ANALYSIS PLAN(V5.0)

- Temperature location (axillary, oral, rectal, ear)
- Administration site (left deltoid, right deltoid, left thigh, right thigh, other)
- Concomitant medication (yes, no)
- Kidney disorder (yes, no)
- Liver disorder (yes, no)
- Pregnancy (yes, no)
- Number of previous Menveo (0, 1, 2, 3)
- Study vaccination number (1, 2, 3, 4)

The n(%) of AEs<sup>†</sup> and its 95% confidence interval will be calculated using the normal approximation and analyzed using  $\chi^2$ - test.If more than 20% of expected frequencies of the cell counts are less than 5, Fisher's exact test will be used instead of the chi-square test.

† AE : AE includes solicited and unsolicited AE (DAY 1-7), medically attended AE (DAY 1-29) and SAE (DAY 1-29).

### **6.2.2.** Analysis of Solicited AE

Frequencies and % of subjects experiencing each adverse event will be presented for each symptom severity. Summary tables showing the occurrence of any local or systemic reaction overall and at each time point will also be presented (see Appendix 1 Table 4.1.3 and 4.2.3).

Post-vaccination adverse events reported from Day 1 to Day 7 will be summarized by maximal severity. The severity of local adverse events for subjects < 6 years of age will be categorized as follows. Injection-site erythema and induration: absent (0 to 9 mm), mild (10 to 25 mm), moderate (26 to 50 mm), severe (> 50 mm); injection-site tenderness: none, mild (minor light reaction to touch), moderate (cried or protested to touch), severe (cried when injected limb was moved). For subjects  $\ge$  6 years, injection-site erythema and induration absent (1 to 24 mm), mild (25 to 50 mm), moderate (51 to 100 mm), severe (>100 mm); pain: none, mild (present but does not interfere with activity), moderate (interferes with activity), severe (prevents daily activity).

For subjects  $\geq$  6 years of age, the severity of systemic adverse events (i.e., chills, nausea, malaise, generalized myalgia, generalized arthralgia, headache) occurring up to 7 days after each vaccination will be categorized as none, mild (present but not interfering with daily activity), moderate (some interference with daily activity), and severe (prevents daily activity) except for rash, which will be



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

07-JUL-2016

Last Update Date

# STATISTICAL ANALYSIS PLAN(V5.0)

categorized as none, urticarial, or other.

For subjects < 6 years of age, the severity of systemic adverse events occurring up to 7 days after each vaccination will be categorized as follows. Change in eating habits: none (no change in appetite), mild (eating less than normal for 1 to feeds), moderate (missed 1 or 2 feeds), severe (missed more than 2 feeds); sleepiness: none (no change in alertness), mild (shows an increased alertness), moderate (sleeps through feeds), severe (sleeps most of the time and it is hard to arouse him/her); irritability: none (no change in child disposition), mild (requires more cudding and he/she is less playful than usual), moderate (more difficult to settle), severe (unable to console); rash: none, urticarial, or other; vomiting: none, mild (1-2 episodes/24 hours), moderate (>2 episodes/24 hours), severe (requires outpatient hydratation); diarrhea: none (fewer than 2 loose stools/24 hours), mild (2-3 loose stools or < 400 gms/24 hours), moderate (4-5 stools or 400-800 gms/24 hours), severe (6 or more watery stools or > 800 gms/24 hours or requires outpatient IV hydration).

Body temperature will be categorized as  $<38^{\circ}$ C (no fever),  $\ge 38^{\circ}$ C (fever) and will be summarized by  $0.5^{\circ}$ C increments from  $36.0^{\circ}$ C up to  $\ge 40^{\circ}$ C. Additionally, no fever vs. fever will be reported.

Each local and systemic adverse event will also be categorized as none vs. any.

### 6.2.3 Analysis of Unsolicited AE

All unsolicited AEs and MAAE recorded in the CRF will be mapped to preferred terms using the most recent MedDRA dictionary and classified by System organ class (SOC) and Preferred Terms (PT). Under the classification standard of MedDRA terms, and all AEs excluding the AEs whose causal relation with the study medication is 'Not Related' shall be treated as AEs whose causal relation cannot be excluded {hereafter "Adverse Drug Reaction(ADR)"}.

- ① The frequency and percentage of unsolicited AE (Day 1-7) and MAAE (Day 8-29) according to the expected, serious, severity, frequency, action taken, outcome, relationship to MenACWY-CRM regarding occurred AE will be calculated.
- ② The frequency of unsolicited AEs (Day 1-7) and MAAE (Day 8-29) will be classified into the preferred terms according to the expected, serious, severity, frequency, action taken, outcome, relationship to MenACWY-CRM.
- 3 The number of subjects and percentage of SAE/Serious ADR (SADR), unexpected AE/ADR,



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

07-JUL-2016

Last Update Date

# STATISTICAL ANALYSIS PLAN(V5.0)

MAAE/ADR, unsolicited AE/ADR and continuous solicited AE/ADR will be calculated according to the preferred terms. And the number of subjects and percentage by study vaccination number of SAE/Serious ADR (SADR), unexpected AE/ADR, MAAE/ADR, unsolicited AE/ADR and continuous solicited AE/ADR will be calculated according to the preferred terms in infants 2 to 23 months.

④ For subjects excluded from safety per protocol set<sup>†</sup>, the number of subjects and the percentage of SAE/Serious ADR (SADR), unexpected AE/ADR, MAAE/ADR, unsolicited AE/ADR and continuous solicited AE/ADR will be calculated according to the preferred terms. And the number of subjects and percentage by study vaccination number of SAE/Serious ADR (SADR), unexpected AE/ADR, MAAE/ADR, unsolicited AE/ADR and continuous solicited AE/ADR will be calculated according to the preferred terms in infants 2 to 23 months.

Subject excluded from safety per protocol set: Except for subjects who didn't receive study vaccination and follow-up failure.

### 6.3 Additional Analyses for DDS (Data Disclosure Shell)

The following will be presented in the Safety set and Safety per Protocol set.

- Frequency and percentage by Age group (2-23 months, 2-11 12-17, 18-64) will be presented.
- Frequency and percentage by study termination and reason not completed will be presented.
- The number of subjects of Non-SAE and the number of Non-SAE incurred shall be calculated, the incidence rate of Non-SAE and its 95% confidence interval will be calculated using the normal approximation.
- The number of death resulting from AE shall be calculated.
- The number of subjects and percentage of Non-SAE will be calculated according to the preferred terms.

### 7. List of Table and Data Listings

### 7.1 Distribution of Subjects

- Number of subjects contracted to the study: The number of subjects are to be collected(under contract) as contracted by the investigator.

# **d**reamc:s


THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

07-JUL-2016

Last Update Date

STATISTICAL ANALYSIS PLAN(V5.0)

- Number of retrieving completed CRFs: Total number of subjects whose completed CRFs.
- Number of safety assessment population: Number of safety assessment population among total number.

### 7.2 Baseline Characteristics

- Mean and standard deviation (SD) or frequency and percentage by gender, age, ethnic origin, weight, height, past diagnosis, pre-Immunization temperature, temperature location, pregnancy
- Frequency and percentage by vaccine site, number of previous Menveo, study vaccination number, concomitant medications.

### 7.3 Safety Analyses

- Incidence rate and the number of AEs according to the baseline characteristics (frequency and percentage).
- The number of the expected serious, severity, frequency, action taken, outcome, relationship to MenACWY-CRM for Unsolicited AE (DAY 1-7) and MAAE (DAY 8-29) (frequency and percentage).
- The number of AEs for the severity, day, fever to MenACWY-CRM according to individual solicited AE (DAY 1-7) (frequency and percentage)..
- Incidence rate and number according to the preferred terms of SAE/SADR, unexpected AE/ADR, MAAE/ADR, unsolicited AE/ADR and continuous solicited AE/ADR (frequency and percentage)
- For subjects excluded from safety per protocol set<sup>†</sup> incidence rate and number according to the preferred terms of SAE/SADR, unexpected AE/ADR, MAAE/ADR, unsolicited AE/ADR and continuous solicited AE/ADR (frequency and percentage).

Subject excluded from safety per protocol set: Except for subjects who didn't receive study mediation and follow-up failure.

### 7.4 Additional Analyses for DDS (Data Disclosure Shell)

- Frequency and percentage by Age group (2-23 months, 2-11 12-17, 18-64)
- Frequency and percentage by study termination and reason not completed
- Incidence rate and the number of Non-SAE
- The number of death resulting from AE (frequency and percentage)



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

07-JUL-2016

Last Update Date

# STATISTICAL ANALYSIS PLAN(V5.0)

- Incidence rate and number according to the preferred terms of Non-SAE (frequency and percentage)

### 8. Notes

- Each statistical analysis will be carried out with SAS Software version 9.4 or more recent version.
- In the descriptive statistics, mean, SD, minimum, median, and maximum will be calculated for continuous variables, and frequency and percentage for categorical variables.
- Data including sign of inequality such as "\ge 20", "\ge 20" will be excluded from analysis.
- All test statistics will be the results of two-sided tests with the statistical significant level of 0.05.
- The followings shall be included only in re-examination report:
  - Analysis by type of concomitant medications
  - Item ② of paragraph 6.2.3
  - Estimation of 95% confidence interval for incidence of AEs by background factors
  - Paragraph 6.3



# STATISTICAL ANALYSIS PLAN

A Multicenter Post Marketing Surveillance Study to Monitor the Safety of GSK Meningococcal ACWY Conjugate Vaccine (MenACWY-CRM)
Administered According to the Prescribing Information to Healthy
Subjects from 2 months to 55 Years of Age in the Republic of South Korea

Product Name : Menveo (MenACWY-CRM)

Protocol No. : V59\_62

Version : V6.0

Effective Date : 23-APR-2018



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY

20-APR-2018

Last U date Date

# STATISTICAL ANALYSIS PLAN(V6.0)

### **Approvals**







THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

20-APR-2018

Last Update Date

# STATISTICAL ANALYSIS PLAN(V6.0)

### **Revisions**

| DATE OF<br>REVISION | INDICATION REVISION | REASON FOR CHANGE | AUTHOR<br>NAME |
|---|---|---|---|
| 22-NOV-2013 | All | Protocol Amendment | PPD |
| | | Modification of tables to include | |
| 10-APR-2014 | Appendix1 | incidence rate of ADR, | PPD |
| | | Fever added to Solicited reaction | |
| 26-JAN-2016 | All | Protocol Amendment | PPD |
| | 6.3 Additional Analyses for DDS | Add the DDS(Data Disclosure | |
| | (Data Disclosure Shell) | Shell) analysis | |
| | 7.4 Additional Analyses for DDS | Add the DDS(Data Disclosure | |
| | (Data Disclosure Shell) | Shell) analysis | |
| 07-JUL-2016 | | Add the DDS(Data Disclosure | PPD |
| | 8. Notes | Shell) analysis in re-examination | |
| | | report | |
| | Ann an din 1 | Add the DDS(Data Disclosure | |
| | Appendix1 | Shell) analysis | |
| | All | Using more appropriate word | |
| | 6.2.3 Analysis of Unsolicited AE | Change the of oritoric MAAF | |
| | 7.3 Safety Analyses | Change the of criteria MAAE | |
| | 6.4 Additional Analyses for AE in | | |
| 20-APR-2018 | the Local Product Document | | PPD |
| | (Unsolicited AE Day 1-29) | Add the analysis requested by | |
| | 7.5 Additional Analyses for AE in | MFDS | |
| | the Local Product Document | | |
| | (Unsolicited AE Day 1-29) | | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

20-APR-2018

Last Update Date

# STATISTICAL ANALYSIS PLAN(V6.0)

### **Table of Contents**

| Revisions | |
|---|---|
| 1. Study Objective | ĺ |
| 2. Study Method and Study Period | ĺ |
| 2.1 Study Period6 | í |
| 2.2 Number of Subjects6 | í |
| 2.3 Study population6 | <u>,</u> |
| 2.3.1 Inclusion criteria | í |
| 2.3.2 Exclusion criteria | 7 |
| 2.4 Study Method | 7 |
| 3. Analysis Sets | ) |
| 3.1 Safety Analysis Sets | ) |
| 3.2 Efficacy Analysis Set | ) |
| 4. Endpoints | ) |
| 4.1 Safety Endpoints 12 | ) |
| 5. Assessment Criteria | ) |
| 5.1 Safety Assessment Criteria | ) |
| 6. Statistical Analyses | , |
| 6.1 Baseline Characteristics | ; |
| 6.2 Safety Analyses | ; |
| 6.2.1 Adverse Events by Baseline Characteristics | ; |
| 6.2.2. Analysis of Solicited AE | ŀ |
| 6.2.3 Analysis of Unsolicited AE | , |
| 6.3 Additional Analyses for DDS (Data Disclosure Shell) | <b>,</b> |
| 6.4 Additional Analyses for AE in the Local Product Label (Unsolicited AE Day 1-29) 16 | í |
| 7. List of Table and Data Listings | 7 |
| 7.1 Distribution of Subjects | 7 |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

20-APR-2018

Last Update Date

# STATISTICAL ANALYSIS PLAN(V6.0)

| | 7.2 Baseline Characteristics | 17 |
|---|---|---|
| | 7.3 Safety Analyses | 17 |
| | 7.4 Additional Analyses for DDS (Data Disclosure Shell) | 18 |
| | 7.5 Additional Analyses for AE in the Local Product Label (Unsolicited AE Day 1-29) | 18 |
| 8 N | Notes | 19 |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

20-APR-2018

Last Update Date

# STATISTICAL ANALYSIS PLAN(V6.0)

### 1. Study Objective

The primary objective of the study is to monitor the safety of a single dose of MenACWY-CRM vaccine in subjects from 2 months to 55 years of age, as evaluated by:

- Local and systemic solicited adverse events reported from study Day 1 (day of vaccination) through study Day 7 post-vaccination.
- All unsolicited Adverse Events (AEs) reported from study Day 1 (day of vaccination) through study Day 7 post-vaccination.
- Medically attended Adverse Events reported from study Day 1 to study termination (Day 29/early termination).
- All Serious Adverse Events (SAEs) reported from study Day 1 to study termination (Day 29/early termination).

### 2. Study Method and Study Period

### 2.1 Study Period

The trial period shall be from market launch date till approximately 22 May 2018.

### 2.2 Number of Subjects

A total of approximately 3,960 subjects are planned for enrolment into this study.

Assuming a 10% drop-out rate, this should provide approximately 3,000 evaluable subjects in the cohort 2 to 55 years of age and 600 in the cohort 2 to 23 months of age. This sample size meets the post-licensure requirements of the MFDS to provide continued safety monitoring in the Korean population.

### 2.3 Study population

### 2.3.1 Inclusion criteria

Individuals eligible for enrolment in this study are those:



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

20-APR-2018

Last Update Date

### STATISTICAL ANALYSIS PLAN(V6.0)

- 1. Male and female subjects from 2 months to 55 years of the age at the time of vaccination (including all 55 years of age subjects, up to one day before their 56<sup>th</sup> year birthday), who are scheduled to receive vaccination with MenACWY-CRM conjugate vaccine, according to the local prescribing information and routine clinical practice
- 2. To whom the nature of the study has been described and the subject or subject's parent/legal representative has provided written informed consent (written assent from minors should be also obtained if required by the relevant IRB);
- 3. Whom the investigator believes that the subject can and will comply with the requirements of the protocol (e.g., completion of the Diary Card);
- 4. Who are in good health as determined by the outcome of medical history, physical assessment and clinical judgment of the investigator

### 2.3.2 Exclusion criteria

- 1. Contraindication, special warnings and/or precautions, as evaluated by the investigators, reported in the MenACWY-CRM conjugate vaccine Korean prescribing information.
- 2. Infants who were already enrolled in this trial for previous vaccination.

### 2.4 Study Method

In order to obtain information on Regulatory PMS data after-market launch, or delegate will create the Regulatory PMS contract with the relevant clinics/hospitals and the physician in charge of the survey shall implement this Regulatory PMS in subjects that receive MenACWY-CRM in the relevant hospital/clinic since the contract date until the number of contracted survey cases, without omission, is reached.

### Overview of Study Design

This is a multicenter post marketing surveillance study to monitor the safety of MenACWY-CRM administered according to the prescribing information to 3,960 healthy subjects from 2 months to 55 years of age in Korea.

Subjects will be enrolled at the time of their visit to a participating clinic or hospital for vaccination with MenACWY-CRM according to the routine clinical care.



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

20-APR-2018

Last Update Date

# STATISTICAL ANALYSIS PLAN(V6.0)

At Visit 1 (Day 1), after obtaining consent from the subjects or subjects' parents/legal representative (and Assent Form, if required by the relevant IRB), the vaccination will be administered. Subjects will remain under observation for at least 30 minutes in the clinic after study immunization.

The subjects or subject's parent/legal representative will be then instructed to complete the Diary Card daily, reporting local and systemic adverse events and all other AEs occurring within 7 days following immunizations, and medically attended AEs or SAEs occurring up to Day 29 within the surveillance period after each study vaccination.

Subjects will also be instructed to return the completed diaries to the study site at Day 29 as follows:

- During a visit at the study center or
- Using the provided pre-addressed stamped envelope (PASE).

At the investigator discretion, the subject or subject's parent/legal representative will be reminded of the date of the study termination by a phone call at Day 29. If any clarification is required after Diary Card retrieval the site staff will follow up by phone, and any additional finding will be recorded on the subject's medical record.

In case the Diary Card is not retrieved within 10 days after Day 29, subject or subject's parent/legal representative will be contacted by phone to assess the occurrence of adverse events, determine the subject's clinical status and complete study termination. All information will be recorded by the site staff on the subject's medical record and collected in the appropriate section of the CRF.

All SAEs will be monitored until resolution and/or the cause is identified. If a SAE remains unresolved at study termination, a clinical assessment will be made by the investigator and the GSK regional physician to determine whether continued follow up of the SAE is needed.

Table 3.1-1: Safety Assessment Table

| Medical History: | From birth, collected at clinic visit |
|---|---|
| All significant past diagnoses including all allergies, major | Day 1 |
| surgeries requiring inpatient hospitalization, other significant | |
| injuries or hospitalizations, any conditions requiring | |
| prescription or chronic medication (i.e., >2 weeks in duration), | |
| or other significant medical conditions based on the | |
| investigator's judgment. | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

20-APR-2018

Last Update Date

# STATISTICAL ANALYSIS PLAN(V6.0)

| Immediate reactions: | For at least 30 minutes after |
|---|---|
| Subjects will be assessed for immediate hypersensitivity | vaccination |
| reactions. | |
| Solicited local adverse events: | Days 1-7 after vaccination |
| < 6 years : injection site erythema, injection site induration, | |
| injection site tenderness | |
| $\geq$ 6 years : injection site erythema, injection site induration, | |
| injection site pain | |
| Solicited systemic adverse events: | Days 1-7 after vaccination |
| < 6 years : change in eating habits, sleepiness, irritability, rash, | |
| vomiting, diarrhea, fever | |
| ≥ 6 years : chills, nausea, malaise, generalized myalgia, | |
| generalized arthralgia, headache, rash, fever | |
| All unsolicited AEs will be collected | Days 1-7 after vaccination |
| Medically attended Adverse Events: | From Day 1 to study termination |
| Events that require a physician's visit or an emergency room | (Day 29/early termination) |
| visit (events that are managed by telephone or means other than | |
| a face-to-face evaluation by a clinician do not qualify as | |
| medically attended AEs). | |
| Serious AEs: | From Day 1 to study termination |
| All SAEs will be collected. | (Day 29/early termination) |
| Medications: | From Day 1 to Day 7 |
| Any medications used to treat any solicited local and systemic | |
| reaction and unsolicited AE be collected. | |
| Medications: | From Day 1 to study termination |
| Any medications used to treat any medically attended AE or | (Day 29/early termination) |
| SAE will be collected. | |



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

20-APR-2018

Last Update Date

# STATISTICAL ANALYSIS PLAN(V6.0)

### 3. Analysis Sets

### 3.1 Safety Analysis Sets

### Safety Set

All subjects who

- have signed an informed consent form, undergone screening procedure(s) and received a subject number,
- received a study vaccination,
- provided post vaccination safety data.

### Safety per protocol set

All subjects in the safety Set with the exclusions of the following cases:

- (1) Subjects administered prior to the contract date.
- (2) Subjects who didn't receive MenACWY-CRM.
- (3) Follow-up failure: The subjects whose safety information cannot be identified due to follow-up loss.
- (4) Not applicable to the indication of study drug [Indication]
  - To prevent invasive meningococcal disease caused by Neisseria meningitides serogroups A, C, Y and W-135 in persons 2 months through 55 years of age.
- (5) Subjects who violate of Protocol: Those who do not meet one item at least of the inclusion/exclusion criteria.

[Inclusion criteria]

- 1) Male and female subjects from 2 months to 55 years of the age at the time of Visit 1 (including all 55 years old subjects, up to one day before their 56<sup>th</sup> year birthday), who are scheduled to receive vaccination with MenACWY-CRM conjugate vaccine, according to the local prescribing information and routine clinical practice.
- 2) To whom the nature of the study has been described and the subject or subject's parent/legal representative has provided written informed consent.
- 3) Whom the investigator believes that the subject can and will comply with the requirements of the protocol.
- 4) Who are in good health as determined by the outcome of medical history, physical



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

20-APR-2018

Last Update Date

STATISTICAL ANALYSIS PLAN(V6.0)

assessment and clinical judgment of the investigator.

[Exclusion criteria]

- 1) Contraindication, special warnings and/or precautions, as evaluated by the investigators, reported in the MenACWY-CRM conjugate vaccine Korean prescribing information
- 2) Infants who were already enrolled in this trial for previous vaccination.
- (6) Subjects who prescribed off-label dosage:
  - Vaccine schedule for children from 2 to 23 months of age :
    - Infants 2 to 6 months of age: Three doses of MenACWY-CRM, each of 0.5 ml, is to be given with an interval of at least 2 months; the fourth dose schedule be administered during the second year of life with an interval of at least 6 months after the third dose.
    - Infants 7 to 23 months of age: MenACWY-CRM is to be administered as two doses, each as single dose (0.5ml), with the second dose administered in the second year of life and at least three months after the first dose.
  - 2 to 55 years of age: MenACWY-CRM is to be administered as a single dose (0.5ml).
  - \* The infant from 2 to 23 months of age may enroll at any point, in the vaccination series, including those subjects who may already initiated vaccination series. According to parental consents, these subjects may be followed up for 29 days within the surveillance period after subsequent vaccination(s) at the same study site.

### Non-Safety per protocol set

Subjects excluded from safety per protocol set except for subjects who did not receive MenACWY-CRM and follow-up failure.

Based on rules for estimation of each number of safety evaluation cases, the following local regulation and Guideline on Standards for re-examination for new drugs, etc of MFDS, non-safety analysis set are excluded from the safety analysis set:

Guideline on Standards for re-examination for new drugs, etc (Chapter II, no. 3) Patient Population for Surveillance:

- A) Patients planned to receive a drug under surveillance by investigator's medical ju dgment shall be subject.
- B) Subject who do not use within approved range shall not be included in the subject in principal.

However, if data of subject whose use is beyond approved range is collected, p erform analysis as a separate item.



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

20-APR-2018

Last Update Date

# STATISTICAL ANALYSIS PLAN(V6.0)

C) Describe actual selection methods of subject in detail.

### 3.2 Efficacy Analysis Set

Not Applicable

### 4. Endpoints

### 4.1 Safety Endpoints

Safety will be assessed after administration of study vaccine in terms of the number and percentage of subjects with:

- Local and systemic solicited adverse events reported from study Day 1 (day of vaccination) through study Day 7 post-vaccination;
- Unsolicited AEs reported from study Day 1 (day of vaccination) through study Day 7 post-vaccination;
- Medically attended AEs reported from study Day 1 to study termination (Day 29/early termination);
- SAEs reported from study Day 1 to study termination (Day 29/early termination).

### 5. Assessment Criteria

### **5.1 Safety Assessment Criteria**

Not Applicable



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

20-APR-2018

Last Update Date

# STATISTICAL ANALYSIS PLAN(V6.0)

### 6. Statistical Analyses

### **6.1 Baseline Characteristics**

Descriptive statistics (mean, standard deviation, median, minimum and maximum) for baseline characteristics such as age, height and weight at enrollment will be calculated in the Safety set and Safety per Protocol set.

The following baseline characteristics will be reported:

- < Subject Baseline Information >
  - gender, age, ethnic origin, children group, weight, height, past diagnosis, kidney disorder, liver disorder, pre-Immunization temperature, temperature location, pregnancy
- < Study Vaccine Information >
  - vaccine site, number of previous Menveo, study vaccination number, concomitant medications

### **6.2 Safety Analyses**

The number of subjects of  $AE^{\dagger}$  and the number of  $AEs^{\dagger}$  incurred shall be calculated, the incidence proportion of  $AEs^{\dagger}$  and its 95% confidence interval will be calculated using the normal approximation on the safety set and safety per protocol set.

† AE : AE includes solicited and unsolicited AE (DAY 1-7), medically attended AE (DAY 1-29) and SAE (DAY 1-29).

### **6.2.1** Adverse Events by Baseline Characteristics

 $AE^{\dagger}s$  (as described below) will be reported (n %) for the following baseline characteristics in the safety set and safety per protocol set :

- Age group (2-23 months, 2-10, 11-18, 19-34, 35-55, 55-64)
- Children group ( $<18, \ge 18$ )
- Gender (male, female)
- Past diagnosis (yes, no)



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

20-APR-2018

Last Update Date

STATISTICAL ANALYSIS PLAN(V6.0)

- Temperature location (axillary, oral, rectal, ear)
- Administration site (left deltoid, right deltoid, left thigh, right thigh, other)
- Concomitant medication (yes, no)
- Kidney disorder (yes, no)
- Liver disorder (yes, no)
- Pregnancy (yes, no)
- Number of previous Menveo (0, 1, 2, 3)
- Study vaccination number (1, 2, 3, 4)

The n(%) of AEs<sup>†</sup> and its 95% confidence interval will be calculated using the normal approximation and analyzed using  $\chi^2$ - test. If more than 20% of expected frequencies of the cell counts are less than 5, Fisher's exact test will be used instead of the chi-square test.

† AE : AE includes solicited and unsolicited AE (DAY 1-7), medically attended AE (DAY 1-29) and SAE (DAY 1-29).

### **6.2.2.** Analysis of Solicited AE

Frequencies and % of subjects experiencing each adverse event will be presented for each symptom severity. Summary tables showing the occurrence of any local or systemic reaction overall and at each time point will also be presented (see Appendix 1 Table 4.1.3 and 4.2.3).

Post-vaccination adverse events reported from Day 1 to Day 7 will be summarized by maximal severity. The severity of local adverse events for subjects < 6 years of age will be categorized as follows. Injection-site erythema and induration: absent (0 to 9 mm), mild (10 to 25 mm), moderate (26 to 50 mm), severe (> 50 mm); injection-site tenderness: none, mild (minor light reaction to touch), moderate (cried or protested to touch), severe (cried when injected limb was moved). For subjects  $\ge$  6 years, injection-site erythema and induration absent (1 to 24 mm), mild (25 to 50 mm), moderate (51 to 100 mm), severe (>100 mm); pain: none, mild (present but does not interfere with activity), moderate (interferes with activity), severe (prevents daily activity).

For subjects  $\geq$  6 years of age, the severity of systemic adverse events (i.e., chills, nausea, malaise, generalized myalgia, generalized arthralgia, headache) occurring up to 7 days after each vaccination will be categorized as none, mild (present but not interfering with daily activity), moderate (some interference with daily activity), and severe (prevents daily activity) except for rash, which will be



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

20-APR-2018

Last Update Date

# STATISTICAL ANALYSIS PLAN(V6.0)

categorized as none, urticarial, or other.

For subjects < 6 years of age, the severity of systemic adverse events occurring up to 7 days after each vaccination will be categorized as follows. Change in eating habits: none (no change in appetite), mild (eating less than normal for 1 to feeds), moderate (missed 1 or 2 feeds), severe (missed more than 2 feeds); sleepiness: none (no change in alertness), mild (shows an increased alertness), moderate (sleeps through feeds), severe (sleeps most of the time and it is hard to arouse him/her); irritability: none (no change in child disposition), mild (requires more cudding and he/she is less playful than usual), moderate (more difficult to settle), severe (unable to console); rash: none, urticarial, or other; vomiting: none, mild (1-2 episodes/24 hours), moderate (>2 episodes/24 hours), severe (requires outpatient hydratation); diarrhea: none (fewer than 2 loose stools/24 hours), mild (2-3 loose stools or < 400 gms/24 hours), moderate (4-5 stools or 400-800 gms/24 hours), severe (6 or more watery stools or > 800 gms/24 hours or requires outpatient IV hydration).

Body temperature will be categorized as  $<38^{\circ}$ C (no fever),  $\ge 38^{\circ}$ C (fever) and will be summarized by 0.5°C increments from 36.0°C up to  $\ge 40^{\circ}$ C. Additionally, no fever vs. fever will be reported.

Each local and systemic adverse event will also be categorized as none vs. any.

### 6.2.3 Analysis of Unsolicited AE

All unsolicited AEs and MAAE recorded in the CRF will be mapped to preferred terms using the most recent MedDRA dictionary and classified by System organ class (SOC) and Preferred Terms (PT). Under the classification standard of MedDRA terms, and all AEs excluding the AEs whose causal relation with the study medication is 'Not Related' shall be treated as AEs whose causal relation cannot be excluded {hereafter "Adverse Drug Reaction(ADR)"}.

- ① The frequency and percentage of unsolicited AE (Day 1-7) and MAAE (Day 1-29) according to the expected, serious, severity, frequency, action taken, outcome, relationship to MenACWY-CRM regarding occurred AE will be calculated.
- ② The frequency of unsolicited AEs (Day 1-7) and MAAE (Day 1-29) will be classified into the preferred terms according to the expected, serious, severity, frequency, action taken, outcome, relationship to MenACWY-CRM.
- 3 The number of subjects and percentage of SAE/Serious ADR (SADR), unexpected AE/ADR,



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

20-APR-2018

Last Update Date

# STATISTICAL ANALYSIS PLAN(V6.0)

MAAE/ADR, unsolicited AE/ADR and continuous solicited AE/ADR will be calculated according to the preferred terms. And the number of subjects and percentage by study vaccination number of SAE/Serious ADR (SADR), unexpected AE/ADR, MAAE/ADR, unsolicited AE/ADR and continuous solicited AE/ADR will be calculated according to the preferred terms in infants 2 to 23 months.

④ For subjects excluded from safety per protocol set<sup>†</sup>, the number of subjects and the percentage of SAE/Serious ADR (SADR), unexpected AE/ADR, MAAE/ADR, unsolicited AE/ADR and continuous solicited AE/ADR will be calculated according to the preferred terms. And the number of subjects and percentage by study vaccination number of SAE/Serious ADR (SADR), unexpected AE/ADR, MAAE/ADR, unsolicited AE/ADR and continuous solicited AE/ADR will be calculated according to the preferred terms in infants 2 to 23 months.

† Subject excluded from safety per protocol set: Except for subjects who didn't receive study vaccination and follow-up failure.

### 6.3 Additional Analyses for DDS (Data Disclosure Shell)

The following will be presented in the Safety set and Safety per Protocol set.

- Frequency and percentage by Age group (2-23 months, 2-10, 11-18, 19-64) will be presented.
- Frequency and percentage by study termination and reason not completed will be presented.
- The number of subjects of Non-SAE and the number of Non-SAE incurred shall be calculated, the incidence proportion of Non-SAE and its 95% confidence interval will be calculated using the normal approximation.
- The number of death resulting from AE shall be calculated.
- The number of subjects and percentage of Non-SAE will be calculated according to the preferred terms.

### 6.4 Additional Analyses for AE in the Local Product Label (Unsolicited AE Day 1-29)

The following will be presented in the Safety set and Safety per Protocol set.

- Preferred terms of Serious AE/ADR, unexpected AE/ADR will be presented respectively according to the proportion of AE in the local product label.



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

20-APR-2018

Last Update Date

STATISTICAL ANALYSIS PLAN(V6.0)

### 7. List of Table and Data Listings

### 7.1 Distribution of Subjects

- Number of subjects contracted to the study: The number of subjects are to be collected (under contract) as contracted by the investigator.
- Number of retrieving completed CRFs: Total number of subjects whose completed CRFs.
- Number of safety assessment population: Number of safety assessment population among total number.

### 7.2 Baseline Characteristics

- Mean and standard deviation (SD) or frequency and percentage by gender, age, ethnic origin, weight, height, past diagnosis, pre-Immunization temperature, temperature location, pregnancy
- Frequency and percentage by vaccine site, number of previous Menveo, study vaccination number, concomitant medications.

### 7.3 Safety Analyses

- Incidence proportion and the number of AEs according to the baseline characteristics (frequency and percentage).
- The number of the expected serious, severity, frequency, action taken, outcome, relationship to MenACWY-CRM for Unsolicited AE (DAY 1-7) and MAAE (DAY 1-29) (frequency and percentage).
- The number of AEs for the severity, day, fever to MenACWY-CRM according to individual solicited AE (DAY 1-7) (frequency and percentage).
- Incidence proportion and number according to the preferred terms of SAE/SADR, unexpected AE/ADR, MAAE/ADR, unsolicited AE/ADR and continuous solicited AE/ADR (frequency and percentage)
- For subjects excluded from safety per protocol set<sup>†</sup> incidence proportion and number according to the preferred terms of SAE/SADR, unexpected AE/ADR, MAAE/ADR, unsolicited AE/ADR and continuous solicited AE/ADR (frequency and percentage).



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

20-APR-2018

Last Update Date

# STATISTICAL ANALYSIS PLAN(V6.0)

† Subject excluded from safety per protocol set: Except for subjects who didn't receive study mediation and follow-up failure.

### 7.4 Additional Analyses for DDS (Data Disclosure Shell)

- Frequency and percentage by Age group (2-23 months, 2-10, 11-18, 19-64)
- Frequency and percentage by study termination and reason not completed
- Incidence proportion and the number of Non-SAE
- The number of death resulting from AE (frequency and percentage)
- Incidence proportion and number according to the preferred terms of Non-SAE (frequency and percentage)

### 7.5 Additional Analyses for AE in the Local Product Label (Unsolicited AE Day 1-29)

- Preferred terms of Serious AE/ADR, unexpected AE/ADR will be presented respectively according to the proportion.



THIS DOCUMENT AND INFORMATION CONTAINED HEREIN IS PROPRIETARY TO COMPANY AND IS NOT TO BE DISCLOSED WITHOUT THE WRITTEN PERMISSION OF COMPANY.

20-APR-2018

Last Update Date

# STATISTICAL ANALYSIS PLAN(V6.0)

### 8. Notes

- Each statistical analysis will be carried out with SAS Software version 9.4 or more recent version.
- In the descriptive statistics, mean, SD, minimum, median, and maximum will be calculated for continuous variables, and frequency and percentage for categorical variables.
- Data including sign of inequality such as "≥20", ">20" will be excluded from analysis.
- All test statistics will be the results of two-sided tests with the statistical significant level of 0.05.
- The followings shall be included only in re-examination report:
  - Analysis by type of concomitant medications
  - Item ② of paragraph 6.2.3
  - Estimation of 95% confidence interval for incidence proportion of AEs by background factors
  - Paragraph 6.3, 6.4